Study alias & e-track number(s): 204812 (RSV F-021) Version: DRAFT1 Date:10-NOV-2016



**Detailed Title:** A Phase II, randomised, observer-blind, controlled,

multi-country study to rank different formulations of GSK Biologicals' investigational RSV vaccine (GSK3003891A), based on immunogenicity, reactogenicity and safety, when administered to

healthy women, aged 18 - 45 years.

**Scope:** All data pertaining to the above study.

**Co-ordinating author:** PPD (Expert Biostatistician)

Other author(s): PPD (Lead Biostatistician)

Reviewed by: (Clinical Research & Development

Leads)

(Clinical Research & Development

Leads)

(Central Safety Physician)

PPD (Lead Statistician)

PPD (Project Statistician)

(Statistical Peer Reviewer)

PPD (Lead Statistical Analyst)

PPD (Lead Sc writer)
PPD (Lead Sc writer)

PPD (Regulatory Affairs

Representative)

Approved by: (Clinical Research & Development

Leads)

(Lead Biostatistician)

PPD (Lead Sc writer)

FORM-9000026972-01 Statistical Analysis Plan Template

Effective date: 01 Jan 2016

GSK SOP Reference: SOP-9000026972 Form Owner: CEG-BSP, PPD


Study alias & e-track number(s): 204812 (RSV F-021)

Version: DRAFT1 Date:10-NOV-2016



#### **TABLE OF CONTENTS**

| | | | | PAGE |
|---|---|---|---|---|
| LIS | T OF A | BBREVIA | TIONS | 4 |
| 1. | DOCUMENT HISTORY6 | | | |
| 2. | STUD | Y DESIGN | N | 6 |
| 3. | OBJE | CTIVES | | 10 |
| 4. | ENDP | OINTS | | 10 |
| 5. | ANAL`<br>5.1.<br>5.2. | Definition 5.1.1. 5.1.2. | Exposed Set (ES) Per-Protocol Set (PPS) for analysis of immunogenicity or eliminating data from Analysis Sets Elimination from Exposed Set (ES) Full Analysis Set (FAS) Elimination from Per-protocol analysis Set (PPS) for | 13<br>13<br>13<br>13<br>13 |
| | 5.3. | Importar<br>protocol | analysis of immunogenicityt protocol deviation not leading to elimination from per-<br>analysis set | |
| 6. | STATI<br>6.1. | | ANALYSES Aphy Analysis of demographics/baseline characteristics planned in the protocol | 15 |
| | <ul><li>6.2.</li><li>6.3.</li><li>6.4.</li><li>6.5.</li></ul> | Analysis<br>Analysis<br>6.4.1.<br>6.4.2. | of immunogenicity | 16<br>2021<br>21 |
| 7. | ANAL' | YSIS INTE | ERPRETATION | 21 |
| 8. | CONDUCT OF ANALYSES | | | |

Study alias & e-track number(s): 204812 (RSV F-021)



| | 8.1. | Sequence of analyses | 22 |
|---|---|---|---|
| | 8.2. | Statistical considerations for interim analyses | 24 |
| 9. | CHAN | GES FROM PLANNED ANALYSES | 24 |
| 10. | LIST C | OF FINAL REPORT TABLES, LISTINGS AND FIGURES | 24 |
| 11. | 11.1.<br>11.2. | X 1: STANDARD DATA DERIVATION RULE AND STAT METHODS | 25<br>25<br>25<br>26 |
| 12. | | X 2: CALCULATION OF INDIVIDUAL AND OVERALL ABILITY INDEX | 32 |
| 12 | ΔNNE. | X 3: STUDY SPECIFIC MOCK TEL | 37 |

Form Owner: CEG-BSP, PPD

Study alias & e-track number(s): 204812 (RSV F-021)




#### LIST OF ABBREVIATIONS

AE Adverse Event

AIDS Acquired Immunodeficiency Syndrome

ANCOVA Analysis of Covariance
ANOVA Analysis of Variance

ALT Alanine Aminotransferase

AST Aspartate Aminotransferase

ATP According-to-Protocol

CDISC Clinical Data Interchange Standards Consortium

CI Confidence Interval

eCRF Electronic Case Report Form

Eli Type Internal GSK database code for type of elimination code

ES Exposed Set

FAS Full Analysis Set

GMC Geometric mean antibody concentration

GMT Geometric mean antibody titer

GSK GlaxoSmithKline

ICH International Conference on Harmonisation
IDMC Independent Data Monitoring Committee

IND Investigational New Drug

iSRC Internal Safety Review Committee

LL Lower Limit of the confidence interval

LLOQ Lower Limit of Quantification

MA-RTI Medically Attended Respiratory Tract Infection
MedDRA Medical Dictionary for Regulatory Activities

FORM-9000026972-01 Statistical Analysis Plan Template

Effective date: 01 Jan 2016

GSK SOP Reference: SOP-9000026972 Form Owner: CEG-BSP, PPD


Study alias & e-track number(s): 204812 (RSV F-021)




NEO Neogenin

PCA Palivizumab Competing Antibodies

PCD Primary completion Date

PCR Polymerase Chain Reaction

PPS Per Protocol Set

PreF Purified recombinant RSV F protein, engineered to preferentially

maintain the pre-fusion conformation

RSV Respiratory syncytial virus

RTI Respiratory Track Infection

SAE Serious adverse event

SAP Statistical Analysis Plan

SAS Statistical Analysis System

SBIR (GSK) Biological's Internet Randomization System

SRT Safety Review Team

TFL Tables Figures and Listings

TOC Table of Content

TVC Total Vaccinated Cohort

UL Upper Limit of the confidence interval

WBC White Blood Cells




#### 1. DOCUMENT HISTORY

| Date | Description | Protocol Version |
|-------------|--------------------------|---------------------|
| 25-AUG-2016 | Version 1: first version | Final – 20-JUL-2016 |

#### 2. STUDY DESIGN

Figure 1. Study design overview



**V** = Visit; **D** = Day; **VACC** = vaccination; **BS** = blood sample; **h/b** = blood sample for haematology/biochemistry; **Imm** = blood sample for immunogenicity; **C** = contact; **RSV** = Respiratory Syncytial Virus; **PCR** = Polymerase Chain Reaction. 1 Safety data up to (minimum) 7 days post-vaccination (including Day 7 haematology and biochemistry parameters) of the first 25% of subjects vaccinated in the study will be reviewed by iSRC.

2 In case of a MA-RTI (e.g. visit to the GP for respiratory symptoms including but not limited to cough, sputum production, difficulty breathing), the subject will be asked to contact the Investigator to enable completion of an event related eCRF and the collection of a nasal swab within 72h after the medical attendance. Vertical lines stand for analysis on all subjects.

• **Experimental design**: Phase II, observer-blind, randomised, controlled, multi-country, study with four parallel groups.

FORM-9000026972-01 Statistical Analysis Plan Template

Effective date: 01 Jan 2016




- **Duration of the study**: the intended duration of the study will be approximately 1 year from Visit 1 to study conclusion (Day 360).
  - Epoch 001: Primary starting at Visit 1 (Day 0) and ending at Visit 5 (Day 90).
  - Epoch 002: Follow-up phase starting one day after Day 90 and ending at Day 360 contact.
- **Primary completion Date (PCD)**: Visit 3 (Day 30).
- End of Study (EoS): Last testing results released of samples collected at Visit 5 (i.e. last testing results released for the assays related to the primary and secondary endpoints).

#### • Study groups:

Table 1 Study groups and epochs foreseen in the study

| Ctudy average | Number of Age (Min/May) | | Epochs | |
|---|---|---|---|---|
| Study groups | subjects | Age (Min/Max) | Epoch 001 | Epoch 002 |
| 30 PreF | ~100 | 18 - 45 years | Х | Х |
| 60 PreF | ~100 | 18 - 45 years | Х | Х |
| 120 PreF | ~100 | 18 - 45 years | Х | Х |
| Control | ~100 | 18 - 45 years | Х | Х |

Table 2 Study groups and treatment foreseen in the study

| Treatment name | Vaccine/ Product | Study Groups | | | |
|---|---|---|---|---|---|
| Treatment name | name | 30 PreF | 60 PreF | 120 PreF | Control |
| 20 ug DroE | PreF-30 | Х | | | |
| 30 µg PreF | NaCl | 1 ^ | | | |
| 60 ug DroF | PreF-60 | | Х | | |
| 60 µg PreF | NaCl | | ^ | | |
| 120 ug DroF | PreF-120 | | | Х | |
| 120 µg PreF | NaCl | | | ^ | |
| Placebo | Formulation buffer S9b | | | | Х |

• Control: Placebo control

• Vaccination schedule: One intramuscular vaccination at Day 0.

Study alias & e-track number(s): 204812 (RSV F-021)




• **Treatment allocation**: Subjects will be randomised using a centralised randomisation system on internet (SBIR) at Day 0. The randomisation algorithm will use a minimisation procedure accounting for age (18 - 32 years or 33 - 45 years) and centre.

The following group and sub-group names will be used for the statistical analyses:

| Group order in tables Group label in tables | | Group definition for footnote |
|---|---|---|
| 1 | 30 PreF | 30 mcg PreF |
| 2 | 60 PreF | 60 mcg PreF |
| 3 | 120 PreF | 120 mcg PreF |
| 4 | Control | Placebo |

Some tables might be presented by age category according to the following description:

| Sub-group | Sub-group order in tables | Sub-group label in tables | Sub-group definition for footnote |
|---|---|---|---|
| Age | 1 | 18-32Y | 18-32 years old subjects |
| | 2 | 33-45Y | 33-45 years old subjects |

• **Blinding**: Observer-blind in Epoch 001 and single-blind in Epoch 002.

Table 3 Blinding of study epochs

| Study Epochs | Blinding |
|--------------|----------------|
| Epoch 001 | observer-blind |
| Epoch 002 | single-blind |

#### • Sampling schedule:

- Blood samples for haematology/biochemistry will be collected (~10 mL) from all subjects at Visit 1 (Day 0), Visit 2 (Day 7), Visit 3 (Day 30), Visit 4 (Day 60) and Visit 5 (Day 90).
- Blood samples for humoral immune response evaluation will be collected (~17 mL) from all subjects at Visit 1 (Day 0), Visit 3 (Day 30), Visit 4 (Day 60) and at Visit 5 (Day 90).
- Nasal swabs will be collected from subjects in case of a medically attended respiratory tract infection from enrolment (Visit 1) until study end (Contact 3).

FORM-9000026972-01 Statistical Analysis Plan Template

Effective date: 01 Jan 2016

GSK SOP Reference: SOP-9000026972 Form Owner: CEG-BSP, PPD


Study alias & e-track number(s): 204812 (RSV F-021)




• Type of study: self-contained

• **Data collection:** Electronic Case Report Form (eCRF).

- Safety monitoring: When the first 25% of subjects (i.e. ~100 subjects; ~25 subjects per study group) have been vaccinated, enrolment will be paused until completion of an unblinded review by a GSK internal Safety Review Committee (iSRC). Continuation of study enrolment will be conditional to a favourable outcome of the iSRC evaluation of all available safety and reactogenicity data collected up to at least 7 days post-vaccination (including Day 7 haematology and biochemistry parameters). In addition, the blinded safety data will be reviewed by GSK Biologicals' Safety Review Team (SRT) on a regular basis throughout the study. Analyses related to iSRC evaluation will be described in a separate document (SAP/TFL for ISRC).
- In case of a MA-RTI (e.g. visit to the GP for respiratory symptoms including but not limited to cough, sputum production, difficulty breathing), the subject will be asked to contact the investigator to enable the collection of a nasal swab within 72 hours after the medical attendance.

Study alias & e-track number(s): 204812 (RSV F-021)




#### 3. OBJECTIVES

#### 3.1 Primary Objective

• To rank different formulations of the investigational RSV vaccine based on safety/reactogenicity and immunogenicity data up to 1 month post-vaccination (Day 30).

#### 3.2 Secondary objectives

- To evaluate the reactogenicity and safety of a single intramuscular dose of the RSV investigational vaccines up to study conclusion.
- To evaluate the immunogenicity of a single intramuscular dose of the RSV investigational vaccines up to 90 days after vaccination (Day 90).
- To further assess the safety of the investigational RSV vaccines by evaluating whether a single dose of the vaccines induces antibodies against the residual host cell protein neogenin (NEO) up to 1 month post-vaccination (Day 30).
- To estimate the incidence of medically attended RSV-associated RTIs up to study conclusion.

### 3.3 Tertiary objective

• If deemed necessary, to further characterize the immune response of a single intramuscular dose of the RSV investigational vaccines.

Refer to Section 5.7.3 Laboratory assays of the Protocol for additional testing proposed to further characterize the immune response to the investigational RSV vaccine.

#### 4. ENDPOINTS

### 4.1 Primary

- Occurrence of AEs from vaccination up to Day 7, for all subjects in each investigational RSV vaccine group:
  - Occurrence of any Grade 2 and Grade 3 general AE (solicited and unsolicited);

FORM-900026972-01 Statistical Analysis Plan Template Effective date: 01 Jan 2016


GlaxoSmithKline

- Occurrence of Grade 2 and Grade 3 fever;
- Occurrence of any vaccine-related SAE.
- Functional antibody titres against RSV at Day 0 and Day 30, for all subjects in each investigational RSV vaccine group.
  - Neutralising antibody titres against RSV-A
- PCA concentrations at Day 0 and Day 30 for all subjects in each investigational RSV vaccine group

#### 4.2 Secondary

- Occurrence of AEs from vaccination up to study conclusion:
  - Occurrence of each solicited local and general AE, during a 7-day follow-up period after vaccination (i.e. the day of vaccination and 6 subsequent days), for all subjects in all groups;
  - Occurrence of any unsolicited AE, during a 30-day follow-up period after vaccination (i.e. the day of vaccination and 29 subsequent days), for all subjects in all groups;
  - Occurrence of any haematological (haemoglobin level, White Blood Cells [WBC], lymphocyte, neutrophil, eosinophil and platelet count) and biochemical (alanine amino-transferase [ALT], aspartate amino-transferase [AST] and creatinine) laboratory abnormality at Day 0, Day 7, Day 30, Day 60 and Day 90 for all subjects in all groups;
  - Occurrence of any SAE, for all subjects in all groups.
- Functional antibody titres against RSV for all subjects in all groups:
  - Neutralising antibody titres against RSV-A at Day 0, Day 30, Day 60 and Day 90;
  - Neutralising antibody titres against RSV-B at Day 0, Day 30, Day 60 and Day 90.
- PCA concentration at Day 0, Day 30, Day 60 and Day 90 for all subjects in all groups.
- Humoral immune response to the residual host cell protein NEO in the investigational RSV vaccine at pre-vaccination (Day 0), and 1 month post-vaccination (Day 30) for all subjects in all groups.

FORM-9000026972-01 Statistical Analysis Plan Template Effective date: 01 Jan 2016

Study alias & e-track number(s): 204812 (RSV F-021)




- Antibody concentrations against NEO
- Occurrence of medically attended RSV-associated RTIs up to study conclusion

### 4.3 Tertiary

See section 5.7.3 of the Protocol for additional testing proposed to further characterize the immune response to the investigational RSV vaccine.

#### 5. ANALYSIS SETS

#### 5.1. Definition

In order to align to ICH and CDISC terminology, the Total Vaccinated Cohort (TVC) and the According To Protocol cohort (ATP) have been renamed Exposed Set (ES) and Per-Protocol Set (PPS) respectively. Two cohorts will be defined for the purpose of the analysis: the Exposed Set (ES) and the Per-Protocol Set (PPS) for analysis of immunogenicity. All analyses will be performed per treatment actually administered.

#### 5.1.1. Exposed Set (ES)

The ES will include all subjects with study vaccine administration documented:

- A safety analysis based on the ES will include all vaccinated subjects
- An **immunogenicity** analysis based on the ES will include all vaccinated subjects for whom immunogenicity data are available.

#### 5.1.2. Per-Protocol Set (PPS) for analysis of immunogenicity

The PPS for immunogenicity will be defined by time point and will include all vaccinated subjects.

- Meeting all eligibility criteria (i.e. no protocol violation linked to the inclusion/ exclusion criteria, including age).
- Who received the study vaccine according to protocol procedures.

FORM-9000026972-01 Statistical Analysis Plan Template Effective date: 01 Jan 2016 GSK SOP Reference: SOP-9000026972

Form Owner: CEG-BSP, PPD

Study alias & e-track number(s): 204812 (RSV F-021)




- Who did not receive a concomitant vaccination/medication/product leading to exclusion from the PPS analysis up to the corresponding timepoint as described in Section 6.6.2 of the Protocol
- Who did not present with an intercurrent medical condition leading to exclusion from the PPS analysis up to the corresponding timepoint, as described in Section 6.7 of the Protocol.
- Who complied with the post-vaccination blood sampling schedule at the corresponding timepoint, as specified in Table 5 of the Protocol.
- For whom post-vaccination immunogenicity results are available for at least 1 assay at the corresponding timepoint.

When presenting different timepoints, the PPS for immunogenicity will be adapted for each timepoint (up to D30 and up to D90).

#### 5.2. Criteria for eliminating data from Analysis Sets

Elimination codes are used to identify subjects to be eliminated from analysis. Detail is provided below for each set.

### 5.2.1. Elimination from Exposed Set (ES)

Code 1030 (Study vaccine not administered at all) and code 900 (invalid informed consent or fraud data) will be used for identifying subjects eliminated from ES.

#### 5.2.2. Full Analysis Set (FAS)

NA

# 5.2.3. Elimination from Per-protocol analysis Set (PPS) for analysis of immunogenicity

A subject will be excluded from the PPS for analysis of immunogenicity analysis under the following conditions

FORM-9000026972-01 Statistical Analysis Plan Template Effective date: 01 Jan 2016

GSK SOP Reference: SOP-9000026972 Form Owner: CEG-BSP, PPD




#### Elimination code from PPS for analysis of immunogenicity Table 4

| Code<br>Eli Type | Condition under which the code is used |
|---|---|
| =M1/M2 | |
| 900 | Invalid informed consent or fraud data |
| 1030 | Study vaccine dose not administered at all but subject number allocated |
| 1040 | Administration of concomitant vaccine(s) forbidden in the protocol up to blood sample at Visit 3/Visit 5 |
| 1050 | Randomisation failure |
| 1060 | Randomisation code broken at the investigator site OR at GSK Safety department |
| 1070 | Study vaccine dose not administered according to protocol: |
| | - Site or route of study vaccine administration wrong or unknown |
| | - Administration not according to protocol for reason specified by the investigator other than side, site and route |
| | - Wrong replacement or study vaccine administered (not compatible with the vaccine regimen associated to the treatment number) |
| 1080 | Vaccine has been administered (effective treatment number) despite a temperature deviation qualified by Status QA GMP NON Use |
| 1090 | Vaccine has been administered (effective treatment number) out of the expiration date at the time of administration |
| 2010 | Protocol violation linked to the inclusion/exclusion criteria |
| 2030 | Biochemistry, haematology and other laboratory values outside normal range before any vaccination |
| 2040 | Administration of any medication forbidden by the protocol up to blood sample at Visit 3/Visit 5 |
| 2050 | Underlying medical condition forbidden by the protocol up to blood sample at Visit 3/Visit 5 |
| 2060 | Concomitant infection related to the vaccine which may influence the immune response up to blood sample at Visit 3/Visit 5 |
| 2070 | Concomitant infection not related to the vaccine which may influence the immune response up to blood sample at Visit 3/Visit 5 |
| 2090 | Non compliance with blood sample schedule at Visit 3/Visit 5 |
| 2100 | Essential serological data missing: serological data missing for all antigens at both sampling time points at Visit 3/Visit 5 |
| 2120 | Obvious incoherence, abnormal serology evolution or error in data (Eg; incoherence between CRF and results, wrong sample labelling) |




M1 for Visit 3 (Day30) analysis and M2 for Visit 5 (Day 90) analysis

Eli type is Internal GSK database code for type of elimination code

# 5.3. Important protocol deviation not leading to elimination from per-protocol analysis set

The following important protocol deviations will be reported by groups:

- Forced randomization: In case of supplies shortage for the next assigned vaccine according to the randomization schedule at the clinical site, the randomization system will use the forced randomization procedure in order to continue to enrol and vaccinate subjects. The system moves seamlessly to the next treatment/randomization number for which vaccine supplies are available. The site will not be aware of the forced randomization event.
- Manual randomization: In case of the randomization system is unavailable, the investigator has the option to perform randomization by selecting supplies available at the site according to a pre-defined rule.
- Short follow-up: subjects who completed the last study contact before the minimum length of follow-up requirement.

#### 6. STATISTICAL ANALYSES

Note that standard data derivation rule and statistical methods are described in Annex 1 and will not be repeated below.

#### 6.1. Demography

# 6.1.1. Analysis of demographics/baseline characteristics planned in the protocol

The analysis of demography will be performed on the ES and on the PPS for immunogenicity.

Demographic characteristics such as age at vaccination in years, race, ethnicity, vital signs and cohort description will be summarised by group using descriptive statistics:

• Frequency tables will be generated for categorical variable such as race.

FORM-9000026972-01 Statistical Analysis Plan Template Effective date: 01 Jan 2016

Study alias & e-track number(s): 204812 (RSV F-021)




• Mean, median, standard error and range will be provided for continuous data such as age.

The distribution of subjects will be tabulated as a whole and per group and for each age category (18 - 32 years and 33 - 45 years).

Withdrawal status will be summarised by group using descriptive statistics:

- The number of subjects enrolled into the study as well as the number of subjects excluded from PPS analyses will be tabulated.
- The number of withdrawn subjects will be tabulated according to the reason for withdrawal.

#### 6.2. Analysis of immunogenicity

The analysis will be performed on the applicable PPS cohort for immunogenicity and, if in any group the percentage of vaccinated subjects with serological results excluded from the PPS for analysis of immunogenicity is  $\geq 5\%$ , a second analysis will be performed on the ES.

#### Within group evaluation

Humoral Immune response to RSV vaccine

For each group, at each timepoint that blood samples are collected and for each assay (unless specified otherwise):

- GMTs/GMCs will be tabulated with 95% CI based on log-transformed values and represented graphically.
- Percentage of subjects above the seropositivity threshold will be tabulated with exact 95% CI.

Percentage of subjects above the seropositivity threshold and GMTs/GMCs will also be tabulated by group for each age category (18 - 32 years and 33 - 45 years).

• Pre- and post-vaccination antibody titres/concentrations will be displayed using reverse cumulative curves.

Study alias & e-track number(s): 204812 (RSV F-021)




- The distributions of **neutralising** antibody titres will be tabulated in the tables with log2 scale (< 7, 7-8, > 8-9, > 9-10, > 10-11, > 11-12, > 12 log2).
- Percentage of responders in terms of **neutralising** antibody titres will be tabulated with exact 95% CI.
- Individual post-vaccination *versus* pre-vaccination results will be plotted using scatter plots. Results of the control group will be used as a reference.
- Geometric mean of ratios of antibody titres/concentrations at each post-vaccination timepoint over pre-vaccination will be tabulated with 95% CI.
- Distribution of the fold increase of **neutralising** antibody titres will be tabulated: by pre-vaccination titre category: < 7, 7-8, > 8-9, > 9-10, > 10-11, > 11-12, > 12 (log2), and by cumulative categories:  $< 7, \ge 7, \ge 8, \ge 9, \ge 10, \ge 11, \ge 12 (log2)$ .
- The kinetics of individual antibody titres/concentrations will be plotted as a function of time for subjects with results available at all timepoints.
- An analysis of variance model for repeated measures will be fitted to calculate GMTs/GMCs using mixed model with treatment group, visit and their interaction as fixed effects.

If deemed necessary, the same analyses may be done by age category (18 - 32 years and 33 - 45 years).

#### **Between group evaluation**

Exploratory comparisons will be performed for **RSV neutralising** antibody titres and PCA concentrations post-vaccination (Day 30, Day 60 and Day 90) between the different RSV vaccine groups.

- Estimation of GMT/GMC ratios between groups with corresponding 95% CI using an ANCOVA model on the logarithm10 transformation of the titres/concentrations. If a statistically significant difference is found (p <0.05), pairwise comparisons will be made using Tukey's multiple comparison adjustment. This model includes:
  - o The vaccine group as the fixed effect
  - The pre-vaccination titre/concentration as the covariate
  - Age groups (18-32 years and 33-45 years) and center as the categorical covariate

FORM-9000026972-01 Statistical Analysis Plan Template

Effective date: 01 Jan 2016

GSK SOP Reference: SOP-9000026972

Form Owner: CEG-BSP, PPD

Study alias & e-track number(s): 204812 (RSV F-021)




- GMT/GMC ratios with corresponding 95% CI will be computed between the RSV vaccine groups
  - o PreF-120 minus PreF-30
  - o PreF-120 minus PreF-60
  - o PreF-60 minus PreF-30

### 6.3. Analysis of safety

The analysis of safety will be performed on the ES.

#### Within group evaluation

The percentage of subjects with at least one **local AE** (solicited and unsolicited), with at least one **general AE** (solicited and unsolicited) and with any AE during the 7-day or 30-day follow-up period after vaccination will be tabulated with exact 95% CI. The same computations will be done for ≥ Grade 2 and Grade 3 AEs, for any AEs considered related to vaccination, for any Grade 3 AEs considered related to vaccination and for AEs resulting in medically attended visit.

The percentage of subjects reporting each individual **solicited local AE** (any grade,  $\geq$  Grade 2, Grade 3, resulting in medically attended visit) during the 7-day follow-up period after vaccination will be tabulated for each study vaccine for each group. The percentage of subjects reporting each individual **solicited general AE** (any grade,  $\geq$  Grade 2, Grade 3, any related,  $\geq$  Grade 2 related, Grade 3 related, resulting in medically attended visit) during the 7-day follow-up period after vaccination will be tabulated for each group.

For fever during the 7-day follow-up period after vaccination, the number and percentage of subjects reporting fever will be reported by half degree (°C) cumulative increments. Similar tabulations will be performed for causally related fever, Grade 3 (> 39.5°C) causally related fever and fever resulting in a medically attended visit. In addition, the prevalence of any and Grade 3 fever will be presented graphically over time after vaccination.

The percentage of subjects with any **unsolicited** symptoms within 30 days after vaccination with its exact 95% CI will be tabulated by group and by Medical Dictionary for Regulatory Activities (MedDRA) preferred term. Similar tabulation will be done for Grade 3 unsolicited symptoms, for any causally related unsolicited symptoms, for Grade




3 causally related unsolicited symptoms and for unsolicited symptoms resulting in a medically attended visit (The verbatim reports of unsolicited symptoms will be reviewed by a physician and the signs and symptoms will be coded according to the MedDRA Dictionary for Adverse Reaction Terminology. Every verbatim term will be matched with the appropriate Preferred Term).

**SAEs** reported throughout the study will be described in detail.

**Pregnancy** exposures throughout the study and pregnancy outcomes will be described in detail (if applicable).

The percentage of subjects using **concomitant medication** (any medication, any antipyretic and any antipyretic taken prophylactically) during the 7-day (Day 0 to Day 6) or 30-day (Day 0 to Day 29) follow-up period after vaccination will be summarised by group.

For all subjects in each group and each **haematology and biochemistry** parameter:

- The percentage of subjects having haematology and biochemistry results below or above the local laboratory normal ranges will be tabulated for each timepoint.
- The maximum grading post-vaccination (from Day 7 to Day 90) versus baseline (Day 0) and the percentage of subjects with laboratory parameters above or equal to Grade 1, Grade 2, Grade 3 and Grade 4 will be tabulated (Grades will be based on the FDA Guidance for Industry "Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials", see APPENDIX D of the Protocol: FDA toxicity grading scale. Those laboratory parameters not included on FDA Toxicity Grading Scale will not be graded).

Assessment of anti-NEO immune response at Day 30 post-vaccination for each group:

- GMCs pre-and post-vaccination will be tabulated with 95% CI and represented graphically.
- Individual post-vaccination *versus* pre-vaccination results will be plotted using scatter plots. Results of the control group will be used as a reference.
- Geometric mean of ratios of antibody concentrations at Day 30 over pre-vaccination will be tabulated with 95% CI.
- Distribution of the antibody concentrations pre-and post-vaccination and of fold increase after vaccination will be tabulated.

FORM-9000026972-01 Statistical Analysis Plan Template Effective date: 01 Jan 2016

Study alias & e-track number(s): 204812 (RSV F-021)




#### Between group evaluation

Exploratory comparisons between each investigational RSV vaccine group and (minus) the control group (*placebo*), and between the RSV vaccine groups will be done in terms of the percentage of subjects reporting any  $\geq$  Grade 2, Grade 3 AE (solicited and unsolicited), and/or any fever > 38.5°C, and/or any vaccine-related SAE during the 7-day follow-up period after vaccination.

- o PreF-30 minus placebo
- o PreF-60 minus placebo
- o PreF-120 minus placebo
- o PreF-120 minus PreF-30
- o PreF-120 minus PreF-60
- o PreF-60 minus PreF-30

The standardised asymptotic 95% CI for the difference between the investigational RSV vaccine groups as well as between the investigational RSV groups and (minus) the control group will be computed.

### 6.4. Analysis for ranking RSV formulations

The totality of data and sum total of evidence for particular dose(s) in terms of safety and immunogenicity will be evaluated by study team in addition to the analyses described in section 6.1 and 6.3 of this document on formulation selection. The desirability index approach described in the section below will be used as a descriptive tool to guide the formulation selection. In addition, any pertinent information from outside this study will be evaluated and may be used by the study team to help to make the final decision on a dose/formulation.

#### 6.4.1. Definition of desirability in the context of Simulations

A desirability approach will be based on safety/reactogenicity and immunogenicity data up to 1 month post-vaccination.




This method is a multi-criteria decision making approach based on desirability functions. The main idea is to identify for each endpoint a desirability function that associates any value to another one between 0 and 1 depending on its desirability ('0' being considered as not desirable at all and '1' as the most desirable). An index with values between 0 and 1 will be created for each endpoint. An overall desirability index can be calculated by computing a weighted geometric mean of the endpoint indexes. By definition, this overall index also takes values between 0 and 1 and characterises the level of desirability of any candidate formulation by a single value [Dewé, 2015].

The desirability index calculations will include reactogenicity and safety data up to Day 7 post vaccination (on the TVC) and immunogenicity data at 30 days post-vaccination (on the ATP cohort for immunogenicity up to Day 30). The formulations will be ranked based on the values obtained with this overall desirability index.

#### 6.4.2. Derived endpoints

The following endpoints will be computed and taken into account in the desirability analysis:

- 1. Incidence rate of any Grade 2 and any Grade 3 general AE (solicited and unsolicited) and any vaccine-related SAE during the 7-day follow-up period after vaccination for each investigational RSV vaccine formulation.
- 2. Incidence rate of Grade 2 and Grade 3 fever during the 7-day follow-up period after vaccination for each investigational RSV vaccine formulation.
- 3. Geometric mean of neutralising antibody titres against RSV-A at Day 30 adjusted for pre-vaccination titres.
- 4. Geometric mean of PCA concentrations at Day 30 adjusted for pre-vaccination titres.

Each individual desirability index will be calculated based on data and tabulated by the treatment group and endpoints above. The details on how to calculate individual desirability index in terms of reactogenicity and immunogenicity and overall desirability index are elaborated in Annex 2.

### 6.5. Analysis of medically attended RTIs

The analysis will be performed on the ES by study group.

FORM-9000026972-01 Statistical Analysis Plan Template Effective date: 01 Jan 2016




The proportion of subjects with at least one medically attended RSV-associated RTI identified by multiplex PCR with 95 % CI will be calculated.

Descriptive analyses (mean, median, min, max, standard deviation) of viral load assessed by the quantitative PCR (RSV-A/B) of RSV-RTI cases will be tabulated for any cases where this assay is performed.

Medically attended RSV-associated RTI co-infected or colonisation with another viral etiology identified by multiplex PCR will be described.

Medically attended RTI with any viral etiology identified by multiplex PCR will be described.

The proportion of subjects with 95% CI with at least one medically attended RTI (all causes) will be calculated by group.

#### 7. ANALYSIS INTERPRETATION

All comparative analyses will be descriptive with the aim to characterise the difference in reactogenicity/immunogenicity between groups. These descriptive analyses should be interpreted with caution considering that there is no adjustment for multiplicity for these comparisons.

#### 8. CONDUCT OF ANALYSES

Any deviation(s) or change(s) from the original statistical plan outlined in this protocol will be described and justified in the final study report.

#### 8.1. Sequence of analyses

The statistical analyses will be performed in several steps:

• In preparation of the planned iSRC evaluation, analysis of safety and reactogenicity data up to at least 7 days post-vaccination of the first 25% of all subjects will be performed (see Section 8.10.2 of the Protocol for more information).

Study alias & e-track number(s): 204812 (RSV F-021)



• The first main analysis on all subjects will be performed when all data up to 30 days post-vaccination are available (primary endpoints). In order to maintain the blind, this analysis by group will be performed by an independent statistician and the results which would lead to the unblinding of some subjects (e.g. a specific AE reported by one subject only) will be blinded (i.e. the group in which this event occurred will not be identified). No individual data listings will be provided.

- A second analysis will be performed when all data up to 90 days post-vaccination are available (secondary endpoints). At this point, the GSK statistician will be unblinded (i.e. will have access to the individual subject treatment assignments), but no individual listings will be provided. Given that summary results may unblind some specific subjects, the study will be conducted in a single-blind manner from this point onwards, with subjects remaining blinded up to study conclusion and the investigators will not have access to the treatment allocation up to study conclusion.
- The final analysis will be performed when all data up to study conclusion are available. All available tertiary endpoints will also be analysed in this step. Individual listings will only be provided at this stage.
- An integrated study report presenting all analyses will be written and made available to the investigators at the time of final analysis.
- If data for tertiary endpoints become available at a later stage, (an) additional analysis/analyses will be performed. These data will be documented in Annex(es) to the study report and will be made available to the investigators at that time.

| Description | Analysis ID | Disclosure Purpose<br>(CTRS=web posting,<br>SR=study report,<br>internal) | Dry run review<br>needed (Y/N) | Study Headline Summary (SHS)requiring expedited communication to upper management (Yes/No) | Reference for TFL |
|---|---|---|---|---|---|
| Final<br>Analysis | E1_01 | Study report<br>CTRS | N | Yes | All tables E1_01 identified in TFL dated xxxxxxx |

FORM-9000026972-01 Statistical Analysis Plan Template

Effective date: 01 Jan 2016

Study alias & e-track number(s): 204812 (RSV F-021)




| ISRC Day 7<br>safety on<br>25% of<br>subjects | E1_02 | Internal | N | Yes | All tables<br>E1_01<br>identified in<br>TFL for ISRC<br>dated xxxxxx |
|---|---|---|---|---|---|
| Analysis of<br>Day 30 | E1_03 | Internal<br>CTRS | N | Yes | All tables<br>E1_03<br>identified in<br>TFL dated<br>xxxxxx |
| Analysis of<br>Day 90 | E1_04 | Internal | N | Yes | All tables<br>E1_04<br>identified in<br>TFL dated<br>xxxxxx |

### 8.2. Statistical considerations for interim analyses

No interim analysis will be performed.

#### 9. CHANGES FROM PLANNED ANALYSES

In order to align to ICH and CDISC terminology the Total Vaccinated Cohort and the According To Protocol cohort have been renamed Exposed Set (ES) and Per-Protocol Set (PPS) respectively.

# 10. LIST OF FINAL REPORT TABLES, LISTINGS AND FIGURES

The TFL TOC provides the list of tables/listings and figures needed for the study report. It also identifies the tables eligible for each analyses and their role (synopsis, in-text, post-text, SHS,...)

Study alias & e-track number(s): 204812 (RSV F-021)

Version: DRAFT1 Date: 10-NOV-2016



#### 11. ANNEX 1 STANDARD DATA DERIVATION RULE AND STAT METHODS

#### 11.1. Statistical method references

The exact two-sided 95% CIs for a proportion within a group will be the Clopper-Pearson exact CI [Clopper CJ, Pearson ES. The use of confidence or fiducial limits illustrated in the case of binomial. *Biometrika*. 1934;26:404-413].

The standardised asymptotic two-sided 95% CI for the group difference in proportions is based on the method described in the following paper:Robert G. Newcombe, interval estimation for the difference between independent proportions: comparison of eleven methods, Statist Med. 1998; 17, 873-890]. The standardised asymptotic method used is the method six

Dewé W, Durand Ch, Marion S et al. A multi-criteria decision making approach to identify a vaccine formulation. Journal of Biopharmaceutical Statistics, 2015; epublication ahead of print: DOI: 10.1080/10543406.2015.1008517.

#### 11.2. Standard data derivation

- SAS date derived from a character date: In case day is missing, 15 is used. In case day and month are missing, 30 June is used.
- Onset day: The onset day for an event will be the number of days between the most recent vaccination and the start of the event. Events occurring on the day of vaccination will have an onset day of 0.
- Duration of events: The duration of an event will be the number of days between the start and stop dates + 1, e.g. an event which starts on 01DEC2014 and ends on 10DEC2014 will have duration of 10 days.

#### 11.2.1. **Demography**

For a given subject and a given demographic variable, missing measurements will not be replaced.

Study alias & e-track number(s): 204812 (RSV F-021)




- Age at vaccination Age will be calculated as the number of complete months between the date of birth and the date of vaccination.
- Height Height will be presented in centimeters. Heights reported in feet and inches will be converted as follows: Height in centimeters = Height in inches \* 2.54 (rounded to the unit no decimal places)
- Weight Weight will be presented in kilograms. Weights reported in pounds will be converted as follows: Weight in kilograms = Weight in pounds / 2.2 (rounded to 2 decimal places).

#### 11.2.2. Immunogenicity

- Any missing or non-evaluable immunogenicity measurement will not be replaced:
  - For the within-group assessment, the descriptive analysis performed for each assay at each timepoint will exclude subjects with a missing or non-evaluable measurement.
  - For the between group assessments, the Analysis of Covariance (ANCOVA)
    model will be fitted based on the subjects having a result at both the baseline and
    the considered timepoint.
- A seronegative subject will be defined as a subject whose antibody titre/concentration is below the cut-off value of the assay. A seropositive subject is a subject whose antibody titre/concentration is greater than or equal to the cut-off value of the assay
- The geometric mean titres (GMTs)/geometric mean concentrations (GMCs) will be computed by taking the anti-logarithm of the arithmetic mean of the log10 transformed titres/concentrations.
  - The 95% CI for the mean of log-transformed titer will be first obtained assuming that log-transformed values were normally distributed with unknown variance. The 95% CI for the GMTs/GMCs will be then obtained by exponential-transformation of the 95% CI for the mean of log-transformed titer.
- Vaccine response in terms of RSV neutralising antibodies will be defined as:
  - At least a 4-fold increase from pre-vaccination if pre-vaccination neutralising antibody titre <7 log2 (<128).</li>

Study alias & e-track number(s): 204812 (RSV F-021)




- At least a 3-fold increase from pre-vaccination if pre-vaccination neutralising antibody titre in [7-8] log2 ([128-256]).
- At least a 2.5-fold increase from pre-vaccination if pre-vaccination neutralising antibody titre in >8-10 log2 (>256-1024).
- At least 1-fold from pre-vaccination if pre-vaccination neutralising antibody titre
   10 log2 (>1024).
- In order to compute fold increase of antibody titres/concentrations (ratio) between post-vaccination and pre-vaccination titres/concentrations, antibody titres/concentrations below the assay cut-off will be given an arbitrary value of half the cut-off.
- For neutralising antibody against RSV-A, the following rules will be applied:

| Raw result | Derivation for<br>seropositivity status | Derivation for GMT calculation | Derivation for fold-increase<br>between Post and Pre-<br>vaccination titres |
|---|---|---|---|
| <8 | NEG | 4 | LLOQ/2 |
| [8-LLOQ[ | POS | 8 | LLOQ/2 |
| ≥LLOQ | POS | Exact value | Exact value |

### 11.2.3. Safety

• Temperature conversion: The conversion of temperature (Fahrenheit to Celsius) will be done as follows and rounded to 1 decimal place:

Temperature (Celsius) =  $((Temperature (Fahrenheit) - 32) \times 5)/9$ 

- Handling of missing data: subjects who missed reporting symptoms
   (solicited/unsolicited or concomitant medications/vaccinations) will be treated as
   subjects without symptoms (solicited/unsolicited or concomitant
   medications/vaccinations, respectively). In case of significant non-compliance of
   study procedures for reporting symptoms, the analysis plan will be reassessed to
   ensure more accurate reporting of study data by further analysis.
- For a given subject and the analysis of solicited symptoms during the 7-day follow-up period after vaccination, missing or non-evaluable measurements will not be replaced. Therefore the analysis of the solicited symptoms based on the ES will

FORM-9000026972-01 Statistical Analysis Plan Template

Effective date: 01 Jan 2016 GSK SOP Reference: SOP-9000026972 Form Owner: CEG-BSP, PPD

Study alias & e-track number(s): 204812 (RSV F-021)




include only vaccinated subjects with documented safety data (i.e., symptom screen completed).

- For analysis of unsolicited AEs, SAEs and for the analysis of concomitant medications, all vaccinated subjects will be considered. Subjects who did not report an event or concomitant medication will be considered as subjects without the event or the concomitant medication respectively.
- For the summary of fever, the occurrence of fever will be reported per 0.5°C cumulative increments starting from 38°C by any route. "All" will including all subjects with a documented temperature of ≥ 38°C/100.4°F by any route and all subjects reporting temperature < 38°C but with missing values (MC) for at least one day during the solicited period).

The preferred route for recording temperature in this study will be oral. For the analysis, temperatures will be coded as follows:

| Grade | Temperature for oral, axillary or tympanic route | Temperature for rectal route |
|---|---|---|
| 0 | < 37.5°C | < 38.0°C |
| 1 | ≥ 37.5°C - ≤ 38.5°C | ≥ 38.0°C - ≤ 39.0°C |
| 2 | > 38.5°C - ≤ 39.5°C | > 39.0°C - ≤ 40.0°C |
| 3 | > 39.5°C | > 40.0°C |

Form Owner: CEG-BSP, PPD

Study alias & e-track number(s): 204812 (RSV F-021)




For the analysis, the intensity scale for the following solicited AEs will be assessed as described:

| Adverse Event | Intensity grade | Parameter |
|---|---|---|
| Pain at injection site 0 | | None |
| | 1 | Mild: Any pain neither interfering with nor preventing normal every day activities. |
| | 2 | Moderate: Painful when limb is moved and interferes with every day activities. |
| | 3 | Severe: Significant pain at rest. Prevents normal every day activities. |
| Redness at injection site | | Record greatest surface diameter in mm |
| Swelling at injection site | | Record greatest surface diameter in mm |
| Fever* | | Record temperature in °C |
| Headache | 0 | Normal |
| | 1 | Mild: Headache that is easily tolerated |
| | 2 | Moderate: Headache that interferes with normal activity |
| | 3 | Severe: Headache that prevents normal activity |
| Fatigue 0 | | Normal |
| | 1 | Mild: Fatigue that is easily tolerated |
| | 2 | Moderate: Fatigue that interferes with normal activity |
| | 3 | Severe: Fatigue that prevents normal activity |
| Gastrointestinal symptoms | ointestinal symptoms 0 Normal | |
| (nausea, vomiting, | omiting, 1 Mild: Gastrointestinal symptoms that are easily tolerated | |
| diarrhoea and/or | and/or 2 Moderate: Gastrointestinal symptoms that interfere with normal activity | |
| abdominal pain) | 3 | Severe: Gastrointestinal symptoms that prevent normal activity |

<sup>\*</sup>Fever is defined as temperature  $\geq$  37.5°C for oral, axillary or tympanic route, or  $\geq$  38.0°C for rectal route. The preferred route for recording temperature in this study will be oral.

The maximum intensity of local injection site redness/swelling will be scored at GSK Biologicals according to the standard GSK Biologicals' scoring system for adults:

< 20 mm

1:  $> 20 \text{ mm to} \le 50 \text{ mm}$ 

2:  $> 50 \text{ mm to} \le 100 \text{ mm}$ 

3. > 100 mm

For clintrial gov and EudraCT posting purposes, a summary of subjects with all combined solicited (regardless of their duration) and unsolicited adverse events will be provided. Solicited adverse events will be coded by MedDRA as per the following codes.




| Solicited symptom | Lower level term name | Lower level term code | Corresponding Primary<br>Term code |
|---|---|---|---|
| Pain | Pain | 10033371 | 10033371 |
| Redness | Erythema | 10015150 | 10015150 |
| Swelling | Swelling | 10042674 | 10042674 |
| Fatigue | Fatigue | 10016256 | 10016256 |
| Fever | Fever | 10016558 | 10037660 |
| Gastroinstestinal symptoms | Gastroinstestinal disorder | 10017944 | 10017944 |
| Headache | Headache | 10019211 | 10019211 |

Note that for all tables described in this section, the way the percentage of subjects will be derived will depend on the event analysed (see table below for details). As a result, the N value will differ from one table to another.

| Event | N used for deriving % per subject for Vaccination phase |
|---|---|
| Concomitant vaccination | All subjects with study vaccine administered |
| Solicited general symptom | All subjects with at least one solicited general symptom documented as either present or absent (i.e., symptom screen completed) |
| Solicited local symptom | All subjects with at least one solicited local symptom documented as either present or absent (i.e., symptom screen completed) |
| Unsolicited symptom | All subjects with study vaccine administered |
| Concomitant medication | All subjects with study vaccine administered |




### 11.3. Number of decimals displayed:

The following decimal description from the decision rules will be used for the demography, immunogenicity and safety/reactogenicity.

| Display Table | Parameters | Number of decimal digits |
|---|---|---|
| All summaries | % of count, including LL & UL of CI | 1 |
| All summaries | % of difference, including LL & UL of CI | 2 |
| Demographic characteristics | Mean, median age, SD (age) | 1 |
| Immunogenicity | Ratio of GMT/GMC | 2 |

Form Owner: CEG-BSP, PPD

Study alias & e-track number(s): 204812 (RSV F-021) Version: DRAFT1

Date: 20-JULY-2016



#### **12**. ANNEX 2 CALCULATION OF INDIVIDUAL AND **OVERALL DESIRABILITY INDEX**

The section below provide the details on how to calculate individual desirability index and overall desirability index score based on Annex E in the Protocol.

#### Reactogenicity

A logistic regression model will be fitted on each reactogenicity endpoint (any Grade 2/3 general AE and any related SAE, Grade 2/3 fever) reported during the 7-day follow-up period after vaccination, including all RSV formulations.

- The vaccine group as the fixed effect
- The age groups (18-32 years and 33-45 years) as the categorical covariant.

The estimation of indication rate will be tabulated by treatment group.

For any Grade 2/3 general AEs and any related SAEs, the incidence rate estimate (1R) will be transformed in a [0,1] desirability index using the following function:

$$DR1 = \frac{\frac{1}{1 + \exp{-50 * 0.25 - IR}}, \quad if \ \mathcal{I}R \le 0.25}{\frac{1}{1 + \exp{-25 * 0.25 - IR}}, \quad if \ \mathcal{I}R \ge 0.25}$$

where *TR* is the incidence rate estimated by the model. This function will allocate a desirability value of 1, 0.5 and 0 to incidence rate equal to 0.1, 0.25 and 0.5 respectively (see ). But the calculation equally weights Grade 2/3 general AEs and any related SAEs.

Study alias & e-track number(s): 204812 (RSV F-021) Version: DRAFT1

Date: 20-JULY-2016



Figure 2 Desirability function for the incidence rate of Grade 2/3 general AEs and related SAEs - for each investigational RSV vaccine formulation



For Grade 2/3 fever, the incidence rate estimate (1R) will be transformed in a [0,1] desirability index using the following function:

$$DR2 = \frac{1}{1 + \exp(-120 * (0.05 - R))}$$

where *IR* is the incidence rate estimated by the model. As illustrated in , the function will allocate desirability values of 1, 0.5 and 0 to incidence rate equal to 0, 0.05 and 0.1 respectively.

Study alias & e-track number(s): 204812 (RSV F-021)

Version: DRAFT1 Date:20-JULY-2016



Figure 3 Desirability function for the incidence rate of Grade 2/3 fever - for each investigational RSV vaccine formulation



Finally, the reactogenicity index will be computed by taking the geometric mean of the 2 indexes:

$$DR = \overline{DR1 * DR2}$$

### Immunogenicity

The ANCOVA model will be fitted on the log-transformed titre for each immune response of neutralising anti-RSV-A and PCA separately including

- The vaccine group as the fixed effect
- The pre-vaccination titre/concentration and age groups (18-32 years and 33-45 years) as the covariates

The mean estimations of GMTs/GMCs for each treatment group at Day 30 and its 95% CI will be provided for immunogenicity desirability calculation. The estimated GMT and LL will be tabulated by treatment group.

As formulations inducing a high immune response will be considered suitable, the lower limit (LL) of the estimated GMT/C adjusted for pre-vaccination titres will be the statistical criterion considered for decision making.

Neutralising anti-RSV-A titres

FORM-9000026972-01 Statistical Analysis Plan Template

Effective date: 01 Jan 2016

Study alias & e-track number(s): 204812 (RSV F-021)

Version: DRAFT1 Date:20-JULY-2016



The LL of the GMT estimate will be transformed into a [0, 1] desirability index using the function:

$$DI1 = \frac{1}{1 + \exp(1.5 * (9.5 - LL))}$$

where LL is the lower limit of the 95% confidence interval of the GMT adjusted for prevaccination titres in log base 2. The function was chosen to have a desirability of 0 at LL value  $\leq 6 \log 2$  (=128), and a desirability of 1 at LL value  $\geq 13 \log 2$ . This function is illustrated in **** 

Figure 4 Desirability function for neutralising anti-RSV-A GMTs - for each investigational RSV vaccine formulation



#### PCA concentrations

The LL of the GMC adjusted for pre-vaccination titres estimate will be transformed using the following function:

$$DI2 = \frac{\frac{1}{1 + \exp 0.05 * 150 - LL}}, \quad if LL \le 150}{\frac{1}{1 + \exp 0.025 * 150 - LL}}, \quad if LL \ge 150}$$

Study alias & e-track number(s): 204812 (RSV F-021)

Version: DRAFT1 Date:20-JULY-2016



As illustrated in ****, a PCA response of 25, 150 and 400  $\mu$ g/mL will have a desirability value of 0, 0.5 and 1 respectively.

Figure 5 Desirability function for PCA concentrations - for each investigational RSV vaccine formulation



Finally, the immunogenicity index will be computed by taking the geometric mean of the 2 indexes:

$$DI = \overline{DI1 * DI2}$$

#### Overall desirability index

The overall desirability index will be obtained by computing the following weighted geometric mean:  $D = DR^{0.4} * DI^{0.6}$ .
### **Statistical Analysis Plan**

Study alias & e-track number(s): 204812 (RSV F-021)

Version: DRAFT1 Date: 20-JULY-2016



### **13**. ANNEX 3: STUDY SPECIFIC MOCK TFL

### Template 46 Descriptive statistics of the viral load assessed by the quantitative PCR (RSV-A/B) of RSV-RTI cases (Total vaccinated cohort)

| | | <each group=""><br/>N =</each> | Total<br>N = |
|-------|------------|--------------------------------|--------------|
| Visit | Parameters | Value | Value |
| | Mean | | |
| | SD | | |
| | Median | | |
| | Minimum | | |
| | Maximum | | |
| | Unknown | | |

<each group>:

30 PreF = 30 mcg PreF Plain

60 PreF = 60 mcg PreF Plain

120 PreF = 120 mcg PreF Plain

Control = Placebo

### Template 47 Desirability index of immunogenicity during the 30-day (Days 0-29) post-vaccination period (ATP cohort for immunogenicity)

| Group | GMT | LL | DI1 | DI2 | DI |
|------------------------|-----|----|-----|-----|----|
| <each group=""></each> | | | | | |

<each group>:

30 PreF = 30 mcg PreF Plain

60 PreF = 60 mcg PreF Plain

120 PreF = 120 mcg PreF Plain

GMT = estimated GMT adjusted for pre-vaccination titres LL

= estimated lower limit adjusted for pre-vaccination titres

DI1 = desirability index for neutralising anti-RSV-A

DI2 = desirability index for PCA concentrations

DI = immunogenicity index

### Template 48 Desirability index of reactogenicity during the 7-day (Days 0-6) postvaccination period (Total vaccination cohort)

| Group | Incidence Rate (IR) | DR1 | DR2 | DR |
|-------|---------------------|-----|-----|----|

FORM-9000026972-01 Statistical Analysis Plan Template

Effective date: 01 Jan 2016

GSK SOP Reference: SOP-9000026972 Form Owner: CEG-BSP, PPD

### Statistical Analysis Plan

Study alias & e-track number(s): 204812 (RSV F-021)

Version: DRAFT1 Date:20-JULY-2016



| <each group=""></each> |
|------------------------|

<each group>:

30 PreF = 30 mcg PreF Plain

60 PreF = 60 mcg PreF Plain

120 PreF = 120 mcg PreF Plain

1R = incidence rate estimated by the model

DR1 = desirability index for any Grade 2/3 general AEs and any related SAEs

DR2 = desirability index for Grade 2/3 fever

DR = reactogenicity index

## Template 49 Desirability index based on reactogenicity and safety (TVC cohort up to Day 7) and immunogenicity (ATP cohort for immunogenicity up to Day 30)

| Group | Reactogenicity Index | Immuno | genicity | Overall Desirability<br>Index<br>DR <sup>0.4</sup> * DI <sup>0.6</sup> |
|---|---|---|---|---|
| | DR1 | DI1 | | |
| <each<br>group&gt;</each<br> | DR2 | DI2 | | |
| | DR | DI | | |

<each group>:

30 PreF = 30 mcg PreF Plain

60 PreF = 60 mcg PreF Plain

120 PreF = 120 mcg PreF Plain

DR1 = desirability index for any Grade 2/3 general AEs and any related SAEs

DR2 = desirability index for Grade 2/3 fever

DR = reactogenicity index

DI1 = desirability index for neutralising anti-RSV-A

DI2 = desirability index for PCA concentrations

DI = immunogenicity index

FORM-9000026972-01 Statistical Analysis Plan Template Effective date: 01 Jan 2016 GSK SOP Reference: SOP-9000026972 Form Owner: CEG-BSP, PPD

204812 (RSV F-021) SAP (associated to IDMC Charter) Amendment 1 Final

| | SAP (associated to IDMC Charter) Amendment 1 Final |
|---|---|
| <b>gsk</b> GlaxoSmithKline | Statistical Analysis Plan |
| Detailed Title: | A Phase II, randomised, observer-blind, controlled, multi-country study to rank different formulations of GSK Biologicals' investigational RSV vaccine (GSK3003891A), based on immunogenicity, reactogenicity and safety, when administered to healthy women, aged 18 – 45 years. |
| eTrack study number and<br>Abbreviated | 204812 (RSV F-021) |
| Scope: | All data pertaining to the above study for review by the IDMC on all subjects with at least Day30 safety and reactogenicity data |
| Date of Statistical Analysis<br>Plan | Amendment 1: 02-May-2017 Version 1: 21-Apr-2017 |
| Co-ordinating author: | (Statistician) |
| Reviewed by: | (Clinical and Epidemiology Project Lead) PPD (Lead statistician) |
| | (Lead statistical analyst) |
| | (SERM physician) |
| | (Independent Statistician) |
| Approved by: | PPD (Clinical & Epidemiological Projects Lead) |
| | (Lead statistician) |
| | (Lead stat analyst) PPD (Lead scientific writer) |
| | (Lead Scientific Writer) |

APP 9000058193 Statistical Analysis Plan Template (Effective date: 14 April 2017)

 02-MAY-2017

204812 (RSV F-021) SAP (associated to IDMC Charter) Amendment 1 Final

### **TABLE OF CONTENTS**

| | | PAGE |
|---|---|---|
| LIS | ST OF ABBREVIATIONS | 7 |
| 1. | DOCUMENT HISTORY | 8 |
| 2. | INTRODUCTION | 8 |
| 3. | STUDY DESIGN | 9 |
| 4. | OBJECTIVES | 10 |
| 5. | ENDPOINTS | 11 |
| 6. | STUDY POPULATION | |
| 7. | STATISTICAL METHODS 7.1. Data to be reviewed 7.2. Group description | 11 |
| 8. | STATISTICAL CALCULATIONS 8.1. Derived and transformed data 8.2. Methodology for computing CI | 13 |
| 9. | CONDUCT OF ANALYSES | 15 |
| 10. | REFERENCES | 15 |
| 11. | LIST OF TABLES AND LISTINGS | 16 |
| 12. | TEMPLATE OF TABLES | 22 |

204812 (RSV F-021) SAP (associated to IDMC Charter) Amendment 1 Final

### **LIST OF TABLES**

| | | PAGE |
|---|---|---|
| Table 1 | Study groups and epochs foreseen in the study | 9 |
| Table 2 | Group order and group label for the blinded and unblinded tables | 12 |
| Table 3 | Grading scales for temperatures, redness and swellings parameters applicable for this study | 13 |
| Table 4 | Toxicity grading scales for hematology and biochemistry parameters applicable for this study | 14 |

02-MAY-2017 

204812 (RSV F-021) SAP (associated to IDMC Charter) Amendment 1 Final

### **LIST OF FIGURES**

| F | PAGE |
|---------------------------|------|
| e 1 Study design overview | 9 |

02-MAY-2017 

204812 (RSV F-021) SAP (associated to IDMC Charter) Amendment 1 Final

### **LIST OF TEMPLATES**

| | P | AGE |
|---|---|---|
| Template 1 | Summary of demographic characteristics (Total vaccinated cohort) | 22 |
| Template 2 | Number of subjects vaccinated, completed and withdrawn with reason for withdrawal (Day 30) (Total vaccinated cohort) | 23 |
| Template 3 | Compliance in returning symptom information (Total vaccinated cohort) | <b>2</b> 3 |
| Template 4 | Incidence of solicited local symptoms reported during the 7-day (Days 0-6) post-vaccination period (Total vaccinated cohort) | 24 |
| Template 5 | Incidence of solicited local symptoms reported during the 7-day (Days 0-6) post-vaccination period by duration (Total vaccinated cohort) | 25 |
| Template 6 | Incidence of solicited general symptoms reported during the 7-day (Days 0-6) post-vaccination period (Total vaccinated cohort) | 26 |
| Template 7 | Incidence of solicited general symptoms reported during the 7-day (Days 0-6) post-vaccination period by duration (Total vaccinated cohort) | 28 |
| Template 8 | Incidence and nature of symptoms (solicited and unsolicited reported during the 7-day (Days 0-6) post-vaccination period (Total vaccinated cohort) | 30 |
| Template 9 | Percentage of subjects reporting the occurrence of unsolicited classified by MedDRA Primary System Organ Class and Preferred Term within the 30-day (Days 0-29) post-vaccination period (Total vaccinated cohort) | 30 |
| Template 10 | Number and percentage of subjects taking a concomitant medication during the 7- day (Days 0-6) post -vaccination period (Total vaccinated cohort) | 31 |
| Template 11 | Listing of SAEs reported up to data lock point (Total vaccinated cohort) | 32 |
| Template 12 | Listing of adverse events, SAEs and solicited symptoms leading to withdrawal from the treatment/study (Total Vaccinated Cohort) | 33 |
| Template 13 | Distribution of change from baseline in haematology and biochemistry with respect to normal laboratory ranges (Total vaccinated cohort). | 33 |

| | 204812 (RS\ | / F-021) |
|---|---|---|
| | SAP (associated to IDMC Charter) Amendmen | t 1 Final |
| Template 14 | Summary of haematology and biochemistry results by maximum grade from VISIT 2 (D7) up to VISIT 5 (D90) versus baseline | |
| | (Total vaccinated cohort) | 34 |
| Template 15 | Summary of haematology change from baseline by maximum grade from VISIT2 (D7) up to VISIT5 (D90) (Total vaccinated | |
| | cohort) | 34 |
| Template 16 | Individuals results of hemoglobin levels outside of the normal ranges in < group> (Total vaccinated cohort) | 35 |

02-MAY-2017 

204812 (RSV F-021)

SAP (associated to IDMC Charter) Amendment 1 Final

### LIST OF ABBREVIATIONS

**AE:** Adverse Event

ALT: Alanine Aminotransferase AST: Aspartate Aminotransferase

**CEPL:** Clinical and Epidemiology Project Lead

**CI:** Confidence Interval

**CRDL:** Clinical Research and Development Lead

**eCRF:** electronic Case Report Form

GP: General Practitioner GSK: GlaxoSmithKline

iSRC: Internal Safety Review Committee
IDMC: Independent Data Monitor Committe
LL: Lower Limit of the confidence interval

MA-RTI: Medically Attended Respiratory Tract Infection MedDRA: Medical Dictionary for Regulatory Activities

**PCR:** Polymerase Chain Reaction

**PreF:** Purified recombinant RSV F protein, engineered to preferentially

maintain the pre-fusion conformation

RSV: Respiratory syncytial virus SAE: Serious Adverse Event SAP: Statistical Analysis Plan

**SBIR:** Randomisation System on Internet

**SRT:** Safety Review Team

**TFL:** Tables Figures and Listing template annexed to SAP

**TVC:** Total Vaccinated Cohort

**UL:** Upper Limit of the confidence interval

**WBC:** White Blood Cells

### 1. DOCUMENT HISTORY

| Date | Version | Description | Protocol Version |
|---|---|---|---|
| 21APR2017 | First Version | Enhanced respiratory disease risk review by IDMC | RSV F-021<br>(204812) Protocol<br>(20-Jul-2016) |
| 02MAY2017 | Amendment 1 | Amendment 1: Description of changes from First Version are as below, - Individual results of levels outside of the normal ranges in each group are generated for all six lab parameters, including hemoglobin, platelets counts, white blood cells counts, ALT, AST, and creatinine to replace individual results of levels in the normal range - Add two tables for AE using maximum grading per subject for each grade - Add two tables for AE on all grades for duration | RSV F-021 (204812) Protocol (20-Jul-2016) |

### 2. INTRODUCTION

This SAP and TFL document presents the analyses of the data of all enrolled subjects up to at least 30 days post administration of the study vaccine or placebo.

- the <u>unblinded</u> analyses and data displays presenting each study group for the Independent Data Monitoring Committee (IDMC).
- the <u>blinded</u> analyses and data displays presenting all groups pooled for the review of safety data by the GSK Safety Review Team (SRT) involved in the project.

Statistical analyses and data displays for the iSRC review, other study analyses and the end of study reporting are not covered in this SAP and will be described in a separate document.

The list of tables, figures and listings to be produced are shown in section 11.

### 3. STUDY DESIGN

Figure 1 Study design overview



- V = Visit; D = Day; VACC = vaccination; BS = blood sample; h/b = blood sample for haematology/biochemistry; lmm = blood sample for immunogenicity; C = contact; RSV = Respiratory Syncytial Virus; PCR = Polymerase Chain Reaction.
- 1 Safety data up to (minimum) 7 days post-vaccination (including Day 7 haematology and biochemistry parameters) of the first 25% of subjects vaccinated in the study will be reviewed by iSRC.
- 2 In case of a MA-RTI (e.g. visit to the GP for respiratory symptoms including but not limited to cough, sputum production, difficulty breathing), the subject will be asked to contact the Investigator to enable completion of an event related eCRF and the collection of a nasal swab within 72h after the medical attendance.
  Vertical lines stand for analysis on all subjects.
- **Experimental design**: Phase II, observer-blind, randomised, controlled, multicountry, study with four parallel groups.
- **Duration of the study**: the intended duration of the study will be approximately 1 year from Visit 1 to study conclusion (Day 360).
  - Epoch 001: Primary starting at Visit 1 (Day 0) and ending at Visit 5 (Day 90).
- Epoch 002: Follow-up phase starting one day after Day 90 and ending at Day 360 contact.

### • Study groups:

Table 1 Study groups and epochs foreseen in the study

| Ctudy groups | Number of aubicate | Ago (Min/Max) Epoch | | ochs |
|---|---|---|---|---|
| Study groups | Number of subjects | Age (Min/Max) | Epoch 001 | Epoch 002 |
| 30 PreF | ~100 | 18 - 45 years | Х | Х |
| 60 PreF | ~100 | 18 - 45 years | Х | Х |
| 120 PreF | ~100 | 18 - 45 years | Х | Х |
| Control | ~100 | 18 - 45 years | Х | Х |

02-MAY-2017 

204812 (RSV F-021)

SAP (associated to IDMC Charter) Amendment 1 Final

- **Treatment allocation**: Subjects will be randomised using a centralised randomisation system on internet (SBIR) at Day 0. The randomisation algorithm will use a minimisation procedure accounting for age (18 32 years or 33 45 years) and centre.
- **Blinding**: Observer-blind in Epoch 001 and single-blind in Epoch 002.

### • Sampling schedule:

- Blood samples for haematology/biochemistry will be collected (~10 mL) from all subjects at Visit 1 (Day 0), Visit 2 (Day 7), Visit 3 (Day 30), Visit 4 (Day 60) and Visit 5 (Day 90).
- Blood samples for humoral immune response evaluation will be collected (~17 mL) from all subjects at Visit 1 (Day 0), Visit 3 (Day 30), Visit 4 (Day 60) and Visit 5 (Day 90).
- Nasal swabs will be collected from subjects in case of a MA-RTIfrom enrolment (Visit 1) until study end (Contact 3).
- Type of study: self-contained
- **Data collection**: Electronic Case Report Form (eCRF).

### • Safety monitoring:

- When the first 25% of subjects are vaccinated in the study, enrolment will be paused until completion of an unblinded review by a GSK iSRC. Continuation of study enrolment will be conditional to a favourable outcome of the iSRC evaluation of all available safety and reactogenicity data collected up to at least 7 days post-vaccination (including Day 7 haematology and biochemistry parameters). In addition, the blinded safety data will be reviewed by GSK Biologicals' SRT on a regular basis throughout the study.
- IDMC will review all available safety and reactogenicity data (including haematology/biochemistry parameters) of all enrolled subjects up to at least 30 days post administration of the study vaccine or placebo. The blinded safety data will also be reviewed by the GSK Biologicals' SRT.
- In case of a MA-RTI (e.g. visit to the GP for respiratory symptoms including but not limited to cough, sputum production, difficulty breathing), the subject will be asked to contact the investigator to enable the collection of a nasal swab within 72 hours after the medical attendance

### 4. OBJECTIVES

This document does not describe the analyses relative to study objectives. This analysis is performed to support the IDMC and SRT reviews of at least Day 30 safety data for all subjects enrolled.

### 5. ENDPOINTS

- Occurrence of AEs from vaccination up to **Day 7**, for all subjects in all groups:
  - Occurrence of any Grade 2 and Grade 3 general AE (solicited and unsolicited);
  - Occurrence of Grade 2 and Grade 3 fever:
  - Occurrence of each solicited local and general AE.
- Occurrence of AEs from vaccination up to **data lock point**, for all subjects in all groups:
  - Occurrence of any unsolicited AE;
  - Occurrence of any haematological (haemoglobin level, White Blood Cells [WBC], lymphocyte, neutrophil, eosinophil and platelet count) and biochemical (alanine amino-transferase [ALT], aspartate amino-transferase [AST] and creatinine) laboratory abnormality at Day 0, Day 7 and Day 30 for all subjects in all groups and at Day 60 and Day 90 for all available subjects in all groups.
- Occurrence of medically attended respiration tract infections (MA-RTIs) up to the data lock point
- Occurrence of any vaccine-related SAE up to the data lock point

### 6. STUDY POPULATION

### 6.1. Study cohorts to be evaluated

The statistical analyses that are described in the document are based on the Total Vaccinated Cohort; i.e. on subjects with at least one vaccine administration.

### 7. STATISTICAL METHODS

### 7.1. Data to be reviewed

The IDMC will review, in an unblinded manner, all available safety and reactogenicity data (including haematology/biochemistry parameters) of all enrolled subjects up to at least 30 days post administration of the study vaccine or placebo and all SAEs reported up to the data lock point.

The following data will be reviewed during the IDMC meeting:

- Demographic characteristics.
- Summary tables containing information on events of interest (any Serious Adverse Events [SAE], any death or life-threatening SAE, any missed visits due to vaccine-related Adverse Event [AE], any AEs causing study withdrawal).

204812 (RSV F-021)

SAP (associated to IDMC Charter) Amendment 1 Final

- Incidence of solicited local AEs (pain, redness, swelling): any, each grade (7-day follow-up period after vaccination).
- Incidence of solicited general AE (fever, headache, fatigue, gastrointestinal symptoms): any, each grade, any related, any Grade 2 related, any Grade 3 related (7-day follow-up period after vaccination).
- Incidence of unsolicited AE: any, Grade 3, any related, Grade 3 related (7-day and 30-day follow-up period after each vaccination).
- Any abnormality in haematological (haemoglobin level, leukocyte, neutrophil, lymphocyte, eosinophil and platelet count) and biochemical (ALT, AST and creatinine) parameters: number and percentage of subjects with parameters outside of the normal ranges, the maximum grading post-vaccination (from Day 7 to data lock point) versus baseline (Day 0) and the percentage of subjects with laboratory parameters above or equal to Grade 1, Grade 2, Grade 3 and Grade 4 (Grades will be based on the Food & Drug Administration [FDA] Guidance for Industry "Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials").
- Additional parameters of interest may be tabulated.

### 7.2. Group description

For the <u>blinded report</u>, the analyses will be presented as one group (RSV groups and Placebo group being pooled) as described in Table 2.

For the <u>unblinded report</u>, the analyses will be presented by group as described in Table 2.

Table 2 Group order and group label for the blinded and unblinded tables

| | Blinded report | | | | Unblinded | report |
|---|---|---|---|---|---|---|
| Study<br>groups | Pooled group order | Pooled group<br>label | Pooled group<br>definition for<br>footnote | Group<br>order | Group<br>label | Group<br>definition for<br>footnote |
| 30 PreF | | 0, 1 | D01/ . D1 . I | 1 | 30 PreF | 30 mcg PreF |
| 60 PreF | 1 | Step 1 | RSV + Placebo | 2 | 60 PreF | 60 mcg PreF |
| 120 PreF | | | | 3 | 120 PreF | 120 mcg PreF |

### 8. STATISTICAL CALCULATIONS

### 8.1. Derived and transformed data

For a given subject and the analysis of solicited symptoms within 7 days post-vaccination, missing or non-evaluable measurements will not be replaced. Therefore the analysis of the solicited symptoms based on the Total Vaccinated Cohort will include only vaccinated subjects for doses with documented safety data (i.e., symptom screen completed). More specifically the following rules will be used:

- Subjects who documented the absence of a solicited symptom after one dose will be considered not having that symptom after that dose.
- Subjects who documented the presence of a solicited symptom and fully or partially recorded daily measurement over the solicited period will be included in the summaries at that dose and classified according to their maximum observed daily recording over the solicited period.
- Subjects who documented the presence of a solicited symptom after one dose without having recorded any daily measurement will be assigned to the lowest intensity category at that dose (i.e., 37.5°C for fever or grade 1 for othersymptoms).
- Doses without symptom sheets documented will be excluded.
- For analyses of unsolicited adverse events, such as serious adverse events or adverse
  events by primary MedDRA term, and for the analysis of concomitant medications,
  all vaccinated subjects will be considered. Subjects who did not report the event or
  the concomitant medication will be considered as subjects without the event or the
  concomitant medication respectively.
- For the analysis, temperatures, redness and swellings will be coded as follows:

Table 3 Grading scales for temperatures, redness and swellings parameters applicable for this study

| | Tempera | | |
|---|---|---|---|
| Grade | Oral, axillary or tympanic route | Rectal route | Redness and swelling |
| 0 | < 37.5°C | < 38.0°C | ≤ 20 mm |
| 1 | ≥ 37.5°C to ≤ 38.5°C | ≥ 38.0°C to ≤ 39.0°C | > 20 mm to ≤ 50 mm |
| 2 | > 38.5°C to ≤ 39.5°C | > 39.0°C to ≤ 40.0°C | > 50 mm to ≤ 100 mm |
| 3 | > 39.5°C | > 40.0°C | > 100 mm |

• Haematology/biochemistry parameters will be graded according to FDA toxicity grading scales

SAP (associated to IDMC Charter) Amendment 1 Final

Table 4 Toxicity grading scales for hematology and biochemistry parameters applicable for this study

| Serum | Mild<br>(Grade 1) | Moderate<br>(Grade 2) | Severe<br>(Grade 3) | Potentially Life<br>Threatening<br>(Grade 4) |
|---|---|---|---|---|
| Creatinine – mg/dL | 1.5 – 1.7 | 1.8 – 2.0 | 2.1 – 2.5 | > 2.5 or requires dialysis |
| Liver Function Tests -ALT, AST increase by factor | 1.1 – 2.5 x ULN | 2.6 – 5.0 x ULN | 5.1 – 10 x ULN | > 10 x ULN |
| Hematology* | Mild<br>(Grade 1) | Moderate<br>(Grade 2) | Severe<br>(Grade 3) | Potentially Life<br>Threatening<br>(Grade 4) |
| Hemoglobin (Female) - gm/dL | 11.0 – 12.0 | 9.5 – 10.9 | 8.0 – 9.4 | < 8.0 |
| Hemoglobin (Female)<br>change from baseline value -<br>gm/dL | Any decrease -<br>1.5 | 1.6 – 2.0 | 2.1 – 5.0 | > 5.0 |
| WBC Increase - cell/mm3 | 10 800 – 15 000 | 15 001 – 20 000 | 20 001 – 25 000 | > 25 000 |
| WBC Decrease - cell/mm3 | 2 500 – 3 500 | 1 500 – 2 499 | 1 000 – 1 499 | < 1 000 |
| Lymphocytes Decrease - cell/mm3 | 750 – 1 000 | 500 – 749 | 250 – 499 | < 250 |
| Neutrophils Decrease - cell/mm3 | 1 500 – 2 000 | 1 000 – 1 499 | 500 – 999 | < 500 |
| Eosinophils - cell/mm3 | 650 – 1 500 | 1 501 - 5 000 | > 5 000 | Hypereosinophilic |
| Platelets Decreased - cell/mm3 | 125 000 –<br>140 000 | 100 000 –<br>124 000 | 25 000 – 99 000 | < 25 000 |

**ULN** = upper limit of the normal range.

• Note that for all tables described in this section, the way the percentage of subjects will be derived will depend on the event analysed (see table below for details). As a result, the N value will differ from one table to another.

| Event | N used for deriving % per subject for Vaccination phase |
|---|---|
| Solicited general | All subjects with at least one solicited general symptom documented as either present or |
| symptom | absent (i.e., symptom screen completed) |
| Solicited local | All subjects with at least one solicited local symptom documented as either present or |
| symptom | absent (i.e., symptom screen completed) |
| Unsolicited symptom | All subjects with study vaccine administered |

### 8.2. Methodology for computing CI

All CI computed will be two-sided 95% CI.

The exact 95% CIs for a proportion within a group will be calculated from Proc StatXact [Clopper CJ, Pearson ES. The use of confidence or fiducial limits illustrated in the case of binomial. *Biometrika*. 1934; 26:404-413].

SAP (associated to IDMC Charter) Amendment 1 Final

### 9. CONDUCT OF ANALYSES

This unblinded analysis will be done by an independent statistician outside GSK to maintain the study team blinded.

| Description | Analysis ID | Disclosure Purpose |
|------------------------|-------------|--------------------|
| IDMC Analysis of Day30 | E1_03 | IDMC |

One unblinded analysis is planned to be reviewed by the IDMC and one blinded analysis is planned to be reviewed by the GSK SRT for the project on all available safety and reactogenicity data (including all available haematology/biochemistry parameters at data lock point) of all enrolled subjects up to at least 30 days post administration of the study vaccine or placebo.

### 10. REFERENCES

Clopper CJ, Pearson ES. The use of confidence or fiducial limits illustrated in the case of binomial. *Biometrika*. 1934; 26:404-413

### 11. LIST OF TABLES AND LISTINGS

### 11.1. List of tables

The tables and figures presented in this section will be created for the unblinded report.

For the blinded report, similar tables/figures will be presented with RSV and Placebo groups being pooled and presented as one group as described in Table 2.

| Template # | Table Title | Output destination | Macro |
|---|---|---|---|
| Template 1 | Summary of demographic characteristics (Total Vaccinated Cohort) | Annex | %DEMOGRA |
| Template 2 | Number of subjects vaccinated, completed and withdrawn with reason for withdrawal ( <b>Day 30</b> ) (Total Vaccinated Cohort) | Annex | %DROP_SUM<br>(OTH=0) |
| Template 2 | Number of subjects vaccinated, completed and withdrawn with reason for withdrawal ( <b>Day 60</b> ) (Total Vaccinated Cohort) | Annex | %DROP_SUM<br>(OTH=0) |
| Template 2 | Number of subjects vaccinated, completed and withdrawn with reason for withdrawal ( <b>Day 90</b> ) (Total Vaccinated Cohort) | Annex | %DROP_SUM<br>(OTH=0) |
| Template 3 | Compliance in returning symptom information (Total Vaccinated Cohort) | Annex | %COMPLI |
| Template 4 | Incidence of solicited <b>local</b> symptoms reported during the 7-day (day 0-6) post-vaccination period (Total Vaccinated Cohort) | Annex | %FREQ |
| Template 5 | Incidence of solicited <b>local</b> symptoms reported during the 7-day (day 0-6) post-vaccination period <b>by duration</b> (Total Vaccinated Cohort) | Annex | %FREQ |
| Template 6 | Incidence of solicited <b>general</b> symptoms reported during the 7-day (day 0-6) post-vaccination period (Total Vaccinated Cohort) | Annex | %FREQ |
| Template 7 | Incidence of solicited <b>general</b> symptoms reported during the 7-day (day 0-6) post-vaccination period <b>by duration</b> (Total Vaccinated Cohort) | Annex | %FREQ |
| Template 8 | Incidence and nature of symptoms (solicited and unsolicited) reported during the 7-day (Days 0-6) post-vaccination period (Total vaccinated cohort) | Annex | %LOCGEN |
| Template 8 | Incidence and nature of symptoms (solicited and unsolicited) considered related to vaccination reported during the 7-day (Days 0-6) post-vaccination period (Total vaccinated cohort) | Annex | %LOCGEN |
| Template 8 | Incidence and nature of symptoms (solicited and unsolicited) with medically attended visit, reported during the 7-day (Days 0-6) post-vaccination period (Total vaccinated cohort) | Annex | %LOCGEN |

| Template # | Table Title | Output | Macro |
|---|---|---|---|
| Template 8 | Incidence and nature of <b>grade 3</b> symptoms | destination<br>Annex | %LOCGEN |
| Template 8 | (solicited and unsolicited) reported during the 7- | Aillex | /0LOCGLIN |
| | day (Days 0-6) post-vaccination period (Total | | |
| | vaccinated cohort) | | |
| Template 8 | Incidence and nature of grade 3 symptoms | Annex | %LOCGEN |
| | (solicited and unsolicited) considered related to | | |
| | vaccination reported during the 7-day (Days 0-6) post-vaccination period (Total vaccinated | | |
| | cohort) | | |
| Template 8 | Incidence and nature of grade 2/3 symptoms | Annex | %LOCGEN |
| | (solicited and unsolicited) reported during the 7- | | |
| | day (Days 0-6) post-vaccination period (Total | | |
| Template 8 | vaccinated cohort) Incidence and nature of symptoms (solicited and | Annex | %LOCGEN |
| Template o | unsolicited) reported during the 30-day (Days 0- | 7 | 702002.1 |
| | 29) post-vaccination period (Total vaccinated | | |
| | cohort) | | |
| Template 8 | Incidence and nature of symptoms (solicited and | Annex | %LOCGEN |
| | unsolicited) <b>considered related to vaccination</b> reported during the 30-day (Days 0-29) post- | | |
| | vaccination period (Total vaccinated cohort) | | |
| Template 8 | Incidence and nature of symptoms (solicited and | Annex | %LOCGEN |
| - | unsolicited) with medically attended visit, | | |
| | reported during the 30-day (Days 0-29) post- | | |
| Townslate 0 | vaccination period (Total vaccinated cohort) | Annov | %LOCGEN |
| Template 8 | Incidence and nature of <b>grade 3</b> symptoms (solicited and unsolicited) reported during the 30- | Annex | %LOCGEN |
| | day (Days 0-29) post-vaccination period (Total | | |
| | vaccinated cohort) | | |
| Template 8 | Incidence and nature of grade 3 symptoms | Annex | %LOCGEN |
| | (solicited and unsolicited) considered related to | | |
| | vaccination reported during the 30-day (Days 0- | | |
| | 29) post-vaccination period (Total vaccinated cohort) | | |
| Template 8 | Incidence and nature of <b>grade 2/3</b> symptoms | Annex | %LOCGEN |
| 2P 2000 | (solicited and unsolicited) reported during the 30- | | |
| | day (Days 0-29) post-vaccination period (Total | | |
| m to a | vaccinated cohort) | A | 0/110001 |
| Template 9 | Percentage of subjects reporting the occurrence | Annex | %UNSOL |
| | of unsolicited symptoms classified by MedDRA Primary System Organ Class and Preferred | | |
| | Term, during the <b>7-day</b> (day 0-6) post- | | |
| | vaccination period (Total Vaccinated Cohort) | | |

| Tomplete # | SAP (associated to IDMC Charter) Amendment 1 | | |
|---|---|---|---|
| Template # | Table Title | Output destination | Macro |
| Template 9 | Percentage of subjects reporting the occurrence of <b>grade 3</b> unsolicited symptoms classified by MedDRA Primary System Organ Class and Preferred Term, during the <b>7-day</b> (day 0-6) post-vaccination period (Total Vaccinated Cohort) | Annex | %UNSOL |
| Template 9 | Percentage of subjects reporting the occurrence of unsolicited symptoms classified by MedDRA Primary System Organ Class and Preferred Term, considered related to vaccination, during the 7-day (day 0-6) post-vaccination period (Total Vaccinated Cohort) | Annex | %UNSOL |
| Template 9 | Percentage of subjects reporting the occurrence of <b>grade 3</b> unsolicited symptoms classified by MedDRA Primary System Organ Class and Preferred Term, <b>considered related to vaccination</b> , during the <b>7-day</b> (day 0-6) post-vaccination period (Total Vaccinated Cohort) | Annex | %UNSOL |
| Template 9 | Percentage of subjects reporting the occurrence of unsolicited symptoms classified by MedDRA Primary System Organ Class and Preferred Term, during the <b>30-day</b> (day 0-29) post-vaccination period (Total Vaccinated Cohort) | Annex | %UNSOL |
| Template 9 | Percentage of subjects reporting the occurrence of <b>grade 3</b> unsolicited symptoms classified by MedDRA Primary System Organ Class and Preferred Term, during the <b>30-day</b> (day 0-29) post-vaccination period (Total Vaccinated Cohort) | Annex | %UNSOL |
| Template 9 | Percentage of subjects reporting the occurrence of unsolicited symptoms classified by MedDRA Primary System Organ Class and Preferred Term, considered related to vaccination, during the 30-day (day 0-29) post-vaccination period (Total Vaccinated Cohort) | Annex | %UNSOL |
| Template 9 | Percentage of subjects reporting the occurrence of <b>grade 3</b> unsolicited symptoms classified by MedDRA Primary System Organ Class and Preferred Term, <b>considered related to vaccination</b> , during the <b>30-day</b> (day 0-29) post-vaccination period (Total Vaccinated Cohort) | Annex | %UNSOL |
| Template 9 | Percentage of subjects reporting the occurrence of medically attended respiration tract infections (MA-RTIs), during the 30-day (day 0-29) post-vaccination period (Total Vaccinated Cohort) | Annex | %UNSOL |
| Template 9 | Percentage of subjects reporting the occurrence of medically attended respiration tract infections (MA-RTIs), during the 60-day (day 0-59) post-vaccination period (Total Vaccinated Cohort) | Annex | %UNSOL |

| Template # | Table Title | Output destination | Macro |
|---|---|---|---|
| Template 9 | Percentage of subjects reporting the occurrence of medically attended respiration tract infections (MA-RTIs), during the 90-day (day 0-89) post-vaccination period (Total Vaccinated Cohort) | Annex | %UNSOL |
| Template 10 | Number and percentage of subjects taking a concomitant medication during the 7- day (Days 0-6) post -vaccination period (Total vaccinated cohort) | Annex | %CMED_INC |
| Template 10 | Number and percentage of subjects taking a concomitant medication during the 30- day (Days 0-29) post -vaccination period (Total vaccinated cohort) | Annex | %CMED_INC |
| Template 11 | Listing of <b>SAEs</b> reported up to data lock point (Total vaccinated cohort) | Annex | %SAE |
| Template 12 | Listing of adverse events, SAEs and solicited symptoms leading to withdrawal from the treatment/study (Total Vaccinated Cohort) | Annex | %DISC_AE |
| Template 13 | Distribution of change from baseline in haematology and biochemistry with respect to normal laboratory ranges (Total vaccinated cohort) | Annex | %HAEMATO_B<br>IOCH |
| Template 14 | Summary of haematology and biochemistry results by maximum grade from VISIT 2 (D7) up to VISIT 5 (D90) versus baseline (Total vaccinated cohort) | Annex | %HAEMATO_<br>BIOCH_GR_<br>CHANGE |
| Template 15 | Summary of haematology change from baseline by maximum grade from VISIT2 (D7) up to VISIT5 (D90) (Total vaccinated cohort) | Annex | %HAEMATO_<br>BIOCH_GR_<br>CHANGE |
| Template 16 | Individuals results of <b>hemoglobin levels</b> outside of the normal ranges in <b>30</b> PreF group (Total vaccinated cohort) | Annex | %HB_PROFIL |
| Template 16 | , | Annex | %HB_PROFIL |
| Template 16 | Individuals results of hemoglobin levels outside of the normal ranges in 120 PreF group (Total vaccinated cohort) | Annex | %HB_PROFIL |
| Template 16 | Individuals results of hemoglobin levels outside of the normal ranges in Control group (Total vaccinated cohort) | Annex | %HB_PROFIL |
| Template 16 | Individuals results of <b>platelets counts</b> outside of<br>the normal ranges in <b>30</b> PreF group (Total<br>vaccinated cohort) | Annex | %HB_PROFIL |

| Template # | Table Title | Output | Macro |
|---|---|---|---|
| T 1 1 1 C | | destination | A/UD DDOE!! |
| Template 16 | Individuals results of platelets counts outside of | Annex | %HB_PROFIL |
| | the normal ranges in 60 PreF group (Total | | |
| <b>m</b> 1 . 14 | vaccinated cohort) | 4 | O/LID DDOE!! |
| Template 16 | Individuals results of platelets counts outside of | Annex | %HB_PROFIL |
| | the normal ranges in <b>120</b> PreF group (Total | | |
| | vaccinated cohort) | 4 | A/UD DDOEU |
| Template 16 | Individuals results of platelets counts outside of | Annex | %HB_PROFIL |
| | the normal ranges in <b>Control</b> group (Total | | |
| <b>m</b> 1 . 16 | vaccinated cohort) | 4 | A/UD DDOEU |
| Template 16 | Individuals results of white blood cells counts | Annex | %HB_PROFIL |
| | outside of the normal ranges in <b>30</b> PreF group | | |
| | (Total vaccinated cohort) | _ | 2/115 556511 |
| Template 16 | Individuals results of white blood cells counts | Annex | %HB_PROFIL |
| | outside of the normal ranges in <b>60</b> PreF group | | |
| | (Total vaccinated cohort) | _ | |
| Template 16 | Individuals results of white blood cells counts | Annex | %HB_PROFIL |
| | outside of the normal ranges in <b>120</b> PreF group | | |
| | (Total vaccinated cohort) | | |
| Template 16 | Individuals results of white blood cells counts | Annex | %HB_PROFIL |
| | outside of the normal ranges in <b>Control</b> group | | |
| | (Total vaccinated cohort) | | |
| Template 16 | Individuals results of <b>ALT levels</b> outside of the | Annex | %HB_PROFIL |
| | normal ranges in <b>30</b> PreF group (Total | | |
| | vaccinated cohort) | | |
| Template 16 | Individuals results of <b>ALT levels</b> outside of the | Annex | %HB_PROFIL |
| | normal ranges in <b>60</b> PreF group (Total | | |
| | vaccinated cohort) | | |
| Template 16 | Individuals results of <b>ALT levels</b> outside of the | Annex | %HB_PROFIL |
| | normal ranges in <b>120</b> PreF group (Total | | |
| | vaccinated cohort) | | |
| Template 16 | Individuals results of <b>ALT levels</b> outside of the | Annex | %HB_PROFIL |
| | normal ranges in <b>Control</b> group (Total | | |
| | vaccinated cohort) | | |
| Template 16 | Individuals results of <b>AST levels</b> outside of the | Annex | %HB_PROFIL |
| • | normal ranges in <b>30</b> PreF group (Total | | |
| | vaccinated cohort) | | |
| Template 16 | Individuals results of <b>AST levels</b> outside of the | Annex | %HB_PROFIL |
| - | normal ranges in <b>60</b> PreF group (Total | | |
| | vaccinated cohort) | | |
| Template 16 | Individuals results of <b>AST levels</b> outside of the | Annex | %HB_PROFIL |
| - | normal ranges in <b>120</b> PreF group (Total | | |
| | vaccinated cohort) | | |
| Template 16 | Individuals results of AST levels outside of the | Annex | %HB_PROFIL |
| • | normal ranges in <b>Control</b> group (Total | | |
| | vaccinated cohort) | | |
| Template 16 | Individuals results of creatinine levels outside of | Annex | %HB_PROFIL |
| - | the newsel render in 20 Dref every (Total | | |
| | the normal ranges in <b>30</b> PreF group (Total | | |

204812 (RSV F-021)

SAP (associated to IDMC Charter) Amendment 1 Final

| Template # | Table Title | Output destination | Macro |
|---|---|---|---|
| Template 16 | Individuals results of <b>creatinine levels</b> outside of<br>the normal ranges in <b>60</b> PreF group (Total<br>vaccinated cohort) | Annex | %HB_PROFIL |
| Template 16 | Individuals results of <b>creatinine levels</b> outside of the normal ranges in <b>120</b> PreF group (Total vaccinated cohort) | Annex | %HB_PROFIL |
| Template 16 | Individuals results of <b>creatinine levels</b> outside of<br>the normal ranges in <b>Control</b> group (Total<br>vaccinated cohort) | Annex | %HB_PROFIL |

### 11.2. List of listings

The listings will present <u>data reported up to the data lock point</u>, of which may be after Visit 3 (Day 30) for some subjects.

For the blinded report, individual data listings are not including the group information.

For the unblinded report individual data listings are including the group in formation (XLS documents).

- APPENDIX TABLE IB DEMOGRAPHY
- APPENDIX TABLE ICII REASON FOR VISIT NOT DONE
- APPENDIX TABLE ID GENERAL MEDICAL HISTORY EXAMINATION
- APPENDIX TABLE II REASON FOR VACCINE NOT ADMINISTERED
- APPENDIX TABLE IIA SOLICITED LOCAL ADVERSE EVENTS
- APPENDIX TABLE IIB SOLICITED GENERAL ADVERSE EVENTS
- APPENDIX TABLE IIC UNSOLICITED ADVERSE EVENTS
- APPENDIX TABLE IID MEDICATION
- APPENDIX TABLE IIEi MA-RTI VISIT INFORMATION
- APPENDIX TABLE IIEii MA-RTI SYMPTOMS INFORMATION
- APPENDIX TABLE IIEiii MA-RTI MICROBIOLOGICAL WORKUP INFORMATION
- APPENDIX TABLE IIEiv CHEST X-RAY OBSERVATIONS AT MA-RTI VISIT
- APPENDIX TABLE IVA HAEMATOLOGY AND BIOCHEMISTRY (ALL VALUES)
- APPENDIX TABLE IVBi RSV
- APPENDIX TABLE IVBii PREGNANCY TEST

### 12. TEMPLATE OF TABLES

### Template 1 Summary of demographic characteristics (Total vaccinated cohort)

| | | <each gr<="" th=""><th>oup&gt; (N=</th><th>Total</th><th>(N=</th></each> | oup> (N= | Total | (N= |
|---|---|---|---|---|---|
| | | Value or | )<br>% | Value or | % |
| Characteristics | Parameters or | n | | n | |
| | Categories | | | | |
| Age (years) at dose 1 | Mean | | | | |
| | SD | | | | |
| | Median | | | | |
| | Minimum | | | | |
| | Maximum | | | | |
| Ethnicity | American Hispanic or Latino | | | | |
| | Not American Hispanic or Latino | | | | |
| Geographic Ancestry | African Heritage / African American | | | | |
| | American Indian or Alaskan Native | | | | |
| | Asian - Central/South Asian Heritage | | | | |
| | Asian - East Asian Heritage | | | | |
| | Asian - Japanese Heritage | | | | |
| | Asian - South East Asian Heritage | | | | |
| | Native Hawaiian or Other Pacific Islander | | | | |
| | White - Arabic / North African Heritage | | | | |
| | White - Caucasian / European Heritage | | | | |
| | Other | | | | |

<each group>:

30 PreF = 30 mcg PreF

60 PreF = 60 mcg PreF

120 PreF =120 mcg PreF

Control = Placebo

N = total number of subjects

n/% = number / percentage of subjects in a given category

Value = value of the considered parameter

SD = standard deviation

204812 (RSV F-021)

SAP (associated to IDMC Charter) Amendment 1 Final

## Template 2 Number of subjects vaccinated, completed and withdrawn with reason for withdrawal (Day 30) (Total vaccinated cohort)

| | <each group=""></each> | Total |
|---|---|---|
| Number of subjects vaccinated | | |
| Number of subjects completed | | |
| Number of subjects withdrawn | | |
| Reasons for withdraw: | | |
| Serious Adverse Event | | |
| Non-serious adverse event | | |
| Protocol violation | | |
| Consent withdrawal (not due to an adverse event) | | |
| Migrated/moved from study area | | |
| Lost to follow-up (subjects with incomplete vaccination course) | | |
| Lost to follow-up (subjects with complete vaccination course) | | |
| Other - <reason></reason> | | |
| Other - <reason></reason> | | |

### <each group>:

30 PreF = 30 mcg PreF

60 PreF = 60 mcg PreF

120 PreF =120 mcg PreF

Control = Placebo

Vaccinated = number of subjects who were vaccinated in the study

Completed = number of subjects who completed up to Day30

withdrawn = number of subjects who did not come up to Day30

Template 3 Compliance in returning symptom information (Total vaccinated cohort)

| Group | Number<br>of<br>doses | Doses NOT according to protocol | Number<br>of<br>general SS | Compliance<br>%<br>general SS | Number<br>of<br>local SS | Compliance<br>%<br>local SS |
|---|---|---|---|---|---|---|
| <each group=""></each> | | | | | | |

### <each group>:

30 PreF = 30 mcg PreF

60 PreF = 60 mcg PreF

120 PreF =120 mcg PreF

Control = Placebo

SS = Symptom screens/sheets used for the collection of local and general solicited AEs

Compliance % = (number of doses with symptom screen/sheet return / number of administered doses) X 100

204812 (RSV F-021)

SAP (associated to IDMC Charter) Amendment 1 Final

## Template 4 Incidence of solicited local symptoms reported during the 7-day (Days 0-6) post-vaccination period (Total vaccinated cohort)

| | | | | <each gro<="" th=""><th>oup&gt;</th><th></th></each> | oup> | |
|---|---|---|---|---|---|---|
| | | | | | 9 | 5 % CI |
| Symptom | Туре | N | n | % | LL | UL |
| Pain | All | | | | | |
| | Grade 1 | | | | | |
| | Grade 2 | | | | | |
| | Grade 3 | | | | | |
| | Onset ≤48h | | | | | |
| | Onset ≤48h * Grade 2 | | | | | |
| | Onset ≤48h * Grade 3 | | | | | |
| Redness<br>(mm) | All | | | | | |
| | >20 and ≤ 50 | | | | | |
| | >50 and ≤ 100 | | | | | |
| | >100 | | | | | |
| | Onset ≤48h | | | | | |
| | Onset ≤48h * >50 and ≤ 100 | | | | | |
| | Onset ≤48h * >100 | | | | | |
| Swelling<br>(mm) | All | | | | | |
| , | >20 and ≤ 50 | | | | | |
| | >50 and ≤ 100 | | | | | |
| | >100 | | | | | |
| | Onset ≤48h | | | | | |
| | Onset ≤48h * >50 and ≤ 100 | | | | | |
| | Onset ≤48h * >100 | | | | | |

### <each group>:

30 PreF = 30 mcg PreF

60 PreF = 60 mcg PreF

120 PreF =120 mcg PreF

Control = Placebo

N= number of subjects with the documented dose

n/%= number/percentage of subjects reporting at least once the symptom

95%CI= Exact 95% confidence interval; LL = lower limit, UL = upper limit

The maximum intensity of local injection site redness/swelling was coded as follows for adults:

0: ≤ 20 mm

1:  $> 20 \text{ mm to} \le 50 \text{ mm}$ 

2:  $> 50 \text{ mm to} \le 100 \text{ mm}$ 

3: > 100 mm

Note: this template is also for the summary by maximum intensity

204812 (RSV F-021)

SAP (associated to IDMC Charter) Amendment 1 Final

Template 5 Incidence of solicited local symptoms reported during the 7-day (Days 0-6) post-vaccination period by duration (Total vaccinated cohort)

| | | | | | <each gro<="" th=""><th>up&gt;</th><th></th></each> | up> | |
|---|---|---|---|---|---|---|---|
| | | | | | | | 5 % CI |
| Symptom | Duration | Туре | N | n | % | LL | UL |
| Pain | =<3 days | All | | | | | |
| | | Grade 1 | | | | | |
| | | Grade 2 | | | | | |
| | | Grade 3 | | | | | |
| | > 3 days | All | | | | | |
| | | Grade 1 | | | | | |
| | | Grade 2 | | | | | |
| | | Grade 3 | | | | | |
| | Total | All | | | | | |
| | | Grade 1 | | | | | |
| | | Grade 2 | | | | | |
| | | Grade 3 | | | | | |
| Redness (mm) | =<3 days | All | | | | | |
| , , | | > 20 and ≤ 50 | | | | | |
| | | > 50 and ≤ 100 | | | | | |
| | | > 100 | | | | | |
| | > 3 days | All | | | | | |
| | , | > 20 and ≤ 50 | | | | | |
| | | > 50 and ≤ 100 | | | | | |
| | | > 100 | | | | | |
| | Total | All | | | | | |
| | | > 20 and ≤ 50 | | | | | |
| | | > 50 and ≤ 100 | | | | | |
| | | > 100 | | | | | |
| Swelling (mm) | =<3 days | All | | | | | |
| <b>3</b> ( ) | , | > 20 and ≤ 50 | | | | | |
| | | > 50 and ≤ 100 | | | | | |
| | | > 100 | | | | | |
| | > 3 days | All | | | | | |
| | , | > 20 and ≤ 50 | | | | | |
| | | > 50 and ≤ 100 | | | | | |
| | | > 100 | | | | | |
| | Total | All | | | | | |
| | | > 20 and ≤ 50 | | | | | |
| | | > 50 and ≤ 100 | | | | | |
| | | > 100 | | | | | |

### <each group>:

30 PreF = 30 mcg PreF

60 PreF = 60 mcg PreF

120 PreF =120 mcg PreF

Control = Placebo

N= number of subjects with the documented dose

n/%= number/percentage of subjects reporting at least once the symptom

95%CI= Exact 95% confidence interval; LL = lower limit, UL = upper limit

The maximum intensity of local injection site redness/swelling was coded as follows for adults:

- 0: ≤20 mm
- 1:  $> 20 \text{ mm to } \le 50 \text{ mm}$
- 2:  $> 50 \text{ mm to} \le 100 \text{ mm}$
- 3: > 100 mm

204812 (RSV F-021)

SAP (associated to IDMC Charter) Amendment 1 Final

# Template 6 Incidence of solicited general symptoms reported during the 7-day (Days 0-6) post-vaccination period (Total vaccinated cohort)

| | | | | <each gi<="" th=""><th></th><th></th></each> | | |
|---|---|---|---|---|---|---|
| | | | | | | 5 % CI |
| Symptom | Туре | N | n | % | LL | UL |
| atigue | All | | | | | |
| · · | Grade 1 | | | | | |
| | Grade 2 | | | | | |
| | Grade 3 | | | | | |
| | Related | | | | | |
| | Grade 2*Related | | | | | |
| | Grade 3*Related | | | | | |
| | Onset ≤48h | | | | | |
| | Onset ≤48h *Grade 2 | | | | | |
| | Onset ≤48h *Grade 3 | | | | | |
| Temperature (Oral) (°C | ) All (≥37.5) | | | | | |
| | >38.0 | | | | | |
| | >38.5 | | | | | |
| | >39.0 | | | | | |
| | >39.5 | | | | | |
| | Related | | | | | |
| | >38.5*Related | | | | | |
| | >39.5*Related | | | | | |
| | Onset ≤48h | | | | | |
| | Onset ≤48h *>38.5 | | | | | |
| | Onset ≤48h *>39.5 | | | | | |
| Gastrointestinal | All | | | | | |
| symptoms | Grade 1 | | | | | |
| Jimptomo | Grade 2 | | | | | |
| | Grade 3 | | | | | |
| | Related | | | | | |
| | Grade 2*Related | | | | | |
| | Grade 3*Related | | | | | |
| | Onset ≤48h | | | | | |
| | Onset ≤48h *Grade 2 | | | | | |
| | Onset ≤48h *Grade 3 | | | | | |
| -leadache | All | | | | | |
| Toddaoilo | Grade 1 | | | | | |
| | Grade 2 | | | | | |
| | Grade 3 | | | | | |
| | Related | | | | | _ |
| | Grade 2*Related | | | | | _ |
| | Grade 3*Related | | | | | |
| | Onset ≤48h | | | | | |
| | Onset ≤48h *Grade 2 | | | | | |
| | Onset ≤48h *Grade 3 | | | | | |

### <each group>:

30 PreF = 30 mcg PreF

60 PreF = 60 mcg PreF

120 PreF =120 mcg PreF

Control = Placebo

N = number of subjects with the documented dose

 $\ensuremath{\text{n}}\xspace/\%$  = number/percentage of subjects reporting the symptom at least once

95%CI = Exact 95% confidence interval; LL = lower limit, UL = upper limit

Temperatures were coded as follows for adults:

204812 (RSV F-021)

SAP (associated to IDMC Charter) Amendment 1 Final

- 0: < 37.5 °C 1: ≥ 37.5 °C to ≤ 38.5 °C 2: > 38.5 °C to ≤ 39.5 °C
- 3: > 39.5°C

Note: this template is also for the summary by maximum intensity

Incidence of solicited general symptoms reported during the 7-day (Days 0-6) post-vaccination period by duration (Total vaccinated Template 7 cohort)

| | | | | ' | <each gr<="" th=""><th></th><th> /</th></each> | | / |
|---|---|---|---|---|---|---|---|
| 0 | D | T= | ., | | 0/ | | 5 % CI |
| Symptom | Duration | Type | N | n | % | LL | UL |
| Fatigue | =<3 days | All | | | | | |
| | | Grade 1 | | | | | |
| | | Grade 2 | | | | | |
| | | Grade 3 | | | | | |
| | | Related | | | | | |
| | | Grade 2*Related | | | | | |
| | | Grade 3*Related | | | | | |
| | > 3 days | All | | | | | |
| | | Grade 1 | | | | | |
| | | Grade 2 | | | | | |
| | | Grade 3 | | | | | |
| | | Related | | | | | |
| | | Grade 2*Related | | | | | |
| | | Grade 3*Related | | | | | |
| | Total | All | | | | | |
| | Total | Grade 1 | | | | | |
| | | Grade 2 | | | | | |
| | | Grade 3 | | | | | |
| | | Related | | | | | |
| | | Grade 2*Related | | | | | |
| | | Grade 3*Related | | | | | |
| Temperature<br>'Oral) (°C) | =<3 days | <i>All (≥37.5)</i> | | | | | |
| , , , | | >38.0 | | | | | |
| | | >38.5 | | | | | |
| | | >39.0 | | | | | |
| | | >39.5 | | | | | |
| | | Related | | | | | |
| | | >38.5*Related | | | | | |
| | | >39.5*Related | | | | | |
| | > 3 days | All (≥37.5) | | | | | |
| | - 5 days | >38.0 | | | | | |
| | | >38.5 | | | | | |
| | | >39.0 | | | | | |
| | | >39.5 | | | | | |
| | | Related | | | | | |
| | | >38.5*Related | | | | | |
| | | >39.5*Related | | | | | |
| | Total | <i>All (≥37.5)</i> | | | | | |
| | | >38.0 | | | | | |
| | | >38.5 | | | | | |
| | | >39.0 | | | | | |
| | | >39.5 | | | | | |
| | | Related | | | | | |
| | | >38.5*Related | | | | | |
| | | >39.5*Related | | | | | |
| Gastrointestinal | =<3 days | All | | | | | |
| ymptoms | 0 30,0 | Grade 1 | | | | | |
| Julipionio | | Grade 2 | | - | | | |

204812 (RSV F-021)

### SAP (associated to IDMC Charter) Amendment 1 Final

| | | | | <each gr<="" th=""><th></th><th></th></each> | | | |
|---|---|---|---|---|---|---|---|
| | | | | | | 9: | 5 % CI |
| Symptom | Duration | Туре | N | n | % | LL | UL |
| | | Grade 3 | | | | | |
| | | Related | | | | | |
| | | Grade 2*Related | | | | | |
| | | Grade 3*Related | | | | | |
| | > 3 days | All | | | | | |
| | | Grade 1 | | | | | |
| | | Grade 2 | | | | | |
| | | Grade 3 | | | | | |
| | | Related | | | | | |
| | | Grade 2*Related | | | | | |
| | | Grade 3*Related | | | | | |
| | Total | All | | | | | |
| | | Grade 1 | | | | | |
| | | Grade 2 | | | | | |
| | | Grade 3 | | | | | |
| | | Related | | | | | |
| | | Grade 2*Related | | | | | |
| | | Grade 3*Related | | | | | |
| -leadache | =<3 days | All | | | | | |
| | | Grade 1 | | | | | |
| | | Grade 2 | | | | | |
| | | Grade 3 | | | | | |
| | | Related | | | | | |
| | | Grade 2*Related | | | | | |
| | | Grade 3*Related | | | | | |
| | > 3 days | All | | | | | |
| | o dayo | Grade 1 | | | | | |
| | | Grade 2 | | | | | |
| | | Grade 3 | | | | | |
| | | Related | | | | | |
| | | Grade 2*Related | | | | | |
| | | Grade 3*Related | | | | | |
| | Total | All | | | | | |
| | | Grade 1 | | | | | |
| | | Grade 2 | | | | | |
| | | Grade 3 | | | | | |
| | | Related | | | | | |
| | | Grade 2*Related | | | | | |
| | | Grade 3*Related | | | | + | |

### <each group>:

30 PreF = 30 mcg PreF

60 PreF = 60 mcg PreF

120 PreF =120 mcg PreF

Control = Placebo

*N* = number of subjects with the documented dose

n/% = number/percentage of subjects reporting the symptom at least once 95%CI = Exact 95% confidence interval; LL = lower limit, UL = upper limit

Temperatures were coded as follows for adults:

0: < 37.5 °C 1: ≥ 37.5 °C to ≤ 38.5 °C

2:  $> 38.5 \text{ °C to} \le 39.5 \text{ °C}$ 

3: > 39.5°C

204812 (RSV F-021)

SAP (associated to IDMC Charter) Amendment 1 Final

# Template 8 Incidence and nature of symptoms (solicited and unsolicited reported during the 7-day (Days 0-6) post-vaccination period (Total vaccinated cohort)

| | Any sy | mptom | | | | General symptoms | | | | | Local symptoms | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | 95% ( | Cl | | | | 95% CI | | | | | 95% CI | |
| Group | N | n | % | LL | UL | N | n | % | LL | UL | N | n | % | LL | UL |
| <each group=""></each> | | | | | | | | | | | | | | | |

### <each group>:

30 PreF = 30 mcg PreF

60 PreF = 60 mcg PreF

120 PreF =120 mcg PreF

Control = Placebo

N = number of subjects with the administered dose

n/% = number/percentage of subjects presenting at least one type of symptom whatever the study vaccine administered

95% CI = exact 95% confidence interval, LL = Lower Limit, UL = Upper Limit

# Template 9 Percentage of subjects reporting the occurrence of unsolicited classified by MedDRA Primary System Organ Class and Preferred Term within the 30-day (Days 0-29) post-vaccination period (Total vaccinated cohort)

| | | <each group=""><br/>N =</each> | | | |
|---|---|---|---|---|---|
| | | | | 95% | CI |
| Primary System Organ Class (CODE) | n | % | LL | UL | |
| At least one symptom | | | | | |
| <each (code)="" soc=""></each> | <each (code)="" pt=""></each> | | | | |

### <each group>:

30 PreF = 30 mcg PreF

60 PreF = 60 mcg PreF

120 PreF =120 mcg PreF

Control = Placebo

At least one symptom = at least one symptom experienced (regardless of the MedDRA Preferred Term)

N = number of subjects with at least one administered dose

n/% = number/percentage of subjects reporting at least once the symptom

95% CI= exact 95% confidence interval; LL = Lower Limit, UL = Upper Limit

204812 (RSV F-021)

SAP (associated to IDMC Charter) Amendment 1 Final

# Template 10 Number and percentage of subjects taking a concomitant medication during the 7- day (Days 0-6) post -vaccination period (Total vaccinated cohort)

| | | | <each ;<="" th=""><th>group&gt;</th><th></th><th></th></each> | group> | |
|---|---|---|---|---|---|
| | | | | | 95% CI |
| | N | n | % | LL | UL |
| Any | | | | | |
| Any antipyretics | | | | | |
| Prophylactic antipyretics | | | | | |

### <each group>:

30 PreF = 30 mcg PreF

60 PreF = 60 mcg PreF

120 PreF =120 mcg PreF

Control = Placebo

N= number of administered doses

n/%= number/percentage of subjects who took the specified concomitant medication at least once during the mentioned period

95% CI = exact 95% confidence interval, LL = Lower Limit, UL = Upper Limit

204812 (RSV F-021)

SAP (associated to IDMC Charter) Amendment 1 Final

### Template 11 Listing of SAEs reported up to data lock point (Total vaccinated cohort)

| Group | Sub.No. Sex | Country | Age at onset (Year) | Verbatim | Primary System Organ<br>Class | MED type | Dose | Day of onset | Duration | Intensity | Causality | Outcome |
|---|---|---|---|---|---|---|---|---|---|---|---|---|

### <each group>:

30 PreF = 30 mcg PreF

60 PreF = 60 mcg PreF

120 PreF =120 mcg PreF

Control = Placebo

02-MAY-2017 

204812 (RSV F-021)

SAP (associated to IDMC Charter) Amendment 1 Final

## Template 12 Listing of adverse events, SAEs and solicited symptoms leading to withdrawal from the treatment/study (Total Vaccinated Cohort)

| Group | Study- | Country | Gender | Race | <b>AE Description</b> | SAE | Causality | Outcome | Type of discontinuation |
|---|---|---|---|---|---|---|---|---|---|
| | Subject No. | | | | | | | | |

<each group>:

30 PreF = 30 mcg PreF 60 PreF = 60 mcg PreF 120 PreF =120 mcg PreF

Control = Placebo

# Template 13 Distribution of change from baseline in haematology and biochemistry with respect to normal laboratory ranges (Total vaccinated cohort)

| | | | <each group=""></each> | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | ng Baseline PRE(D0) | U | Inknown | | Below | | Within | | bove |
| Laboratory parameter | Timing | | n | % | n | % | n | % | n | % |
| Alanine Aminotransferase | PI (D7) | Unknown | | | | | | | | |
| (ALT) | | Below | | | | | | | | |
| | | Within | | | | | | | | |
| | | Above | | | | | | | | |
| | PI (D30) | | | | | | | | | |
| | PI (D60) | | | | | | | | | |
| | PI (D90) | | | | | | | | | |
| Aspartate Aminotransferase | PI (D7) | Unknown | | | | | | | | |
| (AST) | | Below | | | | | | | | |
| | | Within | | | | | | | | |
| | | Above | | | | | | | | |
| | PI (D30) | | | | | | | | | |
| | PI (D60) | | | | | | | | | |
| | PI (D90) | | | | | | | | | |
| Creatinine | | | | | | | | | | |
| Eosinophil | | | | | | | | | | |
| Haemoglobin | | | | | | | | | | |
| Lymphocyte | | | | | | | | | | |
| Neutrophil | | | | | | | | | | |
| Platelet count | | *** | | | | | | | | |
| White Blood Cells (WBC) | | | | | | | | | | |

### <each group>:

30 PreF = 30 mcg PreF

60 PreF = 60 mcg PreF

120 PreF = 120 mcg PreF

Control = Placebo

N = number of subjects with available results for the specified laboratory parameter and timing in a given baseline category

n/% = number/percentage of subjects in the specified category

Below = below the normal laboratory range defined for the specified laboratory parameter

Within = within the normal laboratory range defined for the specified laboratory parameter

Above = above the normal laboratory range defined for the specified laboratory parameter

PI (D7): 7 days post dose 1

PI (D30): 30 days post dose 1

PI(D60) = 60 days post dose 1

PI(D90) = 90 days post dose 1

204812 (RSV F-021)

SAP (associated to IDMC Charter) Amendment 1 Final

# Template 14 Summary of haematology and biochemistry results by maximum grade from VISIT 2 (D7) up to VISIT 5 (D90) versus baseline (Total vaccinated cohort)

| | VISIT2 (D7) up to VISIT5 (D90) | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | <each group=""></each> | | | | | | | | | | | | |
| | | | Unkı | nown | Gra | de 0 | Grad | Grade 1 Grade | | de 2 | 2 Grade 3 | | Grade 4 | |
| Laboratory parameter | Baseline<br>PRE(D0) | N | n | % | n | % | n | % | n | % | n | % | n | % |
| Alanine Aminotransferase (ALT) increase by factor | Unknown | | | | | | | | | | | | | |
| • | Grade 0 | | | | | | | | | | | | | |
| | Grade 1 | | | | | | | | | | | | | |
| | Grade 2 | | | | | | | | | | | | | |
| | Grade 3 | | | | | | | | | | | | | |
| | Grade 4 | | | | | | | | | | | | | |
| | Total | | | | | | | | | | | | | |
| Aspartate Aminotransferase (AST) increase by factor | | | | | | | | | | | | | | |
| Creatinine | | | | | | | | | | | | | | |
| Eosinophils increase | | | | | | | | | | | | | | |
| Hemoglobin decrease | | | | | | | | | | | | | | |
| Lymphocytes decrease | | | | | | | | | | | | | | |
| Neutrophils decrease | | | | | | | | | | | | | | |
| Platelet count decrease | | | | | | | | | | | | | | |
| White Blood Cells (WBC) decrease | | | | | | | | | | | | | | |
| White Blood Cells (WBC) increase | | | | | | | | | | | | | | |

### <each group>:

30 PreF = 30 mcg PreF

60 PreF = 60 mcg PreF

120 PreF = 120 mcg PreF

Control = Placebo

N = number of subjects with at least one available result for the specified laboratory parameter and follow-up period n/% = number/percentage of patients reporting at least once the laboratory event when the maximum grading over the follow-up period is considered

Template 15 Summary of haematology change from baseline by maximum grade from VISIT2 (D7) up to VISIT5 (D90) (Total vaccinated cohort)

| | VISIT2 (D7) up to VISIT5 (D90) | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | <each group=""></each> | | | | | | | | | | | | |
| | | Unkr | nown | Grade 0 | | Grade 1 | | Grade 2 | | Grade 3 | | Grade 4 | |
| Laboratory parameter | | n | % | n | % | n | % | n | % | n | % | n | % |
| Hemoglobin (Change from baseline) | | | | | | | | | | | | | |

### <each group>:

30 PreF = 30 mcg PreF

60 PreF = 60 mcg PreF

120 PreF = 120 mcg PreF

Control = Placebo

N = number of subjects with at least one available result for the specified laboratory parameter and follow-up period n/% = number/percentage of subjects reporting at least once the laboratory event when the maximum grading over the follow-up period is considered
204812 (RSV F-021)

SAP (associated to IDMC Charter) Amendment 1 Final





Note: This figure is shown as an example. For the unblinded report, one figure per group will be performed. For the blinded report, 4 graphs will be performed each of them presenting property subjects regardless of treatment (the first property subjects, from the property to the subject...). The X axis will include Day 0, Day 7 and Day 30. The Y axis will be adapted according to each parameter.

204812 (RSV F-021) Statistical Analysis Plan Amendment 2 Final

| Detailed Title: A Phase II, randomised, observer-blind, controlled multi-country study to rank different formulations GSK Biologicals' investigational RSV vaccine (GSK3003891A), based on immunogenicity, reactogenicity and safety, when administered to healthy women, aged 18 – 45 years. eTrack study number and Abbreviated Scope: All data pertaining to the above study. Date of Statistical Analysis Plan Final: Amendment 2 (09-Nov-2017) Amendment 1 (21-Jul-2017) Version 2.0 (10-Nov-2016) | - |
|---|---|
| multi-country study to rank different formulations GSK Biologicals' investigational RSV vaccine (GSK3003891A), based on immunogenicity, reactogenicity and safety, when administered to healthy women, aged 18 – 45 years. eTrack study number and Abbreviated Scope: All data pertaining to the above study. Date of Statistical Analysis Plan Final: Amendment 2 (09-Nov-2017) Amendment 1 (21-Jul-2017) | - |
| Abbreviated Scope: All data pertaining to the above study. Date of Statistical Analysis Final: Amendment 2 (09-Nov-2017) Plan Amendment 1 (21-Jul-2017) | |
| Date of Statistical Analysis Final: Amendment 2 (09-Nov-2017) Plan Amendment 1 (21-Jul-2017) | |
| Plan Amendment 1 (21-Jul-2017) | |
| intertuncti (21 out 2017) | |
| Version 2.0 (10-Nov-2016) | I |
| | Version 2.0 (10-Nov-2016) |
| Version 1.0 (25-Aug-2016 | Version 1.0 (25-Aug-2016 |
| Co-ordinating author: PPD (Statistician) | |
| Deviewed by: PPD (Clinical and Enidemiology Project | |
| Reviewed by: Clinical and Epidemiology Project Lead) | t |
| Lead) | |
| (Clinical Research and Development Le | ead) |
| (Lead statistician) | |
| (Lead statistical analyst) | |
| PPD (Scientific writer) | (Scientific writer) |
| PPD (Regulatory Affair) | |
| (SERM physician) | |
| (Public disclosure representative) | |
| Approved by: (Clinical Research and Development Lead) | ıt |
| (Lead statistician) | |
| (Lead stat analyst) | |
| (Lead scientific writer) | |

APP 9000058193 Statistical Analysis Plan Template (Effective date: 14 April 2017)

204812 (RSV F-021) Statistical Analysis Plan Amendment 2 Final

# **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| LIS | T OF A | ABBREVIATIONS | 10 |
| 1. | DOC | JMENT HISTORY | 12 |
| 2. | STUE | OY DESIGN | 16 |
| 3. | | CTIVES | 10 |
| J. | 3.1. | Primary Objective | |
| | 3.2. | Secondary objectives | |
| | 3.3. | | |
| 4. | ENDF | POINTS | 19 |
| | 4.1. | Primary | |
| | 4.2. | Secondary | |
| | 4.3. | Tertiary | 20 |
| 5. | ANAL | YSIS SETS | 20 |
| | 5.1. | Definition | |
| | | 5.1.1. Exposed Set (ES) | |
| | | 5.1.2. Per-Protocol Set (PPS) for analysis of immunogenicity | |
| | 5.2. | Criteria for eliminating data from Analysis Sets | |
| | | 5.2.1. Elimination from Exposed Set (ES) | |
| | | 5.2.2. Elimination from Per-protocol analysis Set (PPS) | |
| | | 5.2.2.1. Excluded subjects | 22 |
| | | 5.2.2.2. Right censored Data | 24<br>24 |
| | 5.3. | Important protocol deviation not leading to elimination from per- | 24 |
| | 0.0. | protocol analysis set | 24 |
| 6. | STAT | ISTICAL ANALYSES | 24 |
| • | 6.1. | Demography | |
| | | 6.1.1. Analysis of demographics/baseline characteristics planned | |
| | 0.0 | in the protocol | |
| | 6.2. | Immunogenicity | |
| | | 6.2.1. Analysis of immunogenicity planned in the protocol | |
| | | 6.2.1.2. Between group assessment | |
| | | 6.2.2. Additional considerations | |
| | 6.3. | Analysis of safety | |
| | | 6.3.1. Analysis of safety planned in the protocol | |
| | | 6.3.1.1. Within group analysis | |
| | | 6.3.1.2. Between group assessment | |
| | 6.4. | Analysis for ranking RSV formulations | 30 |
| | | 6.4.1. Definition of desirability in the context of Simulations | |
| | | 6.4.2. Derived endpoints | |
| | 6.5. | Analysis of medically attended RTIs | 31 |
| 7 | ΔΝΔΙ | YSIS INTERPRETATION | 31 |

| | | OOM BENTAL | |
|---|---|---|---|
| | | 204812 (RSV F-<br>Statistical Analysis Plan Amendment 2 | |
| 8. | CONE | OUCT OF ANALYSES | |
| 0. | 8.1. | Sequence of analyses | |
| | 8.2. | Statistical considerations for interim analyses | |
| 0 | CLIAN | ICEC EDOM DI ANNED ANALYOFO | 22 |
| 9. | CHAN | IGES FROM PLANNED ANALYSES | 33 |
| 10. | LIST ( | OF FINAL REPORT TABLES, LISTINGS AND FIGURES | 35 |
| 11 | ΔNNE | X 1 STANDARD DATA DERIVATION RULE AND STATISTICAL | |
| | | IODS | 35 |
| | | Statistical Method References. | |
| | | Standard data derivation | |
| | | 11.2.1. Date derivation | 36 |
| | | 11.2.2. Dose number | 36 |
| | | 11.2.3. Demography | 36 |
| | | 11.2.4. Immunogenicity | 37 |
| | | 11.2.5. Safety | 38 |
| | | 11.2.6. Number of decimals displayed | 41 |
| 12. | ANNE | X 2: SUMMARY ON ELIMINATION CODES | 41 |
| 13. | ANNE<br>INDEX | X 3 CALCULATION OF INDIVIDUAL AND OVERALL DESIRABILITY | 41 |

14. ANNEX 4: STUDY SPECIFIC MOCK TFL 46

204812 (RSV F-021) Statistical Analysis Plan Amendment 2 Final

# **LIST OF TABLES**

| | | PAGE |
|---------|--------------------------------------------------|------|
| Table 1 | Study groups and epochs foreseen in the study | 17 |
| Table 2 | Study groups and treatment foreseen in the study | 17 |
| Table 3 | Blinding of study epochs | 17 |

204812 (RSV F-021) Statistical Analysis Plan Amendment 2 Final

# **LIST OF FIGURES**

| | | PAGE |
|---|---|---|
| Figure 1. | Study design overview | 16 |
| Figure 2 | Desirability function for the incidence rate of Grade 2/3 general AEs and related SAEs - for each investigational RSV vaccine formulation | 42 |
| Figure 3 | Desirability function for the incidence rate of Grade 2/3 fever - for each investigational RSV vaccine formulation | 43 |
| Figure 4 | Desirability function for neutralising anti-RSV-A GMTs - for each investigational RSV vaccine formulation | 44 |
| Figure 5 | Desirability function for PCA concentrations - for each investigational RSV vaccine formulation | 45 |

204812 (RSV F-021) Statistical Analysis Plan Amendment 2 Final

# **LIST OF TEMPLATE**

| | | PAGE |
|---|---|---|
| Template 1 | Number of subjects enrolled into the study as well as the number of subjects excluded from the PPS analyses with reasons for exclusion | 49 |
| Template 2 | Number of subjects vaccinated, completed and withdrawn with reason for withdrawal (Exposed set) | 49 |
| Template 3 | Number of subjects vaccinated, completed and withdrawn with reason for withdrawal (Exposed set) | 50 |
| Template 4 | Number of subjects at each visit and list of withdrawn subjects (Exposed set) | 50 |
| Template 5 | Summary of demographic characteristics (Per Protocol Set) | 51 |
| Template 6 | Summary of demographic characteristics by age category (Exposed set) | 52 |
| Template 7 | Number of subjects by center (Exposed set) | 53 |
| Template 8 | Number of subjects by center for each age category (Exposet) | |
| Template 9 | Number of subjects by country and center (Exposed set) | 53 |
| Template 10 | Deviations from specifications for age and intervals between study visits (Exposed set) | 54 |
| Template 11 | Summary of vital signs characteristics at VISIT 1 (Day 0) (Exposed set) | 55 |
| Template 12 | Study Population (Exposed set) | 56 |
| Template 13 | Number of enrolled subjects by country | 57 |
| Template 14 | Number of enrolled subjects by age category | 57 |
| Template 15 | Minimum and maximum activity dates (Exposed set) | 57 |
| Template 16 | Incidence and nature of symptoms (solicited and unsolicited reported during the 7-day (Days 0-6) post-vaccination period (Exposed set) | 58 |
| Template 17 | Daily prevalence of any fever during the 7-day (Days 0-6) post-vaccination period (Exposed set) | 58 |
| Template 18 | Incidence of solicited local symptoms reported during the 7-day (Days 0-6) post-vaccination period (Exposed set) | 59 |

204812 (RSV F-021)

| Template 19 | Statistical Analysis Plan Amendment Incidence of solicited local symptoms reported during the 7-day | 2 Final |
|---|---|---|
| | (Days 0-6) post-vaccination period by maximum intensity (Exposed set) | 60 |
| Template 20 | Incidence of solicited general symptoms reported during the 7-day (Days 0-6) post-vaccination period (Exposed set) | 61 |
| Template 21 | Femplate 21 Incidence of solicited general symptoms reported during the 7-day (Days 0-6) post-vaccination period by maximum intensity (Exposed set) | |
| Template 22 | Percentage of subjects reporting the occurrence of unsolicited symptoms classified by MedDRA Primary System Organ Class and Preferred Term within the 30-day (Days 0-29) post-vaccination period (Exposed set) | 63 |
| Template 23 | Listing of SAEs reported up to study end (Exposed set) | 63 |
| Template 24 | Number (%) of subjects with serious adverse events up to study end (Exposed set) | 64 |
| Template 25 | Compliance in returning symptom information (Exposed set) | 64 |
| Template 26 | Number and percentage of subjects taking a concomitant medication during the 7- day (Days 0-6) post -vaccination period (Exposed set) | 65 |
| Template 27 | Exploratory comparisons between groups in terms of percentage of subjects reported any Grade 2/3 AE and/or any fever >38.5°C and/or any vaccine-related SAE during the 7-day (Days 0-6) post-vaccination period (Exposed set) | 65 |
| Template 28 | Solicited and unsolicited symptoms experienced by at least 5 % of subjects, classified by MedDRA Primary System Organ Class and Preferred Term within the 30-day (Days 0-29) post-vaccination period including number of events - SAE excluded (Exposed set) | 66 |
| Template 29 | Distribution of change from baseline in haematology and biochemistry with respect to normal laboratory ranges (Exposed set). | 67 |
| Template 30 | Summary of haematology and biochemistry results by maximum grade from VISIT 2 (D7) up to VISIT 3 (D30) versus baseline (Exposed set) | 68 |
| Template 31 | Summary of haematology change from baseline by maximum grade from VISIT2 (D7) up to VISIT3 (D30) (Exposed set) | 69 |
| Template 32 | Individual results of hemoglobin levels outside of the normal ranges in < group> (Exposed set) | 69 |

204812 (RSV F-021)

| Template 33 | Statistical Analysis Plan Amendment 2 Fina Number and percentage of subjects with anti-RSV-A neutralising |
|---|---|
| · | antibody titer equal to or above <cut-off> and GMTs (Per protocol set)</cut-off> |
| Template 34 | Number and percentage of subjects with anti-RSV-A neutralising antibody titer equal to or above <cut-off> and GMTs - by age category (Per protocol set)</cut-off> |
| Template 35 | Geometric mean of the individual ratio of anti-RSV-A neutralising antibody titers at each post-vaccination timepoint compared to pre-vaccination with 95% CI (Per protocol set) |
| Template 36 | GMTs and their 95% CIs for anti-RSV-A neutralising antibody at each timepoint (Per protocol set) |
| Template 37 | Kinetics of GMTs for anti-RSV-A neutralising antibody on subjects with results available at all timepoints (Per protocol set) |
| Template 38 | Distribution of anti-RSV-A neutralising antibody titer (Per protocol set) |
| Template 39 | Distribution of anti-Neogenin antibody concentration (Exposed set) |
| Template 40 | Distribution of fold of anti-RSV-A neutralising antibody titer by pre-vaccination titer category (Per protocol set) |
| Template 41 | Distribution of fold of anti-neogenin antibody concentration (Exposed set) |
| Template 42 | Reverse cumulative distribution curves for anti-RSV-A neutralising antibody titers in each group at <each point="" time=""> (Per protocol set)</each> |
| Template 43 | Individual results of anti-RSV-A neutralising antibody titer at Day <30/60/90> versus pre-vaccination in <each group=""> and Control (Per protocol set)</each> |
| Template 44 | Vaccine response for anti-RSV-A neutralising antibody titer at each post-vaccination timepoint (Per protocol set) |
| Template 45 | Estimated GMTs and 95% CIs for anti-RSV-A neutralising antibody titre (Per protocol set) |
| Template 46 | Exploratory comparisons (GMT ratios) between RSV groups with corresponding 95% confidence interval for anti-RSV A neutralizing antibody titre at Day 30 (Per protocol set) |
| Template 47 | Individual kinetics of anti-neogenin antibody concentrations by group (Exposed set)82 |

| | CONFIDENTIAL | |
|---|---|---|
| | 204812 (RSV | F-021) |
| Template 48 | Statistical Analysis Plan Amendment GM of individual ratios (fold increase post over pre) and their | |
| Template 40 | | |
| | 95% CIs for anti-RSV F IgG1 and IgG total antibody assays and | |
| | each group, at <day xx=""> (Per protocol set)</day> | 83 |
| Template 49 | Exploratory comparisons (GM ratios of fold increase post/pre) | |
| | between RSV groups with corresponding 95% confidence | |
| | interval for anti-RSV F antibody concentrations (IgG Total) at | |
| | Day 30 (Per protocol set) | 84 |
| Template 50 | Comparisons of GM ratios with corresponding 95% confidence | |
| | interval between anti-RSV F antibody concentrations (IgG Total) | |
| | and anti-RSV-A neutralising antibody titers at pre-vaccination | |
| | (Per protocol set) | 84 |
| | (i or processor cos) | |
| Template 51 | Exploratory comparisons (GM ratios of fold increase post/pre) | |
| • | with corresponding 95% confidence interval between anti-RSV F | |
| | antibody concentrations (IgG Total) and anti-RSV-A neutralising | |
| | antibody titers at Day 30 (Per protocol set) | 85 |
| Template 52 | Desirability index of immunogenicity during the 30-day (Days 0- | |
| • | 29) post-vaccination period (Per protocol set) | 85 |
| Template 53 | Desirability index of reactogenicity during the 7-day (Days 0-6) | |
| | post-vaccination period (Exposed set) | 86 |
| Template 54 | Desirability index based on reactogenicity and safety (Exposed | |
| Tompiate 04 | set up to Day 7) and immunogenicity (Per protocol set up to Day | |
| | | 86 |
| | 30) | |

204812 (RSV F-021)

#### Statistical Analysis Plan Amendment 2 Final

#### LIST OF ABBREVIATIONS

AE Adverse Event

AIDS Acquired Immunodeficiency Syndrome

ANCOVA Analysis of Covariance
ANOVA Analysis of Variance

ALT Alanine Aminotransferase
AST Aspartate Aminotransferase

ATP According-to-Protocol

CDISC Clinical Data Interchange Standards Consortium

CI Confidence Interval

eCRF Electronic Case Report Form

Eli Type Internal GSK database code for type of elimination code

ES Exposed Set

FAS Full Analysis Set

GMC Geometric mean antibody concentration

GMT Geometric mean antibody titer

GSK GlaxoSmithKline

ICH International Conference on Harmonisation
IDMC Independent Data Monitoring Committee

IND Investigational New Drug

iSRC Internal Safety Review Committee

LL Lower Limit of the confidence interval

LLOQ Lower Limit of Quantification

MA-RTI Medically Attended Respiratory Tract Infection

MedDRA Medical Dictionary for Regulatory Activities

NEO Neogenin

PCA Palivizumab Competing Antibodies

PCD Primary completion Date
PCR Polymerase Chain Reaction

PPS Per Protocol Set

PreF Purified recombinant RSV F protein, engineered to preferentially

maintain the pre-fusion conformation

RSV Respiratory syncytial virus

204812 (RSV F-021)

Statistical Analysis Plan Amendment 2 Final

RTI Respiratory Track Infection

SAE Serious adverse event

SAP Statistical Analysis Plan

SAS Statistical Analysis System

SBIR (GSK) Biological's Internet Randomization System

SD Standard Deviation

SRT Safety Review Team

TFL Tables Figures and Listings

TOC Table of Content

TVC Total Vaccinated Cohort

UL Upper Limit of the confidence interval

WBC White Blood Cells

# 1. DOCUMENT HISTORY

| Date | Description | Protocol Version |
|---|---|---|
| 25-AUG-2016 | Version1: first version | RSV F-021 (204812)<br>Protocol (20-Jul-2016) |
| 10-NOV-2016<br>21-JUL-2017 | Version2.0: Description of changes from Version 1.0 are as below — The table of elimination code has been modified — Algorithm for handling of data of PCA neutralising antibody concentrations between the LOB and LLOQ was added Amendment 1: Description of changes from | RSV F-021 (204812)<br>Protocol (20-Jul-2016)<br>RSV F-021 (204812) |
| | Version 2.0 are as below: — Use of new template for SAP (Default-APP 9000058193 Statistical Analysis Plan_v1) — In section 6. Statistical Analyses, immunogenicity was moved before safety — For the sequence of analysis, IDMC analysis up to at least Day 30 including haematology and biochemistry parameters was newlyadded — The table of elimination code has been modified for more clarity — In the analysis of immunogenicity section, the distribution of fold increase of the antibody titres against RSV-A/B and concentrations against NEO have been added — In the analysis of safety section, the percentage of subjects reporting each individual solicited local/general AE during the 7-day follow-up period post vaccination based on maximum intensity per subject has been added — Evaluation of last secondary objective 'To estimate the incidence of medically attended RSV-associated RTIs up to study conclusion' will be performed based on MA-RTIs rather than MA-RSV associated RTIs — The cut-off for the updated (qualified) version of the PCA assay will be set at the level of the assay LLOQ (9.60 μg/mL). | Protocol (20-Jul-2016) |

Statistical Analysis Plan Amendment 2 Final

- Algorithm for handling of data of RSV-B neutralising antibody tires between the LOB and LLOQ is defined as similar as for RSV A by considering the LOB for RSV-B is 6
- Addition of analysis of the lgG total and lgG1 subclass
- Addition of analysis of anti-RSV A and anti-PCA in the subset of subjects with IgG/IgG1 data available
- Changes of TFL/TOC
  - In the analysis of safety section, analysis on 'Individuals results of haematological and biochemical parameters outside of the normal ranges in each group' will be reported
  - In the analysis of safety section, the titles in all tables reporting 'incidence and nature of solicited and unsolicited symptoms' have been changed from 'with causal relationship to' to 'considered related to vaccination'
  - In the analysis of safety section, analysis on 'Incidence of solicited local/general symptoms reported during the 7-day post-vaccination period' will also be reported based on maximum intensity per subject for each grade
  - In the analysis of safety section, analysis on 'Number (%) of subjects reporting the occurrence of adverse events within the 7-day and 30-day postvaccination period' will be added
  - In the analysis of safety section, analysis on 'Number (%) of subjects with SAE or SAE considered related to vaccination during the study period' will not be reported
  - In the analysis of safety section, analysis on 'Number and percentage of subjects reporting the occurrence of medically attended respiration tract infections (MA-RTIs), during the 30/60/90-day post-vaccination period and up to study end' will be reported

204812 (RSV F-021) Statistical Analysis Plan Amendment 2 Final

| 1 | Statistical Analysis Plan Amendment 2 Final | |
|---|---|---|
| | <ul> <li>In the analysis of medically attended RTIs, analysis on 'viral load assessed by the quantitative PCR (RSV-A/B) of RSV-RTI cases' will be only listed in the individual listings</li> <li>In the analysis of immunogenicity section, tables/figures related to the analysis of RSV-B will be added</li> <li>In the analysis of immunogenicity section, tables/figures related to the analysis of the IgG total and IgG1 subclass will be added</li> <li>In the analysis of immunogenicity section, tables/figures related to the analysis of anti-RSV A and anti-PCA in the subset of subjects with IgG/IgG1 data available will be added</li> </ul> | |
| 09-NOV-2017 | Amendment 2: Description of changes from Amendment 1 are as below: - PPD (Clinical Research and Development Lead) was added - In the analysis of immunogenicity section, the analysis on GM ratios between anti-RSV F antibody concentrations (IgG Total) and anti-RSV-A neutralising antibody titers at pre-vaccination has been added - In the analysis of immunogenicity section, the analysis on GM ratios of fold increase post/pre (Day 30/Day 0) between anti-RSV F antibody concentrations (IgG Total) and anti-RSV-A neutralising antibody titers has been added - Changes of TFL/TOC • In the analysis of safety section, analysis on 'Individual results of hemoglobin levels beyond grade 2' have been added • In the analysis of safety section, analysis on 'Individual results of white blood cells counts levels lower than LL' and the figures of 'Individual results of white blood cells counts levels higher than UL' have been added | RSV F-021 (204812) Protocol Amendment 1 (21-Aug-2017) |

204812 (RSV F-021)

Statistical Analysis Plan Amendment 2 Final

- In the analysis of immunogenicity section, one new template of "Comparisons of GM ratios with corresponding 95% confidence interval between anti-RSV F antibody concentrations (IgG Total) and anti-RSV-A neutralising antibody titers at prevaccination (Per protocol set) "has been added"
- In the analysis of immunogenicity section, one new template of "Exploratory comparisons (GM ratios of fold increase post/pre) with corresponding 95% confidence interval between anti-RSV F antibody concentrations (IgG Total) and anti-RSV-A neutralising antibody titers at Day 30 (Per protocol set)" has been added

#### 2. STUDY DESIGN

#### Figure 1. Study design overview



- V = Visit; D = Day; VACC = vaccination; BS = blood sample; h/b = blood sample for haematology/biochemistry; lmm = blood sample for immunogenicity; C = contact; RSV = Respiratory Syncytial Virus; PCR = Polymerase Chain Reaction.
- 1 Safety data up to (minimum) 7 days post-vaccination (including Day 7 haematology and biochemistry parameters) of the first 25% of subjects vaccinated in the study will be reviewed by iSRC.
- 2 In case of a MA-RTI (e.g. visit to the GP for respiratory symptoms including but not limited to cough, sputum production, difficulty breathing), the subject will be asked to contact the Investigator to enable completion of an event related eCRF and the collection of a nasal swab within 72h after the medical attendance.

Vertical lines stand for analysis on all subjects.

- **Experimental design**: Phase II, observer-blind, randomised, controlled, multi-country, study with four parallel groups.
  - O **Duration of the study**: the intended duration of the study will be approximately 1 year from Visit 1 to study conclusion (Day 360).
  - o Epoch 001: Primary starting at Visit 1 (Day 0) and ending at Visit 5 (Day 90).
  - Epoch 002: Follow-up phase starting one day after Day 90 and ending at Day 360 contact.
- **Primary Completion Date (PCD)**: Visit 3 (Day 30).
- End of Study (EoS): Last testing results released of samples collected at Visit 5 (i.e. last testing results released for the assays related to the primary and secondary endpoints).
- Study groups:

Statistical Analysis Plan Amendment 2 Final

Table 1 Study groups and epochs foreseen in the study

| Ctudy groups | Number of subjects | Epo | Lumber of subjects Age (Min/Mex) Epochs | ochs |
|---|---|---|---|---|
| Study groups | Number of Subjects | Age (Min/Max) | Epoch 001 | Epoch 002 |
| 30 PreF | ~100 | 18 - 45 years | Х | Х |
| 60 PreF | ~100 | 18 - 45 years | Х | Х |
| 120 PreF | ~100 | 18 - 45 years | Х | Х |
| Control | ~100 | 18 - 45 years | Х | Х |

Table 2 Study groups and treatment foreseen in the study

| Trootmont nome | Vaccine/ Product name | Study Groups | | | |
|---|---|---|---|---|---|
| Treatment name | | 30 PreF | 60 PreF | 120 PreF | Control |
| 30 µg PreF | PreF-30 | Х | | | |
| | NaCl | | | | |
| 60 µg PreF | PreF-60 | | Х | | |
| | NaCl | | ^ | | |
| 120 μg PreF | PreF-120 | | | Х | |
| | NaCl | | | ^ | |
| Placebo | Formulation buffer S9b | | | | Х |

- Control: Placebo control
- Vaccination schedule: One intramuscular vaccination at Day 0.
- **Treatment allocation**: Subjects will be randomised using a centralised randomisation system on internet (SBIR) at Day 0. The randomisation algorithm will use a minimisation procedure accounting for age (18 32 years or 33 45 years) and centre.

The following group and sub-group names will be used for the statistical analyses:

| Group order in tables | Group label in tables | Group definition for footnote |
|---|---|---|
| 1 | 30 PreF | 30 µg PreF |
| 2 | 60 PreF | 60 µg PreF |
| 3 | 120 PreF | 120 μg PreF |
| 4 | Control | Placebo |

Some tables might be presented by age category according to the following description:

| Sub-group | Sub-group order in tables | Sub-group label in tables | Sub-group definition for footnote |
|---|---|---|---|
| Age | 1 | 18-32Y | 18-32 years old subjects |
| | 2 | 33-45Y | 33-45 years old subjects |

• **Blinding**: Observer-blind in Epoch 001 and single-blind in Epoch 002.

Table 3 Blinding of study epochs

| Study Epochs | Blinding |
|--------------|----------------|
| Epoch 001 | observer-blind |
| Epoch 002 | single-blind |

204812 (RSV F-021) Statistical Analysis Plan Amendment 2 Final

### • Sampling schedule:

- o **Blood samples for haematology/biochemistry** will be collected (~10 mL) from all subjects at Visit 1 (Day 0), Visit 2 (Day 7), Visit 3 (Day 30), Visit 4 (Day 60) and Visit 5 (Day 90).
- o **Blood samples for humoral immune response evaluation** will be collected (~17 mL) from all subjects at Visit 1 (Day 0), Visit 3 (Day 30), Visit 4 (Day 60) and at Visit 5 (Day 90).
- o **Nasal swabs** will be collected from subjects in case of a medically attended respiratory tract infection from enrolment (Visit 1) until study end (Contact 3).
- Type of study: self-contained
- **Data collection:** Electronic Case Report Form (eCRF).

#### • Safety monitoring:

- When the first 25% of subjects (i.e. ~100 subjects; ~25 subjects per study group) have been vaccinated, enrolment will be paused until completion of an unblinded review by a GSK internal Safety Review Committee (iSRC). Continuation of study enrolment will be conditional to a favourable outcome of the iSRC evaluation of all available safety and reactogenicity data collected up to at least 7 days post-vaccination (including Day 7 haematology and biochemistry parameters). In addition, the blinded safety data will be reviewed by GSK Biologicals' Safety Review Team (SRT) on a regular basis throughout the study. Analyses related to iSRC evaluation will be described in a separate document (SAP/TFL for iSRC).
- When all subjects have been vaccinated, IDMC will review all available safety and reactogenicity data (including haematology/ biochemistry parameters) of all enrolled subjects up to at least 30 days post administration of the study vaccine or placebo. The blinded safety data will be reviewed by the GSK Biologicals' SRT. Analyses related to IDMC evaluation will be described in a separate document (SAP/TFL for IDMC).
- In case of a MA-RTI (e.g. visit to the GP for respiratory symptoms including but not limited to cough, sputum production, difficulty breathing), the subject will be asked to contact the investigator to enable the collection of a nasal swab within 72 hours after the medical attendance.

#### 3. OBJECTIVES

# 3.1. Primary Objective

• To rank different formulations of the investigational RSV vaccine based on safety/reactogenicity and immunogenicity data up to 1 month post-vaccination (Day 30).

# 3.2. Secondary objectives

- To evaluate the reactogenicity and safety of a single intramuscular dose of the RSV investigational vaccines up to study conclusion.
- To evaluate the immunogenicity of a single intramuscular dose of the RSV investigational vaccines up to 90 days after vaccination (Day 90).
- To further assess the safety of the investigational RSV vaccines by evaluating whether a single dose of the vaccines induces antibodies against the residual host cell protein neogenin (NEO) up to 1 month post-vaccination (Day 30).
- To estimate the incidence of medically attended RSV-associated RTIs up to study conclusion.

# 3.3. Tertiary objective

• If deemed necessary, to further characterize the immune response of a single intramuscular dose of the RSV investigational vaccines.

Refer to Section 5.7.3 Laboratory assays of the Protocol for additional testing proposed to further characterize the immune response to the investigational RSV vaccine.

#### 4. ENDPOINTS

# 4.1. Primary

- Occurrence of AEs from vaccination up to Day 7, for all subjects in each investigational RSV vaccine group:
  - o Occurrence of any Grade 2 and Grade 3 general AE (solicited and unsolicited);
  - o Occurrence of Grade 2 and Grade 3 fever;
  - Occurrence of any vaccine-related SAE.
- Functional antibody titres against RSV at Day 0 and Day 30, for all subjects in each investigational RSV vaccine group.
  - Neutralising antibody titres against RSV-A
- PCA concentrations at Day 0 and Day 30 for all subjects in each investigational RSV vaccine group

# 4.2. Secondary

- Occurrence of AEs from vaccination up to study conclusion:
  - Occurrence of each solicited local and general AE, during a 7-day follow-up period after vaccination (i.e. the day of vaccination and 6 subsequent days), for all subjects in all groups;
  - Occurrence of any unsolicited AE, during a 30-day follow-up period after vaccination (i.e. the day of vaccination and 29 subsequent days), for all subjects in all groups;
  - Occurrence of any haematological (haemoglobin level, White Blood Cells [WBC], lymphocyte, neutrophil, eosinophil and platelet count) and biochemical (alanine amino-transferase [ALT], aspartate amino-transferase [AST] and creatinine) laboratory abnormality at Day 0, Day 7, Day 30, Day 60 and Day 90 for all subjects in all groups;
  - Occurrence of any SAE, for all subjects in all groups.
- Functional antibody titres against RSV for all subjects in all groups:
  - Neutralising antibody titres against RSV-A at Day 0, Day 30, Day 60 and Day 90;
  - Neutralising antibody titres against RSV-B at Day 0, Day 30, Day 60 and Day 90.
- PCA concentration at Day 0, Day 30, Day 60 and Day 90 for all subjects in all groups.
- Humoral immune response to the residual host cell protein NEO in the investigational RSV vaccine at pre-vaccination (Day 0), and 1 month post-vaccination (Day 30) for all subjects in all groups.
  - Antibody concentrations against NEO
- Occurrence of medically attended RSV-associated RTIs up to study conclusion

# 4.3. Tertiary

See section 5.7.3 of the Protocol for additional testing proposed to further characterize the immune response to the investigational RSV vaccine.

### 5. ANALYSIS SETS

#### 5.1. Definition

In order to align to ICH and CDISC terminology, the Total Vaccinated Cohort (TVC) and the According To Protocol cohort (ATP) have been renamed Exposed Set (ES) and Per-Protocol Set (PPS) respectively. Two cohorts will be defined for the purpose of the analysis: the Exposed Set (ES) and the Per-Protocol Set (PPS) for analysis of immunogenicity. All analyses will be performed per treatment actually administered.

Statistical Analysis Plan Amendment 2 Final

## 5.1.1. Exposed Set (ES)

The ES will include all subjects with study vaccine administration documented:

- A **safety** analysis based on the ES will include all vaccinated subjects
- An **immunogenicity** analysis based on the ES will include all vaccinated subjects for whom immunogenicity data are available.

### 5.1.2. Per-Protocol Set (PPS) for analysis of immunogenicity

The PPS for immunogenicity will be defined by time point and will include all vaccinated subjects.

- Meeting all eligibility criteria (i.e. no protocol violation linked to the inclusion/exclusion criteria, including age).
- Who received the study vaccine according to protocol procedures.
- Who did not receive a concomitant vaccination/medication/product leading to exclusion from the PPS analysis up to the corresponding timepoint as described in Section 6.6.2 of the Protocol.
- Who did not present with an intercurrent medical condition leading to exclusion from the PPS analysis up to the corresponding timepoint, as described in Section 6.7 of the Protocol.
- Who complied with the post-vaccination blood sampling schedule at the corresponding timepoint, as specified in Table 5 of the Protocol.
- For whom post-vaccination immunogenicity results are available for at least 1 assay at the corresponding timepoint.

When presenting different timepoints, the PPS for immunogenicity will be adapted for each timepoint (up to D30 and up to D90).

# 5.2. Criteria for eliminating data from Analysis Sets

Elimination codes are used to identify subjects to be eliminated from analysis. Detail is provided below for each sets.

## 5.2.1. Elimination from Exposed Set (ES)

Code 1030 (Study vaccine not administered at all) and code 900 (invalid informed consent or fraud data) will be used for identifying subjects eliminated from ES.

#### 5.2.2. Elimination from Per-protocol analysis Set (PPS)

#### 5.2.2.1. **Excluded subjects**

A subject will be excluded from the PPS analysis under the following conditions.

| | | Applicable Eli Type | |
|---|---|---|---|
| Code | Condition under which the code is used | 'M1' (Applicable<br>up to Visit 3 - Day<br>30) | 'M2' (Applicable<br>up to Visit 5 - Day<br>90) |
| 900 | Invalid informed consent or fraud data (Subjects receiving a code 900 should not receive any other elimination codes) | Applicable | Applicable |
| 1030 | Study vaccine not<br>administered at all<br>(Subjects receiving a code<br>1030 should not receive any<br>other elimination codes) | Applicable | Applicable |
| 1040* | Administration of concomitant vaccine(s) forbidden in the protocol | Applicable<br>(To check up to<br>Visit 3 – Day 30) | Applicable<br>(To check up to<br>Visit 5 – Day 90) |
| 1050 | Randomization failure<br>(subject not randomized<br>in the correct group) | Applicable | Applicable |
| 1060 | Randomization code was broken | Applicable | Applicable |
| 1070** | Subjects got vaccinated with the correct vaccine but containing a lower volume | Applicable | Applicable |
| 1070** | Administration not according to protocol for reason specified by the investigator other than site and route | Applicable | Applicable |
| 1070** | Site or route of study vaccine administration wrong or unknown | Applicable | Applicable |
| 1070** | Wrong or annown Wrong replacement or study vaccine administered (not compatible with the vaccine regimen associated to the treatment number) | Applicable | Applicable |

# 204812 (RSV F-021) Statistical Analysis Plan Amendment 2 Final

| | | Statistical An | alysis Plan Amendme |
|---|---|---|---|
| 1070** | Administered study vaccine reported as being the correct one but is not compatible with the vaccine regimen associated to the treatment number | Applicable | Applicable |
| 1080 | Vaccine temperature deviation | Applicable | Applicable |
| 1090 | Expired vaccine administered | Applicable | Applicable |
| 2010 | Protocol violation<br>(inclusion/exclusion<br>criteria) | Applicable DOB-VAC=18-45 years | Applicable DOB-VAC=18-45 years |
| 2040* | Administration of any medication forbidden by the protocol | Applicable<br>(To check up to<br>Visit 3 – Day 30) | Applicable<br>(To check up to<br>Visit 5 – Day 90) |
| 2050* | Underlying medical condition forbidden by the protocol | Applicable (To check up to Visit 3 – Day 30) | Applicable (To check up to Visit 5 – Day 90) |
| 2060* | Concomitant infection related to the vaccine which may influence the immune response | Applicable<br>(To check up to<br>Visit 3 – Day 30) | Applicable<br>(To check up to<br>Visit 5 – Day 90) |
| 2070* | Concomitant infection not related to the vaccine which may influence the immune response | Applicable<br>(To check up to<br>Visit 3 – Day 30) | Applicable<br>(To check up to<br>Visit 5 – Day 90) |
| 2090 | Subjects did not comply<br>with blood sample<br>schedule | Applicable VAC_1 to SER_2 = 30-44 (days) | Applicable VAC_1 to SER_3 = 56-70 (days) VAC_1 to SER_4 = 86-100 (days) |
| 2100 | Serological results not available post-vaccination | All assay for Day 30 elimination code if ALL are missing v_ID for Neutra RSV-A=3240.001 | All assay for Day60 and Day90 elimination code if ALL are missing v_ID for Neutra RSV-A=3240,001 |
| | | v_ID for Neutra<br>RSV-B=3240.002<br>v_ID for Neutra | v_ID for Neutra RSV-B=3240.002 v ID for Neutra |

204812 (RSV F-021)

Statistical Analysis Plan Amendment 2 Final

| | | PCA=3241.009 | PCA=3241.009 |
|---|---|---|---|
| | | v_ID for IgG<br>total=3241.002 | v_ID for IgG<br>total=3241.002 |
| | | v_ID for IgG<br>I=3241.005 | v_ID for IgG<br>I=3241.005 |
| 2120* | Obvious incoherence or abnormality or error in data*** | All assay for Day<br>30 | All assay for Day<br>60 and Day90 |

<sup>\*</sup> Attribution of these elimcodes to subject need CRDL review of individual data listings

Eli type is Internal GSK database code for type of elimination code M1 for Visit 3 (Day30) analysis; M2 for Visit 5 (Day 90) analysis;

#### 5.2.2.2. Right censored Data

Not applicable

#### 5.2.2.3. Visit-specific censored Data

Not applicable

# 5.3. Important protocol deviation not leading to elimination from per-protocol analysis set

The following important protocol deviations will be reported by groups:

Forced randomization: In case of supplies shortage for the next assigned vaccine according to the randomization schedule at the clinical site, the randomization system will use the forced randomization procedure in order to continue to enrol and vaccinate subjects. The system moves seamlessly to the next treatment/randomization number for which vaccine supplies are available. The site will not be aware of the forced randomization event

Manual randomization: In case of the randomization system is unavailable, the investigator has the option to perform randomization by selecting supplies available at the site according to a pre-defined rule.

Short follow-up: subjects who completed the last study contact before the minimum length of follow-up requirement.

# 6. STATISTICAL ANALYSES

Note that standard data derivation rule and stat methods are described in Annex 1 and will not be repeated below.

<sup>\*\*</sup> Attribution of code 1070 to a subject requires CRDL confirmation

<sup>\*\*\*</sup> Elimination criteria for implausible RSV serum immune responses (neut and/or ELISA): More than 4 fold decrease from pre-vaccination to Day 30; After Day 30, more than 4 fold increase or more than 8 fold decrease within a 30 day period

# 6.1. Demography

# 6.1.1. Analysis of demographics/baseline characteristics planned in the protocol

The analysis of demography will be performed on the ES and on the PPS for immunogenicity.

Demographic characteristics such as age at vaccination in years, race, ethnicity, vital signs and cohort description will be summarised by group using descriptive statistics:

- Frequency tables will be generated for categorical variable such as race.
- Mean, median, standard error and range will be provided for continuous data such as age.

The distribution of subjects will be tabulated as a whole and per group and for each age category (18 - 32 years and 33 - 45 years).

Withdrawal status will be summarised by group using descriptive statistics:

- The number of subjects enrolled into the study as well as the number of subjects excluded from PPS analyses will be tabulated.
- The number of withdrawn subjects will be tabulated according to the reason for withdrawal.

# 6.2. Immunogenicity

# 6.2.1. Analysis of immunogenicity planned in the protocol

The analysis will be performed on the applicable PPS cohort for immunogenicity and, if in any group the percentage of vaccinated subjects with serological results excluded from the PPS for analysis of immunogenicity is  $\geq 5\%$ , a second analysis will be performed on the ES.

#### 6.2.1.1. Within group analysis

Humoral Immune response to RSV vaccine

For each group, at each timepoint that blood samples are collected and for each assay (unless specified otherwise):

204812 (RSV F-021)

Statistical Analysis Plan Amendment 2 Final

- GMTs/GMCs will be tabulated with 95% CI based on log-transformed values and represented graphically.
- Percentage of subjects above the seropositivity threshold will be tabulated with exact 95% CI.
  - Percentage of subjects above the seropositivity threshold and GMTs/GMCs will also be tabulated by group for each age category (18 32 years and 33 45 years).
- Pre- and post-vaccination antibody titres/concentrations will be displayed using reverse cumulative curves.
- The distributions of **neutralising** antibody titres will be tabulated in the tables with log2 scale (< 7, 7-8, > 8-9, > 9-10, > 10-11, > 11-12, > 12 log2).
- Percentage of responders in terms of **neutralising** antibody titres will be tabulated with exact 95% CI.
- Individual post-vaccination *versus* pre-vaccination results will be plotted using scatter plots. Results of the control group will be used as a reference.
- Geometric mean of ratios of antibody titres/concentrations at each post-vaccination timepoint over pre-vaccination will be tabulated with 95% CI.
- Distribution of the fold increase of the antibody titres/concentrations will be tabulated:
  - o For neutralising antibody titres against RSV-A and RSV-B: percentage of subjects with a fold increase equal to or above 1, 2, 2.5, 3, 4, 6, 8 10, 11 and 12 by pre-vaccination titre category: <7, 7-8, ]8-9, ]9-10, ]10-11, ]11-12, >12 log2, and cumulative: <7, ≥7, ≥8, ≥9, ≥10, ≥11, ≥12 log2.
  - For antibody concentrations against NEO: percentage of subjects with a fold increase equal to or above 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5 and 5.
- The kinetics of individual antibody titres/concentrations will be plotted as a function of time for subjects with results available at all timepoints.
- An analysis of variance model for repeated measures will be fitted to calculate GMTs/GMCs with treatment group, visit and their interaction as fixed effects if necessary.

If deemed necessary, the same analyses may be done by age category (18 - 32 years and 33 - 45 years).

### 6.2.1.2. Between group assessment

Exploratory comparisons will be performed for RSV neutralising antibody titres and PCA concentrations post-vaccination (Day 30, Day 60 and Day 90) between the different RSV vaccine groups.

204812 (RSV F-021)

Statistical Analysis Plan Amendment 2 Final

- Estimation of GMT/GMC ratios between groups with corresponding 95% CI using an ANCOVA model on the logarithm10 transformation of the titres/concentrations. If a statistically significant difference is found (p <0.05), pairwise comparisons will be made using Tukey's multiple comparison adjustment. This model includes:
  - The vaccine group as the fixed effect
  - The pre-vaccination titre/concentration as the covariate
  - Age groups (18-32 years and 33-45 years) and center as the categorical covariate if deemed necessary
- GMT/GMC ratios with corresponding 95% CI will be computed between the RSV vaccine groups
  - o PreF-120 minus PreF-30
  - PreF-120 minus PreF-60
  - o PreF-60 minus PreF-30

#### 6.2.2. Additional considerations

In order to add the analysis of the <u>anti-RSV F IgG Total and IgG1 subclass</u> tested at Day 0 and Day 30 in a random subset of 50 subjects per group. The following analysis will be performed on the ATP cohort for immunogenicity analysis for each group and for both assays:

- GMCs with 95% CI will be tabulated.
- Percentage of subjects above the seropositivity threshold will be tabulated with exact 95% CI.
- Geometric mean of ratios of antibody concentrations at each post-vaccination timepoint over pre-vaccination (fold increase) will be tabulated with 95% CI, and represented graphically.
- Individual ratios of antibody concentrations will be displayed using reverse cumulative curves.
- Exploratory comparisons between groups: geometric mean ratios and 95% CIs of fold increase post/pre between the RSV groups:
  - o 120 PreF versus 60 PreF
  - o 120 PreF versus 30 PreF
  - o 60 PreF versus 30 PreF

This will be performed using an ANOVA model on the logarithm 10 transformation of the concentrations including the vaccine group as covariates. If a statistically significant difference is found (p < 0.05), pairwise comparisons will be made using Tukey's multiple comparison adjustment.

In addition, the following immunogenicity analysis will be performed in the subset of subjects with IgG/IgG1data available:

Statistical Analysis Plan Amendment 2 Final

- GMCs will be tabulated with 95% CI for anti-RSV A and anti-PCA
- Percentage of subjects above the seropositivity threshold will be tabulated with exact 95% CI for anti-RSV A and anti-PCA.

# 6.3. Analysis of safety

## 6.3.1. Analysis of safety planned in the protocol

The analysis of safety will be performed on the ES.

#### 6.3.1.1. Within group analysis

The percentage of subjects with at least one **local AE** (solicited and unsolicited), with at least one **general AE** (solicited and unsolicited) and with any AE during the 7-day or 30-day follow-up period after vaccination will be tabulated with exact 95% CI. The same computations will be done for ≥ Grade 2 and Grade 3 AEs, for any AEs considered related to vaccination, for any Grade 3 AEs considered related to vaccination and for AEs resulting in medically attended visit.

The percentage of subjects reporting each individual **solicited local AE** (any grade,  $\geq$  Grade 2, Grade 3, resulting in medically attended visit) during the 7-day follow-up period after vaccination will be tabulated for each study vaccine for each group. The percentage of subjects reporting each individual **solicited general AE** (any grade,  $\geq$  Grade 2, Grade 3, any related,  $\geq$  Grade 2 related, Grade 3 related, resulting in medically attended visit) during the 7-day follow-up period after vaccination will be tabulated for each group.

For fever during the 7-day follow-up period after vaccination, the number and percentage of subjects reporting fever will be reported by half degree (°C) cumulative increments. Similar tabulations will be performed for causally related fever, Grade 3 (> 39.5°C) causally related fever and fever resulting in a medically attended visit. In addition, the prevalence of any and Grade 3 fever will be presented graphically over time after vaccination.

The percentage of subjects with any **unsolicited** symptoms within 30 days after vaccination with its exact 95% CI will be tabulated by group and by Medical Dictionary for Regulatory Activities (MedDRA) preferred term. Similar tabulation will be done for Grade 3 unsolicited symptoms, for any causally related unsolicited symptoms, for Grade 3 causally related unsolicited symptoms and for unsolicited symptoms resulting in a medically attended visit (The verbatim reports of unsolicited symptoms will be reviewed by a physician and the signs and symptoms will be coded according to the MedDRA Dictionary for Adverse Reaction Terminology. Every verbatim term will be matched with the appropriate Preferred Term).

**SAEs** reported throughout the study will be described in detail.

**Pregnancy** exposures throughout the study and pregnancy outcomes will be described in detail (if applicable).

204812 (RSV F-021)

Statistical Analysis Plan Amendment 2 Final

The percentage of subjects using **concomitant medication** (any medication, any antipyretic and any antipyretic taken prophylactically) during the 7-day (Day 0 to Day 6) or 30-day (Day 0 to Day 29) follow-up period after vaccination will be summarised by group.

For all subjects in each group and each **haematology and biochemistry** parameter:

- The percentage of subjects having haematology and biochemistry results below or above the local laboratory normal ranges will be tabulated for each timepoint.
- The maximum grading post-vaccination (from Day 7 to Day 90) versus baseline (Day 0) and the percentage of subjects with laboratory parameters above or equal to Grade 1, Grade 2, Grade 3 and Grade 4 will be tabulated (Grades will be based on the FDA Guidance for Industry "Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials", see APPENDIX D of the Protocol: FDA toxicity grading scale. Those laboratory parameters not included on FDA Toxicity Grading Scale will not be graded).

Assessment of anti-NEO immune response at Day 30 post-vaccination for each group:

- GMCs pre-and post-vaccination will be tabulated with 95% CI and represented graphically.
- Individual post-vaccination *versus* pre-vaccination results will be plotted using scatter plots. Results of the control group will be used as a reference.
- Geometric mean of ratios of antibody concentrations at Day 30 over pre-vaccination will be tabulated with 95% CI.
- Distribution of the antibody concentrations pre-and post-vaccination and of fold increase after vaccination will be tabulated.

#### 6.3.1.2. Between group assessment

Exploratory comparisons between each investigational RSV vaccine group and (minus) the control group (*placebo*), and between the RSV vaccine groups will be done in terms of the percentage of subjects reporting any  $\geq$  Grade 2, Grade 3 AE (solicited and unsolicited), and/or any fever > 38.5°C, and/or any vaccine-related SAE during the 7-day follow-up period after vaccination.

- o PreF-30 minus placebo
- o PreF-60 minus placebo
- o PreF-120 minus placebo
- o PreF-120 minus PreF-30
- o PreF-120 minus PreF-60
- o PreF-60 minus PreF-30

204812 (RSV F-021)

Statistical Analysis Plan Amendment 2 Final

The standardised asymptotic 95% CI for the difference between the investigational RSV vaccine groups as well as between the investigational RSV groups and (minus) the control group will be computed.

# 6.4. Analysis for ranking RSV formulations

The totality of data and sum total of evidence for particular dose(s) in terms of safety and immunogenicity will be evaluated by study team in addition to the analyses described in section 6.1 and 6.3 on formulation selection. The desirability index approach described in the section below will be used as a descriptive tool to guide the formulation selection. In addition, any pertinent information from outside this study will be evaluated and may be used by the study team to help to make the final decision on a dose/formulation.

## 6.4.1. Definition of desirability in the context of Simulations

A desirability approach will be based on safety/reactogenicity and immunogenicity data up to 1 month post-vaccination.

This method is a multi-criteria decision making approach based on desirability functions. The main idea is to identify for each endpoint a desirability function that associates any value to another one between 0 and 1 depending on its desirability ('0' being considered as not desirable at all and '1' as the most desirable). An index with values between 0 and 1 will be created for each endpoint. An overall desirability index can be calculated by computing a weighted geometric mean of the endpoint indexes. By definition, this overall index also takes values between 0 and 1 and characterises the level of desirability of any candidate formulation by a single value [Dewé, 2015].

The desirability index calculations will include reactogenicity and safety data up to Day7 post vaccination (on the TVC) and immunogenicity data at 30 days post-vaccination (on the ATP cohort for immunogenicity up to Day 30). The formulations will be ranked based on the values obtained with this overall desirability index.

#### 6.4.2. Derived endpoints

The following endpoints will be computed and taken into account in the desirability analysis:

- 1. Incidence rate of any Grade 2 and any Grade 3 general AE (solicited and unsolicited) and any vaccine-related SAE during the 7-day follow-up period after vaccination for each investigational RSV vaccine formulation.
- 2. Incidence rate of Grade 2 and Grade 3 fever during the 7-day follow-up periodafter vaccination for each investigational RSV vaccine formulation.
- 3. Geometric mean of neutralising antibody titres against RSV-A at Day 30 adjusted for pre-vaccination titres.
- 4. Geometric mean of PCA concentrations at Day 30 adjusted for pre-vaccination titres.

204812 (RSV F-021)

Statistical Analysis Plan Amendment 2 Final

Each individual desirability index will be calculated based on data and tabulated by the treatment group and endpoints above. The details on how to calculate individual desirability index in terms of reactogenicity and immunogenicity and overall desirability index are elaborated in Annex 2.

# 6.5. Analysis of medically attended RTIs

The analysis will be performed on the ES by study group.

The proportion of subjects with at least one medically attended RSV-associated RTI (with 95 % CI) will be calculated.

Viral load assessed by the quantitative PCR (RSV-A/B) of RSV-RTI cases will be listed for any cases where this assay is performed.

Medically attended RSV-associated RTI co-infected or colonisation with another viral etiology identified by multiplex PCR will be described.

Medically attended RTI with any viral etiology identified by multiplex PCR will be described.

The proportion of subjects (with 95% CI) with at least one medically attended RTI (all causes) will be calculated by group.

#### 7. ANALYSIS INTERPRETATION

All comparative analyses will be descriptive with the aim to characterise the difference in reactogenicity/immunogenicity between groups. These descriptive analyses should be interpreted with caution considering that there is no adjustment for multiplicity for these comparisons.

#### 8. CONDUCT OF ANALYSES

Any deviation(s) or change(s) from the original statistical plan outlined in this protocol will be described and justified in the final study report.

# 8.1. Sequence of analyses

The statistical analyses will be performed in several steps:

- In preparation of the planned iSRC evaluation, analysis of safety and reactogenicity data up to at least 7 days post-vaccination of the first 25% of all subjects will be performed (see Section 8.10.2 of the Protocol for more information).
- In preparation of the planned IDMC evaluation, analysis of safety and reactogenicity data (including haematology/biochemistry parameters) up to at least 30 days post-vaccination of all enrolled subjects will be performed.

204812 (RSV F-021)

Statistical Analysis Plan Amendment 2 Final

- The first main analysis on all subjects will be performed when all data up to 30 days post-vaccination are available (primary endpoints). In order to maintain the blind, this analysis by group will be performed by an independent statistician and the results which would lead to the unblinding of some subjects (e.g. a specific AE reported by one subject only) will be blinded (i.e. the group in which this event occurred will not be identified). No individual data listings will be provided.
- A second analysis will be performed when all data up to 90 days post-vaccination are available (secondary endpoints). At this point, the GSK statistician will be unblinded (i.e. will have access to the individual subject treatment assignments), but no individual listings will be provided. Given that summary results may unblind some specific subjects, the study will be conducted in a single-blind manner from this point onwards, with subjects remaining blinded up to study conclusion and the investigators will not have access to the treatment allocation up to study conclusion.
- The final analysis will be performed when all data up to study conclusion are available. All available tertiary endpoints will also be analysed in this step. Individual listings will only be provided at this stage.
- An integrated study report presenting all analyses will be written and made available to the investigators at the time of final analysis.
- If data for tertiary endpoints become available at a later stage, (an) additional analysis/analyses will be performed. These data will be documented in Annex(es) to the study report and will be made available to the investigators at that time.

| Description | Analysis ID | Disclosure Purpose<br>(CTRS=web posting,<br>SR=study report,<br>internal) | Dry run review<br>needed (Y/N) | Study Headline Summary (SHS)requiring expedited communication to upper management (Yes/No) | Reference for TFL |
|---|---|---|---|---|---|
| Final Analysis | E1_01 | Study report<br>CTRS | N | Yes | All tables from<br>TFL dated<br>13NOV2017 |
| Analysis of<br>Day 30 | E1_04 | Internal<br>CTRS | N | Yes | All tables from<br>TFL dated<br>13NOV2017 |
| Analysis of<br>Day 90 | E1_05 | Internal<br>CTRS | N | Yes | All tables from<br>TFL dated<br>13NOV2017 |

# 8.2. Statistical considerations for interim analyses

No interim analysis will be performed.

#### 9. CHANGES FROM PLANNED ANALYSES

In order to align to ICH and CDISC terminology the Total Vaccinated Cohort and the According To Protocol cohort have been renamed Exposed Set (ES) and Per-Protocol Set (PPS) respectively.

#### Changes in Amendment 1 mainly include the following.

For the sequence of analysis, the IDMC evaluation was newly added to review all available safety and reactogenicity data (including Day 30 haematology and biochemistry parameters) of all enrolled subjects up to at least 30 days post administration of the study vaccine or placebo.

Since the document of criteria for eliminating subjects from analysis will not be used anymore, the table of Elimination codes has been modified for more clarity. Attribution of code 1070 to a subject requires CRDL confirmation. Attribution of these elimcodes including 1040, 2040, 2050, 2060, 2070 and 2120 to subject need CRDL review of individual data listings.

In the analysis of immunogenicity section, the distribution of fold increase of the antibody titres against RSV-A and RSV-B and concentrations against NEO have been added.

For the analysis of safety, the percentage of subjects reporting each individual solicited local AE (any, each grade, resulting in medically attended visit) during the 7-day follow-up period after vaccination will also be tabulated based on maximum intensity per subject for each study vaccine group; the percentage of subjects reporting each individual solicited general AE (any, each grade, any related, any Grade 2 related, any Grade 3 related, resulting in medically attended visit) during the 7-day follow-up period after vaccination will also be based on maximum intensity per subject for each study vaccine group.

Evaluation of last secondary objective 'To estimate the incidence of medically attended RSV-associated RTIs up to study conclusion' will be performed based on MA-RTIs rather than MA-RSV associated RTIs.

The cut-off for the updated (qualified) version of the PCA assay will be set at the level of the assay LLOQ (9.60 µg/mL). Hence the SAP does not need to define handling of data between the LOD and LLOQ anymore, as results will only be provided as of the LLOQ. It only needs to be defined that for results below the cut-off (LLOQ), an arbitrary value of half of the cut-off will be considered for calculation of GMC and fold increase.

Algorithm for handling of data of RSV-B neutralising antibody tires between the LOB and LLOQ is defined as similar as for RSV-A by considering the LOB for RSV-B is 6.

Additional analysis of the IgG total and IgG1 subclass and analysis of anti-RSV A and anti-PCA in the subset of subjects with IgG/IgG1 data have been added.

204812 (RSV F-021)

Statistical Analysis Plan Amendment 2 Final

#### Changes of TFL/TOC

- In the analysis of safety section, figures of 'Individuals results of haematological (haemoglobin level, white blood cells and platelet count) and biochemical (ALT, AST and creatinine) parameters outside of the normal ranges in each group' has been added to replace the figures of 'Mean profile of haematological and biochemical parameters change from baseline (Day 0)';
- In the analysis of safety section, the titles in all tables reporting 'Incidence and nature of symptoms (solicited and unsolicited) during the 7-day and 30-day post-vaccination period' have been changed from 'with causal relationship to' to 'considered related to vaccination';
- In the analysis of safety section, analysis on 'Incidence of solicited local/general symptoms reported during the 7-day post-vaccination period' will be summarized based on maximum intensity for each grade per subject for each group; therefore, analysis on 'incidence of solicited local/general symptoms reported during the 7-day post-vaccination period, including >=grade 2 category' will not be generated.
- In the analysis of safety section, analysis on 'Number (%) of subjects reporting the occurrence of adverse events within the 7-day and 30-day post-vaccination period' will be added.
- In the analysis of safety section, analysis on 'Number (%) of subjects with serious adverse events during the study period including number of events reported' and 'Number (%) of subjects with serious adverse events considered related to vaccination during the study period including number of events reported' by %UNSOL (EVENT=1) will not be reported because %CTR\_SAE macro has been adapted to generate SAE, related SAE, fatal SAE and related fatal SAE.
- In the analysis of safety section, analysis on 'Number and percentage of subjects reporting the occurrence of medically attended respiration tract infections (MA-RTIs), during the 30-day, 60-day or 90-day post-vaccination period and up to study end' will be reported; Therefore, 'Number and percentage of subjects reporting one medically attended RSV-associated RTI and medically attended RTI (all causes) within the 30-day post-vaccination period or throughout the study period' will not be generated;
- In the analysis of medically attended RTIs, viral load assessed by the quantitative PCR (RSV-A/B) of RSV-RTI cases will be only listed in the individual listings; therefore, analysis on 'Descriptive statistics of the viral load assessed by the quantitative PCR (RSV-A/B) of RSV-RTI cases (All vaccinated subjects)' will not be reported;
- In the analysis of immunogenicity section, tables/figures related to the analysis of RSV-B will be added;
- In the analysis of immunogenicity section, tables/figures related to the analysis of the IgG total and IgG1 subclass will be added;
- In the analysis of immunogenicity section, tables related to the analysis of anti-RSV A and anti-PCA in the subset of subjects with IgG/IgG1 data available will be added.

#### Changes in Amendment 2 mainly include the following.

- In the analysis of immunogenicity section, the analysis on GM ratios between anti-RSV F antibody concentrations (IgG Total) and anti-RSV-A neutralising antibody titers at pre-vaccination has been added for Day 90 and final analysis;
- In the analysis of immunogenicity section, the analysis on GM ratios of fold increase post/pre (Day 30/Day 0) between anti-RSV F antibody concentrations (IgG Total) and anti-RSV-A neutralising antibody titers has been added for Day 90 and final analysis.

# Changes of TFL/TOC

- In the analysis of safety section, figures of "Individual results of hemoglobin levels beyond grade 2" will be reported for Day 90 and final analysis to replace the figures of "Individual results of hemoglobin levels outside of normal range";
- In the analysis of safety section, figures of "Individual results of white blood cells counts levels lower than LL" and figures of "Individual results of white blood cells counts levels higher than UL" will be reported for Day 90 and final analysis to replace the figures of "Individual results of white blood cells counts levels outside of normal range".
- In the analysis of immunogenicity section, one new template (Template 50) for "Comparisons of GM ratios with corresponding 95% confidence interval between anti-RSV F antibody concentrations (IgG Total) and anti-RSV-A neutralising antibody titers at pre-vaccination (Per protocol set)" has been added for Day 90 and final analysis;
- In the analysis of immunogenicity section, one new template (Template 51) for "Exploratory comparisons (GM ratios of fold increase post/pre) with corresponding 95% confidence interval between anti-RSV F antibody concentrations (IgG Total) and anti-RSV-A neutralising antibody titers at Day 30 (Per protocol set)" has been added for Day 90 and final analysis;

# 10. LIST OF FINAL REPORT TABLES, LISTINGS AND FIGURES

The TFL TOC provides the list of tables/listings and figures needed for the study report. It also identifies the tables eligible for each analyses and their role (synopsis, in-text, post-text, SHS, CTRS,...).

# 11. ANNEX 1 STANDARD DATA DERIVATION RULE AND STATISTICAL METHODS

#### 11.1. Statistical Method References

The exact two-sided 95% CIs for a proportion within a group will be the Clopper-Pearson exact CI [Clopper CJ, Pearson ES. The use of confidence or fiducial limits illustrated in the case of binomial. *Biometrika*. 1934;26:404-413].
204812 (RSV F-021)

Statistical Analysis Plan Amendment 2 Final

The standardised asymptotic two-sided 95% CI for the group difference in proportions is based on the method described in the following paper:Robert G. Newcombe, interval estimation for the difference between independent proportions: comparison of eleven methods, *Statist Med.* 1998; 17, 873-890]. The standardised asymptotic method used is the method six.

Dewé W, Durand Ch, Marion S *et al*. A multi-criteria decision making approach to identify a vaccine formulation. *Journal of Biopharmaceutical Statistics*, 2015; epublication ahead of print: DOI: 10.1080/10543406.2015.1008517.

#### 11.2. Standard data derivation

#### 11.2.1. Date derivation

- SAS date derived from a character date: In case day is missing, 15 is used. In case day and month are missing, 30 June is used.
- Onset day for an event (ae, medication, vaccination, ...): The onset day is the number of days between the last study vaccination & the start date of the event. This is 0 for an event starting on the same day as a vaccination. See SAS date derived in case the start date of the event is incomplete.
- Duration: Duration of an event is expressed in days. It is the number of days between the start & the stop dates + 1. Therefore duration is 1 day for an event starting & ending on the same day.
- Association of an event to the primary epoch: An adverse event belongs to the primary epoch, if the onset date is before and excluding Visit 5 or the last contact date, whichever is coming first.

#### 11.2.2. Dose number

- The study dose number is defined in reference to the number of study visits at which vaccination occurred.
- Relative dose: the relative dose for an event (AE, medication, vaccination) is the most recent study dose given before an event. In case the event takes place on the day a study dose is given, the related dose will be that of the study dose, even if the event actually took place before vaccination. For instance, if an adverse event begins on the day of the study vaccination but prior to administration of the vaccine, it will be assigned to this dose.

#### 11.2.3. Demography

• Age: Age at the reference activity, computed as the number of units between the date of birth and the reference activity. Note that due to incomplete date, the derived age may be incorrect by 1 month when month is missing from the birthdate. This may lead to apparent inconsistency between the derived age and the eligibility criteria/the age category used for randomization.

204812 (RSV F-021)

Statistical Analysis Plan Amendment 2 Final

• Conversion of weight to kg

The following conversation rule is used:

- Weight in Kilogram = weight in Pounds / 2.2
- Weight in Kilogram = weight in ounces / 35.2

The result is rounded to 2 decimals.

The following conversion rule is used:

- o Weight in Kilogramm= weight in Pounds / 2.2
- Weight in Kilogramm = weight in oncs / 35.2

The result is rounded to 2 decimals.

• Conversion of height to cm

The following conversation rule is used:

- Height in Centimetres = Height in Feet \* 30.48
- Height in Centimetres = Height in Inch \*2.54

The result is rounded to the unit (ie no decimal).

- Height in Centimetres = Height in Feet \* 30.48
- Height in Centimetres = Height in Inch \* 2.54

The result is rounded to the unit (ie no decimal).

• Conversion of temperature to °C

The following conversation rule is used:

Temperature in °Celsius = ((Temperature in °Fahrenheit -32) \*5)/9

The following conversion rule is used:

o Temperature in °Celsius = ((Temperature in °Fahrenheit -32) \*5)/9

The result is rounded to 1 decimal.

#### 11.2.4. Immunogenicity

- For a given subject and given immunogenicity measurement, missing or non-evaluable measurements will not be replaced. Therefore, an analysis will exclude subjects with missing or non-evaluable measurements.
- A seronegative subject is a subject whose antibody titre/concentration is below the cut-off value of the assay. A seropositive subject is a subject whose antibody titre/concentration is greater than or equal to the cut-off value of the assay
- The Geometric Mean Concentrations/Titres (GMC/Ts) calculations are performed by taking the anti-log of the mean of the log titre transformations. Antibody titres below the cut-off of the assay will be given an arbitrary value of half the cut-off of the assay for the purpose of GMT calculation. The cut-off value is defined by the laboratory before the analysis and is described in the protocol.

204812 (RSV F-021)

Statistical Analysis Plan Amendment 2 Final

- In order to compute fold increase of antibody titres/concentrations (ratio) between post-vaccination and pre-vaccination titres/concentrations and for GMC/GMT calculation, antibody titres/concentrations below the assay cut-off will be given an arbitrary value of half the cut-off.
- The cut-off for the updated (qualified) version of the PCA assay will be set at the level of the assay LLOQ (9.60 µg/mL). For results below the cut-off (LLOQ), an arbitrary value of half of the cut-off will be considered for calculation of GMC and fold increase.
- Considering cut-offs or neutralising antibody against RSV-A and RSV-B are below the assays' LLOO, the following rules will be applied:

| Assay | Raw result | Derivation for<br>seropositivity status | Derivation for<br>GMT calculation | Derivation for fold-increase<br>between Post and Pre-<br>vaccination titres |
|---|---|---|---|---|
| Neutra RSV-<br>A | <8 | NEG | 4 | LLOQ/2 |
| | [8-LLOQ[ | POS | 8 | LLOQ/2 |
| | ≥LLOQ | POS | Exact value | Exact value |
| Neutra RSV- | <6 | NEG | 3 | LLOQ/2 |
| В | [6-LLOQ[ | POS | 6 | LLOQ/2 |
| | ≥LLOQ | POS | Exact value | Exact value |

- Vaccine response to the RSV neutralising antibodies (anti-RSV-A and anti-RSV-B) will be defined as:
  - At least a 4-fold increase from pre-vaccination if pre-vaccination neutralising antibody titre <7 log2 (<128).
  - At least a 3-fold increase from pre-vaccination if pre-vaccination neutralising antibody titre in [7-8] log2 ([128-256]).
  - At least a 2.5-fold increase from pre-vaccination if pre-vaccination neutralising antibody titre in >8-10 log2 (>256-1024).
  - At least 1-fold from pre-vaccination if pre-vaccination neutralising antibody titre >10 log2 (>1024).
- All CI computed will be two-sided 95% CI.

#### 11.2.5. Safety

- For a given subject and the analysis of solicited symptoms within 7 days post-vaccination, missing or non-evaluable measurements will not be replaced. Therefore the analysis of the solicited symptoms based on the Total Vaccinated Cohort will include only vaccinated subjects for doses with documented safety data (i.e., symptom screen completed). More specifically the following rules will be used:
  - Subjects who documented the absence of a solicited symptom after one dose will be considered not having that symptom after that dose.

204812 (RSV F-021)

Statistical Analysis Plan Amendment 2 Final

- Subjects who documented the presence of a solicited symptom and fully or
  partially recorded daily measurement over the solicited period will be included in
  the summaries at that dose and classified according to their maximum observed
  daily recording over the solicited period.
- Subjects who documented the presence of a solicited symptom after one dose without having recorded any daily measurement will be assigned to the lowest intensity category at that dose (i.e., 37.5°C for fever or grade 1 for other symptoms).
- o Doses without symptom sheets documented will be excluded.
- For analysis of unsolicited adverse events, such as serious adverse events or adverse
  events by primary MedDRA term, and for the analysis of concomitant medications,
  all vaccinated subjects will be considered. Subjects who did not report the event or
  the concomitant medication will be considered as subjects without the event or the
  concomitant medication respectively.
- The preferred route for recording temperature in this study will be oral. For the analysis, temperatures will be coded as follows:

| Grade | Temperature for oral, axillary or tympanic route | Temperature for rectal route |
|---|---|---|
| 0 | < 37.5°C | < 38.0°C |
| 1 | ≥ 37.5°C - ≤ 38.5°C | ≥ 38.0°C - ≤ 39.0°C |
| 2 | > 38.5°C - ≤ 39.5°C | > 39.0°C - ≤ 40.0°C |
| 3 | > 39.5°C | > 40.0°C |

Note that for all tables described in this section, the way the percentage of subjects will be derived will depend on the event analysed (see table below for details). As a result, the N value will differ from one table to another.

| Event | N used for deriving % per subject for Vaccination phase |
|---|---|
| Concomitant vaccination | All subjects with study vaccine administered |
| Solicited general symptom | All subjects with at least one solicited general symptom documented as either present or absent (i.e., symptom screen completed) |
| Solicited local symptom | All subjects with at least one solicited local symptom documented as either present or absent (i.e., symptom screen completed) |
| Unsolicited symptom | All subjects with study vaccine administered |
| Concomitant medication | All subjects with study vaccine administered |

The intensity scale of the following solicited AEs will be assessed as described:

| Adverse Event | Intensity<br>grade | Parameter |
|---|---|---|
| Pain at injection site | 0 | None |
| | 1 | Mild: Any pain neither interfering with nor preventing normal every day activities. |
| | 2 | Moderate: Painful when limb is moved and interferes with every day activities. |
| | 3 | Severe: Significant pain at rest. Prevents normal every day activities. |
| Redness at injecti | on site | Record greatest surface diameter in mm |
| Swelling at injection | on site | Record greatest surface diameter in mm |
| Fever* | | Record temperature in °C |
| Headache 0 | | Normal |
| | 1 | Mild: Headache that is easily tolerated |
| | 2 | Moderate: Headache that interferes with normal activity |
| | 3 | Severe: Headache that prevents normal activity |
| Fatigue | 0 | Normal |
| | 1 | Mild: Fatigue that is easily tolerated |
| | 2 | Moderate: Fatigue that interferes with normal activity |
| | 3 | Severe: Fatigue that prevents normal activity |
| Gastrointestinal | 0 | Normal |
| symptoms (nausea, | 1 | Mild: Gastrointestinal symptoms that are easily tolerated |
| vomiting, diarrhoea | 2 | Moderate: Gastrointestinal symptoms that interfere with normal activity |
| and/or abdominal pain) | 3 | Severe: Gastrointestinal symptoms that prevent normal activity |

<sup>\*</sup>Fever is defined as temperature  $\geq$  37.5°C for oral, axillary or tympanic route, or  $\geq$  38.0°C for rectal route. The preferred route for recording temperature in this study will be oral.

The maximum intensity of local injection site redness/swelling will be scored at GSK Biologicals according to the standard GSK Biologicals' scoring system for adults:

0:  $\leq 20 \text{ mm}$ 

1:  $> 20 \text{ mm to} \le 50 \text{ mm}$ 

2:  $> 50 \text{ mm to} \le 100 \text{ mm}$ 

3: > 100 mm

The maximum intensity of fever will be scored at GSK Biologicals according to the standard GSK Biologicals' scoring system for adults (via the preferred route for recording temperature in this study which is oral):

0:  $< 37.5 \, ^{\circ}\text{C}$ 

1:  $\geq 37.5 \,^{\circ}\text{C} \text{ to} \leq 38.5 \,^{\circ}\text{C}$ 

2: > 38.5 °C to  $\le 39.5$  °C

3: > 39.5°C

The investigator assessed the maximum intensity that occurred over the duration of the event for all unsolicited AEs (including SAEs) recorded during the study. The assessment was based on the investigator's clinical judgement.

For clintrial gov and EudraCT posting purposes, a summary of subjects with all combined solicited (regardless of their duration) and unsolicited adverse events will be provided. Solicited adverse events will be coded by MedDRA as per the following codes.

204812 (RSV F-021)

Statistical Analysis Plan Amendment 2 Final

| Solicited symptom | Lower level term name | Lower level term code | Corresponding Primary<br>Term code |
|---|---|---|---|
| Pain | Pain | 10033371 | 10033371 |
| Redness | Erythema | 10015150 | 10015150 |
| Swelling | Swelling | 10042674 | 10042674 |
| Fatigue | Fatigue | 10016256 | 10016256 |
| Fever | Fever | 10016558 | 10037660 |
| Gastroinstestinal symptoms | Gastroinstestinal disorder | 10017944 | 10017944 |
| Headache | Headache | 10019211 | 10019211 |

#### 11.2.6. Number of decimals displayed

The following decimal description from the decision rules will be used for the demography, immunogenicity and safety/reactogenicity.

| Display Table | Parameters | Number of decimal digits |
|---|---|---|
| All summaries | % of count, including LL & UL of CI | 1 |
| All summaries | % of difference, including LL & UL of CI | 2 |
| Demographic characteristics | Mean, median age, SD (age) | 1 |
| Reactogenicity | Mean, Min, Q1, Median, Q3, Max for duration | 1 |
| Immunogenicity | Ratio of GMT/GMC | 2 |

#### 12. ANNEX 2: SUMMARY ON ELIMINATION CODES

Refer to section 5.2

## 13. ANNEX 3 CALCULATION OF INDIVIDUAL AND OVERALL DESIRABILITY INDEX

The section below provide the details on how to calculate individual desirability index and overall desirability index score based on Annex E in the Protocol.

#### Reactogenicity

A logistic regression model will be fitted on each reactogenicity endpoint (any Grade 2/3 general AE and any related SAE, Grade 2/3 fever) reported during the 7-day follow-up period after vaccination, including all RSV formulations.

- o The vaccine group as the fixed effect
- The age groups (18-32 years and 33-45 years) as the categorical covariant if deemed necessary.

The estimation of indication rate will be tabulated by treatment group. The SAS codes can be used as reference:

```
proc logistic data=React;
  class Treatment AgeGroup / param=glm;
  model response (event='AE')= Treatment| AgeGroup;
  lsmeans Treatment / ILINK e diff oddsratio adjust=bon cl;
run;
```

For any Grade 2/3 general AEs and any related SAEs, the incidence rate estimate (IR) will be transformed in a [0,1] desirability index using the following function:

$$DR1 = \begin{cases} \frac{1}{1 + \exp(-50 * (0.25 - IR))}, & \text{if } IR \le 0.25 \\ \frac{1}{1 + \exp(-25 * (0.25 - IR))}, & \text{if } IR \ge 0.25 \end{cases}$$

where IR is the incidence rate estimated by the model. This function will allocate a desirability value of 1, 0.5 and 0 to incidence rate equal to 0.1, 0.25 and 0.5 respectively (see Figure 2). But the calculation equally weights Grade 2/3 general AEs and any related SAEs.

Figure 2 Desirability function for the incidence rate of Grade 2/3 general AEs and related SAEs - for each investigational RSV vaccine formulation



For Grade 2/3 fever, the incidence rate estimate (**FR**) will be transformed in a [0,1] desirability index using the following function:

$$DR2 = \frac{1}{1 + \exp(-120 * (0.05 - IR))}$$

where **IR** is the incidence rate estimated by the model. As illustrated in Figure 3, the function will allocate desirability values of 1, 0.5 and 0 to incidence rate equal to 0, 0.05 and 0.1 respectively.

Figure 3 Desirability function for the incidence rate of Grade 2/3 fever - for each investigational RSV vaccine formulation



Finally, the reactogenicity index will be computed by taking the geometric mean of the 2 indexes:

$$DR = \sqrt{DR1 * DR2}$$

#### **Immunogenicity**

The ANCOVA model will be fitted on the log-transformed titre for each immune response of neutralising anti-RSV-A and PCA separately including

- o The vaccine group as the fixed effect
- The pre-vaccination titre/concentration and age groups (18-32 years and 33-45 years) as the covariates if deemed necessary

The mean estimations of GMTs/GMCs for each treatment group at Day 30 and its 95% CI will be provided for immunogenicity desirability calculation. The estimated GMT and LL will be tabulated by treatment group.

As formulations inducing a high immune response will be considered suitable, the lower limit (LL) of the estimated GMT/C adjusted for pre-vaccination titres will be the statistical criterion considered for decision making.

Neutralising anti-RSV-A titres

The LL of the GMT estimate will be transformed into a [0, 1] desirability index using the function:

DI1 = 
$$\frac{1}{1 + \exp(1.5 * (9.5 - LL))}$$

where LL is the lower limit of the 95% confidence interval of the GMT adjusted for prevaccination titres in log base 2. The function was chosen to have a desirability of 0 at LL value  $\leq$  6 log2 (=128), and a desirability of 1 at LL value  $\geq$  13 log2. This function is illustrated in Figure 4.

Figure 4 Desirability function for neutralising anti-RSV-A GMTs - for each investigational RSV vaccine formulation



PCA concentrations

The LL of the GMC adjusted for pre-vaccination titres estimate will be transformed using the following function:

DI2 = 
$$\frac{\frac{1}{1 + \exp(0.05 * (150 - LL))}}, \quad \text{if LL} \le 150$$
$$\frac{1}{1 + \exp(0.025 * (150 - LL))}, \quad \text{if LL} \ge 150$$

As illustrated in Figure 5, a PCA response of 25, 150 and 400 μg/mL will have a desirability value of 0, 0.5 and 1 respectively.

Figure 5 Desirability function for PCA concentrations - for each investigational RSV vaccine formulation



Finally, the immunogenicity index will be computed by taking the geometric mean of the 2 indexes:

$$DI = \sqrt{DI1 * DI2}$$

### Overall desirability index

The overall desirability index for each formulation will be obtained by computing the following weighted geometric mean:  $D = DR^{0.4} * DI^{0.6}$ .

#### 14. ANNEX 4: STUDY SPECIFIC MOCK TFL

The following draft study specific mock TFLs will be used. The data display, title and footnote are for illustration purpose and will be adapted to the study specificity as indicated in the TFL TOC.

Note that there may be few changes between the study specific SAP mock TFL and the final TFLs. These editorial/minor changes will not lead to a SAP amendment.

| Template # | Table Title | Macro |
|---|---|---|
| Template 1 | Number of subjects enrolled into the study as well as the number of subject excluded from ATP analysis with reasons for exclusion | %ELIMLIST |
| Template 2 | Number of subjects vaccinated, completed and withdrawn with reason for withdrawal (Exposed set) | %DROP_SUM (OTH=1) |
| Template 3 | Number of subjects vaccinated, completed and withdrawn with reason for withdrawal (Exposed set) | %DROP_SUM (OTH=0) |
| Template 4 | Number of subjects at each visit and list of withdrawn subjects (Exposed set) | %DROPOUT |
| Template 5 | Summary of demographic characteristics (Exposed set) | %DEMOGRA |
| Template 6 | Summary of demographic characteristics by age category (Exposed set) | %DEMOGRA |
| Template 7 | Number of subjects by center (Exposed set) | %CENTER |
| Template 8 | Number of subjects by center for each age category (Exposed set) | %CENTER |
| Template 9 | Number of subjects by country and center (Exposed set) | %CENTER |
| Template 10 | Deviations from specifications for age and intervals between study visits (Exposed set) | %INT_VAL |
| Template 11 | Summary of vital signs characteristics (Exposed set) | %VITAL_SIGNS |
| Template 16 | Study Population (Exposed set) | %CTR_DEMOG |
| Template 17 | Number of enrolled subjects by country | %FREQ_DIS |
| Template 23 | Number of enrolled subjects by age category | %FREQ_DIS |
| Template 24 | Minimum and maximum activity dates (Exposed set) | %DATE |
| Template 25 | Incidence and nature of symptoms (solicited and unsolicited) reported during the <b>7-day</b> (Days 0-6) post-vaccination period (Exposed set) | %LOCGEN |
| Template 26 | Daily prevalence of <b>any fever</b> during the 7-day (Days 0-6) post-vaccination period (Exposed set) | %SYMPLOT |
| Template 27 | Incidence of solicited <b>local</b> symptoms reported during the 7-day (Days 0-6) post-vaccination period (Exposed set) | %FREQ |
| Template 28 | Incidence of solicited <b>local</b> symptoms reported during the 7-day (Days 0-6) post-vaccination period by <b>maximum intensity</b> (Exposed set) | %FREQ |
| Template 34 | Incidence of solicited <b>general</b> symptoms reported during the 7-day (Days 0-6) post-vaccination period (Exposed set) | %FREQ |
| Template 35 | Incidence of solicited <b>general</b> symptoms reported during the 7- | %FREQ |

## 204812 (RSV F-021) Statistical Analysis Plan Amendment 2 Final

| | | llysis Plan Amendment 2 Final |
|---|---|---|
| | day (Days 0-6) post-vaccination period <b>by maximum intensity</b> (Exposed set) | |
| Template 36 | Percentage of subjects reporting the occurrence of unsolicited symptoms classified by MedDRA Primary System Organ Class and Preferred Term, during the <b>30-day</b> (Days 0-29) post-vaccination period (Exposed set) | %UNSOL |
| Template 37 | Listing of <b>SAEs</b> reported up to study end (Exposed set) | %SAE |
| Template 38 | Number (%) of subjects with serious adverse events up <b>Day 7</b> (Exposed set) | %CTR_SAE |
| Template 40 | Compliance in returning symptom information (Exposed set) | % COMPLI |
| Template 41 | Number and percentage of subjects taking a <b>concomitant medication</b> during the <b>7- day</b> (Days 0-6) post -vaccination period (Exposed set) | %CMED_INC |
| Template 42 | Exploratory comparisons between groups in terms of percentage of subjects reported any <b>Grade 2/3 AE</b> and/or <b>any fever &gt;38.5°C</b> and/or <b>any vaccine-related SAE</b> during the <b>7 day</b> (Days 0-6) Post- vaccination period (Exposed set) | %COMP_FQ_AE |
| Template 43 | Solicited and unsolicited symptoms experienced by <b>at least 5</b> % <b>of subjects</b> , classified by MedDRA Primary System Organ Class and Preferred Term within the <b>30-day</b> (Days 0-29) post-vaccination period including number of events - SAE excluded (Exposed set) | %UNSOL (NIH=5, EVENT=1) |
| Template 44 | Distribution of change from baseline in haematology and biochemistry with respect to normal laboratory ranges (Exposed set) | %HAEMATO_BIOCH |
| Template 45 | Summary of haematology and biochemistry results by maximum grade from VISIT 2 (D7) up to VISIT 3 (D30) versus baseline (Exposed set) | %HAEMATO_BIOCH_GR_CHAN<br>GE |
| Template 46 | Summary of haematology change from baseline by maximum grade from VISIT2 (D7) up to VISIT 3 (D30) (Exposed set) | %HAEMATO_BIOCH_GR_CHAN<br>GE |
| Template 32 | Individual results of <b>hemoglobin</b> levels <b>outside of the normal</b> ranges in < <i>group</i> > (Exposed set) | %HB_PROFIL |
| Template 48 | Number and percentage of subjects with anti-RSV-A neutralising antibody titer equal to or above <cut-off> and GMTs (Per protocol set)</cut-off> | %GMT |
| Template 34 | Number and percentage of subjects with anti-RSV-A neutralising antibody titer equal to or above <cut-off> and GMTs - by age category (Per protocol set)</cut-off> | %GMT |
| Template 35 | Geometric mean of the individual ratio of <b>anti-RSV-A</b> neutralising antibody titers at each post-vaccination timepoint compared to pre-vaccination with 95% CI (Per protocol set) | %GMRACT |
| Template 36 | GMTs and their 95% CIs for <b>anti-RSV-A</b> neutralising antibody at each timepoint (Per protocol set) | %GMTPLOT* |
| Template 37 | Kinetics of GMTs for <b>anti-RSV-A</b> neutralising antibody on subjects with results available at all timepoints (Per protocol set) | %KIN_GM* |
| Template 38 | Distribution of <b>anti-RSV-A</b> neutralising antibody titer (Per protocol set) | %DIS |
| Template 39 | Distribution of <b>anti-neogenin</b> antibody concentration (Exposed set) | %DIS |
| Template 40 | Distribution of fold of <b>anti-RSV-A</b> neutralising antibody titer by pre-vaccination titer category (Per protocol set) | %DIS |
| Template 41 | Distribution of fold of anti-neogenin antibody concentration (Exposed set) | %DIS |
| Template 42 | Reverse cumulative distribution curves for anti-RSV-A | %REVCUM |

## 204812 (RSV F-021) Statistical Analysis Plan Amendment 2 Final

| | neutralising antibody titers in each group at pre-vaccination (Per protocol set) | ayor Harry Wilding High |
|---|---|---|
| Template 43 | Individual results of <b>anti-RSV-A</b> neutralising antibody titer at Day <30/60/90> versus pre-vaccination in <each group=""> and Control (Per protocol set)</each> | %SCATTERPLOT* |
| Template 44 | Vaccine response for <b>anti-RSV-A</b> neutralising antibody titer at each post-vaccination timepoint (Per protocol set) | %HUM_RESP* |
| Template 45 | Estimated GMTs and 95% CIs for <b>anti-RSV-A</b> neutralising antibody titre (Per protocol set) | %GMT_ANOVA |
| Template 46 | Exploratory comparisons (GMT ratios) between RSV groups with corresponding 95% confidence interval for <b>anti-RSV A</b> neutralizing antibody titre at <b>Day 30</b> (Per protocol set) | %GMT_RATIO |
| Template 47 | Individual kinetics of <b>anti-neogenin</b> antibody concentrations by group (Exposed set) | %NEO_INDKIN* |
| Template 48 | GM of individual ratios (fold increase post over pre) and their 95% Cls for <b>anti-RSV F lgG1 and lgG total</b> antibody assays and each group, at <b>Day 30</b> (Per protocol set) | %GMRPLOT* |
| Template 49 | Exploratory comparisons (GM ratios of fold increase post/pre) between RSV groups with corresponding 95% confidence interval for <b>anti-RSV F IgG1</b> antibody concentrations at <b>Day 30</b> (Per protocol set) | %GMF_RATIO* |
| Template 50 | Comparisons of GM ratios with corresponding 95% confidence interval between anti-RSV F antibody concentrations (IgG Total) and anti-RSV-A neutralising antibody titers at pre-vaccination (Per protocol set) | %GM_RATIO_PRE.SAS** |
| Template 51 | Exploratory comparisons (GM ratios of fold increase post/pre) with corresponding 95% confidence interval between anti-RSV F antibody concentrations (IgG Total) and anti-RSV-A neutralising antibody titers at Day 30 (Per protocol set) | %GM_RATIO_FI.SAS** |
| Template 52 | Desirability index of immunogenicity during the 30-day (Days 0-29) post-vaccination period (Per protocol set) | %lmmuno_DI** |
| Template 53 | Desirability index of reactogenicity during the 7-day (Days 0-6) post-vaccination period (Exposed set) | %Reacto_DI** |
| Template 54 | Desirability index based on reactogenicity and safety (Exposed set up to Day 7) and immunogenicity (Per protocol set up to Day 30) | %Overall_DI** |

<sup>\*</sup> Name of specific macros created in study RSV F-001 (116969) and RSV F-020 (201510) \*\* Name of specific macros newly created in study RSV F-021 (204812)

204812 (RSV F-021)

Statistical Analysis Plan Amendment 2 Final

## Template 1 Number of subjects enrolled into the study as well as the number of subjects excluded from the PPS analyses with reasons for exclusion

| | Total <e< th=""><th><each g<="" th=""><th>roup&gt;</th></each></th></e<> | | <each g<="" th=""><th>roup&gt;</th></each> | roup> | |
|---|---|---|---|---|---|
| Title | n | S | % | n | S |
| Total enrolled cohort | | | | | |
| Study vaccine dose not administered at all but subject number allocated (code 1030) | | | | | |
| Exposed set | | | | | |
| <reason &="" code="" elimination="" for=""></reason> | | | | | |
| <reason &="" code="" elimination="" for=""></reason> | | | | | |
| Per protocol set for immunogenicity | | | | | |

#### <each group>:

30 PreF = 30 µg PreF

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

Note: Subjects may have more than one elimination code assigned

n = number of subjects with the elimination code assigned excluding subjects who have been assigned a lower elimination code number

s = number of subjects with the elimination code assigned

% = percentage of subjects in the considered Per protocol set relative to the Exposed set

### Template 2 Number of subjects vaccinated, completed and withdrawn with reason for withdrawal (Exposed set)

| | <each group=""></each> | Total |
|---|---|---|
| Number of subjects vaccinated | | |
| Number of subjects completed | | |
| Number of subjects withdrawn | | |
| Reasons for withdraw: | | |
| Serious Adverse Event | | |
| Non-serious adverse event | | |
| Protocol violation | | |
| Consent withdrawal (not due to an adverse event) | | |
| Migrated/moved from study area | | |
| Lost to follow-up (subjects with incomplete vaccination course) | | |
| Lost to follow-up (subjects with complete vaccination course) | | |
| Others | | |

#### <each group>:

30 PreF = 30 µg PreF

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

Vaccinated = number of subjects who were vaccinated in the study

Completed = number of subjects who completed last study visit

withdrawn = number of subjects who did not come for the last study visit

204812 (RSV F-021)

Statistical Analysis Plan Amendment 2 Final

## Template 3 Number of subjects vaccinated, completed and withdrawn with reason for withdrawal (Exposed set)

| | <each group=""></each> | Total |
|---|---|---|
| Number of subjects vaccinated | | |
| Number of subjects completed | | |
| Number of subjects withdrawn | | |
| Reasons for withdrawal : | | |
| Serious Adverse Event | | |
| Non-Serious Adverse Event | | |
| Protocol violation | | |
| Consent withdrawal (not due to an adverse event) | | |
| Migrated/moved from study area | | |
| Lost to follow-up (subjects with incomplete vaccination course) | | |
| Lost to follow-up (subjects with complete vaccination course) | | |
| Sponsor study termination | | |
| Other - <reason></reason> | | |
| Other - <reason></reason> | | |

#### <each group>:

30 PreF = 30  $\mu$ g PreF

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

Vaccinated = number of subjects who were vaccinated in the study

Completed = number of subjects who completed last study visit

Withdrawn = number of subjects who did not come for the last study visit

Template 4 Number of subjects at each visit and list of withdrawn subjects (Exposed set)

| Group | Visit | N | Withdrawn Subject number | Reason for withdrawal |
|---|---|---|---|---|
| <each group=""></each> | VISIT 1 (D0) | | | |
| | VISIT 2 (D7) | | | |
| | VISIT 3 (D30) | | | |
| | VISIT 4 (D60) | | | |
| | VISIT 5 (D90) | | | |

#### <each group>:

 $30 \text{ PreF} = 30 \mu \text{g PreF}$ 

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

N = Number of subjects who are still in the study up to the visit

Withdrawn = Subject who did not return after the visit

204812 (RSV F-021)

Statistical Analysis Plan Amendment 2 Final

### Template 5 Summary of demographic characteristics (Per Protocol Set)

| | | <each group=""><br/>(N=)</each> | | Total<br>(N= ) | |
|---|---|---|---|---|---|
| Characteristics | Parameters or | Value<br>or n | % | Value<br>or n | % |
| Onura de Cristios | Categories | 0 | | 01 11 | |
| Age (years) at vaccination | Mean | | | | |
| | SD | | | | |
| | Median | | | | |
| | Minimum | | | | |
| | Maximum | | | | |
| Ethnicity | American Hispanic or Latino | | | | |
| | Not American Hispanic or Latino | | | | |
| Geographic Ancestry | African Heritage / African American | | | | |
| | American Indian or Alaskan Native | | | | |
| | Asian - Central/South Asian Heritage | | | | |
| | Asian - East Asian Heritage | | | | |
| | Asian - Japanese Heritage | | | | |
| | Asian - South East Asian Heritage | | | | |
| | Native Hawaiian or Other Pacific Islander | | | | |
| | White - Arabic / North African Heritage | | | | |
| | White - Caucasian / European Heritage | | | | |
| | Other | | | | |

#### <each group>:

 $30 \text{ PreF} = 30 \mu \text{g PreF}$ 

60 PreF = 60 μg PreF

120 PreF = 120 µg PreF

Control = Placebo

N = total number of subjects

n/% = number / percentage of subjects in a given category

Value = value of the considered parameter

SD = standard deviation

204812 (RSV F-021)

Statistical Analysis Plan Amendment 2 Final

## Template 6 Summary of demographic characteristics by age category (Exposed set)

| | | <each group=""><br/>(N=)</each> | | | | | otal<br>l= ) | | |
|---|---|---|---|---|---|---|---|---|---|
| | | <sub< th=""><th>group&gt;</th><th><sub< th=""><th>group&gt;</th><th><sub< th=""><th>group&gt;</th><th><sub< th=""><th>group&gt;</th></sub<></th></sub<></th></sub<></th></sub<> | group> | <sub< th=""><th>group&gt;</th><th><sub< th=""><th>group&gt;</th><th><sub< th=""><th>group&gt;</th></sub<></th></sub<></th></sub<> | group> | <sub< th=""><th>group&gt;</th><th><sub< th=""><th>group&gt;</th></sub<></th></sub<> | group> | <sub< th=""><th>group&gt;</th></sub<> | group> |
| Characteristics | Parameters or<br>Categories | Value<br>or n | % | Value<br>or n | % | Value<br>or n | % | Value<br>or n | % |
| Age (years) at | Mean<br>SD | | | | | | | | |
| vaccination | Median | | | | | | | | |
| | Minimum<br>Maximum | | | | | | | | |
| Ethnicity | American Hispanic or Latino | | | | | | | | |
| Geographic<br>Ancestry | Not American Hispanic or Latino African Heritage / African American | | | | | | | | |
| , | American Indian or Alaskan Native Asian - Central/South Asian Heritage | | | | | | | | |
| | Asian - East Asian Heritage | | | | | | | | |
| | Asian - Japanese Heritage Asian - South East Asian Heritage | | | | | | | | |
| | Native Hawaiian or Other Pacific Islander | | | | | | | | |
| | White - Arabic / North African<br>Heritage | | | | | | | | |
| | White - Caucasian / European<br>Heritage | | | | | | | | |
| | Other | | | | | | | | |

#### <each group>:

30 PreF = 30 μg PreF

60 PreF = 60 µg PreF

120 PreF = 120 µg PreF

Control = Placebo

N = total number of subjects

n/% = number / percentage of subjects in a given category

Value = value of the considered parameter

SD = standard deviation

#### <subgroup> by age category:

18-32Y = 18-32 years old subjects

33-45Y = 33-45 years old subjects

204812 (RSV F-021)

Statistical Analysis Plan Amendment 2 Final

#### Template 7 Number of subjects by center (Exposed set)

| | | <each group=""></each> | To | tal |
|--------|---|------------------------|----|-----|
| Center | • | n | n | % |
| PPD | | | | |
| All | | | | |

#### <each group>:

30 PreF = 30 µg PreF

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

n = number of subjects included in each group or in total for a given center or for all centers

All = sum of all subjects in each group or in total (sum of all groups)

 $% = n/AII \times 100$ 

Center = GSK Biologicals assigned center number

#### Template 8 Number of subjects by center for each age category (Exposed set)

| | • • • | PreF | • • • • | PreF | | PreF | | itrol | | To | tal | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 18-32Y | 33-45Y | 18-32Y | 33-45Y | 18-32Y | 33-45Y | 18-32Y | 33-45Y | 18-3 | 2Y | 33-4 | 5Y |
| Center | n | n | n | n | n | n | n | n | n | % | n | % |

 $30 \text{ PreF} = 30 \mu \text{g PreF}$ 

60 PreF = 60 µg PreF

120 PreF = 120 µg PreF

Control = Placebo

18-32Y = 18-32 years old subjects

33-45Y = 33-45 years old subjects

n = number of subjects included in each group or in total for a given center or for all centers

All = sum of all subjects in each group or in total (sum of all groups)

 $% = n/AII \times 100$ 

Center = GSK Biologicals assigned center number

#### Template 9 Number of subjects by country and center (Exposed set)

| | | <each group=""></each> | | Total |
|---------|--------|------------------------|---|-------|
| Country | Center | n | n | % |
| | All | | | |
| All | All | | | |

#### <each group>:

 $30 \text{ PreF} = 30 \mu \text{g PreF}$ 

60 PreF = 60 µg PreF

120 PreF = 120 µg PreF

Control = Placebo

n = number of subjects included in each group or in total for a given center or for all centers

All = sum of all subjects in each group or in total (sum of all groups)

 $% = n/AII \times 100$ 

Center = GSK Biologicals assigned center number

204812 (RSV F-021)

Statistical Analysis Plan Amendment 2 Final

## Template 10 Deviations from specifications for age and intervals between study visits (Exposed set)

| | | Age | Dose:1-PI (D30) | Dose:1-PI (D60) | Dose:1-PI (D90) | Dose:1-<br>CONCLUSION |
|---|---|---|---|---|---|---|
| Group | | Protocol | Protocol | Protocol | Protocol | Protocol |
| | | from 18 to 45 years | from 30 to 44 days | from 56 to 70 days | from 86 to 100 days | from 330 to 390<br>days |
| <each<br>group&gt;</each<br> | n | | | | | |
| | N | | | | | |
| | % | | | | | |
| | range | | | | | |

#### <each group>:

30 PreF = 30 μg PreF

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

N = total number of subjects with available results

n/% = number / percentage of subjects with results outside of the interval

range = minimum-maximum for age and intervals

PI(D30) = Post-vaccination at Day 30

PI(D60) = Post-vaccination at Day 60

PI(D90) = Post-vaccination at Day 90

204812 (RSV F-021)

Statistical Analysis Plan Amendment 2 Final

## Template 11 Summary of vital signs characteristics at VISIT 1 (Day 0) (Exposed set)

| | | <each group=""><br/>N =</each> | Total<br>N = |
|---|---|---|---|
| Characteristics | Parameters | Value | Value |
| Height (Cm) | Mean | | |
| | SD | | |
| | Median | | |
| | Minimum | | |
| | Maximum | | |
| | Unknown | | |
| Weight (Kg) | Mean | | |
| | SD | | |
| | Median | | |
| | Minimum | | |
| | Maximum | | |
| | Unknown | | |
| Heart rate (Beats per minute) | Mean | | |
| , , | SD | | |
| | Median | | |
| | Minimum | | |
| | Maximum | | |
| | Unknown | | |
| Respiratory rate (Breadth per minute) | Mean | | |
| | SD | | |
| | Median | | |
| | Minimum | | |
| | Maximum | | |
| | Unknown | | |
| Systolic blood pressure (Mmhg) | Mean | | |
| | SD | | |
| | Median | | |
| | Minimum | | |
| | Maximum | | |
| | Unknown | | |
| Diastolic blood pressure (Mmhg) | Mean | | |
| | SD | | |
| | Median | | |
| | Minimum | | |
| | Maximum | | |
| | Unknown | | |

#### <each group>:

 $30 \text{ PreF} = 30 \mu \text{g PreF}$ 

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 μg PreF

Control = Placebo

N = total number of subjects

Value = value of the considered parameter

SD = standard deviation

204812 (RSV F-021)

#### Statistical Analysis Plan Amendment 2 Final

### **Template 12 Study Population (Exposed set)**

| Number of subjects | <each group=""></each> | Total |
|---|---|---|
| Planned, N | | |
| Randomised, N (Exposed set) | | |
| Completed, n (%) | | |
| Demographics | <each group=""></each> | Total |
| N (Exposed set) | | |
| Females:Males | | |
| Mean Age, years (SD) | | |
| Median Age, years (minimum, maximum) | | |
| White - caucasian / european heritage, n (%) | | |
| Asian – South East Asian heritage, n (%) | | |

<each group>: 30 PreF = 30 μg PreF

60 PreF = 60 µg PreF 120 PreF = 120 µg PreF Control = Placebo

204812 (RSV F-021)

Statistical Analysis Plan Amendment 2 Final

#### Template 13 Number of enrolled subjects by country

| | | <each group=""><br/>N =</each> | Total<br>N = |
|---|---|---|---|
| Characteristics | Categories | n | n |
| Country | Czech Republic | | |
| | Australia | | |

<each group>:

 $30 \text{ PreF} = 30 \mu \text{g PreF}$ 

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

N = Number of enrolled subjects

n= number of enrolled subjects included in each group or in total for a given country or for all countries

#### Template 14 Number of enrolled subjects by age category

| | | <each group=""> N =</each> | Total |
|-----------------|----------------------|----------------------------|-------|
| Characteristics | Categories | n | n |
| Age category | Adults (18-45 years) | | |
| | Missing | | |

<each group>:

 $30 \text{ PreF} = 30 \mu \text{g PreF}$ 

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

N = Number of enrolled subjects

n= number of enrolled subjects included in each group or in total for a given age category or for all age categories Missing = age at dose 1 unknown

#### Template 15 Minimum and maximum activity dates (Exposed set)

| Group | Activity | <b>Activity Description</b> | Minimum date | Maximum date |
|---|---|---|---|---|
| | number | | | |
| <each group=""></each> | 10 | VISIT 1 (DAY 0) | | |
| | 20 | VISIT 2 (M 1) | | |
| | 30 | VISIT 3 (M 2) | | |
| | 40 | VISIT 4 (M 3) | | |

<each group>:

 $30 \text{ PreF} = 30 \mu \text{g PreF}$ 

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

204812 (RSV F-021)

Statistical Analysis Plan Amendment 2 Final

# Template 16 Incidence and nature of symptoms (solicited and unsolicited reported during the 7-day (Days 0-6) post-vaccination period (Exposed set)

| | Any sy | y symptom 95% CI | | | | General symptoms | | | | | Local symptoms | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | 95% ( | CI | | | | 95% C | Cl | | | | 95% | CI |
| Group | N | n | % | LL | UL | N | n | % | LL | UL | N | n | % | LL | UL |
| <each group=""></each> | | | | | | | | | | | | | | | |

#### <each group>:

30 PreF = 30 µg PreF

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

N = number of subjects with the administered dose

n/% = number/percentage of subjects presenting at least one type of symptom whatever the study vaccine administered

95% CI = exact 95% confidence interval, LL = Lower Limit, UL = Upper Limit

Note: the same table will be generated by group/sub-group, with sub-group= age category (see SAP).

Template 17 Daily prevalence of any fever during the 7-day (Days 0-6) post-vaccination period (Exposed set)



30 PreF = 30 µg PreF 60 PreF = 60 µg PreF 120 PreF = 120 µg PreF Control = Placebo

204812 (RSV F-021)

Statistical Analysis Plan Amendment 2 Final

### Template 18 Incidence of solicited local symptoms reported during the 7-day (Days 0-6) post-vaccination period (Exposed set)

| | | | | <each gro<="" th=""><th>up&gt;</th><th></th></each> | up> | |
|---|---|---|---|---|---|---|
| | | | | | | 95 % CI |
| Symptom | Туре | N | n | % | LL | UL |
| Pain | All | | | | | |
| | Grade 1 | | | | | |
| | Grade 2 | | | | | |
| | Grade 3 | | | | | |
| | Onset ≤48h | | | | | |
| | Medical advice | | | | | |
| Redness (mm) | All | | | | | |
| eaness (mm) | >20 and ≤ 50 | | | | | |
| | >50 and ≤ 100 | | | | | |
| | >100 | | | | | |
| | Onset ≤48h | | | | | |
| | Medical advice | | | | | |
| Swelling (mm) | All | | | | | |
| | >20 and ≤ 50 | | | | | |
| | >50 and ≤ 100 | | | | | |
| | >100 | | | | | |
| | Onset ≤48h | | | | | |
| | Medical advice | | | | | |

#### <each group>:

 $30 \text{ PreF} = 30 \mu \text{g PreF}$ 

60 PreF = 60 µg PreF

120 PreF =120 µg PreF

Control = Placebo

N= number of subjects with the documented dose

n/%= number/percentage of subjects reporting at least once the symptom

95%CI= Exact 95% confidence interval; LL = lower limit, UL = upper limit

The maximum intensity of local injection site redness/swelling was coded as follows for adults:

- $0: \leq 20 \text{ mm}$
- 1:  $> 20 \text{ mm to} \le 50 \text{ mm}$
- 2:  $> 50 \text{ mm to} \le 100 \text{ mm}$
- 3: > 100 mm

204812 (RSV F-021)

Statistical Analysis Plan Amendment 2 Final

## Template 19 Incidence of solicited local symptoms reported during the 7-day (Days 0-6) post-vaccination period by maximum intensity (Exposed set)

| | | | < | each gro | oup> | |
|---------------|----------------|---|---|----------|------|--------|
| | | | | | | 5 % CI |
| Symptom | Туре | N | n | % | LL | UL |
| Pain | All | | | | | |
| | Grade 1 | | | | | |
| | Grade 2 | | | | | |
| | Grade 3 | | | | | |
| | Onset ≤48h | | | | | |
| | Medical advice | | | | | |
| Redness (mm) | All | | | | | |
| | >20 and ≤50 | | | | | |
| | >50 and ≤100 | | | | | |
| | >100 | | | | | |
| | Onset ≤48h | | | | | |
| | Medical advice | | | | | |
| Swelling (mm) | All | | | | | |
| <b>3</b> ( ) | >20 and ≤50 | | | | | |
| | >50 and ≤100 | | | | | |
| | >100 | | | | | |
| | Onset ≤48h | | | | | |
| | Medical advice | | | | | |

#### <each group>:

30 Pre $\overline{F}$  = 30  $\mu$ g Pre $\overline{F}$ 

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

Type=Max grade & onset

All=any severity >Grade 0 for pain and any diameter >20mm for redness and swelling

N=number of vaccinated subjects who returned the diary card

n/% = number/percentage of subjects reporting the AE at least once. Maximum intensity only

95%CI = Exact 95% confidence interval; LL = lower limit, UL = upper limit

The maximum intensity of local injection site redness/swelling was coded as follows for adults:

0: ≤ 20 mm

1:  $> 20 \text{ mm to} \le 50 \text{ mm}$ 

 $2: > 50 \text{ mm to} \le 100 \text{ mm}$ 

3: > 100 mm

204812 (RSV F-021)

Statistical Analysis Plan Amendment 2 Final

### Template 20 Incidence of solicited general symptoms reported during the 7-day (Days 0-6) post-vaccination period (Exposed set)

| | | | | <each gi<="" th=""><th>roup&gt;</th><th></th></each> | roup> | |
|---|---|---|---|---|---|---|
| | | | | | 9: | 5 % CI |
| Symptom | Туре | N | n | % | LL | UL |
| Fatigue | All | | | | | |
| - | Grade 1 | | | | | |
| | Grade 2 | | | | | |
| | Grade 3 | | | | | |
| | Related | | | | | |
| | Grade 2 Related | | | | | |
| | Grade 3 Related | | | | | |
| | Onset ≤48h | | | | | |
| | Medical advice | | | | | |
| Temperature (Oral)<br>(°C) | All (≥37.5) | | | | | |
| ( ) | >38.0 | | | | | |
| | >38.5 | | | | | |
| | >39.0 | | | | | |
| | >39.5 | | | | | |
| | Related | | | | | |
| | >38.5 Related | | | | | |
| | >39.5 Related | | | | | |
| | Onset ≤48h | | | | | |
| | Medical advice | | | | | |
| Gastrointestinal | All | | | | | |
| symptoms | Grade 1 | | | | | |
| -, | Grade 2 | | | | | |
| | Grade 3 | | | | | |
| | Related | | | | | |
| | Grade 2 Related | | | | | |
| | Grade 3 Related | | | | | |
| | Onset ≤48h | | | | | |
| | Medical advice | | | | | |
| Headache | All | | | | | |
| | Grade 1 | | | | | |
| | Grade 2 | | | | | |
| | Grade 3 | | | | | |
| | Related | | | | | |
| | Grade 2 Related | | | | | |
| | Grade 3 Related | | | | | |
| | Onset ≤48h | | | | | |
| | Medical advice | | | | | |

#### <each group>:

30 PreF = 30 μg PreF

60 PreF = 60 µg PreF

120 PreF =120 µg PreF

Control = Placebo

N = number of subjects with the documented dose

n/% = number/percentage of subjects reporting the symptom at least once 95%CI = Exact 95% confidence interval; LL = lower limit, UL = upper limit

Temperatures were coded as follows for adults:

0: < 37.5 °C

1:  $\geq$  37.5 °C to  $\leq$  38.5 °C

2: > 38.5 °C to  $\leq 39.5$  °C

3: > 39.5°C

204812 (RSV F-021)

Statistical Analysis Plan Amendment 2 Final

## Template 21 Incidence of solicited general symptoms reported during the 7-day (Days 0-6) post-vaccination period by maximum intensity (Exposed set)

| | | <each group=""></each> | | | | |
|---|---|---|---|---|---|---|
| | | | | | | 5 % CI |
| Symptom | Туре | N | n | % | LL | UL |
| Fatigue | All | | | | | |
| · · | Grade 1 | | | | | |
| | Grade 2 | | | | | |
| | Grade 3 | | | | | |
| | Related* | | | | | |
| | Grade 2 Related | | | | | |
| | Grade 3 Related | | | | | |
| | Onset ≤48h | | | | | |
| | Medical advice | | | | | |
| Gastrointestinal | All | | | | | |
| symptoms | | | | | | |
| yp. | Grade 1 | | | | | |
| | Grade 2 | | | | | |
| | Grade 3 | | | | | |
| | Related* | | | | | |
| | Grade 2 Related | | | | | |
| | Grade 3 Related | | | | | |
| | Onset ≤48h | | | | | |
| | Medical advice | | | | | |
| Headache | All | | | | | |
| | Grade 1 | | | | | |
| | Grade 2 | | | | | |
| | Grade 3 | | | | | |
| | Related* | | | | | |
| | Grade 2 Related | | | | | |
| | Grade 3 Related | | | | | |
| | Onset ≤48h | | | | | |
| | Medical advice | | | | | |
| Fever/(Oral) (°C) | All | | | | | |
| | >38.0 | | | | | |
| | >38.5 | | | | | |
| | >39.0 | | | | | |
| | >39.5 | | | | | |
| | Related* | | | | | |
| | >38.5 Related | | | | | |
| | >39.5 Related | | | | | |
| | Medical advice | | | | | |
| | Modical advice | | | | | |

#### <each group>:

 $30 \text{ PreF} = 30 \mu \text{g PreF}$ 

60 PreF = 60 µg PreF

120 PreF = 120 µg PreF

Control = Placebo

All=any grade>0 for Fatigue, Gastrointestinal symptoms, Headache and any >37.5°C for Temperature/(Oral)

Related\*= any grade>0 for Fatigue, Gastrointestinal symptoms, Headache and any >37.5°C for Temperature/(Oral) considered related to vaccination by the investigator

N=number of vaccinated subjects who returned the diary card

n/% = number/percentage of subjects reporting the AE at least once. Maximum intensity only

95%CI = Exact 95% confidence interval; LL = lower limit, UL = upper limit

Temperatures were coded as follows for adults:

204812 (RSV F-021)

Statistical Analysis Plan Amendment 2 Final

0: < 37.5 °C

1: ≥ 37.5 °C to ≤ 38.5 °C

 $2: > 38.5 \,^{\circ}\text{C} \text{ to} \le 39.5 \,^{\circ}\text{C}$ 

3: > 39.5°C

# Template 22 Percentage of subjects reporting the occurrence of unsolicited symptoms classified by MedDRA Primary System Organ Class and Preferred Term within the 30-day (Days 0-29) post-vaccination period (Exposed set)

| | | | <eac< th=""><th>h group<br/>N =</th><th>&gt;</th></eac<> | h group<br>N = | > |
|---|---|---|---|---|---|
| | | | | 95% | CI |
| Primary System Organ Class (CODE) | Preferred Term (CODE) | n | % | LL | UL |
| At least one symptom | | | | | |
| <each (code)="" soc=""></each> | <each (code)="" pt=""></each> | | | | |

#### <each group>:

30 PreF = 30 µg PreF

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

At least one symptom = at least one symptom experienced (regardless of the MedDRA Preferred Term)

N = number of subjects with at least one administered dose

n/% = number/percentage of subjects reporting at least once the symptom

95% CI= exact 95% confidence interval; LL = Lower Limit, UL = Upper Limit

#### Template 23 Listing of SAEs reported up to study end (Exposed set)

| Group | Sub. | Sex | Country | Race | Age | Verbatim | Preferred | Primary | MED | Dose | Day | Duration | Intensity | Causality | Outcome |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | No. | | | | at | | | System | type | | of | | | | |
| | | | | | onset<br>(Year) | | | Organ<br>Class | | | onset | | | | |
| <each group=""></each> | | | | | | | | | | | | | | | |

#### <each group>:

30 PreF = 30 μg PreF

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

204812 (RSV F-021)

Statistical Analysis Plan Amendment 2 Final

## Template 24 Number (%) of subjects with serious adverse events up to study end (Exposed set)

| | | | <ea< th=""><th>ch gro<br/>N =</th><th>up&gt;</th></ea<> | ch gro<br>N = | up> |
|---|---|---|---|---|---|
| Type of Event | Primary System Organ Class | Preferred Term (CODE) | n* | n | % |
| SAE | At least one symptom | | | | |
| | <each soc=""></each> | <each pt="" term=""></each> | | | |
| Related SAE | At least one symptom | | | | |
| | <each soc=""></each> | <each pt="" term=""></each> | | | |
| Fatal SAE | At least one symptom | | | | |
| | <each soc=""></each> | <each pt="" term=""></each> | | | |
| Related fatal SAE | At least one symptom | | | | |
| | <each soc=""></each> | <each pt="" term=""></each> | | | |

#### <each group>:

30 PreF = 30  $\mu$ g PreF

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

N = number of subjects with the administered dose

n\* = number of events reported

n/% = number/percentage of subjects reporting the symptom at least once

#### **Template 25 Compliance in returning symptom information (Exposed set)**

| Group | Number | Doses | Number | Compliance | Number | Compliance |
|---|---|---|---|---|---|---|
| | of | NOT | of | % | of | % |
| | doses | according to | general SS | general SS | local SS | local SS |
| | | protocol | | | | |
| <each group=""></each> | | | | | | |

#### <each group>:

 $30 \text{ PreF} = 30 \mu \text{g PreF}$ 

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

SS = Symptom screens/sheets used for the collection of local and general solicited AEs

Compliance % = (number of doses with symptom screen/sheet return / number of administered doses) X 100

204812 (RSV F-021)

Statistical Analysis Plan Amendment 2 Final

## Template 26 Number and percentage of subjects taking a concomitant medication during the 7- day (Days 0-6) post -vaccination period (Exposed set)

| | | | <each group<="" th=""><th>&gt;</th><th></th></each> | > | |
|---|---|---|---|---|---|
| | | | | 95% | CI |
| | N | n | % | LL | UL |
| Any | | | | | |
| Any antipyretics | | | | | |
| Prophylactic antipyretics | | | | | |

#### <each group>:

30 PreF = 30 µg PreF

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

N= number of administered doses

n/%= number/percentage of subjects who took the specified concomitant medication at least once during the mentioned period

95% CI = exact 95% confidence interval, LL = Lower Limit, UL = Upper Limit

Template 27 Exploratory comparisons between groups in terms of percentage of subjects reported any Grade 2/3 AE and/or any fever >38.5°C and/or any vaccine-related SAE during the 7-day (Days 0-6) post-vaccination period (Exposed set)

| | | | | | | | | Difference in<br>(Group 1 min | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | | 95 | % CI |
| Group 1 | N | n | % | Group 2 | N | n | % | Difference | % | LL | UL |
| 30 PreF | | | | Control | | | | 30 PreF - Control | | | |
| 60 PreF | | | | Control | | | | 60 PreF - Control | | | |
| 120 PreF | | | | Control | | | | 120 PreF - Control | | | |
| 60 PreF | | | | 30 PreF | | | | 60 PreF - 30 PreF | | | |
| 120 PreF | | | | 30 PreF | | | | 120 PreF - 30 PreF | | | |
| 120 PreF | | | | 60 PreF | | | | 120 PreF - 60 PreF | | | |

#### <each group>:

30 PreF = 30 µg PreF

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

N = Number of subjects with the administered dose

n/% = number/percentage of subjects reporting a specified symptom

95% CI = Standardized asymptotic 95% confidence interval, LL = Lower Limit, UL = Upper Limit

204812 (RSV F-021)

Statistical Analysis Plan Amendment 2 Final

Template 28 Solicited and unsolicited symptoms experienced by at least 5 % of subjects, classified by MedDRA Primary System Organ Class and Preferred Term within the 30-day (Days 0-29) post-vaccination period including number of events - SAE excluded (Exposed set)

| | | <e< th=""><th>ach g<br/>N =</th><th>roup&gt;</th></e<> | ach g<br>N = | roup> |
|---|---|---|---|---|
| Primary System<br>Organ Class<br>(CODE) | Preferred Term<br>(CODE) | n* | n | % |
| At least one symptom | | | | |
| <each soc=""></each> | <each pt="" term=""></each> | | | |

#### <each group>:

 $30 \text{ PreF} = 30 \mu \text{g PreF}$ 

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

At least one symptom = at least one symptom experienced (regardless of the MedDRA Preferred Term)

N = number of subjects with the administered dose

n\* = number of events reported

n/% = number/percentage of subjects reporting the symptom at least once

204812 (RSV F-021)

Statistical Analysis Plan Amendment 2 Final

## Template 29 Distribution of change from baseline in haematology and biochemistry with respect to normal laboratory ranges (Exposed set)

| | | | | | <e< th=""><th>ас</th><th>h gro</th><th>up</th><th>&gt;</th><th></th></e<> | ас | h gro | up | > | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | Uı | | | | | | Α | bove |
| Laboratory parameter | Timing | | N | n | % | n | % | n | % | n | % |
| Alanine Aminotransferase | PI(D7) | Unknown | | | | | | | | | |
| (ALT) | | Below | | | | | | | | | |
| (/ (= 1) | | Within | | | | | | | | | |
| | | Above | | | | | | | | | |
| | PI(D30) | | | | | | | | | | |
| | PI(D60) | | | | | | | | | | |
| | PI(D90) | | | | | | | | | | |
| Aspartate Aminotransferase | PI(D7) | Unknown | | | | | | | | | |
| (AST) | | Below | | | | | | | | | |
| | | Above | | | | | | | | | |
| | PRE(D0) | | | | | | | | | | |
| Creatinine | | | | | | | | | | | |
| Eosinophils | | | | | | | | | | | |
| Haemoglobin | | | | | | | | | | | |
| Lymphocytes | | | | | | | | | | | |
| Neutrophils | | | | | | | | | | | |
| Platelet count | | | | | | | | | | | |
| White Blood Cells (WBC) | | | | | | | | | | | |

#### <each group>:

 $30 \text{ PreF} = 30 \mu \text{g PreF}$ 

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

N = number of subjects with available results for the specified laboratory parameter and timing in a given baseline category

n/% = number/percentage of subjects in the specified category

Below = below the normal laboratory range defined for the specified laboratory parameter

Within = within the normal laboratory range defined for the specified laboratory parameter

Above = above the normal laboratory range defined for the specified laboratory parameter

PI(D7) = Post-vaccination at Day 7

PI(D30) = Post-vaccination at Day 30

PI(D60) = Post-vaccination at Day 60

PI(D90) = Post-vaccination at Day 90

204812 (RSV F-021)

Statistical Analysis Plan Amendment 2 Final

# Template 30 Summary of haematology and biochemistry results by maximum grade from VISIT 2 (D7) up to VISIT 3 (D30) versus baseline (Exposed set)

| | | | | | VIS | SIT2 | (D7) u | | | | 90) | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | <eac< th=""><th></th><th></th><th></th><th></th><th></th><th></th><th></th></eac<> | | | | | | | |
| | | | Unkı | nown | Gra | de 0 | Grad | de 1 | Gra | de 2 | Gra | de 3 | Gra | de 4 |
| Laboratory parameter | Baseline PRE(D0) | N | n | % | n | % | n | % | n | % | n | % | n | % |
| Alanine Aminotransferase (ALT) increase by factor | Unknown | | | | | | | | | | | | | |
| • | Grade 0 | | | | | | | | | | | | | |
| | Grade 1 | | | | | | | | | | | | | |
| | Grade 2 | | | | | | | | | | | | | |
| | Grade 3 | | | | | | | | | | | | | |
| | Grade 4 | | | | | | | | | | | | | |
| | Total | | | | | | | | | | | | | |
| Aspartate Aminotransferase (AST) increase by factor | | | | | | | | | | | | | | |
| Creatinine | | | | | | | | | | | | | | |
| | | | | | | - | | | | | | | | |
| Eosinophils increase | | | | | | | | | | | | | | |
| Hemoglobin decrease | | | | | | | | | | | | | | |
| Lymphocytes decrease | | | | | | | | | | | | | | |
| Neutrophils decrease | | | | | | | | | | | | | | |
| Platelet count decrease | | | | | | | | | | | | | | |
| White Blood Cells (WBC) decrease | | | | | | | | | | | | | | |
| White Blood Cells (WBC) increase | | | | | | | | | | | | | | |

#### <each group>:

 $30 \text{ PreF} = 30 \mu \text{g PreF}$ 

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

N = number of subjects with at least one available result for the specified laboratory parameter and follow-up period n/% = number/percentage of patients reporting at least once the laboratory event when the maximum grading over the follow-up period is considered

204812 (RSV F-021)

Statistical Analysis Plan Amendment 2 Final

## Template 31 Summary of haematology change from baseline by maximum grade from VISIT2 (D7) up to VISIT3 (D30) (Exposed set)

| | | | | VIS | IT2 ( | D7) u | p to | VISI | T5 (D | 90) | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | <each group=""></each> | | | | | | | | | | | |
| | | Unkr | nown | Grad | de 0 | Grad | de 1 | Grade 2 | | Grade 3 | | Grade 4 | |
| Laboratory parameter | N | n | % | n | % | n | % | n | % | n | % | n | % |
| Hemoglobin (Change from baseline) | | | | | | | | | | | | | |

#### <each group>:

 $30 \text{ PreF} = 30 \mu \text{g PreF}$ 

60 PreF = 60 µg PreF

120 PreF = 120  $\mu$ g PreF

Control = Placebo

N = number of subjects with at least one available result for the specified laboratory parameter and follow-up period n/% = number/percentage of subjects reporting at least once the laboratory event when the maximum grading over the follow-up period is considered

## Template 32 Individual results of hemoglobin levels outside of the normal ranges in < group> (Exposed set)



**Note:** This figure is shown as an example. For the unblinded report, one figure per group will be performed. For the blinded report, 4 graphs will be performed each of them presenting pp subjects regardless of treatment (the first pp subjects, from the pp th subject...). The X axis will include Day 0, Day 7 and Day 30. The Y axis will be adapted according to each parameter.

204812 (RSV F-021)

Statistical Analysis Plan Amendment 2 Final

## Template 33 Number and percentage of subjects with anti-RSV-A neutralising antibody titer equal to or above <cut-off> and GMTs (Per protocol set)

| Antibody | | | | ≥cut-off GMT | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | 959 | % CI | | 95% CI | | | |
| | Group | Timing | N | n | % | LL | UL | value | LL | UL | Min | Max |
| Anti-RSV-A<br>Neutralizing<br>Antibody | | PRE | | | | | | | | | | |
| • | | PI(D30) | | | | | | | | | | |
| | | PI(D60) | | | | | | | | | | |
| | | PI(D90) | | | | | | | | | | |

#### <each group>:

 $30 \text{ PreF} = 30 \mu \text{g PreF}$ 

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

GMT = geometric mean antibody titer calculated on all subjects

N = Number of subjects with available results

95% CI = 95% confidence interval; LL = lower limit, UL = upper limit

n/% = number/percentage of subjects with titer equal to or above specified value

MIN/MAX = Minimum/Maximum

PRE= Pre-vaccination at Day 0

PI(D30) = Post-vaccination at Day 30

PI(D60) = Post-vaccination at Day 60

PI(D90) = Post-vaccination at Day 90

204812 (RSV F-021)

Statistical Analysis Plan Amendment 2 Final

## Template 34 Number and percentage of subjects with anti-RSV-A neutralising antibody titer equal to or above <cut-off> and GMTs - by age category (Per protocol set)

| Antibody | | | | | ≥cut-off | | | | | GMT | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | N | | | 95% CI | | | 95% CI | | | |
| | Group | Sub-<br>Group | Timing | | n | % | LL | UL | value | LL | UL | Min | Max |
| Anti-RSV-A<br>Neutralizing<br>Antibody | <each<br>group&gt;</each<br> | 18-32Y | PRE<br>PI(D30)<br>PI(D60)<br>PI(D90) | | | | | | | | | | |
| | | 33-45Y | PRE<br>PI(D30)<br>PI(D60)<br>PI(D90) | | | | | | | | | | |

#### <each group>:

 $30 \text{ PreF} = 30 \mu \text{g PreF}$ 

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

18-32Y = 18-32 years old subjects

33-45Y = 33-45 years old subjects

GMT = geometric mean antibody titer calculated on all subjects

N = Number of subjects with available results

95% CI = 95% confidence interval; LL = lower limit, UL = upper limit

n/% = number/percentage of subjects with titer equal to or above specified value

MIN/MAX = Minimum/Maximum

PRE= Pre-vaccination at Day 0

PI(D30) = Post-vaccination at Day 30

PI(D60) = Post-vaccination at Day 60

PI(D90) = Post-vaccination at Day 90
204812 (RSV F-021)

Statistical Analysis Plan Amendment 2 Final

# Template 35 Geometric mean of the individual ratio of anti-RSV-A neutralising antibody titers at each post-vaccination timepoint compared to prevaccination with 95% CI (Per protocol set)

| | | | | | | | GMT rati | 0 | |
|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | 9 | 5% CI |
| Group | N | Time point description | GMT | Time point description | GMT | Ratio order | Value | LL | UL |
| <each group=""></each> | | PI(D30) | | PRE | | PI(D30) / PRE | | | |
| | | PI(D60) | | PRE | | PI(D60) / PRE | | | |
| | | PI(D90) | | PRE | | PI(D90) / PRE | | | |

#### <each group>:

 $30 \text{ PreF} = 30 \mu \text{g PreF}$ 

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 μg PreF

Control = Placebo

GMT = geometric mean antibody titer

N = Number of subjects with available results at the two considered time points

95% CI = 95% confidence interval; LL = Lower Limit, UL = Upper Limit

PRE= Pre-vaccination at Day 0

PI(D30) = Post-vaccination at Day 30

PI(D60) = Post-vaccination at Day 60

PI(D90) = Post-vaccination at Day 90

Statistical Analysis Plan Amendment 2 Final

Template 36 GMTs and their 95% Cls for anti-RSV-A neutralising antibody at each timepoint (Per protocol set)



 $30 \text{ PreF} = 30 \mu \text{g PreF}$ 

60 PreF = 60 µg PreF

120 PreF = 120 µg PreF

Control = Placebo

GMT = geometric mean antibody titer calculated on all subjects

95% CI = 95% confidence interval

Note: This graph is provided as an example. For each assay separately, this graph will display the 4 groups and the 4 immuno timepoints: PRE, PI(D30), PI(D60) and PI(D90)

Statistical Analysis Plan Amendment 2 Final

Template 37 Kinetics of GMTs for anti-RSV-A neutralising antibody on subjects with results available at all timepoints (Per protocol set)



30 PreF = 30 µg PreF 60 PreF = 60 µg PreF 120 PreF = 120 µg PreF Control = Placebo

GMT = geometric mean antibody titer calculated on subjects with results available at all timepoints **Note:** 

- This graph is provided as an example. For each assay separately, this graph will display the 4 groups and the 4 immuno timepoints PRE, PI(D30), PI(D60) and PI(D90)
- For the kinetic of the estimated GMTs, footnote will be adapted as: GMT = geometric mean antibody titer estimated by the ANOVA model for repeated measures

204812 (RSV F-021)

Statistical Analysis Plan Amendment 2 Final

## Template 38 Distribution of anti-RSV-A neutralising antibody titer (Per protocol set)

| | | | | | <7<br>og2 | | ≥7<br>og2 | | ≥8<br>og2 | _ | ≥9<br>og2 | | :10<br>og2 | | 11<br>og2 | _ | 12<br>g2 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Antibody | Group | Timing | N | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Anti-RSV A Neutralizing Antibody | <each group=""></each> | PRE | | | | | | | | | | | | | | | |
| | | PI(D30) | | | | | | | | | | | | | | | |
| | | PI(D60) | | | | | | | | | | | | | | | |
| | | PI(D90) | | | | | | | | | | | | | | | |

#### <each group>:

 $30 \text{ PreF} = 30 \mu \text{g PreF}$ 

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

N = number of subjects with available results

n/% = number/percentage of subjects with titre within the specified range

PRE = Pre-vaccination at Day 0

PI(D30) = Post-vaccination at Day 30

PI(D60) = Post-vaccination at Day 60

PI(D90) = Post-vaccination at Day 90

#### Template 39 Distribution of anti-Neogenin antibody concentration (Exposed set)

| | | | | | <55<br>g/ml | | ≥55<br>g/ml | | :100<br>g/ml | | 150<br>g/ml | | 200<br>g/ml | | 250<br>g/ml | | 300<br>g/ml |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Antibody | Group | Timing | N | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Anti-neogenin antibody | <each<br>group&gt;</each<br> | PRE | | | | | | | | | | | | | | | |
| , | | PI(D30) | | | | | | | | | | | | | | | |
| | | PI(D60) | | | | | | | | | | | | | | | |
| | | PI(D90) | | | | | | | | | | | | | | | |

#### <each group>:

30 PreF = 30 µg PreF

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

N = number of subjects with available results

n/% = number/percentage of subjects with concentration within the specified range

PRE = Pre-vaccination at Day 0

PI(D30) = Post-vaccination at Day 30

PI(D60) = Post-vaccination at Day 60

PI(D90) = Post-vaccination at Day 90

204812 (RSV F-021) Statistical Analysis Plan Amendment 2 Final

## Template 40 Distribution of fold of anti-RSV-A neutralising antibody titer by pre-vaccination titer category (Per protocol set)

| A (!! ! | | | - · | | <1 | | ≥1 | , | 22 | ≥ | 2.5 | 2 | 3 | ≥4 | + | ≥6 | <u> </u> | <b>∠</b> ୪ | 2 | IU | 21 | 1 | 21 | 2 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Antibody | Group | Sub-group | Timing | N | n S | % I | n የ | / <sub>0</sub> | n 🏸 | n | % | n | % | 'n | % | n % | r | ۱ % | n | % | n ' | % | n ' | % |
| Anti-RSV A Neutralizing | 30 PreF | <7 | PI (D30) | | | | | | | | | | | | | | | | | | | | Ш | |
| Antibody | | | PI (D60) | | | | | | | | | | | | | | | | | | | | Ш | |
| | | | PI (D90) | | | | | | | | | | | | | | | | | | | | Ш | _ |
| | | [7-8] | PI (D30) | | | | | | | | | | | | | | | | | | | | Ш | |
| | | | PI (D60) | | | | | | | | | | | | | | | | | | | | Ш | |
| | | | PI (D90) | | | | | | | | | | | | | | | | | | | | Ш | |
| | | ]8-9] | PI (D30) | | | | | | | | | | | | | | | | | | | | Ш | |
| | | | PI (D60) | | | | | | | | | | | | | | | | | | | | lacksquare | |
| | | 10.401 | PI (D90) | | | | | | | | | | | | | | | | | | | | $\vdash$ | |
| | | ]9-10] | PI (D30) | | | | | | | | | | | | | | | | | | | | $\vdash$ | |
| | | | PI (D60) | | | | | | | | | | | | | | | | | | | | | |
| | | 140 441 | PI (D90) | | | | | | | | | | | | | | | | | | | | lacksquare | _ |
| | | ]10-11] | PI (D30) | | | | | | | | | | | | | | | | | | | | H | |
| | | | PI (D60) | | | | | | | | | | | | | | | | | | | | H | |
| | | 144 401 | PI (D90) | | | | | | | | | | | | | | | | | | | | H | |
| | | ]11-12] | PI (D30) | | | | | | | | | | | | | | | | | | | | $\vdash$ | |
| | | | PI (D60) | | | | | | | | | | | | | | | | | | | | $\vdash$ | |
| | | . 40 | PI (D90) | | | | | | | | | | | | | | | | | | | | H | |
| | | > 12 | PI (D30) | | | | | | | | | | | | | | | | | | | | H | |
| | | | PI (D60)<br>PI (D90) | | | | | | | | | | | | | | | | | | | | H | |
| | | Tatal | | | | | | | | | | | | | | | | | | | | | $\vdash$ | |
| | | Total | PI (D30) | | | | | | | | | | | | | | | | | | | | $\vdash$ | |
| | | | PI (D60) | | | | | | | | | | | | | | | | | | | | H | |
| | 60 D==E | 47 | PI (D90)<br>PI (D30) | | | | | | | | | | | | | | | - | | | | | H | |
| | 60 PreF | <7 | PI (D30) | | | | | | | | | | | | | | | - | | | | | H | |
| | | | | | | | | | | | | | | | | | | - | | | | | H | |
| | | [7 0] | PI (D90) | | | | | | | | | | | | | | | | | | | | H | |
| | | [7-8] | PI (D30) | | | | | | | | | | | | | | | | | | | | H | |
| | | | PI (D60) | | | | | | | | | | | | | | | - | | | | | H | |
| | | 10.01 | PI (D90) | | | | | | | | | | | | | | | - | | | | | H | |
| | | ]8-9] | PI (D30)<br>PI (D60) | | | | | | | | | | | | | | | - | | | | | H | |
| | | | | | | | | | | | | | | | | | | | | | | | H | |
| | | 10.401 | PI (D90) | | | | | | | | | | | | | | | | | | | | H | |
| | | ]9-10] | PI (D30) | | | | | | | | | | | | | | | - | | | | | H | |
| | | | PI (D60) | | | | | | | | | | | | | | | | | | | | $\vdash$ | |
| | | 140 441 | PI (D90)<br>PI (D30) | | + | | | | | | | | | | | | | | | | | | H | |
| | | ]10-11] | PI (D30) | | + | | | | | | | | | | | | | | | | | | H | _ |
| | | | PI (D00) | | + | | | | | | | | | | | | | | | | | | H | _ |
| | | 144 401 | PI (D30) | | | | | | | | | | | | | | | | | | | | $\vdash$ | |
| | | ]11-12] | PI (D30) | | | | | | | | | | | | | | | | | | | | $\vdash$ | |
| | | | PI (D00) | | + | | | | | | | | | | | | | | | | | | H | _ |
| | | > 12 | PI (D90) | $\vdash$ | + | - | | + | + | | | | | $\dashv$ | | | - | + | - | | H | | H | |
| | | <i>&gt;</i> 12 | PI (D30) | H | + | - | | + | + | 1 | | | | $\dashv$ | | | + | - | - | 1 | $\vdash$ | | $\vdash$ | |
| | | | PI (D00) | $\vdash$ | + | - | - | - | + | | | | | - | | | + | + | | - | H | | H | |
| | | Total | PI (D90) | H | + | - | | + | + | 1 | | | | $\dashv$ | | | + | - | - | 1 | $\vdash$ | | $\vdash$ | |
| | | Total | PI (D30) | $\vdash$ | + | - | + | + | + | + | | | | | | | + | + | | - | | | H | |
| | | | PI (D60) | | $\perp$ | - | | | $\perp$ | | | | | - | | | | + | - | | | | $\vdash$ | |

204812 (RSV F-021)

Statistical Analysis Plan Amendment 2 Final

| | | | | | < | 1 | ≥ | 1 | ≥2 | 2 ≥ | 2.5 | ; ≥ | ≥3 | ≥ | 4 | ≥ | 6 | ≥ | :8 | ≥′ | 10 | ≥1 | 1 | ≥′ |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Antibody | Group | Sub-group | Timing | N | | | | | | | 1 % | | | | | | | | | | | | | |
| | 120 PreF | <7 | PI (D30) | | 1 | | | | | - | | T | 1 | | | | | | | | | | - | |
| | 1201101 | ' | PI (D60) | | 1 | | | | | | | | | | | | | H | | Ħ | | H | | |
| | | | PI (D90) | | + | | | | | | | | | | | | | H | | H | | H | | |
| | | [7-8] | PI (D30) | H | - | | | | | | | | | | | | | H | | H | | H | | |
| | | [1-0] | PI (D60) | | | | | | | | | | | | | | | H | | H | | H | | _ |
| | | | PI (D00) | $\vdash$ | | | | | | | | + | | | | | | | <u> </u> | | - | | _ | _ |
| | | 10.01 | | | | | | | | | | | - | | | | | Щ | | Н | | Н | _ | _ |
| | | ]8-9] | PI (D30) | | _ | | | | | | | - | | | | | | | _ | | - | | | _ |
| | | | PI (D60) | | | | | | | | | | | | | | | Ш | | Ш | | Ш | | _ |
| | | | PI (D90) | | | | | | | | | | | | | | | | | Ш | L | Ш | | _ |
| | | ]9-10] | PI (D30) | | | | | | | | | | | | | | | | | | L | | | _ |
| | | | PI (D60) | | | | | | | | | | | | | | | | | Ш | L | Ш | | - |
| | | | PI (D90) | | | | | | | | | | | | | | | | L | | | | | _ |
| | | ]10-11] | PI (D30) | | | | | | | | | | | | | | | | | | | | | |
| | | | PI (D60) | | | | | | | | | | | | | | | | | | | | | _ |
| | | | PI (D90) | | | | | | | | | | | | | | | | | | | | | |
| | | ]11-12] | PI (D30) | | | | | | | | | | | | | | | | | | | | | |
| | | | PI (D60) | | | | | | | | | | | | | | | | | | | | | ì |
| | | | PI (D90) | | | | | | | | | | | | | | | | | | | | | |
| | | > 12 | PI (D30) | | | | | | | | | | | | | | | | | П | | | | |
| | | | PI (D60) | | | | | | | | | | | | | | | | | | | | | Τ |
| | | | PI (D90) | | | | | | | | | | | | | | | | | П | | П | | _ |
| | | Total | PI (D30) | | | | | | | | | T | | | | | | | | | | | | _ |
| | | | PI (D60) | | | | | | | | | | | | | | | | | П | | П | | _ |
| | | | PI (D90) | | | | | | | | | | | | | | | | | H | | | | |
| | Control | <7 | PI (D30) | | | | | | | | | | | | | | | | | H | | | | |
| | Control | 1 | PI (D60) | | | | | | | | | + | | | | | | | | H | | | _ | _ |
| | | | PI (D90) | H | - | | | | | | | | | | | | | H | | H | | H | | |
| | | [7-8] | PI (D30) | H | - | | | | | | | | | | | | | H | | H | | H | | |
| | | [1-0] | PI (D60) | | + | | = | | | | | + | 1 | | | | | H | _ | H | | H | _ | |
| | | | PI (D00) | | | | | | | | | | | | | | | H | | H | | H | _ | _ |
| | | 10.01 | PI (D30) | | | | | | | | | | | | | | | H | | H | | H | _ | _ |
| | | ]8-9] | | $\vdash$ | | | | | | | | + | | | | | | | <u> </u> | | - | | _ | _ |
| | | | PI (D60) | | _ | | | | | | | - | | | | | | | _ | | | | | |
| | | 10.401 | PI (D90) | | _ | | | | | | | - | | | | | | | _ | | | | | _ |
| | | ]9-10] | PI (D30) | | | | | | | | | | | | | | | Ш | | Ш | | Ш | | |
| | | | PI (D60) | | | | | | | | | | | | | | | | _ | | | | | |
| | | | PI (D90) | | | | | | | | | | | | | | | | | | L | | | |
| | | ]10-11] | PI (D30) | | | | | | | | | | | | | | | | | Ш | L | Ш | | - |
| | | | PI (D60) | | | | | | | | | | | | | | | | L | | | | | |
| | | | PI (D90) | | | | | | | | | | | | | | | | | | | | | <u> </u> |
| | | ]11-12] | PI (D30) | | | | | | | | | | | | | | | | | | | | | |
| | | | PI (D60) | | | | | | | | | | | | | | | | | | | | | |
| | | | PI (D90) | | | | | | | | | | | | | | | | | | | | | ı |
| | | > 12 | PI (D30) | | | | | | | | | | | | | | | | | | | | | |
| | | | PI (D60) | | T | | | | | | | | | | | | | | | П | | | | |
| | | | PI (D90) | | T | | | | | 1 | | T | | П | | | | | | П | | П | | |
| | | Total | PI (D30) | H | T | | Ħ | | | t | | T | | | | | | Ħ | | Ħ | | П | | |
| | | | PI (D60) | | 1 | | | | | | $\top$ | | | H | | | | Ħ | | Н | | Н | | _ |
| | | | PI (D90) | Н | + | | Ħ | | $\dashv$ | 1 | + | t | 1 | H | | П | | H | | H | | H | | |

#### <each group>:

30 PreF = 30 μg PreF 60 PreF = 60 μg PreF 120 PreF = 120 μg PreF

Control = Placebo

N = number of subjects with available results

Statistical Analysis Plan Amendment 2 Final

n/% = number/percentage of subjects with titer within the specified range

PI(D30) = Post-vaccination at Day 30

PI(D60) = Post-vaccination at Day 60

PI(D90) = Post-vaccination at Day 90

## Template 41 Distribution of fold of anti-neogenin antibody concentration (Exposed set)

| | | | | • | <1 | > | =1 | >= | =1.5 | > | =2 | >= | 2.5 | > | =3 | >= | 3.5 | >: | =4 | >= | 4.5 | > | =5 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Antibody | Group | Timing | N | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Anti-neogenin antibody | <each group=""></each> | PI(D30) | | | | | | | | | | | | | | | | | | | | | |
| | | PI(D60) | | | | | | | | | | | | | | | | | | | | | |
| | | PI(D90) | | | | | | | | | | | | | | | | | | | | | |

#### <each group>:

30 PreF = 30 µg PreF

60 PreF = 60 µg PreF

120 PreF = 120 µg PreF

Control = Placebo

N = number of subjects with available results

n/% = number/percentage of subjects with concentration within the specified range

PI(D30) = Post-vaccination at Day 30

PI(D60) = Post-vaccination at Day 60

PI(D90) = Post-vaccination at Day 90

Template 42 Reverse cumulative distribution curves for anti-RSV-A neutralising antibody titers in each group at <each time point> (Per protocol set)



30 PreF = 30 µg PreF

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

Note: This graph is provided as an example. The same graph will be provided for each time point and each assay comparing the values of the groups:30 PreF, 60 PreF, 120 PreF and Control.

204812 (RSV F-021)

Statistical Analysis Plan Amendment 2 Final

Template 43 Individual results of anti-RSV-A neutralising antibody titer at Day <30/60/90> versus pre-vaccination in <each group> and Control (Per protocol set)



#### <each group>:

30 PreF = 30 μg PreF

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

Note: This graph is provided as an example. The same graph will be generated for each assay and each timepoint separately (Day 30, 60, 90):

204812 (RSV F-021)

Statistical Analysis Plan Amendment 2 Final

## Template 44 Vaccine response for anti-RSV-A neutralising antibody titer at each post-vaccination timepoint (Per protocol set)

| | | | | | | Vaccine | respon | se* |
|---|---|---|---|---|---|---|---|---|
| | | | | | | | 9 | 5% CI |
| Antibody | Group | Post-vaccination timing | Pre-vaccination category (log2) | N | n | % | LL | UL |
| <each<br>antibody&gt;</each<br> | <each group=""></each> | PI(D30) | <7 | | | | | |
| | | | [7-8] | | | | | |
| | | | ]8-10] | | | | | |
| | | | >10 | | | | | |
| | | | Total | | | | | |
| | | PI(D60) | <7 | | | | | |
| | | | [7-8] | | | | | |
| | | | ]8-10] | | | | | |
| | | | >10 | | | | | |
| | | | Total | | | | | |
| | | PI(D90) | <7 | | | | | |
| | | | [7-8] | | | | | |
| | | | ]8-10] | | | | | |
| | | | >10 | | | | | |
| | | | Total | | | | | |

#### <each group>:

30 PreF = 30 µg PreF

60 PreF = 60 µg PreF

120 PreF = 120 µg PreF

Control = Placebo

Total = all subjects with pre-vaccination result available

\*Vaccine response defined as:

For subjects with pre-vaccination titer <7 log2: antibody titer at post-vaccination>= 4 fold the pre-vaccination antibody titer For subjects with pre-vaccination titer in [7-8] log2: antibody titer at post-vaccination >= 3 fold the pre-vaccination antibody titer For subjects with pre-vaccination titer in [8-10] log2: antibody titer at post-vaccination >= 2.5 fold the pre-vaccination antibody titer For subjects with pre-vaccination titer >10 log2: antibody titer at post-vaccination >= 1 fold the pre-vaccination antibody titer

N = number of subjects with both pre- and post-vaccination results available

n/% = number/percentage of responders

95% CI = exact 95% confidence interval, LL = Lower Limit, UL = Upper Limit

PI(D30) = Post-vaccination at Day 30

PI(D60) = Post-vaccination at Day 60

PI(D90) = Post-vaccination at Day 90

204812 (RSV F-021)

Statistical Analysis Plan Amendment 2 Final

## Template 45 Estimated GMTs and 95% CIs for anti-RSV-A neutralising antibody titre (Per protocol set)

| | | | | Est | imate | d GMT |
|---|---|---|---|---|---|---|
| | | | | | 9 | 5% CI |
| Antibody | Group | Timing | N | value | LL | UL |
| Anti-RSV-A | <each< td=""><td>PRE</td><td></td><td></td><td></td><td></td></each<> | PRE | | | | |
| Neutralizing | group> | | | | | |
| Antibody | | | | | | |
| | | PI(D30) | | | | |
| | | PI(D60) | | | | |
| | | PI(D90) | | | | |

<each group>:

 $30 \text{ PreF} = 30 \mu \text{g PreF}$ 

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

GMT = geometric mean antibody titer estimated by the ANOVA model for repeated measures

N = Number of subjects with available results

95% CI = 95% confidence interval (ANOVA model); LL = lower limit, UL = upper limit

PRE= Pre-vaccination at Day 0

PI(D30) = Post-vaccination at Day 30

PI(D60) = Post-vaccination at Day 60

PI(D90) = Post-vaccination at Day 90

## Template 46 Exploratory comparisons (GMT ratios) between RSV groups with corresponding 95% confidence interval for anti-RSV A neutralizing antibody titre at Day 30 (Per protocol set)

| | | | | | | | | GI | /IT ratio | 0 | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | | Tukey's | 95% CI |
| Antibody | Timepoint | Group | N | <b>GMT</b> | Group | N | <b>GMT</b> | Ratio order | Value | LL | UL |
| | - | description | | | description | | | | | | |
| Anti-RSV A | PI(D30) | 120 PreF | | | 30 PreF | | | 120 PreF/30 PreF | | | |
| Neutralizing | , , | 120 PreF | | | 60 PreF | | | 120 PreF/60 PreF | | | |
| Antibody | | 60 PreF | | | 30 PreF | | | 60 PreF/30 PreF | | | |

30 PreF = 30 µg PreF

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

antibody titre estimated by the ANCOVA model

N = Number of subjects with pre-vaccination results available

Tukey's 95% CI = 95% confidence interval for the GMT ratio (ANCOVA model, Tukey's adjustment), LL = lower limit, UL = upper limit

Pvalue of ANCOVA model is xxxx

PI(D30) = Post-vaccination at Day 30

Statistical Analysis Plan Amendment 2 Final

Template 47 Individual kinetics of anti-neogenin antibody concentrations by group (Exposed set)



 $30 \text{ PreF} = 30 \mu \text{g PreF}$ 

60 PreF = 60 µg PreF

120 PreF = 120 µg PreF

Control = Placebo

Note: This graph is provided as an example. This graph will display the 4 groups and the 4 immuno timepoints: PRE, PI(D30), PI(D60) and PI(D90)

204812 (RSV F-021)

Statistical Analysis Plan Amendment 2 Final

# Template 48 GM of individual ratios (fold increase post over pre) and their 95% Cls for anti-RSV F IgG1 and IgG total antibody assays and each group, at <Day xx> (Per protocol set)



30 PreF = 30 μg PreF 60 PreF = 60 μg PreF

120 PreF = 120 µg PreF

Control = Placebo

Note: this graph is provided as an example. It will be adapted to display IgG total and Ig1 only, and the 4 groups: 30 PreF, 60 PreF, 120 PreF, Control.

204812 (RSV F-021)

Statistical Analysis Plan Amendment 2 Final

# Template 49 Exploratory comparisons (GM ratios of fold increase post/pre) between RSV groups with corresponding 95% confidence interval for anti-RSV F antibody concentrations (IgG Total) at Day 30 (Per protocol set)

| | | | | | | | G | MF rati | 0 | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | | ukey s<br>5% Cl |
| Antibody | Timepoint | Group description | N | Group description | N | GMF | Ratio order | Value | LL | UL |
| anti-RSV F antibody<br>(IgG Total) | PI(D30) | 120 PreF | | 60 PreF | | | 120 Pre/60<br>PreF | | | |
| , | | 120 PreF | | 30 PreF | | | 120 PreF/30<br>PreF | | | |
| | | 60 PreF | | 30 PreF | | | 60 PreF/30<br>PreF | | | |

30 PreF = 30 µg PreF

60 PreF = 60 µg PreF

120 PreF = 120 µg PreF

Antibody concentration estimated by the ANOVA model

GMF = Geometric mean of fold increase

N = Number of subjects with pre-vaccination results available

Tukey's 95% CI = 95% confidence interval for the GMF ratio (ANOVA model, Tukey's adjustment), LL = lower limit, UL = upper limit

Pvalue of ANOVA model at PI(D30) is: xxxx

PI(D30) = Post-vaccination at Day 30

Template 50 Comparisons of GM ratios with corresponding 95% confidence interval between anti-RSV F antibody concentrations (IgG Total) and anti-RSV-A neutralising antibody titers at pre-vaccination (Per protocol set)

| | | | | | | | | | GI | / rati | 0 |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | 95% | √ CI | | 95% | 6 CI | | 95% | % CI |
| Timing | Group<br>description | N | IgG Total<br>GMC | LL | UL | RSV-A neut<br>GMT | LL | UL | Value | LL | UL |
| PRE(D0) | <each group=""></each> | | | | | | | | | | |
| PRE(D0) | | | | | | | | | | | |
| PRE(D0) | | | | | | | | | | | |
| PRE(D0) | | | | | | | | | | | |

<each group>:

30 PreF = 30 µg PreF

60 PreF = 60 μg PreF

120 PreF = 120 µg PreF

Control = Placebo

N = Number of subjects with available results at Day30 and pre-vaccination for IgG Total and RSV-A neut

GMC = Geometric mean antibody concentration calculated on all subjects for IgG Total

GMT = Geometric mean antibody titre calculated on all subjects for RSV-A neut

GM Ratio=Geometric mean of individual ratio of IgG Total to RSV-A neut for each group

95% CI = 95% confidence interval; LL = lower limit, UL = upper limit

PRE= Pre-vaccination at Day 0

204812 (RSV F-021)

Statistical Analysis Plan Amendment 2 Final

# Template 51 Exploratory comparisons (GM ratios of fold increase post/pre) with corresponding 95% confidence interval between anti-RSV F antibody concentrations (IgG Total) and anti-RSV-A neutralising antibody titers at Day 30 (Per protocol set)

| | | | | | | | | | GN | IF Ra | tio |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | | 95 | % CI |
| Timepoint | Group | N | IgG Total | 95% | CI | RSV-A neut | 95% | | Value | LL | UL |
| - | - | | ĞMF | LL | UL | GMF | LL | UL | | | |
| PI(D30)/PRE | <each group=""></each> | | | | | | | | | | |
| PI(D30)/PRE | | | | | | | | | | | |
| PI(D30)/PRE | | | | | | | | | | | |
| PI(D30)/PRE | | | | | | | | | | | |

<each group>:

30 PreF = 30 μg PreF

60 PreF = 60 µg PreF

120 PreF = 120 µg PreF

Control = Placebo

N = Number of subjects with available results at the two considered time points for lgG Total and anti-RSV-A GMF = Geometric mean of fold increase

GMF Ratio= Geometric mean of individual ratio of fold increase for each group

95% CI = 95% confidence interval; LL = lower limit, UL = upper limit

PRE= Pre-vaccination at Day 0

PI(D30) = Post-vaccination at Day 30

Template 52 Desirability index of immunogenicity during the 30-day (Days 0-29) post-vaccination period (Per protocol set)

| Group | GMT | LL1 | DI1 | GMC | LL2 | DI2 | DI |
|------------------------|-----|-----|-----|-----|-----|-----|----|
| <each group=""></each> | | | | | | | |

<each group>:

30 PreF = 30 μg PreF

60 PreF = 60 µg PreF

120 PreF = 120 µg PreF

Control = Placebo

GMT = estimated log2-scale GMT adjusted for pre-vaccination titres for neutralising anti-RSV-A

GMC = estimated log10-scale GMC adjusted for pre-vaccination concentrations for PCA

LL1 = estimated log2-scale lower limit adjusted for pre-vaccination titres for neutralising anti-RSV-A

LL2 = estimated log10-scale lower limit adjusted for pre-vaccination concentrations for PCA

DI1 = desirability index for neutralising anti-RSV-A

DI2 = desirability index for PCA concentrations

DI = immunogenicity index

204812 (RSV F-021)

Statistical Analysis Plan Amendment 2 Final

## Template 53 Desirability index of reactogenicity during the 7-day (Days 0-6) post-vaccination period (Exposed set)

| Group | Incidence Rate<br>(I民 ) | Incidence Rate<br>(IR2) | DR1 | DR2 | DR |
|---|---|---|---|---|---|
| <each group=""></each> | | | | | |

<each group>:

30 PreF = 30 μg PreF

 $60 \text{ PreF} = 60 \mu\text{gPreF}$ 

120 PreF = 120 μg PreF

Control = Placebo

IR = incidence rate estimated by the model for any Grade 2/3 general AEs and any related SAEs

IR2 = incidence rate estimated by the model for Grade 2/3 fever

DR1 = desirability index for any Grade 2/3 general AEs and any related SAEs

DR2 = desirability index for Grade 2/3 fever

DR = reactogenicity index

## Template 54 Desirability index based on reactogenicity and safety (Exposed set up to Day 7) and immunogenicity (Per protocol set up to Day 30)

| Group | Reactogenicity Index | | Immunogenicity Index | | Index | Overall Desirability Index | |
|---|---|---|---|---|---|---|---|
| | DR1 | DR2 | DR | DI1 | DI2 | DI | DR <sup>0.4</sup> * DI <sup>0.6</sup> |
| <each group=""></each> | | | | | | | |

<each group>:

30 PreF = 30 μg PreF

60 PreF = 60 µg PreF

120 PreF = 120 µg PreF

Control = Placebo

DR1 = desirability index for any Grade 2/3 general AEs and any related SAEs

DR2 = desirability index for Grade 2/3 fever

DR = reactogenicity index

DI1 = desirability index for neutralising anti-RSV-A

DI2 = desirability index for PCA concentrations

DI = immunogenicity index

| | Statistical Analysis Plan Amendment 3 Final |
|---|---|
| <b>gsk</b> GlaxoSmithKline | Statistical Analysis Plan |
| Detailed Title: | A Phase II, randomised, observer-blind, controlled, multi-country study to rank different formulations of GSK Biologicals' investigational RSV vaccine (GSK3003891A), based on immunogenicity, reactogenicity and safety, when administered to healthy women, aged 18 – 45 years. |
| eTrack study number and<br>Abbreviated | 204812 (RSV F-021) |
| Scope: | All data pertaining to the above study. |
| <b>Date of Statistical Analysis</b> | Final: Amendment 3 (15-Mar-2018) |
| Plan | Amendment 2 (09-Nov-2017) |
| | Amendment 1 (21-Jul-2017) |
| | Version 2.0 (10-Nov-2016) |
| | Version 1.0 (25-Aug-2016 |
| Co-ordinating author: | PPD (Statistician) |
| Reviewed by: | (Clinical and Epidemiology Project Lead) |
| | (Clinical Research and Development Lead) |
| | (Lead statistician) |
| | (Lead statistical analyst) |
| | (Scientific writer) |
| | (Regulatory Affair) |
| | (SERM physician) |
| | (Public disclosure representative) |
| Approved by: | PPD (Clinical Research and Development Lead) |
| | (Lead statistician) |
| | (Lead stat analyst) |
| | (Lead scientific writer) |

APP 9000058193 Statistical Analysis Plan Template (Effective date: 14 April 2017)

204812 (RSV F-021) Statistical Analysis Plan Amendment 3 Final

#### **TABLE OF CONTENTS**

| | | | | | PAGE |
|---|---|---|---|---|---|
| LIS | T OF A | BBREVIA <sup>-</sup> | TIONS | | 10 |
| 1. | DOCU | MENT HIS | STORY | | 12 |
| 2. | STUD | Y DESIGN | ١ | | 17 |
| 3. | OBJEC | CTIVES | | | 20 |
| 0. | 3.1. | | | | |
| | 3.2. | , | , | S | |
| | 3.3. | | | | |
| 4. | ENDP | OINTS | | | 20 |
| | 4.1. | Primary. | | | 20 |
| | 4.2. | Seconda | ry | | 21 |
| | 4.3. | Tertiary. | | | 21 |
| 5. | ANALY | SIS SET | S | | 21 |
| | 5.1. | Definition | າ | | 21 |
| | | 5.1.1. | | Set (ES) | |
| | | 5.1.2. | | col Set (PPS) for analysis of immunogenicity | |
| | 5.2. | | | ng data from Analysis Sets | |
| | | 5.2.1. | | from Exposed Set (ES) | |
| | | 5.2.2. | | from Per-protocol analysis Set (PPS) | |
| | | | 5.2.2.1. | | |
| | | | | Right censored Data | |
| | <b>5</b> 0 | 1 | 5.2.2.3. | Visit-specific censored Data | 25 |
| | 5.3. | | | eviation not leading to elimination from per- | 25 |
| _ | OT 4 TU | 071041 4 | | | 0.5 |
| 6. | | | | | |
| | 6.1. | | apny | follows a way being the analysis and a way be wishing a barrow of | 26 |
| | | 6.1.1. | | f demographics/baseline characteristics planned | 26 |
| | 6.2. | Immunoc | • | | |
| | 0.2. | 6.2.1. | | f immunogenicity planned in the protocol | |
| | | 0.2 | 6.2.1.1. | Within group analysis | |
| | | | 6.2.1.2. | Between group assessment | |
| | | 6.2.2. | - | considerations | |
| | 6.3. | Analysis | | | |
| | | 6.3.1. | | f safety planned in the protocol | |
| | | | | Within group analysis | |
| | | | 6.3.1.2. | Between group assessment | |
| | 6.4. | Analysis | for ranking | RSV formulations | 31 |
| | | 6.4.1. | | of desirability in the context of Simulations | |
| | | 6.4.2. | | ndpoints | |
| | 6.5. | Analysis | of medically | y attended RTIs | 32 |
| 7. | ANALY | SIS INTE | RPRETAT | ION | 32 |

| | | | | 204812 (RSV I | |
|---|---|---|---|---|---|
| _ | | | | Statistical Analysis Plan Amendment 3 | |
| 8. | | | | | |
| | 8.1.<br>8.2. | | | analyses | |
| | 0.2. | Statistica | a considerations for interim | analyses | აა |
| 9. | CHAN | GES FRO | )M PLANNED ANALYSES. | | 34 |
| 10. | LIST C | F FINAL | REPORT TABLES, LISTIN | GS AND FIGURES | 37 |
| 11. | ANNE | X 1 STAN | IDARD DATA DERIVATION | NRULE AND STATISTICAL | |
| | METH | | | | 38 |
| | 11.1. | Statistica | al Method References | | 38 |
| | 11.2. | | | | |
| | | 11.2.1. | | | |
| | | 11.2.2.<br>11.2.3. | | | |
| | | 11.2.3. | | | |
| | | 11.2.5. | | | |
| | | 11.2.6. | | yed | |
| 12. | ANNE | X 2: SUM | MARY ON ELIMINATION C | CODES | 43 |
| 13. | | | | AND OVERALL DESIRABILITY | 12 |
| | INDEX | ٠ | | | 43 |
| 14. | ANNE | X 4: STUI | DY SPECIFIC MOCK TFL | | 48 |

204812 (RSV F-021) Statistical Analysis Plan Amendment 3 Final

#### **LIST OF TABLES**

| | | PAGE |
|---------|--------------------------------------------------|------|
| Table 1 | Study groups and epochs foreseen in the study | 18 |
| Table 2 | Study groups and treatment foreseen in the study | 18 |
| Table 3 | Blinding of study epochs | 18 |

204812 (RSV F-021) Statistical Analysis Plan Amendment 3 Final

#### **LIST OF FIGURES**

| | | PAGE |
|---|---|---|
| Figure 1 | Study design overview | 17 |
| Figure 2 | Desirability function for the incidence rate of Grade 2/3 general AEs and related SAEs - for each investigational RSV vaccine formulation | 44 |
| Figure 3 | Desirability function for the incidence rate of Grade 2/3 fever - for each investigational RSV vaccine formulation | 45 |
| Figure 4 | Desirability function for neutralising anti-RSV-A GMTs - for each investigational RSV vaccine formulation | 46 |
| Figure 5 | Desirability function for PCA concentrations - for each investigational RSV vaccine formulation | 47 |

204812 (RSV F-021) Statistical Analysis Plan Amendment 3 Final

#### **LIST OF TEMPLATE**

| | PA | GE |
|---|---|---|
| Template 1 | Number of subjects enrolled into the study as well as the number of subjects excluded from the PPS analyses with reasons for exclusion | .51 |
| Template 2 | Number of subjects vaccinated, completed and withdrawn with reason for withdrawal (Exposed set) | .51 |
| Template 3 | Number of subjects vaccinated, completed and withdrawn with reason for withdrawal (Exposed set) | . 52 |
| Template 4 | Number of subjects at each visit and list of withdrawn subjects (Exposed set) | . 52 |
| Template 5 | Summary of demographic characteristics (Per Protocol Set) | . 53 |
| Template 6 | Summary of demographic characteristics by age category (Exposed set) | . 54 |
| Template 7 | Number of subjects by center (Exposed set) | . 55 |
| Template 8 | Number of subjects by center for each age category (Exposed set) | |
| Template 9 | Number of subjects by country and center (Exposed set) | . 55 |
| Template 10 | Deviations from specifications for age and intervals between study visits (Exposed set) | . 56 |
| Template 11 | Summary of vital signs characteristics at VISIT 1 (Day 0) (Exposed set) | . 57 |
| Template 12 | Study Population (Exposed set) | . 58 |
| Template 13 | Number of enrolled subjects by country | . 59 |
| Template 14 | Number of enrolled subjects by age category | . 59 |
| Template 15 | Minimum and maximum activity dates (Exposed set) | . 59 |
| Template 16 | Incidence and nature of symptoms (solicited and unsolicited reported during the 7-day (Days 0-6) post-vaccination period (Exposed set) | .60 |
| Template 17 | Daily prevalence of any fever during the 7-day (Days 0-6) post-vaccination period (Exposed set) | .60 |
| Template 18 | Incidence of solicited local symptoms reported during the 7-day (Days 0-6) post-vaccination period (Exposed set) | .61 |

204812 (RSV F-021)

| Template 19 | Statistical Analysis Plan Amendment 3 Fina Incidence of solicited local symptoms reported during the 7-day |
|---|---|
| remplate re | (Days 0-6) post-vaccination period by maximum intensity (Exposed set) |
| Template 20 | Incidence of solicited general symptoms reported during the 7-day (Days 0-6) post-vaccination period (Exposed set)6 |
| Template 21 | Incidence of solicited general symptoms reported during the 7-day (Days 0-6) post-vaccination period by maximum intensity (Exposed set) |
| Template 22 | Percentage of subjects reporting the occurrence of unsolicited symptoms classified by MedDRA Primary System Organ Class and Preferred Term within the 30-day (Days 0-29) post-vaccination period (Exposed set) |
| Template 23 | Percentage of subjects reporting the occurrence of unsolicited symptoms classified by MedDRA Primary System Organ Class and Preferred Term within the 30-day (Days 0-29) post-vaccination period (Exposed set) |
| Template 24 | Listing of SAEs reported up to study end (Exposed set)6 |
| Template 25 | Number (%) of subjects with serious adverse events up to Day 7 (Exposed set)6 |
| Template 26 | Compliance in returning symptom information (Exposed set)6 |
| Template 27 | Number and percentage of subjects taking a concomitant medication during the 7- day (Days 0-6) post -vaccination period (Exposed set) |
| Template 28 | Exploratory comparisons between groups in terms of percentage of subjects reported any Grade 2/3 AE and/or any fever >38.5°C and/or any vaccine-related SAE during the 7-day (Days 0-6) post-vaccination period (Exposed set) |
| Template 29 | Solicited and unsolicited symptoms experienced by at least 5 % of subjects, classified by MedDRA Primary System Organ Class and Preferred Term within the 30-day (Days 0-29) post-vaccination period including number of events - SAE excluded (Exposed set) |
| Template 30 | Distribution of change from baseline in haematology and biochemistry with respect to normal laboratory ranges (Exposed set) |
| Template 31 | Summary of haematology and biochemistry results by maximum grade from VISIT 2 (D7) up to VISIT 3 (D30) versus baseline (Exposed set) |

204812 (RSV F-021)

| | Statistical Analysis Plan Amendment 3 Fina |
|---|---|
| Template 32 | Summary of haematology and biochemistry results by maximum grade in the specified category from VISIT 2 (D7) up to VISIT 3 (D30) versus baseline (Exposed set) |
| Template 33 | Summary of haematology change from baseline by maximum grade from VISIT2 (D7) up to VISIT3 (D30) (Exposed set) |
| Template 34 | Summary of haematology change from baseline by maximum grade in the specified category from VISIT2 (D7) up to VISIT3 (D30) (Exposed set) |
| Template 35 | Individual results of hemoglobin levels outside of the normal ranges in < group> (Exposed set) |
| Template 36 | Number and percentage of subjects with anti-RSV-A neutralising antibody titer equal to or above <cut-off> and GMTs (Per protocol set)</cut-off> |
| Template 37 | Number and percentage of subjects with anti-RSV-A neutralising antibody titer equal to or above <cut-off> and GMTs - by age category (Per protocol set)</cut-off> |
| Template 38 | Geometric mean of the individual ratio of anti-RSV-A neutralising antibody titers at each post-vaccination timepoint compared to pre-vaccination with 95% CI (Per protocol set) |
| Template 39 | GMTs and their 95% CIs for anti-RSV-A neutralising antibody at each timepoint (Per protocol set) |
| Template 40 | Kinetics of GMTs for anti-RSV-A neutralising antibody on subjects with results available at all timepoints (Per protocol set)81 |
| Template 41 | Distribution of anti-Neogenin antibody concentration (Exposed set) |
| Template 42 | Distribution of fold of anti-neogenin antibody concentration (Exposed set)82 |
| Template 43 | Distribution of anti-RSV-A neutralising antibody titer (Per protocol set)83 |
| Template 44 | Distribution of fold of anti-RSV-A neutralising antibody titer by pre-vaccination titer category (Per protocol set)84 |
| Template 45 | Distribution of fold of anti-RSV-A neutralising antibody titer by cumulative pre-vaccination titer category (Per protocol set) |
| Template 46 | Reverse cumulative distribution curves for anti-RSV-A neutralising antibody titers in each group at <each point="" time=""> (Per protocol set)</each> |

204812 (RSV F-021)

| | Statistical Analysis Plan Amendment 3 | |
|---|---|---|
| Template 47 | Individual results of anti-RSV-A neutralising antibody titer at Day <30/60/90> versus pre-vaccination in <each group=""> and Control (Per protocol set)</each> | |
| Template 48 | Vaccine response for anti-RSV-A neutralising antibody titer at each post-vaccination timepoint (Per protocol set) | 91 |
| Template 49 | Estimated GMTs and 95% CIs for anti-RSV-A neutralising antibody titre (Per protocol set) | 92 |
| Template 50 | Exploratory comparisons (GMT ratios) between RSV groups with corresponding 95% confidence interval for anti-RSV A neutralizing antibody titre at Day 30 (Per protocol set) | 92 |
| Template 51 | Individual kinetics of anti-neogenin antibody concentrations by group (Exposed set) | 93 |
| Template 52 | GM of individual ratios (fold increase post over pre) and their 95% CIs for anti-RSV F IgG1 and IgG total antibody assays and each group, at <day xx=""> (Per protocol set)</day> | 94 |
| Template 53 | Exploratory comparisons (GM ratios of fold increase post/pre) between RSV groups with corresponding 95% confidence interval for anti-RSV F antibody concentrations (IgG Total) at Day 30 (Per protocol set) | 95 |
| Template 54 | Comparisons of GM ratios with corresponding 95% confidence interval between anti-RSV F antibody concentrations (IgG Total) and anti-RSV-A neutralising antibody titers at pre-vaccination (Per protocol set) | 96 |
| Template 55 | Exploratory comparisons (GM ratios of fold increase post/pre) with corresponding 95% confidence interval between anti-RSV F antibody concentrations (IgG Total) and anti-RSV-A neutralising antibody titers at Day 30 (Per protocol set) | 97 |
| Template 56 | Desirability index of immunogenicity during the 30-day (Days 0-29) post-vaccination period (Per protocol set) | 98 |
| Template 57 | Desirability index of reactogenicity during the 7-day (Days 0-6) post-vaccination period (Exposed set) | 98 |
| Template 58 | Desirability index based on reactogenicity and safety (Exposed set up to Day 7) and immunogenicity (Per protocol set up to Day 30) | 99 |
| Template 59 | Percentage of subjects reporting solicited local symptoms (any grade / grade 3) during the 7-day post-vaccination period (Exposed set) | 100 |
| | · | |

204812 (RSV F-021)

Statistical Analysis Plan Amendment 3 Final

#### **LIST OF ABBREVIATIONS**

AE Adverse Event

AIDS Acquired Immunodeficiency Syndrome

ANCOVA Analysis of Covariance
ANOVA Analysis of Variance

ALT Alanine Aminotransferase
AST Aspartate Aminotransferase

ATP According-to-Protocol

CDISC Clinical Data Interchange Standards Consortium

CI Confidence Interval

eCRF Electronic Case Report Form

Eli Type Internal GSK database code for type of elimination code

ES Exposed Set

FAS Full Analysis Set

GMC Geometric mean antibody concentration

GMT Geometric mean antibody titer

GSK GlaxoSmithKline

ICH International Conference on Harmonisation
IDMC Independent Data Monitoring Committee

IND Investigational New Drug

iSRC Internal Safety Review Committee

LL Lower Limit of the confidence interval

LLOQ Lower Limit of Quantification

MA-RTI Medically Attended Respiratory Tract Infection

MedDRA Medical Dictionary for Regulatory Activities

NEO Neogenin

PCA Palivizumab Competing Antibodies

PCD Primary completion Date
PCR Polymerase Chain Reaction

PPS Per Protocol Set

PreF Purified recombinant RSV F protein, engineered to preferentially

maintain the pre-fusion conformation

RSV Respiratory syncytial virus

204812 (RSV F-021)

Statistical Analysis Plan Amendment 3 Final

RTI Respiratory Track Infection

SAE Serious adverse event

SAP Statistical Analysis Plan

SAS Statistical Analysis System

SBIR (GSK) Biological's Internet Randomization System

SD Standard Deviation

SRT Safety Review Team

TFL Tables Figures and Listings

TOC Table of Content

TVC Total Vaccinated Cohort

UL Upper Limit of the confidence interval

WBC White Blood Cells

#### 1. DOCUMENT HISTORY

| Date | Description | Protocol Version |
|---|---|---|
| 25-AUG-2016 | Version1: first version | RSV F-021 (204812)<br>Protocol (20-Jul-2016) |
| 10-NOV-2016 | Version2.0: Description of changes from Version 1.0 are as below 1. The table of elimination code has been modified 2 Algorithm for handling of data of PCA neutralising antibody concentrations between the LOB and LLOQ was added | RSV F-021 (204812)<br>Protocol (20-Jul-2016) |
| 21-JUL-2017 | Amendment 1: Description of changes from Version 2.0 are as below: - Use of new template for SAP (Default-APP 9000058193 Statistical Analysis Plan_v1) - In section 6. Statistical Analyses, immunogenicity was moved before safety - For the sequence of analysis, IDMC analysis up to at least Day 30 including haematology and biochemistry parameters was newly-added - The table of elimination code has been modified for more clarity - In the analysis of immunogenicity section, the distribution of fold increase of the antibody titres against RSV-A/B and concentrations against NEO have been added - In the analysis of safety section, the percentage of subjects reporting each individual solicited local/general AE during the 7-day follow-up period post vaccination based on maximum intensity per subject has been added - Evaluation of last secondary objective 'To estimate the incidence of medically attended RSV-associated RTIs up to study conclusion' will be performed based on MA-RTIs rather than MA-RSV associated RTIs - The cut-off for the updated (qualified) version of the PCA assay will be set at the level of the assay LLOQ (9.60 µg/mL). | RSV F-021 (204812)<br>Protocol (20-Jul-2016) |

Statistical Analysis Plan Amendment 3 Final

- Algorithm for handling of data of RSV-B neutralising antibody tires between the LOB and LLOQ is defined as similar as for RSV A by considering the LOB for RSV-B is 6
- Addition of analysis of the IgG total and IgG1 subclass
- Addition of analysis of anti-RSV A and anti-PCA in the subset of subjects with IgG/IgG1 data available
- Changes of TFL/TOC
  - In the analysis of safety section, analysis on 'Individuals results of haematological and biochemical parameters outside of the normal ranges in each group' will be reported
  - In the analysis of safety section, the titles in all tables reporting 'incidence and nature of solicited and unsolicited symptoms' have been changed from 'with causal relationship to' to 'considered related to vaccination'
  - In the analysis of safety section, analysis on 'Incidence of solicited local/general symptoms reported during the 7-day post-vaccination period' will also be reported based on maximum intensity per subject for each grade
  - In the analysis of safety section, analysis on 'Number (%) of subjects reporting the occurrence of adverse events within the 7-day and 30-day postvaccination period' will be added
  - In the analysis of safety section, analysis on 'Number (%) of subjects with SAE or SAE considered related to vaccination during the study period' will not be reported
  - In the analysis of safety section, analysis on 'Number and percentage of subjects reporting the occurrence of medically attended respiration tract infections (MA-RTIs), during the 30/60/90-day post-vaccination period and up to study end' will be reported

204812 (RSV F-021) Statistical Analysis Plan Amendment 3 Final

| 1 | Statistical Analysis Plan Amendment 3 Final | |
|---|---|---|
| | <ul> <li>In the analysis of medically attended</li> </ul> | |
| | RTIs, analysis on 'viral load assessed by | |
| | the quantitative PCR (RSV-A/B) of RSV- | |
| | RTI cases' will be only listed in the | |
| | individual listings | |
| | In the analysis of immunogenicity | |
| | section, tables/figures related to the | |
| | analysis of RSV-B will be added | |
| | In the analysis of immunogenicity | |
| | section, tables/figures related to the | |
| | analysis of the IgG total and IgG1 | |
| | subclass will be added | |
| | In the analysis of immunogenicity | |
| | section, tables/figures related to the | |
| | analysis of anti-RSV A and anti-PCA in | |
| | the subset of subjects with IgG/IgG1 | |
| | data available will be added | |
| 09-NOV-2017 | Amendment 2: Description of changes from | RSV F-021 (204812) |
| | Amendment 1 are as below: | Protocol Amendment 1 |
| | - PPD (Clinical Research and | (21-Aug-2017) |
| | Development Lead) was added | |
| | - In the analysis of immunogenicity section, | |
| | the analysis on GM ratios between anti-RSV | |
| | F antibody concentrations (IgG Total) and | |
| | anti-RSV-A neutralising antibody titers at | |
| | pre-vaccination has been added | |
| | - In the analysis of immunogenicity section, | |
| | the analysis on GM ratios of fold increase | |
| | post/pre (Day 30/Day 0) between anti-RSV F | |
| | antibody concentrations (IgG Total) and anti- | |
| | RSV-A neutralising antibody titers has been | |
| | added | |
| | - Changes of TFL/TOC | |
| | In the analysis of safety section, | |
| | analysis on 'Individual results of | |
| | hemoglobin levels beyond grade 2' have | |
| | been added | |
| | <ul> <li>In the analysis of safety section,</li> </ul> | |
| | analysis on 'Individual results of white | |
| | blood cells counts levels lower than LL' | |
| | and the figures of 'Individual results of | |
| | white blood cells counts levels higher | |
| | than UL' have been added | |
| | ulali OL ilave pecli auded | |

204812 (RSV F-021)

Statistical Analysis Plan Amendment 3 Final

- In the analysis of immunogenicity section, one new template of "Comparisons of GM ratios with corresponding 95% confidence interval between anti-RSV F antibody concentrations (IgG Total) and anti-RSV-A neutralising antibody titers at prevaccination (Per protocol set)"has been added
- In the analysis of immunogenicity section, one new template of "Exploratory comparisons (GM ratios of fold increase post/pre) with corresponding 95% confidence interval between anti-RSV F antibody concentrations (IgG Total) and anti-RSV-A neutralising antibody titers at Day 30 (Per protocol set)" has been added

204812 (RSV F-021) Statistical Analysis Plan Amendment 3 Final

| | Statistical Analysis Fran Americanical String | |
|---|---|---|
| 15-Mar-2018 | Amendment 3: Description of changes from | RSV F-021 (204812) |
| | Amendment 2 are as below: | Protocol Amendment 1 |
| | For final analysis, | (21-Aug-2017) |
| | Some tables have been updated including | |
| | removing to Annex, creating new | |
| | corresponding in-text table by deleting or | |
| | collapsing some columns/rows; | |
| | Two figures of 'percentage of subjects | |
| | reporting solicited local/general symptoms | |
| | (any grade / grade 3) during the 7-day post- | |
| | vaccination period' have been newly | |
| | generated for the final analysis, respectively; | |
| | The table of 'Distribution of change from | |
| | baseline in haematology and biochemistry | |
| | with respect to normal laboratory ranges' | |
| | has been splitted and modified into three in- | |
| | text tables for Alanine Aminotransferase | |
| | (ALT)/ Aspartate Aminotransferase | |
| | (AST)/Eosinophils, Creatinine/Lymphocytes/ | |
| | White Blood Cells (WBC), | |
| | Haemoglobin/platelet count/Neutrophils, | |
| | separately; | |
| | Two new in-text tables of 'Summary of | |
| | haematology and biochemistry results by | |
| | maximum grade in the specified category' | |
| | and 'Summary of haematology change from | |
| | baseline by maximum grade in the specified | |
| | category' have been generated; | |
| | Some figures of Individual results for each | |
| | parameter have been modified. | |

#### 2. STUDY DESIGN

#### Figure 1. Study design overview



- V = Visit; D = Day; VACC = vaccination; BS = blood sample; h/b = blood sample for haematology/biochemistry; lmm = blood sample for immunogenicity; C = contact; RSV = Respiratory Syncytial Virus; PCR = Polymerase Chain Reaction.
- 1 Safety data up to (minimum) 7 days post-vaccination (including Day 7 haematology and biochemistry parameters) of the first 25% of subjects vaccinated in the study will be reviewed by iSRC.
- 2 In case of a MA-RTI (e.g. visit to the GP for respiratory symptoms including but not limited to cough, sputum production, difficulty breathing), the subject will be asked to contact the Investigator to enable completion of an event related eCRF and the collection of a nasal swab within 72h after the medical attendance. Vertical lines stand for analysis on all subjects.
- **Experimental design**: Phase II, observer-blind, randomised, controlled, multicountry, study with four parallel groups.
  - O **Duration of the study**: the intended duration of the study will be approximately 1 year from Visit 1 to study conclusion (Day 360).
  - o Epoch 001: Primary starting at Visit 1 (Day 0) and ending at Visit 5 (Day 90).
  - Epoch 002: Follow-up phase starting one day after Day 90 and ending at Day 360 contact.
- **Primary Completion Date (PCD)**: Visit 3 (Day 30).
- End of Study (EoS): Last testing results released of samples collected at Visit 5 (i.e. last testing results released for the assays related to the primary and secondary endpoints).
- Study groups:

Statistical Analysis Plan Amendment 3 Final

Table 1 Study groups and epochs foreseen in the study

| Ctudy around | Number of outlinets | Age (Min/Mey) | Epo | ochs |
|--------------|---------------------|---------------|-----------|-----------|
| Study groups | Number of subjects | Age (Min/Max) | Epoch 001 | Epoch 002 |
| 30 PreF | ~100 | 18 - 45 years | Х | Х |
| 60 PreF | ~100 | 18 - 45 years | Х | Х |
| 120 PreF | ~100 | 18 - 45 years | Х | Х |
| Control | ~100 | 18 - 45 years | Х | Х |

Table 2 Study groups and treatment foreseen in the study

| Tractment name | Vaccina/ Draduct name | | Study ( | Groups | |
|---|---|---|---|---|---|
| Treatment name | Vaccine/ Product name | 30 PreF | 60 PreF | 120 PreF | Control |
| 20 ug DroE | PreF-30 | V | Х | | |
| 30 µg PreF | NaCl | ^ | | | |
| CO D E | PreF-60 | | V | | |
| 60 µg PreF | NaCl | | Х | ^ | |
| 120 µg PreF | PreF-120 | | | Х | |
| | NaCl | | | ۸ | |
| Placebo | Formulation buffer S9b | | | | Х |

- Control: Placebo control
- Vaccination schedule: One intramuscular vaccination at Day 0.
- **Treatment allocation**: Subjects will be randomised using a centralised randomisation system on internet (SBIR) at Day 0. The randomisation algorithm will use a minimisation procedure accounting for age (18 32 years or 33 45 years) and centre.

The following group and sub-group names will be used for the statistical analyses:

| Group order in tables | Group label in tables | Group definition for footnote |
|---|---|---|
| 1 | 30 PreF | 30 µg PreF |
| 2 | 60 PreF | 60 µg PreF |
| 3 | 120 PreF | 120 μg PreF |
| 4 | Control | Placebo |

Some tables might be presented by age category according to the following description:

| Sub-group | Sub-group order in tables | Sub-group label in tables | Sub-group definition for footnote |
|---|---|---|---|
| Age | 1 | 18-32Y | 18-32 years old subjects |
| | 2 | 33-45Y | 33-45 years old subjects |

• **Blinding**: Observer-blind in Epoch 001 and single-blind in Epoch 002.

Table 3 Blinding of study epochs

| Study Epochs | Blinding |
|--------------|----------------|
| Epoch 001 | observer-blind |
| Epoch 002 | single-blind |

204812 (RSV F-021) Statistical Analysis Plan Amendment 3 Final

#### • Sampling schedule:

- o **Blood samples for haematology/biochemistry** will be collected (~10 mL) from all subjects at Visit 1 (Day 0), Visit 2 (Day 7), Visit 3 (Day 30), Visit 4 (Day 60) and Visit 5 (Day 90).
- o **Blood samples for humoral immune response evaluation** will be collected (~17 mL) from all subjects at Visit 1 (Day 0), Visit 3 (Day 30), Visit 4 (Day 60) and at Visit 5 (Day 90).
- Nasal swabs will be collected from subjects in case of a medically attended respiratory tract infection from enrolment (Visit 1) until study end (Contact 3).
- Type of study: self-contained
- **Data collection:** Electronic Case Report Form (eCRF).

#### • Safety monitoring:

- When the first 25% of subjects (i.e. ~100 subjects; ~25 subjects per study group) have been vaccinated, enrolment will be paused until completion of an unblinded review by a GSK internal Safety Review Committee (iSRC). Continuation of study enrolment will be conditional to a favourable outcome of the iSRC evaluation of all available safety and reactogenicity data collected up to at least 7 days post-vaccination (including Day 7 haematology and biochemistry parameters). In addition, the blinded safety data will be reviewed by GSK Biologicals' Safety Review Team (SRT) on a regular basis throughout the study. Analyses related to iSRC evaluation will be described in a separate document (SAP/TFL for iSRC).
- When all subjects have been vaccinated, IDMC will review all available safety and reactogenicity data (including haematology/ biochemistry parameters) of all enrolled subjects up to at least 30 days post administration of the study vaccine or placebo. The blinded safety data will be reviewed by the GSK Biologicals' SRT. Analyses related to IDMC evaluation will be described in a separate document (SAP/TFL for IDMC).
- In case of a MA-RTI (e.g. visit to the GP for respiratory symptoms including but not limited to cough, sputum production, difficulty breathing), the subject will be asked to contact the investigator to enable the collection of a nasal swab within 72 hours after the medical attendance.

#### 3. OBJECTIVES

#### 3.1. Primary Objective

• To rank different formulations of the investigational RSV vaccine based on safety/reactogenicity and immunogenicity data up to 1 month post-vaccination (Day 30).

#### 3.2. Secondary objectives

- To evaluate the reactogenicity and safety of a single intramuscular dose of the RSV investigational vaccines up to study conclusion.
- To evaluate the immunogenicity of a single intramuscular dose of the RSV investigational vaccines up to 90 days after vaccination (Day 90).
- To further assess the safety of the investigational RSV vaccines by evaluating whether a single dose of the vaccines induces antibodies against the residual host cell protein neogenin (NEO) up to 1 month post-vaccination (Day 30).
- To estimate the incidence of medically attended RSV-associated RTIs up to study conclusion.

#### 3.3. Tertiary objective

• If deemed necessary, to further characterize the immune response of a single intramuscular dose of the RSV investigational vaccines.

Refer to Section 5.7.3 Laboratory assays of the Protocol for additional testing proposed to further characterize the immune response to the investigational RSV vaccine.

#### 4. ENDPOINTS

#### 4.1. Primary

- Occurrence of AEs from vaccination up to Day 7, for all subjects in each investigational RSV vaccine group:
  - o Occurrence of any Grade 2 and Grade 3 general AE (solicited and unsolicited);
  - o Occurrence of Grade 2 and Grade 3 fever;
  - Occurrence of any vaccine-related SAE.
- Functional antibody titres against RSV at Day 0 and Day 30, for all subjects in each investigational RSV vaccine group.
  - o Neutralising antibody titres against RSV-A
- PCA concentrations at Day 0 and Day 30 for all subjects in each investigational RSV vaccine group

#### 4.2. Secondary

- Occurrence of AEs from vaccination up to study conclusion:
  - Occurrence of each solicited local and general AE, during a 7-day follow-up period after vaccination (i.e. the day of vaccination and 6 subsequent days), for all subjects in all groups;
  - Occurrence of any unsolicited AE, during a 30-day follow-up period after vaccination (i.e. the day of vaccination and 29 subsequent days), for all subjects in all groups;
  - Occurrence of any haematological (haemoglobin level, White Blood Cells [WBC], lymphocyte, neutrophil, eosinophil and platelet count) and biochemical (alanine amino-transferase [ALT], aspartate amino-transferase [AST] and creatinine) laboratory abnormality at Day 0, Day 7, Day 30, Day 60 and Day 90 for all subjects in all groups;
  - Occurrence of any SAE, for all subjects in all groups.
- Functional antibody titres against RSV for all subjects in all groups:
  - Neutralising antibody titres against RSV-A at Day 0, Day 30, Day 60 and Day 90;
  - Neutralising antibody titres against RSV-B at Day 0, Day 30, Day 60 and Day 90
- PCA concentration at Day 0, Day 30, Day 60 and Day 90 for all subjects in all groups.
- Humoral immune response to the residual host cell protein NEO in the investigational RSV vaccine at pre-vaccination (Day 0), and 1 month post-vaccination (Day 30) for all subjects in all groups.
  - Antibody concentrations against NEO
- Occurrence of medically attended RSV-associated RTIs up to study conclusion

#### 4.3. Tertiary

See section 5.7.3 of the Protocol for additional testing proposed to further characterize the immune response to the investigational RSV vaccine.

#### 5. ANALYSIS SETS

#### 5.1. Definition

In order to align to ICH and CDISC terminology, the Total Vaccinated Cohort (TVC) and the According To Protocol cohort (ATP) have been renamed Exposed Set (ES) and Per-Protocol Set (PPS) respectively. Two cohorts will be defined for the purpose of the analysis: the Exposed Set (ES) and the Per-Protocol Set (PPS) for analysis of immunogenicity. All analyses will be performed per treatment actually administered.
# 5.1.1. Exposed Set (ES)

The ES will include all subjects with study vaccine administration documented:

- A safety analysis based on the ES will include all vaccinated subjects
- An **immunogenicity** analysis based on the ES will include all vaccinated subjects for whom immunogenicity data are available.

### 5.1.2. Per-Protocol Set (PPS) for analysis of immunogenicity

The PPS for immunogenicity will be defined by time point and will include all vaccinated subjects.

- Meeting all eligibility criteria (i.e. no protocol violation linked to the inclusion/ exclusion criteria, including age).
- Who received the study vaccine according to protocol procedures.
- Who did not receive a concomitant vaccination/medication/product leading to exclusion from the PPS analysis up to the corresponding timepoint as described in Section 6.6.2 of the Protocol.
- Who did not present with an intercurrent medical condition leading to exclusion from the PPS analysis up to the corresponding timepoint, as described in Section 6.7 of the Protocol.
- Who complied with the post-vaccination blood sampling schedule at the corresponding timepoint, as specified in Table 5 of the Protocol.
- For whom post-vaccination immunogenicity results are available for at least 1 assay at the corresponding timepoint.

When presenting different timepoints, the PPS for immunogenicity will be adapted for each timepoint (up to D30 and up to D90).

# 5.2. Criteria for eliminating data from Analysis Sets

Elimination codes are used to identify subjects to be eliminated from analysis. Detail is provided below for each sets.

## 5.2.1. Elimination from Exposed Set (ES)

Code 1030 (Study vaccine not administered at all) and code 900 (invalid informed consent or fraud data) will be used for identifying subjects eliminated from ES.

#### 5.2.2. **Elimination from Per-protocol analysis Set (PPS)**

#### 5.2.2.1. **Excluded subjects**

A subject will be excluded from the PPS analysis under the following conditions.

| | | Applicable Eli Type | |
|---|---|---|---|
| Code | Condition under which the code is used | 'M1' (Applicable<br>up to Visit 3 - Day<br>30) | 'M2' (Applicable<br>up to Visit 5 - Day<br>90) |
| 900 | Invalid informed consent or fraud data (Subjects receiving a code 900 should not receive any other elimination codes) | Applicable | Applicable |
| 1030 | Study vaccine not<br>administered at all<br>(Subjects receiving a code<br>1030 should not receive any<br>other elimination codes) | Applicable | Applicable |
| 1040* | Administration of concomitant vaccine(s) forbidden in the protocol | Applicable<br>(To check up to<br>Visit 3 – Day 30) | Applicable<br>(To check up to<br>Visit 5 – Day 90) |
| 1050 | Randomization failure<br>(subject not randomized<br>in the correct group) | Applicable | Applicable |
| 1060 | Randomization code was broken | Applicable | Applicable |
| 1070** | Subjects got vaccinated with the correct vaccine but containing a lower volume | Applicable | Applicable |
| 1070** | Administration not according to protocol for reason specified by the investigator other than site and route | Applicable | Applicable |
| 1070** | Site or route of study vaccine administration wrong or unknown | Applicable | Applicable |
| 1070** | Wrong replacement or study vaccine administered (not compatible with the vaccine regimen associated to the treatment number) | Applicable | Applicable |

| | | Statistical Att | alysis Plan Amendme |
|---|---|---|---|
| 1070** | Administered study vaccine reported as being the correct one but is not compatible with the vaccine regimen associated to the treatment number | Applicable | Applicable |
| 1080 | Vaccine temperature deviation | Applicable | Applicable |
| 1090 | Expired vaccine administered | Applicable | Applicable |
| 2010 | Protocol violation<br>(inclusion/exclusion<br>criteria) | Applicable DOB-VAC=18-45 years | Applicable DOB-VAC=18-45 years |
| 2040* | Administration of any medication forbidden by the protocol | Applicable<br>(To check up to<br>Visit 3 – Day 30) | Applicable<br>(To check up to<br>Visit 5 – Day 90) |
| 2050* | Underlying medical condition forbidden by the protocol | Applicable<br>(To check up to<br>Visit 3 – Day 30) | Applicable<br>(To check up to<br>Visit 5 – Day 90) |
| 2060* | Concomitant infection related to the vaccine which may influence the immune response | Applicable<br>(To check up to<br>Visit 3 – Day 30) | Applicable<br>(To check up to<br>Visit 5 – Day 90) |
| 2070* | Concomitant infection not related to the vaccine which may influence the immune response | Applicable<br>(To check up to<br>Visit 3 – Day 30) | Applicable<br>(To check up to<br>Visit 5 – Day 90) |
| 2090 | Subjects did not comply<br>with blood sample<br>schedule | Applicable VAC_1 to SER_2 = 30-44 (days) | Applicable VAC_1 to SER_3 = 56-70 (days) VAC_1 to SER_4 = 86-100 (days) |
| 2100 | Serological results not available post-vaccination | All assay for Day<br>30<br>elimination code<br>if ALL are | All assay for Day60 and Day90 elimination code if ALL are |
| | | missing v_ID for Neutra RSV-A=3240.001 v_ID for Neutra RSV-B=3240.002 | missing v_ID for Neutra RSV-A=3240.001 v_ID for Neutra RSV-B=3240.002 |
| | | v_ID for Neutra | v_ID for Neutra |

204812 (RSV F-021)

Statistical Analysis Plan Amendment 3 Final

| | | PCA=3241.009 | PCA=3241.009 |
|---|---|---|---|
| | | v_ID for IgG<br>total=3241.002 | v_ID for IgG<br>total=3241.002 |
| | | v_ID for IgG<br>I=3241.005 | v_ID for IgG<br>1=3241.005 |
| 2120* | Obvious incoherence or abnormality or error in data*** | All assay for Day<br>30 | All assay for Day<br>60 and Day90 |

<sup>\*</sup> Attribution of these elimcodes to subject need CRDL review of individual data listings

Eli type is Internal GSK database code for type of elimination code M1 for Visit 3 (Day30) analysis; M2 for Visit 5 (Day 90) analysis;

#### 5.2.2.2. Right censored Data

Not applicable

#### 5.2.2.3. Visit-specific censored Data

Not applicable

# 5.3. Important protocol deviation not leading to elimination from per-protocol analysis set

The following important protocol deviations will be reported by groups:

Forced randomization: In case of supplies shortage for the next assigned vaccine according to the randomization schedule at the clinical site, the randomization system will use the forced randomization procedure in order to continue to enrol and vaccinate subjects. The system moves seamlessly to the next treatment/randomization number for which vaccine supplies are available. The site will not be aware of the forced randomization event

Manual randomization: In case of the randomization system is unavailable, the investigator has the option to perform randomization by selecting supplies available at the site according to a pre-defined rule.

Short follow-up: subjects who completed the last study contact before the minimum length of follow-up requirement.

#### 6. STATISTICAL ANALYSES

Note that standard data derivation rule and stat methods are described in Annex 1 and will not be repeated below.

<sup>\*\*</sup> Attribution of code 1070 to a subject requires CRDL confirmation

<sup>\*\*\*</sup> Elimination criteria for implausible RSV serum immune responses (neut and/or ELISA): More than 4 fold decrease from pre-vaccination to Day 30; After Day 30, more than 4 fold increase or more than 8 fold decrease within a 30 day period

# 6.1. Demography

# 6.1.1. Analysis of demographics/baseline characteristics planned in the protocol

The analysis of demography will be performed on the ES and on the PPS for immunogenicity.

Demographic characteristics such as age at vaccination in years, race, ethnicity, vital signs and cohort description will be summarised by group using descriptive statistics:

- Frequency tables will be generated for categorical variable such as race.
- Mean, median, standard error and range will be provided for continuous data such as age.

The distribution of subjects will be tabulated as a whole and per group and for each age category (18 - 32 years and 33 - 45 years).

Withdrawal status will be summarised by group using descriptive statistics:

- The number of subjects enrolled into the study as well as the number of subjects excluded from PPS analyses will be tabulated.
- The number of withdrawn subjects will be tabulated according to the reason for withdrawal.

# 6.2. Immunogenicity

# 6.2.1. Analysis of immunogenicity planned in the protocol

The analysis will be performed on the applicable PPS cohort for immunogenicity and, if in any group the percentage of vaccinated subjects with serological results excluded from the PPS for analysis of immunogenicity is  $\geq 5\%$ , a second analysis will be performed on the ES

#### 6.2.1.1. Within group analysis

Humoral Immune response to RSV vaccine

For each group, at each timepoint that blood samples are collected and for each assay (unless specified otherwise):

204812 (RSV F-021)

Statistical Analysis Plan Amendment 3 Final

- GMTs/GMCs will be tabulated with 95% CI based on log-transformed values and represented graphically.
- Percentage of subjects above the seropositivity threshold will be tabulated with exact 95% CI.
  - Percentage of subjects above the seropositivity threshold and GMTs/GMCs will also be tabulated by group for each age category (18 32 years and 33 45 years).
- Pre- and post-vaccination antibody titres/concentrations will be displayed using reverse cumulative curves.
- The distributions of **neutralising** antibody titres will be tabulated in the tables with  $\log 2$  scale (< 7, 7-8, > 8-9, > 9-10, > 10-11, > 11-12, > 12  $\log 2$ ).
- Percentage of responders in terms of **neutralising** antibody titres will be tabulated with exact 95% CI.
- Individual post-vaccination *versus* pre-vaccination results will be plotted using scatter plots. Results of the control group will be used as a reference.
- Geometric mean of ratios of antibody titres/concentrations at each post-vaccination timepoint over pre-vaccination will be tabulated with 95% CI.
- Distribution of the fold increase of the antibody titres/concentrations will be tabulated:
  - o For neutralising antibody titres against RSV-A and RSV-B: percentage of subjects with a fold increase equal to or above 1, 2, 2.5, 3, 4, 6, 8 10, 11 and 12 by pre-vaccination titre category: <7, 7-8, ]8-9, ]9-10, ]10-11, ]11-12, >12 log2, and cumulative: <7, ≥7, ≥8, ≥9, ≥10, ≥11, ≥12 log2.
  - For antibody concentrations against NEO: percentage of subjects with a fold increase equal to or above 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5 and 5.
- The kinetics of individual antibody titres/concentrations will be plotted as a function of time for subjects with results available at all timepoints.
- An analysis of variance model for repeated measures will be fitted to calculate GMTs/GMCs with treatment group, visit and their interaction as fixed effects if necessary.

If deemed necessary, the same analyses may be done by age category (18 - 32 years and 33 - 45 years).

#### 6.2.1.2. Between group assessment

Exploratory comparisons will be performed for RSV neutralising antibody titres and PCA concentrations post-vaccination (Day 30, Day 60 and Day 90) between the different RSV vaccine groups.

204812 (RSV F-021)

Statistical Analysis Plan Amendment 3 Final

- Estimation of GMT/GMC ratios between groups with corresponding 95% CI using an ANCOVA model on the logarithm10 transformation of the titres/concentrations. If a statistically significant difference is found (p <0.05), pairwise comparisons will be made using Tukey's multiple comparison adjustment. This model includes:
  - o The vaccine group as the fixed effect
  - The pre-vaccination titre/concentration as the covariate
  - Age groups (18-32 years and 33-45 years) and center as the categorical covariate if deemed necessary
- GMT/GMC ratios with corresponding 95% CI will be computed between the RSV vaccine groups
  - o PreF-120 minus PreF-30
  - o PreF-120 minus PreF-60
  - o PreF-60 minus PreF-30

#### 6.2.2. Additional considerations

In order to add the analysis of the <u>anti-RSV F IgG Total and IgG1 subclass</u> tested at Day 0 and Day 30 in a random subset of 50 subjects per group. The following analysis will be performed on the Per-Protocol Set (PPS) for analysis of immunogenicity for each group and for both assays:

- GMCs with 95% CI will be tabulated.
- Percentage of subjects above the seropositivity threshold will be tabulated with exact 95% CI.
- Geometric mean of ratios of antibody concentrations at each post-vaccination timepoint over pre-vaccination (fold increase) will be tabulated with 95% CI, and represented graphically.
- Individual ratios of antibody concentrations will be displayed using reverse cumulative curves.
- Exploratory comparisons between groups: geometric mean ratios and 95% CIs of fold increase post/pre between the RSV groups:
  - o 120 PreF versus 60 PreF
  - o 120 PreF versus 30 PreF
  - o 60 PreF versus 30 PreF

This will be performed using an ANOVA model on the logarithm 10 transformation of the concentrations including the vaccine group as covariates. If a statistically significant difference is found (p < 0.05), pairwise comparisons will be made using Tukey's multiple comparison adjustment.

In addition, the following immunogenicity analysis will be performed in the subset of subjects with IgG/IgG1data available:

Statistical Analysis Plan Amendment 3 Final

- GMCs will be tabulated with 95% CI for anti-RSV A and anti-PCA
- Percentage of subjects above the seropositivity threshold will be tabulated with exact 95% CI for anti-RSV A and anti-PCA.

# 6.3. Analysis of safety

# 6.3.1. Analysis of safety planned in the protocol

The analysis of safety will be performed on the ES.

#### 6.3.1.1. Within group analysis

The percentage of subjects with at least one **local AE** (solicited and unsolicited), with at least one **general AE** (solicited and unsolicited) and with any AE during the 7-day or 30-day follow-up period after vaccination will be tabulated with exact 95% CI. The same computations will be done for ≥ Grade 2 and Grade 3 AEs, for any AEs considered related to vaccination, for any Grade 3 AEs considered related to vaccination and for AEs resulting in medically attended visit.

The percentage of subjects reporting each individual **solicited local AE** (any grade,  $\geq$  Grade 2, Grade 3, resulting in medically attended visit) during the 7-day follow-up period after vaccination will be tabulated for each study vaccine for each group. The percentage of subjects reporting each individual **solicited general AE** (any grade,  $\geq$  Grade 2, Grade 3, any related,  $\geq$  Grade 2 related, Grade 3 related, resulting in medically attended visit) during the 7-day follow-up period after vaccination will be tabulated for each group.

For fever during the 7-day follow-up period after vaccination, the number and percentage of subjects reporting fever will be reported by half degree (°C) cumulative increments. Similar tabulations will be performed for causally related fever, Grade 3 (> 39.5°C) causally related fever and fever resulting in a medically attended visit. In addition, the prevalence of any and Grade 3 fever will be presented graphically over time after vaccination.

The percentage of subjects with any **unsolicited** symptoms within 30 days after vaccination with its exact 95% CI will be tabulated by group and by Medical Dictionary for Regulatory Activities (MedDRA) preferred term. Similar tabulation will be done for Grade 3 unsolicited symptoms, for any causally related unsolicited symptoms, for Grade 3 causally related unsolicited symptoms and for unsolicited symptoms resulting in a medically attended visit (The verbatim reports of unsolicited symptoms will be reviewed by a physician and the signs and symptoms will be coded according to the MedDRA Dictionary for Adverse Reaction Terminology. Every verbatim term will be matched with the appropriate Preferred Term).

**SAEs** reported throughout the study will be described in detail.

**Pregnancy** exposures throughout the study and pregnancy outcomes will be described in detail (if applicable).

204812 (RSV F-021)

Statistical Analysis Plan Amendment 3 Final

The percentage of subjects using **concomitant medication** (any medication, any antipyretic and any antipyretic taken prophylactically) during the 7-day (Day 0 to Day 6) or 30-day (Day 0 to Day 29) follow-up period after vaccination will be summarised by group.

For all subjects in each group and each **haematology and biochemistry** parameter:

- The percentage of subjects having haematology and biochemistry results below or above the local laboratory normal ranges will be tabulated for each timepoint.
- The maximum grading post-vaccination (from Day 7 to Day 90) versus baseline (Day 0) and the percentage of subjects with laboratory parameters above or equal to Grade 1, Grade 2, Grade 3 and Grade 4 will be tabulated (Grades will be based on the FDA Guidance for Industry "Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials", see APPENDIX D of the Protocol: FDA toxicity grading scale. Those laboratory parameters not included on FDA Toxicity Grading Scale will not be graded).

Assessment of anti-NEO immune response at Day 30 post-vaccination for each group:

- GMCs pre-and post-vaccination will be tabulated with 95% CI and represented graphically.
- Individual post-vaccination *versus* pre-vaccination results will be plotted using scatter plots. Results of the control group will be used as a reference.
- Geometric mean of ratios of antibody concentrations at Day 30 over pre-vaccination will be tabulated with 95% CI.
- Distribution of the antibody concentrations pre-and post-vaccination and of fold increase after vaccination will be tabulated.

#### 6.3.1.2. Between group assessment

Exploratory comparisons between each investigational RSV vaccine group and (minus) the control group (*placebo*), and between the RSV vaccine groups will be done in terms of the percentage of subjects reporting any  $\geq$  Grade 2, Grade 3 AE (solicited and unsolicited), and/or any fever > 38.5°C, and/or any vaccine-related SAE during the 7-day follow-up period after vaccination.

- o PreF-30 minus placebo
- o PreF-60 minus placebo
- o PreF-120 minus placebo
- o PreF-120 minus PreF-30
- o PreF-120 minus PreF-60
- o PreF-60 minus PreF-30

204812 (RSV F-021)

Statistical Analysis Plan Amendment 3 Final

The standardised asymptotic 95% CI for the difference between the investigational RSV vaccine groups as well as between the investigational RSV groups and (minus) the control group will be computed.

# 6.4. Analysis for ranking RSV formulations

The totality of data and sum total of evidence for particular dose(s) in terms of safety and immunogenicity will be evaluated by study team in addition to the analyses described in section 6.1 and 6.3 on formulation selection. The desirability index approach described in the section below will be used as a descriptive tool to guide the formulation selection. In addition, any pertinent information from outside this study will be evaluated and may be used by the study team to help to make the final decision on a dose/formulation.

### 6.4.1. Definition of desirability in the context of Simulations

A desirability approach will be based on safety/reactogenicity and immunogenicity data up to 1 month post-vaccination.

This method is a multi-criteria decision making approach based on desirability functions. The main idea is to identify for each endpoint a desirability function that associates any value to another one between 0 and 1 depending on its desirability ('0' being considered as not desirable at all and '1' as the most desirable). An index with values between 0 and 1 will be created for each endpoint. An overall desirability index can be calculated by computing a weighted geometric mean of the endpoint indexes. By definition, this overall index also takes values between 0 and 1 and characterises the level of desirability of any candidate formulation by a single value [Dewé, 2015].

The desirability index calculations will include reactogenicity and safety data up to Day 7 post vaccination (on the TVC) and immunogenicity data at 30 days post-vaccination (on the ATP cohort for immunogenicity up to Day 30). The formulations will be ranked based on the values obtained with this overall desirability index.

#### 6.4.2. Derived endpoints

The following endpoints will be computed and taken into account in the desirability analysis:

- 1. Incidence rate of any Grade 2 and any Grade 3 general AE (solicited and unsolicited) and any vaccine-related SAE during the 7-day follow-up period after vaccination for each investigational RSV vaccine formulation.
- 2. Incidence rate of Grade 2 and Grade 3 fever during the 7-day follow-up period after vaccination for each investigational RSV vaccine formulation.
- 3. Geometric mean of neutralising antibody titres against RSV-A at Day 30 adjusted for pre-vaccination titres.
- 4. Geometric mean of PCA concentrations at Day 30 adjusted for pre-vaccination titres.

204812 (RSV F-021)

Statistical Analysis Plan Amendment 3 Final

Each individual desirability index will be calculated based on data and tabulated by the treatment group and endpoints above. The details on how to calculate individual desirability index in terms of reactogenicity and immunogenicity and overall desirability index are elaborated in Annex 2.

# 6.5. Analysis of medically attended RTIs

The analysis will be performed on the ES by study group.

The proportion of subjects (with 95% CI) with at least one medically attended RTI (all causes) will be calculated by group.

Viral load assessed by the quantitative PCR (RSV-A/B) of RSV-RTI cases will be listed for any cases where this assay is performed.

Medically attended RSV-associated RTI co-infected or colonisation with another viral etiology identified by multiplex PCR will be described.

Medically attended RTI with any viral etiology identified by multiplex PCR will be described.

### 7. ANALYSIS INTERPRETATION

All comparative analyses will be descriptive with the aim to characterise the difference in reactogenicity/immunogenicity between groups. These descriptive analyses should be interpreted with caution considering that there is no adjustment for multiplicity for these comparisons.

#### 8. CONDUCT OF ANALYSES

Any deviation(s) or change(s) from the original statistical plan outlined in this protocol will be described and justified in the final study report.

# 8.1. Sequence of analyses

The statistical analyses will be performed in several steps:

- In preparation of the planned iSRC evaluation, analysis of safety and reactogenicity data up to at least 7 days post-vaccination of the first 25% of all subjects will be performed (see Section 8.10.2 of the Protocol for more information).
- In preparation of the planned IDMC evaluation, analysis of safety and reactogenicity data (including haematology/ biochemistry parameters) up to at least 30 days post-vaccination of all enrolled subjects will be performed.

204812 (RSV F-021)

Statistical Analysis Plan Amendment 3 Final

- The first main analysis on all subjects will be performed when all data up to 30 days post-vaccination are available (primary endpoints). In order to maintain the blind, this analysis by group will be performed by an independent statistician and the results which would lead to the unblinding of some subjects (e.g. a specific AE reported by one subject only) will be blinded (i.e. the group in which this event occurred will not be identified). No individual data listings will be provided.
- A second analysis will be performed when all data up to 90 days post-vaccination are available (secondary endpoints). At this point, the GSK statistician will be unblinded (i.e. will have access to the individual subject treatment assignments), but no individual listings will be provided. Given that summary results may unblind some specific subjects, the study will be conducted in a single-blind manner from this point onwards, with subjects remaining blinded up to study conclusion and the investigators will not have access to the treatment allocation up to study conclusion.
- The final analysis will be performed when all data up to study conclusion are available. All available tertiary endpoints will also be analysed in this step. Individual listings will only be provided at this stage.
- An integrated study report presenting all analyses will be written and made available to the investigators at the time of final analysis.
- If data for tertiary endpoints become available at a later stage, (an) additional analysis/analyses will be performed. These data will be documented in Annex(es) to the study report and will be made available to the investigators at that time.

| Description | Analysis ID | Disclosure Purpose<br>(CTRS=web posting,<br>SR=study report,<br>internal) | Dry run review<br>needed (Y/N) | Study Headline Summary (SHS)requiring expedited communication to upper management (Yes/No) | Reference for TFL |
|---|---|---|---|---|---|
| Final Analysis | E1_01 | Study report<br>CTRS | N | Yes | All tables from<br>TFL dated<br>15MAR2018 |
| Analysis of<br>Day 30 | E1_04 | Internal<br>CTRS | N | Yes | All tables from<br>TFL dated<br>13NOV2017 |
| Analysis of<br>Day 90 | E1_05 | Internal<br>CTRS | N | Yes | All tables from<br>TFL dated<br>13NOV2017 |

# 8.2. Statistical considerations for interim analyses

No interim analysis will be performed.

#### 9. CHANGES FROM PLANNED ANALYSES

In order to align to ICH and CDISC terminology the Total Vaccinated Cohort and the According To Protocol cohort have been renamed Exposed Set (ES) and Per-Protocol Set (PPS) respectively.

#### Changes in Amendment 1 mainly include the following.

For the sequence of analysis, the IDMC evaluation was newly added to review all available safety and reactogenicity data (including Day 30 haematology and biochemistry parameters) of all enrolled subjects up to at least 30 days post administration of the study vaccine or placebo.

Since the document of criteria for eliminating subjects from analysis will not be used anymore, the table of Elimination codes has been modified for more clarity. Attribution of code 1070 to a subject requires CRDL confirmation. Attribution of these elimcodes including 1040, 2040, 2050, 2060, 2070 and 2120 to subject need CRDL review of individual data listings.

In the analysis of immunogenicity section, the distribution of fold increase of the antibody titres against RSV-A and RSV-B and concentrations against NEO have been added.

For the analysis of safety, the percentage of subjects reporting each individual solicited local AE (any, each grade, resulting in medically attended visit) during the 7-day follow-up period after vaccination will also be tabulated based on maximum intensity per subject for each study vaccine group; the percentage of subjects reporting each individual solicited general AE (any, each grade, any related, any Grade 2 related, any Grade 3 related, resulting in medically attended visit) during the 7-day follow-up period after vaccination will also be based on maximum intensity per subject for each study vaccine group.

Evaluation of last secondary objective 'To estimate the incidence of medically attended RSV-associated RTIs up to study conclusion' will be performed based on MA-RTIs rather than MA-RSV associated RTIs.

The cut-off for the updated (qualified) version of the PCA assay will be set at the level of the assay LLOQ (9.60 µg/mL). Hence the SAP does not need to define handling of data between the LOD and LLOQ anymore, as results will only be provided as of the LLOQ. It only needs to be defined that for results below the cut-off (LLOQ), an arbitrary value of half of the cut-off will be considered for calculation of GMC and fold increase.

Algorithm for handling of data of RSV-B neutralising antibody tires between the LOB and LLOQ is defined as similar as for RSV-A by considering the LOB for RSV-B is 6.

Additional analysis of the IgG total and IgG1 subclass and analysis of anti-RSV A and anti-PCA in the subset of subjects with IgG/IgG1 data have been added.

204812 (RSV F-021)

Statistical Analysis Plan Amendment 3 Final

#### Changes of TFL/TOC

- In the analysis of safety section, figures of 'Individuals results of haematological (haemoglobin level, white blood cells and platelet count) and biochemical (ALT, AST and creatinine) parameters outside of the normal ranges in each group' has been added to replace the figures of 'Mean profile of haematological and biochemical parameters change from baseline (Day 0)';
- In the analysis of safety section, the titles in all tables reporting 'Incidence and nature of symptoms (solicited and unsolicited) during the 7-day and 30-day post-vaccination period' have been changed from 'with causal relationship to' to 'considered related to vaccination';
- In the analysis of safety section, analysis on 'Incidence of solicited local/general symptoms reported during the 7-day post-vaccination period' will be summarized based on maximum intensity for each grade per subject for each group; therefore, analysis on 'incidence of solicited local/general symptoms reported during the 7-day post-vaccination period, including >=grade 2 category' will not be generated.
- In the analysis of safety section, analysis on 'Number (%) of subjects reporting the occurrence of adverse events within the 7-day and 30-day post-vaccination period' will be added.
- In the analysis of safety section, analysis on 'Number (%) of subjects with serious adverse events during the study period including number of events reported' and 'Number (%) of subjects with serious adverse events considered related to vaccination during the study period including number of events reported' by %UNSOL (EVENT=1) will not be reported because %CTR\_SAE macro has been adapted to generate SAE, related SAE, fatal SAE and related fatal SAE.
- In the analysis of safety section, analysis on 'Number and percentage of subjects reporting the occurrence of medically attended respiration tract infections (MA-RTIs), during the 30-day, 60-day or 90-day post-vaccination period and up to study end' will be reported; Therefore, 'Number and percentage of subjects reporting one medically attended RSV-associated RTI and medically attended RTI (all causes) within the 30-day post-vaccination period or throughout the study period' will not be generated;
- In the analysis of medically attended RTIs, viral load assessed by the quantitative PCR (RSV-A/B) of RSV-RTI cases will be only listed in the individual listings; therefore, analysis on 'Descriptive statistics of the viral load assessed by the quantitative PCR (RSV-A/B) of RSV-RTI cases (All vaccinated subjects)' will not be reported;
- In the analysis of immunogenicity section, tables/figures related to the analysis of RSV-B will be added;
- In the analysis of immunogenicity section, tables/figures related to the analysis of the IgG total and IgG1 subclass will be added;
- In the analysis of immunogenicity section, tables related to the analysis of anti-RSV A and anti-PCA in the subset of subjects with IgG/IgG1 data available will be added.

204812 (RSV F-021)

Statistical Analysis Plan Amendment 3 Final

### Changes in Amendment 2 mainly include the following.

- In the analysis of immunogenicity section, the analysis on GM ratios between anti-RSV F antibody concentrations (IgG Total) and anti-RSV-A neutralising antibody titers at pre-vaccination has been added for Day 90 and final analysis;
- In the analysis of immunogenicity section, the analysis on GM ratios of fold increase post/pre (Day 30/Day 0) between anti-RSV F antibody concentrations (IgG Total) and anti-RSV-A neutralising antibody titers has been added for Day 90 and final analysis.

### Changes of TFL/TOC

- In the analysis of safety section, figures of "Individual results of hemoglobin levels beyond grade 2" will be reported for Day 90 and final analysis to replace the figures of "Individual results of hemoglobin levels outside of normal range";
- In the analysis of safety section, figures of "Individual results of white blood cells counts levels lower than LL" and figures of "Individual results of white blood cells counts levels higher than UL" will be reported for Day 90 and final analysis to replace the figures of "Individual results of white blood cells counts levels outside of normal range".
- In the analysis of immunogenicity section, one new template (Template 54) for "Comparisons of GM ratios with corresponding 95% confidence interval between anti-RSV F antibody concentrations (IgG Total) and anti-RSV-A neutralising antibody titers at pre-vaccination (Per protocol set)" has been added for Day 90 and final analysis;
- In the analysis of immunogenicity section, one new template (Template 55) for "Exploratory comparisons (GM ratios of fold increase post/pre) with corresponding 95% confidence interval between anti-RSV F antibody concentrations (IgG Total) and anti-RSV-A neutralising antibody titers at Day 30 (Per protocol set)" has been added for Day 90 and final analysis;

#### Changes in Amendment 3 mainly include the following.

## Changes of TFL/TOC for final analysis

- All tables concerned with 'Incidence and nature of symptoms (solicited and unsolicited)' have been moved to Annex; such tables for Grade 3 are kept as in-text tables;
- Tables of 'Incidence of solicited local/general symptoms reported during the 7-day (Days 0-6) post-vaccination period' have been moved to Annex; such tables by maximum intensity are kept as in-text tables and corresponding figures have been newly generated for the final analysis, that is, 'Percentage of subjects reporting solicited local/general symptoms (any grade / grade 3) during the 7-day post-vaccination period';
- All tables concerned with 'Percentage of subjects reporting the occurrence of unsolicited symptoms' have been moved to Annex; Such tables for Grade 3 and/or considered related to vaccination are kept as in-text tables with the simplification by removing the columns of LL and UL;

Statistical Analysis Plan Amendment 3 Final

- Tables of 'Percentage of subjects reporting the occurrence of SAE within the 30-day (Days 0-29) post-vaccination period/throughout the study period' are kept as in-text tables with the simplification by removing the columns of LL and UL;
- All tables concerned with 'Number (%) of subjects reporting the occurrence of adverse events' have been moved to Annex;
- All tables of 'Number and percentage of subjects reporting the occurrence of medically attended respiration tract infections (MA-RTIs)' have been moved to Annex; MA-RTIs reported up to DBF of final analysis is kept as one in-text table with the simplification by removing the columns of LL and UL;
- The table of 'Compliance in returning symptom information' and all tables concerned with 'Number and percentage of subjects taking a concomitant medication' have been moved to Annex;
- The table of 'Exploratory comparisons between groups in terms of percentage of subjects reported any Grade 2/3 AE and/or any fever >38.5°C and/or any vaccine-related SAE during the 7 day (Days 0-6) Post-vaccination period' will not be reported in the final analysis;
- The table of 'Distribution of change from baseline in haematology and biochemistry with respect to normal laboratory ranges' has been moved to Annex; Three splitted in-text tables for ALT/AST /Eosinophils, Creatinine/Lymphocytes/White Blood Cells and Haemoglobin/ platelet count/ Neutrophils have been generated, separately;
- The table of 'Summary of haematology and biochemistry results by maximum grade' has been moved to Annex; One newly formatted in-text table of 'Summary of haematology and biochemistry results by maximum grade in the specified category' has been generated by collapsing the categories of unknown/grade 0 and grade 1 then renaming the new category of 'other', keeping grade 2, 3 and 4 column, and removing the column of n;
- The table of 'Summary of haematology change from baseline by maximum grade' has been moved to Annex; One newly formatted in-text table of 'Summary of haematology change from baseline by maximum grade in the specified category' has been generated by collapsing the categories of unknown/grade 0 and grade 1 then renaming the new category of 'other', keeping grade 2, 3 and 4 column, and removing the column of n;

# 10. LIST OF FINAL REPORT TABLES, LISTINGS AND FIGURES

The TFL TOC provides the list of tables/listings and figures needed for the study report. It also identifies the tables eligible for each analyses and their role (synopsis, in-text, post-text, SHS, CTRS,...).

Statistical Analysis Plan Amendment 3 Final

# 11. ANNEX 1 STANDARD DATA DERIVATION RULE AND STATISTICAL METHODS

#### 11.1. Statistical Method References

The exact two-sided 95% CIs for a proportion within a group will be the Clopper-Pearson exact CI [Clopper CJ, Pearson ES. The use of confidence or fiducial limits illustrated in the case of binomial. *Biometrika*. 1934;26:404-413].

The standardised asymptotic two-sided 95% CI for the group difference in proportions is based on the method described in the following paper:Robert G. Newcombe, interval estimation for the difference between independent proportions: comparison of eleven methods, *Statist Med.* 1998; 17, 873-890]. The standardised asymptotic method used is the method six.

Dewé W, Durand Ch, Marion S *et al*. A multi-criteria decision making approach to identify a vaccine formulation. *Journal of Biopharmaceutical Statistics*, 2015; epublication ahead of print: DOI: 10.1080/10543406.2015.1008517.

#### 11.2. Standard data derivation

#### 11.2.1. Date derivation

- SAS date derived from a character date: In case day is missing, 15 is used. In case day and month are missing, 30 June is used.
- Onset day for an event (ae, medication, vaccination, ...): The onset day is the number of days between the last study vaccination & the start date of the event. This is 0 for an event starting on the same day as a vaccination. See SAS date derived in case the start date of the event is incomplete.
- Duration: Duration of an event is expressed in days. It is the number of days between the start & the stop dates + 1. Therefore duration is 1 day for an event starting & ending on the same day.
- Association of an event to the primary epoch: An adverse event belongs to the primary epoch, if the onset date is before and excluding Visit 5 or the last contact date, whichever is coming first.

#### 11.2.2. Dose number

- The study dose number is defined in reference to the number of study visits at which vaccination occurred.
- Relative dose: the relative dose for an event (AE, medication, vaccination) is the most recent study dose given before an event. In case the event takes place on the day a study dose is given, the related dose will be that of the study dose, even if the event actually took place before vaccination. For instance, if an adverse event begins

204812 (RSV F-021)

Statistical Analysis Plan Amendment 3 Final

on the day of the study vaccination but prior to administration of the vaccine, it will be assigned to this dose.

### 11.2.3. Demography

- Age: Age at the reference activity, computed as the number of units between the date of birth and the reference activity. Note that due to incomplete date, the derived age may be incorrect by 1 month when month is missing from the birthdate. This may lead to apparent inconsistency between the derived age and the eligibility criteria/the age category used for randomization.
- Conversion of weight to kg

The following conversation rule is used:

- Weight in Kilogram = weight in Pounds / 2.2
- Weight in Kilogram = weight in ounces / 35.2

The result is rounded to 2 decimals.

• Conversion of height to cm

The following conversation rule is used:

- Height in Centimetres = Height in Feet \* 30.48
- Height in Centimetres = Height in Inch \* 2.54

The result is rounded to the unit (ie no decimal).

• Conversion of temperature to °C

The following conversion rule is used:

o Temperature in °Celsius = ((Temperature in °Fahrenheit -32) \*5)/9

The result is rounded to 1 decimal.

### 11.2.4. Immunogenicity

- For a given subject and given immunogenicity measurement, missing or non-evaluable measurements will not be replaced. Therefore, an analysis will exclude subjects with missing or non-evaluable measurements.
- A seronegative subject is a subject whose antibody titre/concentration is below the cut-off value of the assay. A seropositive subject is a subject whose antibody titre/concentration is greater than or equal to the cut-off value of the assay
- The Geometric Mean Concentrations/Titres (GMC/Ts) calculations are performed by taking the anti-log of the mean of the log titre transformations. Antibody titres below the cut-off of the assay will be given an arbitrary value of half the cut-off of the assay for the purpose of GMT calculation. The cut-off value is defined by the laboratory before the analysis and is described in the protocol.

Statistical Analysis Plan Amendment 3 Final

- In order to compute fold increase of antibody titres/concentrations (ratio) between post-vaccination and pre-vaccination titres/concentrations and for GMC/GMT calculation, antibody titres/concentrations below the assay cut-off will be given an arbitrary value of half the cut-off.
- The cut-off for the updated (qualified) version of the PCA assay will be set at the level of the assay LLOQ (9.60 µg/mL). For results below the cut-off (LLOQ), an arbitrary value of half of the cut-off will be considered for calculation of GMC and fold increase.
- Considering cut-offs or neutralising antibody against RSV-A and RSV-B are below the assays' LLOO, the following rules will be applied:

| Assay | Raw result | Derivation for<br>seropositivity status | Derivation for<br>GMT calculation | Derivation for fold-increase<br>between Post and Pre-<br>vaccination titres |
|---|---|---|---|---|
| Neutra RSV-<br>A | <8 | NEG | 4 | LLOQ/2 |
| | [8-LLOQ[ | POS | 8 | LLOQ/2 |
| | ≥LLOQ | POS | Exact value | Exact value |
| Neutra RSV- | <6 | NEG | 3 | LLOQ/2 |
| В | [6-LLOQ[ | POS | 6 | LLOQ/2 |
| | ≥LLOQ | POS | Exact value | Exact value |

- Vaccine response to the RSV neutralising antibodies (anti-RSV-A and anti-RSV-B) will be defined as:
  - At least a 4-fold increase from pre-vaccination if pre-vaccination neutralising antibody titre <7 log2 (<128).
  - At least a 3-fold increase from pre-vaccination if pre-vaccination neutralising antibody titre in [7-8] log2 ([128-256]).
  - At least a 2.5-fold increase from pre-vaccination if pre-vaccination neutralising antibody titre in >8-10 log2 (>256-1024).
  - At least 1-fold from pre-vaccination if pre-vaccination neutralising antibody titre >10 log2 (>1024).
- All CI computed will be two-sided 95% CI.

### 11.2.5. Safety

- For a given subject and the analysis of solicited symptoms within 7 days post-vaccination, missing or non-evaluable measurements will not be replaced. Therefore the analysis of the solicited symptoms based on the Total Vaccinated Cohort will include only vaccinated subjects for doses with documented safety data (i.e., symptom screen completed). More specifically the following rules will be used:
  - Subjects who documented the absence of a solicited symptom after one dose will be considered not having that symptom after that dose.

204812 (RSV F-021)

Statistical Analysis Plan Amendment 3 Final

- Subjects who documented the presence of a solicited symptom and fully or
  partially recorded daily measurement over the solicited period will be included in
  the summaries at that dose and classified according to their maximum observed
  daily recording over the solicited period.
- O Subjects who documented the presence of a solicited symptom after one dose without having recorded any daily measurement will be assigned to the lowest intensity category at that dose (i.e., 37.5°C for fever or grade 1 for other symptoms).
- o Doses without symptom sheets documented will be excluded.
- For analysis of unsolicited adverse events, such as serious adverse events or adverse
  events by primary MedDRA term, and for the analysis of concomitant medications,
  all vaccinated subjects will be considered. Subjects who did not report the event or
  the concomitant medication will be considered as subjects without the event or the
  concomitant medication respectively.
- The preferred route for recording temperature in this study will be oral. For the analysis, temperatures will be coded as follows:

| Grade | Temperature for oral, axillary | Temperature for rectal |
|-------|--------------------------------|------------------------|
| | or tympanic route | route |
| 0 | < 37.5°C | < 38.0°C |
| 1 | ≥ 37.5°C - ≤ 38.5°C | ≥ 38.0°C - ≤ 39.0°C |
| 2 | > 38.5°C - ≤ 39.5°C | > 39.0°C - ≤ 40.0°C |
| 3 | > 39.5°C | > 40.0°C |

Note that for all tables described in this section, the way the percentage of subjects will be derived will depend on the event analysed (see table below for details). As a result, the N value will differ from one table to another.

| Event | N used for deriving % per subject for Vaccination phase |
|---|---|
| Concomitant vaccination | All subjects with study vaccine administered |
| Solicited general symptom Solicited local symptom | All subjects with at least one solicited general symptom documented as either present or absent (i.e., symptom screen completed) All subjects with at least one solicited local symptom documented as either present or |
| Solicited local symptom | absent (i.e., symptom screen completed) |
| Unsolicited symptom | All subjects with study vaccine administered |
| Concomitant medication | All subjects with study vaccine administered |

The intensity scale of the following solicited AEs will be assessed as described:

| Adverse Event | Intensity<br>grade | Parameter |
|---|---|---|
| Pain at injection site | 0 | None |
| | 1 | Mild: Any pain neither interfering with nor preventing normal every day activities. |
| | 2 | Moderate: Painful when limb is moved and interferes with every day activities. |
| | 3 | Severe: Significant pain at rest. Prevents normal every day activities. |
| Redness at injecti | on site | Record greatest surface diameter in mm |
| Swelling at injection | on site | Record greatest surface diameter in mm |
| Fever* | | Record temperature in °C |
| Headache | 0 | Normal |
| | 1 | Mild: Headache that is easily tolerated |
| | 2 | Moderate: Headache that interferes with normal activity |
| | 3 Severe: Headache that prevents normal activity | |
| Fatigue | 0 | Normal |
| | 1 | Mild: Fatigue that is easily tolerated |
| | 2 | Moderate: Fatigue that interferes with normal activity |
| | 3 | Severe: Fatigue that prevents normal activity |
| Gastrointestinal | 0 | Normal |
| symptoms (nausea, 1 Mild: Gastrointestinal symptoms that are easily tolerated | | Mild: Gastrointestinal symptoms that are easily tolerated |
| vomiting, diarrhoea | 2 | Moderate: Gastrointestinal symptoms that interfere with normal activity |
| and/or abdominal pain) | 3 | Severe: Gastrointestinal symptoms that prevent normal activity |

<sup>\*</sup>Fever is defined as temperature  $\geq$  37.5°C for oral, axillary or tympanic route, or  $\geq$  38.0°C for rectal route. The preferred route for recording temperature in this study will be oral.

The maximum intensity of local injection site redness/swelling will be scored at GSK Biologicals according to the standard GSK Biologicals' scoring system for adults:

0:  $\leq$  20 mm

1:  $> 20 \text{ mm to} \le 50 \text{ mm}$ 

2:  $> 50 \text{ mm to} \le 100 \text{ mm}$ 

3: > 100 mm

The maximum intensity of fever will be scored at GSK Biologicals according to the standard GSK Biologicals' scoring system for adults (via the preferred route for recording temperature in this study which is oral):

0:  $< 37.5 \, ^{\circ}\text{C}$ 

1:  $\geq 37.5 \,^{\circ}\text{C} \text{ to} \leq 38.5 \,^{\circ}\text{C}$ 

2: > 38.5 °C to  $\le 39.5$  °C

3: > 39.5°C

The investigator assessed the maximum intensity that occurred over the duration of the event for all unsolicited AEs (including SAEs) recorded during the study. The assessment was based on the investigator's clinical judgement.

For clintrial.gov and EudraCT posting purposes, a summary of subjects with all combined solicited (regardless of their duration) and unsolicited adverse events will be provided. Solicited adverse events will be coded by MedDRA as per the following codes.

204812 (RSV F-021)

Statistical Analysis Plan Amendment 3 Final

| Solicited symptom | Lower level term name | Lower level term code | Corresponding Primary Term code |
|---|---|---|---|
| Pain | Pain | 10033371 | 10033371 |
| Redness | Erythema | 10015150 | 10015150 |
| Swelling | Swelling | 10042674 | 10042674 |
| Fatigue | Fatigue | 10016256 | 10016256 |
| Fever | Fever | 10016558 | 10037660 |
| Gastroinstestinal symptoms | Gastroinstestinal disorder | 10017944 | 10017944 |
| Headache | Headache | 10019211 | 10019211 |

### 11.2.6. Number of decimals displayed

The following decimal description from the decision rules will be used for the demography, immunogenicity and safety/reactogenicity.

| Display Table | Parameters | Number of |
|---|---|---|
| | | decimal digits |
| All summaries | % of count, including LL & UL of CI | 1 |
| All summaries | % of difference, including LL & UL of CI | 2 |
| Demographic | Mean, median age, SD (age) | 1 |
| characteristics | | |
| Reactogenicity | Mean, Min, Q1, Median, Q3, Max for duration | 1 |
| Immunogenicity | Ratio of GMT/GMC | 2 |

## 12. ANNEX 2: SUMMARY ON ELIMINATION CODES

Refer to section 5.2

# 13. ANNEX 3 CALCULATION OF INDIVIDUAL AND OVERALL DESIRABILITY INDEX

The section below provide the details on how to calculate individual desirability index and overall desirability index score based on Annex E in the Protocol.

#### Reactogenicity

A logistic regression model will be fitted on each reactogenicity endpoint (any Grade 2/3 general AE and any related SAE, Grade 2/3 fever) reported during the 7-day follow-up period after vaccination, including all RSV formulations.

- o The vaccine group as the fixed effect
- The age groups (18-32 years and 33-45 years) as the categorical covariant if deemed necessary.

The estimation of indication rate will be tabulated by treatment group. The SAS codes can be used as reference:

Statistical Analysis Plan Amendment 3 Final

```
proc logistic data=React;
  class Treatment AgeGroup / param=glm;
  model response (event='AE')= Treatment| AgeGroup;
  lsmeans Treatment / ILINK e diff oddsratio adjust=bon cl;
run;
```

For any Grade 2/3 general AEs and any related SAEs, the incidence rate estimate (1R) will be transformed in a [0,1] desirability index using the following function:

$$DR1 = \frac{1}{1 + \exp -50 * 0.25 - IR}, \quad if \ TR \le 0.25$$

$$\frac{1}{1 + \exp -25 * 0.25 - IR}, \quad if \ TR \ge 0.25$$

where *1R* is the incidence rate estimated by the model. This function will allocate a desirability value of 1, 0.5 and 0 to incidence rate equal to 0.1, 0.25 and 0.5 respectively (see Figure 2). But the calculation equally weights Grade 2/3 general AEs and any related SAEs.

Figure 2 Desirability function for the incidence rate of Grade 2/3 general AEs and related SAEs - for each investigational RSV vaccine formulation



For Grade 2/3 fever, the incidence rate estimate (1R) will be transformed in a [0,1] desirability index using the following function:

$$DR2 = \frac{1}{1 + \exp(-120 * (0.05 - R))}$$

Statistical Analysis Plan Amendment 3 Final

where *fR* is the incidence rate estimated by the model. As illustrated in Figure 3, the function will allocate desirability values of 1, 0.5 and 0 to incidence rate equal to 0, 0.05 and 0.1 respectively.

Figure 3 Desirability function for the incidence rate of Grade 2/3 fever - for each investigational RSV vaccine formulation



Finally, the reactogenicity index will be computed by taking the geometric mean of the 2 indexes:

$$DR = \sqrt{DR1 * DR2}$$

#### **Immunogenicity**

The ANCOVA model will be fitted on the log-transformed titre for each immune response of neutralising anti-RSV-A and PCA separately including

- o The vaccine group as the fixed effect
- o The pre-vaccination titre/concentration and age groups (18-32 years and 33-45 years) as the covariates if deemed necessary

The mean estimations of GMTs/GMCs for each treatment group at Day 30 and its 95% CI will be provided for immunogenicity desirability calculation. The estimated GMT and LL will be tabulated by treatment group.

As formulations inducing a high immune response will be considered suitable, the lower limit (LL) of the estimated GMT/C adjusted for pre-vaccination titres will be the statistical criterion considered for decision making.

Neutralising anti-RSV-A titres

The LL of the GMT estimate will be transformed into a [0, 1] desirability index using the function:

$$DI1 = \frac{1}{1 + \exp(4.5 * (9.5 - LL))}$$

where LL is the lower limit of the 95% confidence interval of the GMT adjusted for prevaccination titres in log base 2. The function was chosen to have a desirability of 0 at LL value  $\leq 6 \log 2$  (=128), and a desirability of 1 at LL value  $\geq 13 \log 2$ . This function is illustrated in Figure 4.

Figure 4 Desirability function for neutralising anti-RSV-A GMTs - for each investigational RSV vaccine formulation



PCA concentrations

The LL of the GMC adjusted for pre-vaccination titres estimate will be transformed using the following function:

$$DI2 = \begin{array}{c} \frac{1}{1 + \exp 0.05 * 150 - LL}, & if \ LL \le 150 \\ \frac{1}{1 + \exp 0.025 * 150 - LL}, & if \ LL \ge 150 \end{array}$$

As illustrated in Figure 5, a PCA response of 25, 150 and 400 μg/mL will have a desirability value of 0, 0.5 and 1 respectively.

Statistical Analysis Plan Amendment 3 Final

Figure 5 Desirability function for PCA concentrations - for each investigational RSV vaccine formulation



Finally, the immunogenicity index will be computed by taking the geometric mean of the 2 indexes:

$$DI = \overline{DI1 * DI2}$$

# Overall desirability index

The overall desirability index for each formulation will be obtained by computing the following weighted geometric mean:  $D = DR^{0.4} * DI^{0.6}$ .

# 14. ANNEX 4: STUDY SPECIFIC MOCK TFL

The following draft study specific mock TFLs will be used. The data display, title and footnote are for illustration purpose and will be adapted to the study specificity as indicated in the TFL TOC.

Note that there may be few changes between the study specific SAP mock TFL and the final TFLs. These editorial/minor changes will not lead to a SAP amendment.

| Template # | Table Title | Macro |
|---|---|---|
| Template 1 | Number of subjects enrolled into the study as well as the number of subject excluded from PPS analysis with reasons for exclusion | %ELIMLIST |
| Template 2 | Number of subjects vaccinated, completed and withdrawn with reason for withdrawal (Exposed set) | %DROP_SUM (OTH=1) |
| Template 3 | Number of subjects vaccinated, completed and withdrawn with reason for withdrawal (Exposed set) | %DROP_SUM (OTH=0) |
| Template 4 | Number of subjects at each visit and list of withdrawn subjects (Exposed set) | %DROPOUT |
| Template 5 | Summary of demographic characteristics (Exposed set) | %DEMOGRA |
| Template 6 | Summary of demographic characteristics by age category (Exposed set) | %DEMOGRA |
| Template 7 | Number of subjects by center (Exposed set) | %CENTER |
| Template 8 | Number of subjects by center for each age category (Exposed set) | %CENTER |
| Template 9 | Number of subjects by country and center (Exposed set) | %CENTER |
| Template 10 | Deviations from specifications for age and intervals between study visits (Exposed set) | %INT_VAL |
| Template 11 | Summary of vital signs characteristics (Exposed set) | %VITAL_SIGNS |
| Template 16 | Study Population (Exposed set) | %CTR_DEMOG |
| Template 17 | Number of enrolled subjects by country | %FREQ_DIS |
| Error! Not a valid result for table. | Number of enrolled subjects by age category | %FREQ_DIS |
| Error! Not a valid result for table. | Minimum and maximum activity dates (Exposed set) | %DATE |
| Template 26 | Incidence and nature of symptoms (solicited and unsolicited) reported during the <b>7-day</b> (Days 0-6) post-vaccination period (Exposed set) | %LOCGEN |
| Template 27 | Daily prevalence of <b>any fever</b> during the 7-day (Days 0-6) post-vaccination period (Exposed set) | %SYMPLOT |
| Template 28 | Incidence of solicited <b>local</b> symptoms reported during the 7-day (Days 0-6) post-vaccination period (Exposed set) | %FREQ |
| Template 29 | Incidence of solicited <b>local</b> symptoms reported during the 7-day (Days 0-6) post-vaccination period by <b>maximum intensity</b> (Exposed set) | %FREQ |
| Template 37 | Incidence of solicited <b>general</b> symptoms reported during the 7-day (Days 0-6) post-vaccination period (Exposed set) | %FREQ |

| | | llysis Plan Amendment 3 Final |
|---|---|---|
| Template 38 | Incidence of solicited <b>general</b> symptoms reported during the 7-day (Days 0-6) post-vaccination period <b>by maximum intensity</b> (Exposed set) | %FREQ |
| Template 39 | Percentage of subjects reporting the occurrence of unsolicited symptoms classified by MedDRA Primary System Organ Class and Preferred Term, during the <b>30-day</b> (Days 0-29) post-vaccination period (Exposed set) | %UNSOL |
| Template 39<br>*** | Percentage of subjects reporting the occurrence of unsolicited symptoms classified by MedDRA Primary System Organ Class and Preferred Term, during the 30-day (Days 0-29) post-vaccination period (Exposed set) | %UNSOL |
| Template 40 | Listing of <b>SAEs</b> reported up to study end (Exposed set) | %SAE |
| Template 41 Dist ribution of anti- Neogenin antibody concentratio n (Exposed set) Antibody | Number (%) of subjects with serious adverse events up <b>Day 7</b> (Exposed set) | %CTR_SAE |
| Anti-neogenin<br>antibody | | |
| <each group="">: 30 PreF = 30 μg PreF 60 PreF = 60 μg PreF 120 PreF = 120 μg PreF Control = Placebo N = number of subjects with available results n/% = number/perce ntage of subjects with concentration within the specified range PRE = Pre- vaccination at</each> | | |

204812 (RSV F-021) Statistical Analysis Plan Amendment 3 Final Day 0 PI(D30) = Postvaccination at Day 30 PI(D60) = Postvaccination at Day 60 PI(D90) = Postvaccination at Day 90 **Template** 

| | Statistical Alla | ilysis Plan Amendment 3 Final |
|---|---|---|
| <pre></pre> | | |
| 11223 | | |
| - - | | |
| 5 5 | | |
| ri | | |
| $ \hspace{.06cm} $ | | |
| $ \hspace{.06cm} $ | | |

| | Statistical Arial | iysis Plan Amendment 3 Finai |
|---|---|---|
| nel ta( iic - h3 n 0 eg) or go eu np i n a n t ii b o d d yy II ( 66 0 ) | Statistical Alfa | ysis Plan Amendment 3 Final |
| concentr | | |

| | Statistical Ana | llysis Plan Amendment 3 Final |
|---|---|---|
| ation within the specified range PI(D30) = Post- vaccinati on at Day 30 PI(D60) = Post- vaccinati on at Day 60 PI(D90) = Post- vaccinati on at Day 90 | | |
| Template<br>43 | | |
| Template 44 | Compliance in returning symptom information (Exposed set) | % COMPLI |
| Error!<br>Reference<br>source not<br>found. | Number and percentage of subjects taking a <b>concomitant medication</b> during the <b>7- day</b> (Days 0-6) post -vaccination period (Exposed set) | %CMED_INC |
| Template 45 Dist ribution of fold of anti- RSV-A neutralising antibody titer by cumulative pre- vaccination titer category (Per protocol set) Antibody Anti-RSV A Neu Antibody | Exploratory comparisons between groups in terms of percentage of subjects reported any Grade 2/3 AE and/or any fever >38.5°C and/or any vaccine-related SAE during the 7 day (Days 0-6) Post- vaccination period (Exposed set) | %COMP_FQ_AE |

204812 (RSV F-021)

| | | | | , - | - , | , |
|-------------|------------|------|------|----------|---------|---|
| Statistical | l Analysis | Plan | Amer | ndment 3 | 3 Final | l |

| | | Statis | ticai | Ana | ilysis | s Plar | 1 A | mei | nar | nen | (3 h | -ın | aı |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | PI(D90) | | | | | | | | | | | | |
| ≥8 | 9 PI(D30) | | | | | | | | | | | | |
| | PI(D60) | | | | | | | | | | | | |
| | PI(D90) | | | | | | | | | | + | $\top$ | |
| >9 | | | | | | | | | | | + | + | +- |
| | PI(D60) | | | | | | | | | | + | - | - |
| | | | | | | | | | | | - | + | - |
| | PI(D90) | | | | | | | | | | | + | ₩ |
| ≥1 | 10 PI(D30) | | | | | | | | | | $\bot$ | 4 | |
| | PI(D60) | | | | | | | | | | | | |
| | PI(D90) | | | | | | | | | | | | |
| ≥1 | | | | | | | | | | | | | |
| | PI(D60) | | | | | | | | | | | | |
| | PI(D90) | | | | | | | | | | | | |
| To | otal PI(D30) | | | | | | | | | | ++ | | - |
| | PI(D60) | | | | | | | | | | ++ | + | - |
| | D(D00) | | | | | | | | | | + | + | - |
| 00 5 5 5 | PI(D90) | | | | | | | | | | $\vdash$ | 4 | _ |
| 60 PreF <7 | | $\bot \bot \bot$ | | | | | $\perp$ | Ш | | | 44 | $\perp$ | $\perp$ |
| | PI(D60) | | | | | | | | | | | | |
| | PI(D90) | | | | | | | | | | | | 1 |
| ≥7 | 7 PI(D30) | | | | | | | | | | | | |
| | PI(D60) | | | | | | | | | | | $\top$ | |
| | PI(D90) | | | | | | | | | | ++ | | + |
| ≥8 | | | | | | | | | | | + | - | - |
| | PI(D60) | | | | | | | | | | - | + | - |
| | | | | | | | | | | | | + | |
| | PI(D90) | | | | | | | | | | ₩. | 4 | - |
| ≥9 | | | | | | | | | | | | | |
| | PI(D60) | | | | | | | | | | | | |
| | PI(D90) | | | | | | | | | | | | |
| ≥1 | 10 PI(D30) | | | | | | | | | | | | |
| | PI(D60) | | | | | | | | | | | | |
| | PI(D90) | | | | | | | | | | 1 | + | |
| To | otal PI(D30) | | | | | | | | | | ++ | + | +- |
| | PI(D60) | | | | | | | | | | +- | + | - |
| | D(D00) | | | | | | | | | | + | + | - |
| 100 | PI(D90) | | | | | | | | | | | + | ₩ |
| 120_ <7 | 7 PI(D30) | | | | | | | | | | | | |
| PreF | | | | | | | | | | | | | |
| | PI(D60) | | | | | | | | | | | | |
| | PI(D90) | | | | | | | | | | | | |
| ≥7 | | | | | | | | | | | | | T |
| | PI(D60) | | | | | | | | | | $\Box$ | $\top$ | T |
| | PI(D90) | | | | | | | H | | | + | + | + |
| <u>≥</u> 8 | | | | | | | + | H | - | | + | + | <del> </del> |
| | PI(D60) | | | | | | | | | | - | + | - |
| | | | | | | | | | | | | + | - |
| | PI(D90) | | | | | | | | | | Ш | | |
| ≥9 | 9 PI(D30) | | | | | | | | | | | | |
| | PI(D60) | | | | | | | | | | | | |
| | PI(D90) | | | | | | | I | | | | | |
| ≥1 | | | | | | | | | | | П | | |
| | PI(D60) | | | | | | $\top$ | H | | | T | + | T |
| | PI(D90) | | | | | | + | + | | | + | + | $\vdash$ |
| 1 1 | 1 I(D30) | | | | | ++ | - | $\vdash$ | | | + | + | $\vdash$ |
| | | | | | | | - | $\vdash$ | | $\vdash$ | + | + | ₩ |
| ≥1 | 11 PI(D30) | | | | | | | | | | | | |
| ≥1 | PI(D60) | | | | | | | | | | Ш | - | +- |
| | PI(D60)<br>PI(D90) | | | | | | | | | | | I | |
| | PI(D60)<br>PI(D90)<br>otal PI(D30) | | | | | | | | | | | Ŧ | |
| | PI(D60)<br>PI(D90) | | | | | | | | | | | | |

| | | | | Stati | stica | ıl An | alys | is Pl | an / | ٩m | en | dme | ent | 3 I | -in | al |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Control | <7 | PI(D30) | | | | | | | | | | | | | |
| | | | PI(D60) | | | | | | | | | | | | | |
| | | | PI(D90) | | | | | | | | | | | | | |
| | | ≥7 | PI(D30) | | | | | | | | + | | | | + | |
| | | <u>-1</u> | DI(DGO) | | | | - | | | | | | | | | |
| | | | PI(D60) | | | | | | | | | | | | | |
| | | | PI(D90) | | | | | | | | | | | | | |
| | | ≥8 | PI(D30) | | | | | | | | | | | | | |
| | | | PI(D60) | | | | | | | | | | | | | |
| | | | PI(D90) | | | | | | | | | | | | | |
| | | ≥9 | PI(D30) | | | | | | | | П | | | | | |
| | | | PI(D60) | | | | | | | | | | | | | |
| | | | PI(D90) | | | | | | | | | | | | | |
| | | ≥10 | PI(D30) | | | | | | | | | | | | | <u> </u> |
| | | ≥10 | | | | | | | | _ | | | | | | _ |
| | | | PI(D60) | | | | | | | | | | | | | |
| | | | PI(D90) | | | | | | | | | | | | | |
| | | Total | PI(D30) | | | | | | | | | | | | | |
| | | | PI(D60) | | | | | | | | | | | | | |
| | | | PI(D90) | | | | | | | | П | | | | | |
| 30 PreF = 30 | | | 1 1(- 5 5) | | | | | | | | | | | !_ | | <u> </u> |
| μg PreF | | | | | | | | | | | | | | | | |
| 60 PreF = 60 | | | | | | | | | | | | | | | | |
| μg PreF | | | | | | | | | | | | | | | | |
| 120 PreF = | | | | | | | | | | | | | | | | |
| 120 µg PreF | | | | | | | | | | | | | | | | |
| Control = | | | | | | | | | | | | | | | | |
| Placebo | | | | | | | | | | | | | | | | |
| <7 = Log2 | | | | | | | | | | | | | | | | |
| results are | | | | | | | | | | | | | | | | |
| less than 7 at | | | | | | | | | | | | | | | | |
| pre- | | | | | | | | | | | | | | | | |
| vaccination | | | | | | | | | | | | | | | | |
| ≥7 = Log2 | | | | | | | | | | | | | | | | |
| results are ≥7 | | | | | | | | | | | | | | | | |
| at pre- | | | | | | | | | | | | | | | | |
| vaccination | | | | | | | | | | | | | | | | |
| ≥8 = Log2 | | | | | | | | | | | | | | | | |
| results are ≥8 | | | | | | | | | | | | | | | | |
| at pre- | | | | | | | | | | | | | | | | |
| vaccination | | | | | | | | | | | | | | | | |
| ≥9 = Log2 | | | | | | | | | | | | | | | | |
| results are ≥9 | | | | | | | | | | | | | | | | |
| at pre- | | | | | | | | | | | | | | | | |
| vaccination | | | | | | | | | | | | | | | | |
| ≥10 = Log2 | | | | | | | | | | | | | | | | |
| results are | | | | | | | | | | | | | | | | |
| ≥10 at pre- | | | | | | | | | | | | | | | | |
| vaccination | | | | | | | | | | | | | | | | |
| ≥11 = Log2 | | | | | | | | | | | | | | | | |
| results are | | | | | | | | | | | | | | | | |
| ≥11 at pre- | | | | | | | | | | | | | | | | |
| vaccination | | | | | | | | | | | | | | | | |
| Total = all | | | | | | | | | | | | | | | | |
| subjects with | | | | | | | | | | | | | | | | |
| pre- | | | | | | | | | | | | | | | | |
| vaccination | | | | | | | | | | | | | | | | |
| result | | | | | | | | | | | | | | | | |
| available | | | | | | | | | | | | | | | | |
| I CIVCHICIUIT | | | | | | | | | | | | | | | | |

| | Statistical Ana | alysis Plan Amendment 3 Final |
|---|---|---|
| N = number of<br>subjects with<br>available<br>results<br>n/% =<br>number/perce<br>ntage of<br>subjects with<br>titre within the<br>specified<br>range | Statistical Ana | lysis Plan Amendment 3 Final |
| PI(D30) = Post- vaccination at Day 30 PI(D60) = Post- | | |
| vaccination at Day 60 PI(D90) = Post- vaccination at Day 90 | | |
| Template 46 | Solicited and unsolicited symptoms experienced by <b>at least 5</b> | %UNSOL (NIH=5, EVENT=1) |
| Template 47 | % of subjects, classified by MedDRA Primary System Organ Class and Preferred Term within the 30-day (Days 0-29) post-vaccination period including number of events - SAE excluded (Exposed set) | 7,001,002 (HIII 0, 2 v2 HI 1) |
| Template 48 | Distribution of change from baseline in haematology and biochemistry with respect to normal laboratory ranges (Exposed set) | %HAEMATO_BIOCH |
| Template 49 | Summary of haematology and biochemistry results by maximum grade from VISIT 2 (D7) up to VISIT 3 (D30) versus baseline (Exposed set) | %HAEMATO_BIOCH_GR_CHAN<br>GE |
| Template 32 | Summary of haematology and biochemistry results by maximum grade in the specified category from VISIT 2 (D7) up to VISIT 3 (D30) versus baseline (Exposed set) | %freq_dis |
| Template 50 | Summary of <b>haematology</b> change from baseline by maximum grade from <b>VISIT2 (D7) up to VISIT 3 (D30)</b> (Exposed set) | %HAEMATO_BIOCH_GR_CHAN<br>GE |
| Template 34 | Summary of haematology change from baseline by maximum grade in the specified category from VISIT2 (D7) up to VISIT3 (D30) (Exposed set) | %freq_dis |
| Template 35 | Individual results of <b>hemoglobin</b> levels <b>outside of the normal</b> ranges in < <i>group</i> > (Exposed set) | %HB_PROFIL |
| Template 52 | Number and percentage of subjects with anti-RSV-A neutralising antibody titer equal to or above <cut-off> and GMTs (Per protocol set)</cut-off> | %GMT |
| Template 7 | Number and percentage of subjects with anti-RSV-A neutralising antibody titer equal to or above <cut-off> and GMTs - by age category (Per protocol set)</cut-off> | %GMT |

| | | alysis Plan Amendment 3 Final |
|---|---|---|
| Template | Geometric mean of the individual ratio of anti-RSV-A | %GMRACT |
| | neutralising antibody titers at each post-vaccination timepoint | |
| | compared to pre-vaccination with 95% CI (Per protocol set) | |
| Template | GMTs and their 95% Cls for <b>anti-RSV-A</b> neutralising antibody | %GMTPLOT* |
| Tompiato | at each timepoint (Per protocol set) | 700WTT 201 |
| Template | Kinetics of GMTs for anti-RSV-A neutralising antibody on | %KIN GM* |
| remplate | | /ortin_Givi |
| | subjects with results available at all timepoints (Per protocol | |
| | set) | |
| Error! | Distribution of anti-neogenin antibody concentration (Exposed | %DIS |
| Reference | set) | |
| source not | | |
| found.1 | | |
| Error! | Distribution of fold of anti-neogenin antibody concentration | %DIS |
| Reference | (Exposed set) | |
| source not | | |
| found. | | |
| | Distribution of <b>anti-RSV-A</b> neutralising antibody titer (Per | %DIS |
| Tamonlata 11 | protocol set) | 70510 |
| Template 41 | protocor set) | |
| Dist | | |
| ribution of | | |
| anti- | | |
| Neogenin | | |
| antibody | | |
| concentratio | | |
| n (Exposed | | |
| ` ' | | |
| set) | | |
| Antibody | | |
| Anti-neogenin | | |
| antibody | | |
| Jan 1812 C Lly | | |
| <each< td=""><td></td><td></td></each<> | | |
| group>: | | |
| 30 PreF = 30 | | |
| µg PreF | | |
| 60 PreF = 60 | | |
| µg PreF | | |
| 120 PreF = | | |
| 120 µg PreF | | |
| Control = | | |
| Placebo | | |
| N = number of | | |
| subjects with | | |
| available | | |
| results | | |
| n/% = | | |
| number/perce | | |
| ntage of | | |
| subjects with | | |
| concentration | | |
| within the | | |
| specified | | |
204812 (RSV F-021) Statistical Analysis Plan Amendment 3 Final range PRE = Prevaccination at Day 0 PI(D30) = Postvaccination at Day 30 PI(D60) = Postvaccination at Day 60 PI(D90) = Postvaccination at Day 90 **Template** 

| | Statistical Ana | llysis Plan Amendment 3 Final |
|-------------------|-----------------|-------------------------------|
| 1 1 = = = | | |
| 1 1 2 2 3 | | |

| t t i i i i i i i i | ıaı |
|---------------------------------------|-----|
| d | nai |
| group>: | |
| μg PreF | |

| | Statistical Ana | llysis Plan Amendment 3 Final |
|---|---|---|
| results | | |
| n/% = | | |
| number/p | | |
| ercentag | | |
| e of | | |
| subjects | | |
| with | | |
| concentr | | |
| ation | | |
| within the | | |
| specified | | |
| range | | |
| PI(D30) = | | |
| Post- | | |
| vaccinati | | |
| on at Day<br>30 | | |
| PI(D60) = | | |
| Pi(D60) =<br>Post- | | |
| vaccinati | | |
| on at Day | | |
| 60 | | |
| PI(D90) = | | |
| Post- | | |
| vaccinati | | |
| on at Day | | |
| 90 | | |
| 30 | | |
| Template | | |
| Template | Distribution of fold of anti-RSV-A neutralising antibody titer by | %DIS |
| | pre-vaccination titer category (Per protocol set) | |
| Template 45 | Distribution of fold of anti-RSV-A neutralising antibody titer by | %DIS |
| | cumulative pre-vaccination titer category (Per protocol set) | A/== |
| Template 45 | Reverse cumulative distribution curves for anti-RSV-A | %REVCUM |
| Dist | neutralising antibody titers in each group at pre-vaccination | |
| ribution of | (Per protocol set) | |
| fold of anti- | | |
| RSV-A | | |
| neutralising | | |
| antibody | | |
| titer by | | |
| cumulative | | |
| pre- | | |
| vaccination | | |
| titer | | |
| category | | |
| (Per | | |
| protocol | | |
| set) | | |
| Antibody | | |
| Anti-RSV A Neu | | |
| Antibody | | |

| | | 204812 (RSV F-02 |
|-------------|------------|-------------------------------------------|
| | | Statistical Analysis Plan Amendment 3 Fir |
| | | PI(D60) |
| | | PI(D90) |
| | ≥7 | PI(D30) |
| | | PI(D60) |
| | | PI(D90) |
| | ≥8 | PI(D30) |
| | | PI(D60) |
| | | PI(D90) |
| | ≥9 | PI(D30) |
| | _3 | PI(D60) |
| | | PI(D90) |
| | > 40 | PI(D30) |
| | ≥10 | PI(D30) |
| | | PI(D60) |
| | | PI(D90) |
| | ≥11 | PI(D30) |
| | | PI(D60) |
| | | PI(D90) |
| | Total | PI(D30) |
| | Total | PI(D60) |
| | | PI(D90) |
| 60 D== E | <7 | PI(D30) |
| 60 PreF | <1 | |
| | | PI(D60) |
| | | PI(D90) |
| | ≥7 | PI(D30) |
| | | PI(D60) |
| | | PI(D90) |
| | ≥8 | PI(D30) |
| | | PI(D60) |
| | | PI(D90) |
| | ≥9 | PI(D30) |
| | _5 | PI(D60) |
| | | DI(D00) |
| | . 40 | PI(D90) |
| | ≥10 | PI(D30) |
| | | PI(D60) |
| | | PI(D90) |
| | Total | PI(D30) |
| | | PI(D60) |
| | | PI(D90) |
| 120<br>PreF | <7 | PI(D30) |
| 101 | | PI(D60) |
| | | PI(D90) |
| | ≥7 | PI(D30) |
| | <b>=</b> 1 | DI/DEO) |
| | | PI(D60) |
| | | PI(D90) |
| | ≥8 | PI(D30) |
| | | PI(D60) |
| | | PI(D90) |
| | ≥9 | PI(D30) |
| | | PI(D60) |
| | | PI(D90) |
| | ≥10 | PI(D30) |
| | -10 | PI(D60) |
| | | PI(D90) |
| | _11 | |
| | ≥11 | PI(D30) |
| 1 | | PI(D60) |

PI(D60)

204812 (RSV F-021)

| | | | | Stati | stica | l An | alys | is P | | | dme | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | PI(D90) | | | | | | | | | | | |
| | | Total | PI(D30) | | | | | | | | | | | |
| | | | PI(D60) | | | | | | | | | | | |
| | | | PI(D90) | | | | | | | | | | | |
| | Control | <7 | PI(D30) | | | | | | | | | | | |
| | 000. | | PI(D60) | | | | | | | | | | | |
| | | | PI(D90) | | | | | | | | | | | |
| | | ≥7 | PI(D30) | | | | | | | | | | | |
| | | <u>-1</u> | | | | | | | | | | | | |
| | | | PI(D60) | | | | | | | | | _ | | |
| | | | PI(D90) | | | | | | | | | _ | _ | |
| | | ≥8 | PI(D30) | | | | | | | | | | | |
| | | | PI(D60) | | | | | | | | | | | |
| | | | PI(D90) | | | | | | | | | | | |
| | | ≥9 | PI(D30) | | | | | | | | | | | |
| | | | PI(D60) | | | | | | | | | | | |
| | | | PI(D90) | | | | | | | | | | | |
| | | ≥10 | PI(D30) | | + | + | + | + | + | + | + | $\dashv$ | + | |
| | | | PI(D60) | | ++ | ++ | ++ | ++ | + | + | | $\dashv$ | + | |
| | | | PI(D00) | | | ++ | + | ++ | + | + | | - | - | + |
| | | Total | | | | ++ | + | + | - | + | + | - | - | $\vdash$ |
| | | Total | PI(D30) | | | | + | + | - | | | _ | - | $\perp$ |
| | | | PI(D60) | | | | | | | | | _ | | Щ |
| 0 PreF = 30 | | | PI(D90) | | | | | | | | | | | |
| results are ess than 7 at ore- vaccination ≥7 = Log2 results are ≥7 at pre- vaccination ≥8 = Log2 results are ≥8 at pre- vaccination ≥9 = Log2 results are ≥9 at pre- vaccination ≥10 = Log2 results are ≥10 at pre- | | | | | | | | | | | | | | |
| accination | | | | | | | | | | | | | | |

| | Statistical Arte | alysis Plan Amendment 3 Final |
|---|---|---|
| pre- | | |
| vaccination | | |
| result | | |
| available | | |
| N = number of | | |
| subjects with | | |
| available | | |
| results | | |
| n/% = | | |
| number/perce | | |
| ntage of | | |
| subjects with | | |
| titre within the | | |
| specified | | |
| range | | |
| PI(D30) = | | |
| , , | | |
| Post- | | |
| vaccination at | | |
| Day 30 | | |
| PI(D60) = | | |
| Post- | | |
| vaccination at | | |
| Day 60 | | |
| PI(D90) = | | |
| Post- | | |
| vaccination at | | |
| Day 90 | | |
| 24,00 | | |
| Tamanlata | | |
| Template | | |
| | Individual results of anti-RSV-A neutralising antibody titer at | %SCATTERPLOT* |
| Template | Day <30/60/90> versus pre-vaccination in <each group=""> and</each> | |
| | Control (Per protocol set) | |
| Template | Vaccine response for anti-RSV-A neutralising antibody titer at | %HUM RESP* |
| · | each post-vaccination timepoint (Per protocol set) | |
| Template 49 | Estimated GMTs and 95% CIs for anti-RSV-A neutralising | %GMT ANOVA |
| ,p | antibody titre (Per protocol set) | |
| Template | Exploratory comparisons (GMT ratios) between RSV groups | %GMT_RATIO |
| Template | | ///OIVIT_IVATIO |
| | with corresponding 95% confidence interval for anti-RSV A | |
| T 1 . | neutralizing antibody titre at <b>Day 30</b> (Per protocol set) | WALEO INDICATE |
| Template | Individual kinetics of <b>anti-neogenin</b> antibody concentrations | %NEO_INDKIN* |
| | by group (Exposed set) | |
| Template | GM of individual ratios (fold increase post over pre) and their | %GMRPLOT* |
| | 95% Cls for anti-RSV F IgG1 and IgG total antibody assays | |
| | and each group, at <b>Day 30</b> (Per protocol set) | |
| Template | Exploratory comparisons (GM ratios of fold increase post/pre) | %GMF_RATIO* |
| ' | between RSV groups with corresponding 95% confidence | _ |
| | interval for anti-RSV F IgG1 antibody concentrations at Day | |
| | 30 (Per protocol set) | |
| | Comparisons of GM ratios with corresponding 95% | %GM_RATIO_PRE.SAS** |
| Tomplete | | /0GWI_NATIO_FRE.SAS |
| Template | confidence interval between anti-RSV F antibody | |
| | concentrations (IgG Total) and anti-RSV-A neutralising | |
| | antibody titers at pre-vaccination (Per protocol set) | |
| Template | Exploratory comparisons (GM ratios of fold increase | %GM_RATIO_FI.SAS** |
| | post/pre) with corresponding 95% confidence interval | |
| | between anti-RSV F antibody concentrations (IgG Total) | |
| | and anti-RSV-A neutralising antibody titers at Day 30 (Per | |

| | protocol set) | |
|---|---|---|
| Template | Desirability index of immunogenicity during the 30-day (Days 0-29) post-vaccination period (Per protocol set) | %Immuno_DI** |
| | Desirability index of reactogenicity during the 7-day (Days 0-6) post-vaccination period (Exposed set) | %Reacto_DI** |
| Template | Desirability index based on reactogenicity and safety (Exposed set up to Day 7) and immunogenicity (Per protocol set up to Day 30) | %Overall_DI** |
| Template 59 | Percentage of subjects reporting solicited local symptoms (any grade / grade 3) during the 7-day post-vaccination period (Exposed set) | %GFREQ |

<sup>\*</sup> Name of specific macros created in study RSV F-001 (116969), RSV F-020 (201510)

\*\* Name of specific macros created in study RSV F-021 (204812)

\*\*\* It is the simplified version of Template 22 added in in-text tables for the final analysis

204812 (RSV F-021)

Statistical Analysis Plan Amendment 3 Final

### Template 1 Number of subjects enrolled into the study as well as the number of subjects excluded from the PPS analyses with reasons for exclusion

| | | Tota | | <each g<="" th=""><th>group&gt;</th></each> | group> |
|---|---|---|---|---|---|
| Title | n | S | % | n | S |
| Total enrolled cohort | | | | | |
| Study vaccine dose not administered at all but subject number allocated (code 1030) | | | | | |
| Exposed set | | | | | |
| <reason &="" code="" elimination="" for=""></reason> | | | | | |
| <reason &="" code="" elimination="" for=""></reason> | | | | | |
| Per protocol set for immunogenicity | | | | | |

#### <each group>:

30 PreF = 30 μg PreF

60 PreF = 60 µg PreF

120 PreF = 120 µg PreF

Control = Placebo

Note: Subjects may have more than one elimination code assigned

n = number of subjects with the elimination code assigned excluding subjects who have been assigned a lower elimination code number

s = number of subjects with the elimination code assigned

% = percentage of subjects in the considered Per protocol set relative to the Exposed set

### Template 2 Number of subjects vaccinated, completed and withdrawn with reason for withdrawal (Exposed set)

| | <each group=""></each> | Total |
|---|---|---|
| Number of subjects vaccinated | | |
| Number of subjects completed | | |
| Number of subjects withdrawn | | |
| Reasons for withdraw: | | |
| Serious Adverse Event | | |
| Non-serious adverse event | | |
| Protocol violation | | |
| Consent withdrawal (not due to an adverse event) | | |
| Migrated/moved from study area | | |
| Lost to follow-up (subjects with incomplete vaccination course) | | |
| Lost to follow-up (subjects with complete vaccination course) | | |
| Others | | |

#### <each group>:

30 PreF = 30 µg PreF

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

Vaccinated = number of subjects who were vaccinated in the study

Completed = number of subjects who completed last study visit

withdrawn = number of subjects who did not come for the last study visit

204812 (RSV F-021)

Statistical Analysis Plan Amendment 3 Final

### Template 3 Number of subjects vaccinated, completed and withdrawn with reason for withdrawal (Exposed set)

| | <each group=""></each> | Total |
|---|---|---|
| Number of subjects vaccinated | | |
| Number of subjects completed | | |
| Number of subjects withdrawn | | |
| Reasons for withdrawal : | | |
| Serious Adverse Event | | |
| Non-Serious Adverse Event | | |
| Protocol violation | | |
| Consent withdrawal (not due to an adverse event) | | |
| Migrated/moved from study area | | |
| Lost to follow-up (subjects with incomplete vaccination course) | | |
| Lost to follow-up (subjects with complete vaccination course) | | |
| Sponsor study termination | | |
| Other - <reason></reason> | | |
| Other - <reason></reason> | | |

#### <each group>:

30 PreF = 30 μg PreF

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

Vaccinated = number of subjects who were vaccinated in the study

Completed = number of subjects who completed last study visit

Withdrawn = number of subjects who did not come for the last study visit

Template 4 Number of subjects at each visit and list of withdrawn subjects (Exposed set)

| Group | Visit | N | Withdrawn Subject number | Reason for withdrawal |
|---|---|---|---|---|
| <each group=""></each> | VISIT 1 (D0) | | | |
| | VISIT 2 (D7) | | | |
| | VISIT 3 (D30) | | | |
| | VISIT 4 (D60) | | | |
| | VISIT 5 (D90) | | | |

#### <each group>:

 $30 \text{ PreF} = 30 \mu \text{g PreF}$ 

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

N = Number of subjects who are still in the study up to the visit

Withdrawn = Subject who did not return after the visit

204812 (RSV F-021)

Statistical Analysis Plan Amendment 3 Final

#### Template 5 Summary of demographic characteristics (Per Protocol Set)

| | | <each group=""><br/>(N=)</each> | | Total<br>(N= ) | |
|---|---|---|---|---|---|
| Characteristics | Parameters or<br>Categories | Value<br>or n | % | Value<br>or n | % |
| Age (years) at vaccination | Mean | | | | |
| | SD | | | | |
| | Median | | | | |
| | Minimum | | | | |
| | Maximum | | | | |
| Ethnicity | American Hispanic or Latino | | | | |
| | Not American Hispanic or Latino | | | | |
| Geographic Ancestry | African Heritage / African American | | | | |
| | American Indian or Alaskan Native | | | | |
| | Asian - Central/South Asian Heritage | | | | |
| | Asian - East Asian Heritage | | | | |
| | Asian - Japanese Heritage | | | | |
| | Asian - South East Asian Heritage | | | | |
| | Native Hawaiian or Other Pacific Islander | | | | |
| | White - Arabic / North African Heritage | | | | |
| | White - Caucasian / European Heritage | | | | |
| | Other | | | | |

#### <each group>:

 $30 \text{ PreF} = 30 \mu \text{g PreF}$ 

60 PreF = 60 μg PreF

120 PreF = 120 μg PreF

Control = Placebo

N = total number of subjects

n/% = number / percentage of subjects in a given category

Value = value of the considered parameter

SD = standard deviation

204812 (RSV F-021)

Statistical Analysis Plan Amendment 3 Final

### Template 6 Summary of demographic characteristics by age category (Exposed set)

| | | | | group><br> = ) | • | | | otal<br>l= ) | |
|---|---|---|---|---|---|---|---|---|---|
| | | <sub< th=""><th>group&gt;</th><th><sub< th=""><th>group&gt;</th><th><sub< th=""><th>group&gt;</th><th><sub< th=""><th>group&gt;</th></sub<></th></sub<></th></sub<></th></sub<> | group> | <sub< th=""><th>group&gt;</th><th><sub< th=""><th>group&gt;</th><th><sub< th=""><th>group&gt;</th></sub<></th></sub<></th></sub<> | group> | <sub< th=""><th>group&gt;</th><th><sub< th=""><th>group&gt;</th></sub<></th></sub<> | group> | <sub< th=""><th>group&gt;</th></sub<> | group> |
| Characteristics | Parameters or | Value or n | % | Value or n | % | Value or n | % | Value or n | % |
| | Categories | | | | | | | | |
| Age (years) at | Mean | | | | | | | | |
| vaccination | SD | | | | | | | | |
| | Median | | | | | | | | |
| | Minimum | | | | | | | | |
| | Maximum | | | | | | | | |
| Ethnicity | American Hispanic or Latino | | | | | | | | |
| • | Not American Hispanic or Latino | | | | | | | | |
| Geographic | African Heritage / African American | | | | | | | | |
| Ancestry | American Indian or Alaskan Native | | | | | | | | |
| | Asian - Central/South Asian Heritage | | | | | | | | |
| | Asian - East Asian Heritage | | | | | | | | |
| | Asian - Japanese Heritage | | | | | | | | |
| | Asian - South East Asian Heritage | | | | | | | | |
| | Native Hawaiian or Other Pacific | | | | | | | | |
| | Islander | | | | | | | | |
| | White - Arabic / North African | | | | | | | | |
| | Heritage | | | | | | | | |
| | White - Caucasian / European | | | | | | | | |
| | Heritage | | | | | | | | |
| | Other | | | | | | | | |

#### <each group>:

 $30 \text{ PreF} = 30 \mu \text{g PreF}$ 

60 PreF = 60 μg PreF

120 PreF = 120 μg PreF

Control = Placebo

N = total number of subjects

n/% = number / percentage of subjects in a given category

Value = value of the considered parameter

SD = standard deviation

#### <subgroup> by age category:

18-32Y = 18-32 years old subjects

33-45Y = 33-45 years old subjects

Statistical Analysis Plan Amendment 3 Final

#### Template 7 Number of subjects by center (Exposed set)

| | <each group=""></each> | | Total |
|--------|------------------------|---|-------|
| Center | n | n | % |
| PPD | | | |
| PPD | | | |
| All | | | |

#### <each group>:

30 PreF = 30 µg PreF

60 PreF = 60 µg PreF

120 PreF = 120 µg PreF

Control = Placebo

n = number of subjects included in each group or in total for a given center or for all centers

All = sum of all subjects in each group or in total (sum of all groups)

 $% = n/AII \times 100$ 

Center = GSK Biologicals assigned center number

#### Template 8 Number of subjects by center for each age category (Exposed set)

| | 30 F | PreF | 60 F | PreF | 120 | PreF | Cor | itrol | Total | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 18-32Y | 33-45Y | 18-32Y | 33-45Y | 18-32Y | 33-45Y | 18-32Y | 33-45Y | 18-3 | 2Y | 33-4 | 5Y |
| Center | n | n | n | n | n | n | n | n | n | % | n | % |

30 PreF = 30 µg PreF

60 PreF = 60 µg PreF

120 PreF = 120 µg PreF

Control = Placebo

18-32Y = 18-32 years old subjects

33-45Y = 33-45 years old subjects

n = number of subjects included in each group or in total for a given center or for all centers

All = sum of all subjects in each group or in total (sum of all groups)

 $% = n/AII \times 100$ 

Center = GSK Biologicals assigned center number

#### Template 9 Number of subjects by country and center (Exposed set)

| | | <each group=""></each> | | Total |
|---------|--------|------------------------|---|-------|
| Country | Center | n | n | % |
| | All | | | |
| All | All | | | |

#### <each group>:

30 PreF = 30 µg PreF

60 PreF = 60 µg PreF

120 PreF = 120 µg PreF

Control = Placebo

n = number of subjects included in each group or in total for a given center or for all centers

All = sum of all subjects in each group or in total (sum of all groups)

 $% = n/AII \times 100$ 

Center = GSK Biologicals assigned center number

204812 (RSV F-021)

Statistical Analysis Plan Amendment 3 Final

### Template 10 Deviations from specifications for age and intervals between study visits (Exposed set)

| | | Age | Dose:1-PI (D30) | Dose:1-PI (D60) | Dose:1-PI (D90) | Dose:1-<br>CONCLUSION |
|---|---|---|---|---|---|---|
| Group | | Protocol | Protocol | Protocol | Protocol | Protocol |
| | | from 18 to 45 years | from 30 to 44 days | from 56 to 70 days | from 86 to 100<br>days | from 330 to 390 days |
| <each group=""></each> | n | | | | | |
| | N | | | | | |
| | % | | | | | |
| | range | | | | | |

#### <each group>:

30 PreF = 30 μg PreF

60 PreF = 60 µg PreF

120 PreF = 120 µg PreF

Control = Placebo

N = total number of subjects with available results

n/% = number / percentage of subjects with results outside of the interval

range = minimum-maximum for age and intervals

PI(D30) = Post-vaccination at Day 30

PI(D60) = Post-vaccination at Day 60

PI(D90) = Post-vaccination at Day 90

204812 (RSV F-021)

Statistical Analysis Plan Amendment 3 Final

### Template 11 Summary of vital signs characteristics at VISIT 1 (Day 0) (Exposed set)

| | | <each group=""></each> | Total<br>N = |
|---|---|---|---|
| Characteristics | Parameters | Value | Value |
| Height (Cm) | Mean | arameters lean D ledian linimum laximum nknown lean D ledian linimum laximum laximum nknown lean D ledian linimum laximum laximum nknown lean D ledian linimum laximum nknown lean D | |
| | SD | | |
| | Median | | |
| | Minimum | | |
| | Maximum | | |
| | Unknown | | |
| Weight (Kg) | Mean SD Median Minimum Maximum Unknown Mean SD Median Minimum Maximum Unknown Mean SD Median Minimum Maximum Unknown Mean SD Median Minimum Maximum Unknown Maximum Unknown Mean SD Median Minimum Maximum Unknown Mean SD Median Minimum Maximum Unknown Mean SD Median Minimum Maximum Unknown Mean SD Median Minimum Maximum Unknown Mean SD Median Minimum Maximum Unknown Mean Minimum Maximum Unknown Mean Minimum Maximum Maximum Unknown Mean | | |
| | SD | | |
| | Median | | |
| | Minimum | | |
| | Maximum | | |
| | Unknown | | |
| Heart rate (Beats per minute) | Parameters Mean SD Median Minimum Maximum Unknown | | |
| | SD | | |
| | Median | | |
| | Minimum | | |
| | Maximum | | |
| | Unknown | | |
| Respiratory rate (Breadth per minute) | Mean | | |
| | SD | | |
| | Median | | |
| | Minimum | | |
| | Maximum | | |
| | Unknown | | |
| Systolic blood pressure (Mmhg) | Mean | | |
| | SD | | |
| | Median | | |
| | Minimum | | |
| | Maximum | | |
| | Unknown | | |
| Diastolic blood pressure (Mmhg) | Mean | | |
| | Median | | |
| | Minimum | | |
| | Maximum | | |
| | Unknown | | |

#### <each group>:

30 PreF = 30 μg PreF

60 PreF = 60 μg PreF

120 PreF = 120 µg PreF

Control = Placebo

N = total number of subjects

Value = value of the considered parameter

SD = standard deviation

## 204812 (RSV F-021) Statistical Analysis Plan Amendment 3 Final

#### **Template 12 Study Population (Exposed set)**

| Number of subjects | <each group=""></each> | Total |
|---|---|---|
| Planned, N | | |
| Randomised, N (Exposed set) | | |
| Completed, n (%) | | |
| Demographics | <each group=""></each> | Total |
| N (Exposed set) | | |
| Females:Males | | |
| Mean Age, years (SD) | | |
| Median Age, years (minimum, maximum) | | |
| White - caucasian / european heritage, n (%) | | |
| Asian – South East Asian heritage, n (%) | | |

<each group>:
30 PreF = 30 μg PreF
60 PreF = 60 μg PreF
120 PreF = 120 μg PreF
Control = Placebo

204812 (RSV F-021)

Statistical Analysis Plan Amendment 3 Final

#### Template 13 Number of enrolled subjects by country

| | | <each group=""><br/>N =</each> | Total<br>N = |
|---|---|---|---|
| Characteristics | Categories | n | n |
| Country | Czech Republic | | |
| - | Australia | | |

#### <each group>:

 $30 \text{ PreF} = 30 \mu \text{g PreF}$ 

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

N = Number of enrolled subjects

n= number of enrolled subjects included in each group or in total for a given country or for all countries

#### Template 14 Number of enrolled subjects by age category

| | | <each group=""><br/>N =</each> | Total<br>N = |
|---|---|---|---|
| Characteristics | Categories | n | n |
| Age category | Adults (18-45 years) | | |
| | Missing | | |

#### <each group>:

30 PreF = 30 µg PreF

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

N = Number of enrolled subjects

n= number of enrolled subjects included in each group or in total for a given age category or for all age categories Missing = age at dose 1 unknown

#### Template 15 Minimum and maximum activity dates (Exposed set)

| Group | Activity | <b>Activity Description</b> | Minimum date | Maximum date |
|---|---|---|---|---|
| | number | | | |
| <each group=""></each> | 10 | VISIT 1 (DAY 0) | | |
| | 20 | VISIT 2 (M 1) | | |
| | 30 | VISIT 3 (M 2) | | |
| | 40 | VISIT 4 (M 3) | | |

#### <each group>:

 $30 \text{ PreF} = 30 \mu \text{g PreF}$ 

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

204812 (RSV F-021)

Statistical Analysis Plan Amendment 3 Final

## Template 16 Incidence and nature of symptoms (solicited and unsolicited reported during the 7-day (Days 0-6) post-vaccination period (Exposed set)

| | Any sy | mptom | | | | Genera | ıl sympt | toms | | | Local s | ymptor | ns | | - |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | 95% ( | Cl | | | | 95% C | Cl | | | | 95% | CI |
| Group | N | n | % | LL | UL | N | n | % | LL | UL | N | n | % | LL | UL |
| <each group=""></each> | | | | | | | | | | | | | | | |

#### <each group>:

30 PreF = 30 µg PreF

60 PreF = 60 µg PreF

120 PreF = 120 µg PreF

Control = Placebo

N = number of subjects with the administered dose

n/% = number/percentage of subjects presenting at least one type of symptom whatever the study vaccine administered

95% CI = exact 95% confidence interval, LL = Lower Limit, UL = Upper Limit

**Note:** the same table will be generated by group/sub-group, with sub-group= age category (see SAP).

Template 17 Daily prevalence of any fever during the 7-day (Days 0-6) post-vaccination period (Exposed set)



30 PreF = 30 μg PreF 60 PreF = 60 μg PreF

120 PreF = 120 µg PreF

Control = Placebo

204812 (RSV F-021)

Statistical Analysis Plan Amendment 3 Final

### Template 18 Incidence of solicited local symptoms reported during the 7-day (Days 0-6) post-vaccination period (Exposed set)

| | | | | <each gro<="" th=""><th>up&gt;</th><th></th></each> | up> | |
|---|---|---|---|---|---|---|
| | | | | | | 95 % CI |
| Symptom | Туре | N | n | % | LL | UL |
| Pain | All | | | | | |
| | Grade 1 | | | | | |
| | Grade 2 | | | | | |
| | Grade 3 | | | | | |
| | Onset ≤48h | | | | | |
| | Medical advice | | | | | |
| Redness (mm) | All | | | | | |
| , , | >20 and ≤ 50 | | | | | |
| | >50 and ≤ 100 | | | | | |
| | >100 | | | | | |
| | Onset ≤48h | | | | | |
| | Medical advice | | | | | |
| Swelling (mm) | All | | | | | |
| | >20 and ≤ 50 | | | | | |
| | >50 and ≤ 100 | | | | | |
| | >100 | | | | | |
| | Onset ≤48h | | | | | |
| | Medical advice | | | | | |

#### <each group>:

30 PreF = 30 μg PreF

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF =120 µg PreF

Control = Placebo

N= number of subjects with the documented dose

n/%= number/percentage of subjects reporting at least once the symptom

95%CI= Exact 95% confidence interval; LL = lower limit, UL = upper limit

The maximum intensity of local injection site redness/swelling was coded as follows for adults:

- 0:  $\leq$  20 mm
- 1: > 20 mm to  $\leq$  50 mm
- 2:  $> 50 \text{ mm to} \le 100 \text{ mm}$
- 3: > 100 mm

204812 (RSV F-021)

Statistical Analysis Plan Amendment 3 Final

## Template 19 Incidence of solicited local symptoms reported during the 7-day (Days 0-6) post-vaccination period by maximum intensity (Exposed set)

| | | | < | each gro | oup> | |
|---------------|----------------|---|---|----------|------|--------|
| | | | | | | 5 % CI |
| Symptom | Туре | N | n | % | LL | UL |
| Pain | All | | | | | |
| | Grade 1 | | | | | |
| | Grade 2 | | | | | |
| | Grade 3 | | | | | |
| | Onset ≤48h | | | | | |
| | Medical advice | | | | | |
| Redness (mm) | All | | | | | |
| , , | >20 and ≤50 | | | | | |
| | >50 and ≤100 | | | | | |
| | >100 | | | | | |
| | Onset ≤48h | | | | | |
| | Medical advice | | | | | |
| Swelling (mm) | All | | | | | |
| | >20 and ≤50 | | | | | |
| | >50 and ≤100 | | | | | |
| | >100 | | | | | |
| | Onset ≤48h | | | | | |
| | Medical advice | | | | | |

#### <each group>:

 $30 \text{ PreF} = 30 \mu \text{g PreF}$ 

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

Type=Max grade & onset

All=any severity >Grade 0 for pain and any diameter >20mm for redness and swelling

N=number of vaccinated subjects who returned the diary card

n/% = number/percentage of subjects reporting the AE at least once. Maximum intensity only

95%CI = Exact 95% confidence interval; LL = lower limit, UL = upper limit

The maximum intensity of local injection site redness/swelling was coded as follows for adults:

0: ≤ 20 mm

- 1: > 20 mm to  $\leq$  50 mm
- $2: > 50 \text{ mm to} \le 100 \text{ mm}$
- 3: > 100 mm

204812 (RSV F-021)

Statistical Analysis Plan Amendment 3 Final

#### Template 20 Incidence of solicited general symptoms reported during the 7-day (Days 0-6) post-vaccination period (Exposed set)

| | | | | <each gi<="" th=""><th></th><th></th></each> | | |
|---|---|---|---|---|---|---|
| | | | | | | 5 % CI |
| Symptom | Туре | N | n | % | LL | UL |
| Fatigue | All | | | | | |
| J | Grade 1 | | | | | |
| | Grade 2 | | | | | |
| | Grade 3 | | | | | |
| | Related | | | | | |
| | Grade 2 Related | | | | | |
| | Grade 3 Related | | | | | |
| | Onset ≤48h | | | | | |
| | Medical advice | | | | | |
| Temperature (Oral)<br>(°C) | All (≥37.5) | | | | | |
| ( ) | >38.0 | | | | | |
| | >38.5 | | | | | |
| | >39.0 | | | | | |
| | >39.5 | | | | | |
| | Related | | | | | |
| | >38.5 Related | | | | | |
| | >39.5 Related | | | | | |
| | Onset ≤48h | | | | | |
| | Medical advice | | | | | |
| Gastrointestinal | All | | | | | |
| symptoms | Grade 1 | | | | | |
| oyp.tomo | Grade 2 | | | | | |
| | Grade 3 | | | | | |
| | Related | | | | | |
| | Grade 2 Related | | | | | |
| | Grade 3 Related | | | | | |
| | Onset ≤48h | | | | | |
| | Medical advice | | | | | |
| Headache | All | | | | | |
| | Grade 1 | | | | | |
| | Grade 2 | | | | | |
| | Grade 3 | | | | | |
| | Related | | | | | |
| | Grade 2 Related | | | | | |
| | Grade 3 Related | | | | | |
| | Onset ≤48h | | | | | |
| | Medical advice | | | | | |

#### <each group>:

30 PreF = 30 μg PreF

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF =120 µg PreF

Control = Placebo

N = number of subjects with the documented dose

n/% = number/percentage of subjects reporting the symptom at least once

95%CI = Exact 95% confidence interval; LL = lower limit, UL = upper limit

Temperatures were coded as follows for adults:

0: < 37.5 °C

1:  $\geq 37.5 \,^{\circ}\text{C} \text{ to} \leq 38.5 \,^{\circ}\text{C}$ 

2: > 38.5 °C to ≤ 39.5°C 3: > 39.5°C

204812 (RSV F-021)

Statistical Analysis Plan Amendment 3 Final

## Template 21 Incidence of solicited general symptoms reported during the 7-day (Days 0-6) post-vaccination period by maximum intensity (Exposed set)

| | | <each group=""></each> | | | | |
|---|---|---|---|---|---|---|
| | | | | <u> </u> | | 5 % CI |
| Symptom | Туре | N | n | % | LL | UL |
| Fatigue | All | | | | | |
| • | Grade 1 | | | | | |
| | Grade 2 | | | | | |
| | Grade 3 | | | | | |
| | Related* | | | | | |
| | Grade 2 Related | | | | | |
| | Grade 3 Related | | | | | |
| | Onset ≤48h | | | | | |
| | Medical advice | | | | | |
| Gastrointestinal | All | | | | | |
| symptoms | | | | | | |
| | Grade 1 | | | | | |
| | Grade 2 | | | | | |
| | Grade 3 | | | | | |
| | Related* | | | | | |
| | Grade 2 Related | | | | | |
| | Grade 3 Related | | | | | |
| | Onset ≤48h | | | | | |
| | Medical advice | | | | | |
| Headache | All | | | | | |
| | Grade 1 | | | | | |
| | Grade 2 | | | | | |
| | Grade 3 | | | | | |
| | Related* | | | | | |
| | Grade 2 Related | | | | | |
| | Grade 3 Related | | | | | |
| | Onset ≤48h | | | | | |
| | Medical advice | | | | | |
| Fever/(Oral) (°C) | All | | | | | |
| ( / ( / | >38.0 | | | | | |
| | >38.5 | | | | | |
| | >39.0 | | | | | |
| | >39.5 | | | | | |
| | Related* | | | | | |
| | >38.5 Related | | | | | |
| | >39.5 Related | | | | | |
| | Medical advice | | | | | |

#### <each group>:

 $30 \text{ PreF} = 30 \mu \text{g PreF}$ 

60 PreF = 60 µg PreF

120 PreF = 120 µg PreF

Control = Placebo

All=any grade>0 for Fatigue, Gastrointestinal symptoms, Headache and any >37.5°C for Temperature/(Oral)

Related\*= any grade>0 for Fatigue, Gastrointestinal symptoms, Headache and any >37.5°C for Temperature/(Oral) considered related to vaccination by the investigator

N=number of vaccinated subjects who returned the diary card

n/% = number/percentage of subjects reporting the AE at least once. Maximum intensity only

95%CI = Exact 95% confidence interval; LL = lower limit, UL = upper limit

Temperatures were coded as follows for adults:

204812 (RSV F-021) Statistical Analysis Plan Amendment 3 Final

0: < 37.5 °C

1: ≥ 37.5 °C to ≤ 38.5 °C

2: > 38.5 °C to ≤ 39.5 °C

3: > 39.5°C

204812 (RSV F-021)

Statistical Analysis Plan Amendment 3 Final

# Template 22 Percentage of subjects reporting the occurrence of unsolicited symptoms classified by MedDRA Primary System Organ Class and Preferred Term within the 30-day (Days 0-29) post-vaccination period (Exposed set)

| | | | <each group=""><br/>N =</each> | | |
|---|---|---|---|---|---|
| | | | | 95% | CI |
| Primary System Organ Class (CODE) | Preferred Term (CODE) | n | % | LL | UL |
| At least one symptom | | | | | |
| <each (code)="" soc=""></each> | <each (code)="" pt=""></each> | | | | |

#### <each group>:

30 PreF = 30 µg PreF

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

At least one symptom = at least one symptom experienced (regardless of the MedDRA Preferred Term)

N = number of subjects with at least one administered dose

n/% = number/percentage of subjects reporting at least once the symptom

95% CI= exact 95% confidence interval; LL = Lower Limit, UL = Upper Limit

Template 23 Percentage of subjects reporting the occurrence of unsolicited symptoms classified by MedDRA Primary System Organ Class and Preferred Term within the 30-day (Days 0-29) post-vaccination period (Exposed set)

| | | | group><br> = |
|---|---|---|---|
| Primary System Organ Class (CODE) | Preferred Term (CODE) | n | % |
| At least one symptom | | | |
| <each (code)="" soc=""></each> | <each (code)="" pt=""></each> | | |

#### <each group>:

30 PreF = 30 μg PreF

60 PreF = 60 μg PreF

120 PreF = 120 μg PreF

Control = Placebo

At least one symptom = at least one symptom experienced (regardless of the MedDRA Preferred Term)

*N* = number of subjects with at least one administered dose

n/% = number/percentage of subjects reporting at least once the symptom

Note: It is the simplified version of Template 22 added as one in-text tables for final analysis

#### Template 24 Listing of SAEs reported up to study end (Exposed set)

| Group | Sub.<br>No. | Sex | Country | Race | Age at onset (Year) | Verbatim | Preferred<br>term | Primary<br>System<br>Organ<br>Class | MED<br>type | Dose | Day of onset | Duration | Intensity | Causality | Outcome |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| <each< td=""><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td></each<> | | | | | | | | | | | | | | | |
| group> | | | | | | | | | | | | | | | |

<each group>:

30 PreF = 30 μg PreF 60 PreF = 60 μg PreF 120 PreF = 120 μg PreF

Control = Placebo

204812 (RSV F-021)

Statistical Analysis Plan Amendment 3 Final

### Template 25 Number (%) of subjects with serious adverse events up to study end (Exposed set)

| | | | <each group=""> N =</each> | | |
|---|---|---|---|---|---|
| Type of Event | Primary System Organ Class | Preferred Term (CODE) | n* | n | % |
| SAE | At least one symptom | | | | |
| | <each soc=""></each> | <each pt="" term=""></each> | | | |
| Related SAE | At least one symptom | | | | |
| | <each soc=""></each> | <each pt="" term=""></each> | | | |
| Fatal SAE | At least one symptom | | | | |
| | <each soc=""></each> | <each pt="" term=""></each> | | | |
| Related fatal SAE | At least one symptom | | | | |
| | <each soc=""></each> | <each pt="" term=""></each> | | | |

#### <each group>:

 $30 \text{ PreF} = 30 \mu \text{g PreF}$ 

60 PreF = 60 μg PreF

120 PreF = 120 μg PreF

Control = Placebo

N = number of subjects with the administered dose

n\* = number of events reported

n/% = number/percentage of subjects reporting the symptom at least once

#### Template 26 Compliance in returning symptom information (Exposed set)

| Group | Number | Doses | Number | Compliance | Number | Compliance |
|---|---|---|---|---|---|---|
| | of | NOT | of | % | of | % |
| | doses | according to | general SS | general SS | local SS | local SS |
| | | protocol | | | | |
| <each group=""></each> | | | | | | |

#### <each group>:

 $30 \text{ PreF} = 30 \mu \text{g PreF}$ 

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

SS = Symptom screens/sheets used for the collection of local and general solicited AEs

Compliance % = (number of doses with symptom screen/sheet return / number of administered doses) X 100

204812 (RSV F-021)

Statistical Analysis Plan Amendment 3 Final

## Template 27 Number and percentage of subjects taking a concomitant medication during the 7- day (Days 0-6) post -vaccination period (Exposed set)

| | | | <each group<="" th=""><th>&gt;</th><th></th></each> | > | |
|---|---|---|---|---|---|
| | | | | 95% | CI |
| | N | n | % | LL | UL |
| Any | | | | | |
| Any antipyretics | | | | | |
| Prophylactic antipyretics | | | | | |

#### <each group>:

30 PreF = 30 µg PreF

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

N= number of administered doses

n/%= number/percentage of subjects who took the specified concomitant medication at least once during the mentioned period

95% CI = exact 95% confidence interval, LL = Lower Limit, UL = Upper Limit

Template 28 Exploratory comparisons between groups in terms of percentage of subjects reported any Grade 2/3 AE and/or any fever >38.5°C and/or any vaccine-related SAE during the 7-day (Days 0-6) post-vaccination period (Exposed set)

| | | | | | | | | Difference in<br>(Group 1 min | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | | 95 | % CI |
| Group 1 | N | n | % | Group 2 | N | n | % | Difference | % | LL | UL |
| 30 PreF | | | | Control | | | | 30 PreF - Control | | | |
| 60 PreF | | | | Control | | | | 60 PreF - Control | | | |
| 120 PreF | | | | Control | | | | 120 PreF - Control | | | |
| 60 PreF | | | | 30 PreF | | | | 60 PreF - 30 PreF | | | |
| 120 PreF | | | | 30 PreF | | | | 120 PreF - 30 PreF | | | |
| 120 PreF | | | | 60 PreF | | | | 120 PreF - 60 PreF | | | |

#### <each group>:

30 PreF = 30 µg PreF

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

N = Number of subjects with the administered dose

n/% = number/percentage of subjects reporting a specified symptom

95% CI = Standardized asymptotic 95% confidence interval, LL = Lower Limit, UL = Upper Limit

204812 (RSV F-021)

Statistical Analysis Plan Amendment 3 Final

Template 29 Solicited and unsolicited symptoms experienced by at least 5 % of subjects, classified by MedDRA Primary System Organ Class and Preferred Term within the 30-day (Days 0-29) post-vaccination period including number of events - SAE excluded (Exposed set)

| | | <e< th=""><th>ach gi<br/>N =</th><th></th></e<> | ach gi<br>N = | |
|---|---|---|---|---|
| Primary System<br>Organ Class<br>(CODE) | Preferred Term<br>(CODE) | n* | n | % |
| At least one | | | | |
| symptom | | | | |
| <each soc=""></each> | <each pt="" term=""></each> | | | |

#### <each group>:

 $30 \text{ PreF} = 30 \mu \text{g PreF}$ 

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

At least one symptom = at least one symptom experienced (regardless of the MedDRA Preferred Term)

N = number of subjects with the administered dose

n\* = number of events reported

n/% = number/percentage of subjects reporting the symptom at least once

204812 (RSV F-021)

Statistical Analysis Plan Amendment 3 Final

### Template 30 Distribution of change from baseline in haematology and biochemistry with respect to normal laboratory ranges (Exposed set)

| | | | | | <e< th=""><th>ас</th><th>h gro</th><th>oup</th><th>&gt;</th><th></th><th></th></e<> | ас | h gro | oup | > | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | Ur | known | В | elow | Ŵ | ithin | Α | bove |
| Laboratory parameter | Timing | Baseline PRE(D0) | N | | % | _ | % | | % | | % |
| Alanine Aminotransferase | PI(D7) | Unknown | | | | | | | | | |
| (ALT) | , | Below | | | | | | | | | |
| , | | Within | | | | | | | | | |
| | | Above | | | | | | | | | |
| | PI(D30) | | | | | | | | | | |
| | PI(D60) | | | | | | | | | | |
| | PI(D90) | | | | | | | | | | |
| Aspartate Aminotransferase | PI(D7) | Unknown | | | | | | | | | |
| (AST) | | Below | | | | | | | | | |
| | | Within | | | | | | | | | |
| | | Above | | | | | | | | | |
| | PI(D30) | | | | | | | | | | |
| | PI(D60) | | | | | | | | | | |
| | PI(D90) | | | | | | | | | | |
| Creatinine | | | | | | | | | | | |
| Eosinophils | | | | | | | | | | | |
| Haemoglobin | | | | | | | | | | | |
| Lymphocytes | | | | | | | | | | | |
| Neutrophils | | | | | | | | | | | |
| Platelet count | | | | | | | | | | | |
| White Blood Cells (WBC) | | | | | | | | | | | |

#### <each group>:

30 PreF = 30 µg PreF

60 PreF = 60 µg PreF

120 PreF = 120 µg PreF

Control = Placebo

N = number of subjects with available results for the specified laboratory parameter and timing in a given baseline category

n/% = number/percentage of subjects in the specified category

Below = below the normal laboratory range defined for the specified laboratory parameter

Within = within the normal laboratory range defined for the specified laboratory parameter

Above = above the normal laboratory range defined for the specified laboratory parameter

PI(D7) = Post-vaccination at Day 7

PI(D30) = Post-vaccination at Day 30

PI(D60) = Post-vaccination at Day 60

PI(D90) = Post-vaccination at Day 90

Note: For the final analysis, three newly added in-text tables of 'Distribution of change from baseline in ALT, AST and Eosinophil's with respect to normal laboratory ranges (Exposed set)', 'Distribution of change from baseline in Creatinine, Lymphocytes and White Blood Cells (WBC) with respect to normal laboratory ranges (Exposed set)' and 'Distribution of change from baseline in Hemoglobin, Neutrophils and Platelet count with respect to normal laboratory ranges (Exposed set)' will use Template 30.

204812 (RSV F-021)

Statistical Analysis Plan Amendment 3 Final

## Template 24 Summary of haematology and biochemistry results by maximum grade from VISIT 2 (D7) up to VISIT 3 (D30) versus baseline (Exposed set)

| | | VISIT2 (D7) up to VISIT3 (D30) | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | <eacl< th=""><th>h gro</th><th>up &gt;</th><th>1</th><th></th><th></th><th></th><th></th></eacl<> | h gro | up > | 1 | | | | |
| | | | Unknown Grade 0 Grade 1 Grade 2 Grade | | | | | de 3 | Grade 4 | | | | | |
| Laboratory parameter | Baseline<br>PRE(D0) | N | n | % | n | % | n | % | n | % | n | % | n | % |
| Alanine Aminotransferase (ALT) increase by factor | Unknown | | | | | | | | | | | | | |
| | Grade 0 | | | | | | | | | | | | | |
| | Grade 1 | | | | | | | | | | | | | |
| | Grade 2 | | | | | | | | | | | | | |
| | Grade 3 | | | | | | | | | | | | | |
| | Grade 4 | | | | | | | | | | | | | |
| | Total | | | | | | | | | | | | | |
| Aspartate Aminotransferase (AST) increase by factor | | | | | | | | | | | | | | |
| Creatinine | | | | | | | | | | | | | | |
| Eosinophils increase | | | | | | | | | | | | | | |
| Hemoglobin decrease | | | | | | | | | | | | | | |
| Lymphocytes decrease | | | | | | | | | | | | | | |
| Neutrophils decrease | | | | | | | | | | | | | | |
| Platelet count decrease | | | | | | | | | | | | | | |
| White Blood Cells (WBC) decrease | | | | | | | | | | | | | | |
| White Blood Cells (WBC) increase | | | | | | | | | | | | | | |

#### <each group>:

 $30 \text{ PreF} = 30 \mu \text{g PreF}$ 

60 PreF = 60 µg PreF

120 PreF = 120 µg PreF

Control = Placebo

N = number of subjects with at least one available result for the specified laboratory parameter and follow-up period n/% = number/percentage of patients reporting at least once the laboratory event when the maximum grading over the follow-up period is considered

ALT/AST increase by factor: Grade 1 is 1.1-2.5xULN, Grade 2 is 2.6-5.0xULN, Grade 3 is 5.1-10xULN, Grade 4 is >10ULN; ULN is upper limit of the normal range.

204812 (RSV F-021)

Statistical Analysis Plan Amendment 3 Final

## Template 25 Summary of haematology and biochemistry results by maximum grade in the specified category from VISIT 2 (D7) up to VISIT 3 (D30) (Exposed set)

| | | <each group<br="">N =</each> | |
|---|---|---|---|
| Laboratory parameter | Maximum grade | n | % |
| Alanine Aminotransferase(ALT) increase by factor | Other | | |
| • | Grade 2 | | |
| | Grade 3 | | |
| | Grade 4 | | |
| Aspartate Aminotransferase(AST) increase by factor | Other | | |
| | Grade 2 | | |
| | Grade 3 | | |
| | Grade 4 | | |
| Creatinine | Other | | |
| | Grade 2 | | |
| | Grade 3 | | |
| | Grade 4 | | |
| Eosinophils increase | Other | | |
| • | Grade 2 | | |
| | Grade 3 | | |
| | Grade 4 | | |
| Hemoglobin decrease | Other | | |
| <b>3</b> | Grade 2 | | |
| | Grade 3 | | |
| | Grade 4 | | |
| Lymphocytes decrease | Other | | |
| | Grade 2 | | |
| | Grade 3 | | |
| | Grade 4 | | |
| Neutrophils decrease | Other | | |
| | Grade 2 | | |
| | Grade 3 | | |
| | Grade 4 | | |
| Platelet count decrease | Other | | |
| | Grade 2 | | |
| | Grade 3 | | |
| | Grade 4 | | |
| White Blood Cells (WBC) decrease | Other | | |
| Time Block Cone (Tibe) decirates | Grade 2 | | |
| | Grade 3 | | |
| | Grade 4 | | |
| White Blood Cells (WBC) increase | Other | | |
| Time Dioda della (TIDO) illoredae | Grade 2 | | |
| | Grade 3 | | |
| | Grade 4 | | |

<each group>:

30 PreF = 30 μg PreF

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 μg PreF

Control = Placebo

*N* = number of subjects with the administered dose

n = number of subjects in the specified category

% = n / Number of subjects with available results x 100

Other=all Unknown, Grade 0 and Grade 1

204812 (RSV F-021)

Statistical Analysis Plan Amendment 3 Final

ALT/AST increase by factor: Grade 1 is 1.1-2.5xULN, Grade 2 is 2.6-5.0xULN, Grade 3 is 5.1-10xULN, Grade 4 is >10ULN; ULN is upper limit of the normal range.

Template 26 Summary of haematology change from baseline by maximum grade from VISIT2 (D7) up to VISIT3 (D30) (Exposed set)

| | <b>\</b> | . , ~, | • •• | • • • • • | , | | , ,— | ,,,,,, | | | , -, | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | VISIT2 (D7) up to VISIT3 (D30) <each group=""> Unknown Grade 0 Grade 1 Grade 2 Grade 3 Grade 2 Grade 3 Grade 3 </each> | | | | | | | | | | | |
| | | <each group=""></each> | | | | | | | | | | | |
| | | Unkr | nown | Grade 0 | | Grade 1 | | Grade 2 | | Grade 3 | | Gra | de 4 |
| Laboratory parameter | N | n | % | n | % | n | % | n | % | n | % | n | % |
| Hemoglobin (Change from baseline) | | | | | | | | | | | | | |

#### <each group>:

30 PreF = 30 μg PreF

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

N = number of subjects with at least one available result for the specified laboratory parameter and follow-up period n/% = number/percentage of subjects reporting at least once the laboratory event when the maximum grading over the follow-up period is considered

Hemoglobin (Female) change from baseline value (gm/dL): Grade 1 is any decrease-1.5, Grade 2 is 1.6-2.0, Grade 3 is 2.1-5.0 and Grade 4 is >5.0.

204812 (RSV F-021)

Statistical Analysis Plan Amendment 3 Final

## Template 34 Summary of haematology change from baseline by maximum grade in the specified category from VISIT2 (D7) up to VISIT3 (D30) (Exposed set)

| | | <each group=""> N =</each> | |
|---|---|---|---|
| Laboratory parameter | Maximum grade | n | % |
| Hemoglobin (Change from baseline) | Other | | |
| | Grade 2 | | |
| | Grade 3 | | |
| | Grade 4 | | |

<each group>:

 $30 \text{ PreF} = 30 \mu \text{g PreF}$ 

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

*N* = number of subjects with the administered dose

n= number of subjects in the specified category

% = n / Number of subjects with available results x 100

Other=all Unknown, Grade 0 and Grade 1

Hemoglobin (Female) change from baseline value (gm/dL): Grade 1 is any decrease-1.5, Grade 2 is 1.6-2.0,

Grade 3 is 2.1-5.0 and Grade 4 is >5.0.

Statistical Analysis Plan Amendment 3 Final

Template 35 Individual results of hemoglobin levels outside of the normal ranges in < group> (Exposed set)



**Note:** This figure is shown as an example. For the unblinded report, one figure per group will be performed. For the blinded report, 4 graphs will be performed each of them presenting 25 subjects regardless of treatment (the first 25 subjects, from the 26<sup>th</sup> to the 50<sup>th</sup> subject...). The X axis will include Day 0, Day 7 and Day 30. The Y axis will be adapted according to each parameter.

204812 (RSV F-021)

Statistical Analysis Plan Amendment 3 Final

## Template 36 Number and percentage of subjects with anti-RSV-A neutralising antibody titer equal to or above <cut-off> and GMTs (Per protocol set)

| | Group | | | | ≥cı | ıt-off | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Antibody | | | | | | 959 | % CI | | 95% CI | | | |
| | | Timing | N | n | % | LL | UL | value | LL | UL | Min | Max |
| Anti-RSV-A | <each< td=""><td>PRE</td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td></each<> | PRE | | | | | | | | | | |
| Neutralizing | group> | | | | | | | | | | | |
| Antibody | | | | | | | | | | | | |
| • | | PI(D30) | | | | | | | | | | |
| | | PI(D60) | | | | | | | | | | |
| | | PI(D90) | | | | | | | | | | |

#### <each group>:

 $30 \text{ PreF} = 30 \mu \text{g PreF}$ 

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

GMT = geometric mean antibody titer calculated on all subjects

N = Number of subjects with available results

95% CI = 95% confidence interval; LL = lower limit, UL = upper limit

n/% = number/percentage of subjects with titer equal to or above specified value

MIN/MAX = Minimum/Maximum

PRE= Pre-vaccination at Day 0

PI(D30) = Post-vaccination at Day 30

PI(D60) = Post-vaccination at Day 60

PI(D90) = Post-vaccination at Day 90

204812 (RSV F-021)

Statistical Analysis Plan Amendment 3 Final

## Template 37 Number and percentage of subjects with anti-RSV-A neutralising antibody titer equal to or above <cut-off> and GMTs - by age category (Per protocol set)

| | | | | | | ≥cı | ıt-off | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Antibody | | | Timing | N | | | | % CI | | 95% CI | | | |
| | Group | Sub-<br>Group | | | n | % | LL | UL | value | LL | UL | Min | Max |
| Anti-RSV-A<br>Neutralizing<br>Antibody | <each<br>group&gt;</each<br> | 18-32Y | PRE | | | | | | | | | | |
| | | | PI(D30) | | | | | | | | | | |
| | | | PI(D60) | | | | | | | | | | |
| | | | PI(D90) | | | | | | | | | | |
| | | 33-45Y | PRE | | | | | | | | | | |
| | | | PI(D30) | | | | | | | | | | |
| | | | PI(D60) | | | | | | | | | | |
| | | | PI(D90) | | | | | | | | | | |

#### <each group>:

 $30 \text{ PreF} = 30 \mu \text{g PreF}$ 

60 PreF = 60 µg PreF

120 PreF = 120 µg PreF

Control = Placebo

18-32Y = 18-32 years old subjects

33-45Y = 33-45 years old subjects

GMT = geometric mean antibody titer calculated on all subjects

N = Number of subjects with available results

95% CI = 95% confidence interval; LL = lower limit, UL = upper limit

n/% = number/percentage of subjects with titer equal to or above specified value

MIN/MAX = Minimum/Maximum

PRE= Pre-vaccination at Day 0

PI(D30) = Post-vaccination at Day 30

PI(D60) = Post-vaccination at Day 60

PI(D90) = Post-vaccination at Day 90
204812 (RSV F-021)

Statistical Analysis Plan Amendment 3 Final

## Template 38 Geometric mean of the individual ratio of anti-RSV-A neutralising antibody titers at each post-vaccination timepoint compared to prevaccination with 95% CI (Per protocol set)

| | | | | | | | GMT rati | 0 | |
|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | 9 | 5% CI |
| Group | N | Time point | GMT | Time point | GMT | Ratio order | Value | LL | UL |
| | | description | | description | | | | | |
| <each group=""></each> | | PI(D30) | | PRE | | PI(D30) / PRE | | | |
| | | PI(D60) | | PRE | | PI(D60) / PRE | | | |
| | | PI(D90) | | PRE | | PI(D90) / PRE | | | |

#### <each group>:

30 PreF = 30 µg PreF

60 PreF = 60 µg PreF

120 PreF = 120 µg PreF

Control = Placebo

GMT = geometric mean antibody titer

N = Number of subjects with available results at the two considered time points

95% CI = 95% confidence interval; LL = Lower Limit, UL = Upper Limit

PRE= Pre-vaccination at Day 0

PI(D30) = Post-vaccination at Day 30

PI(D60) = Post-vaccination at Day 60

PI(D90) = Post-vaccination at Day 90

Statistical Analysis Plan Amendment 3 Final

Template 39 GMTs and their 95% Cls for anti-RSV-A neutralising antibody at each timepoint (Per protocol set)



30 PreF = 30 µg PreF

60 PreF = 60 µg PreF

120 PreF = 120 µg PreF

Control = Placebo

GMT = geometric mean antibody titer calculated on all subjects

95% CI = 95% confidence interval

Note: This graph is provided as an example. For each assay separately, this graph will display the 4 groups and the 4 immuno timepoints: PRE, PI(D30), PI(D60) and PI(D90)

Statistical Analysis Plan Amendment 3 Final

Template 40 Kinetics of GMTs for anti-RSV-A neutralising antibody on subjects with results available at all timepoints (Per protocol set)



30 PreF = 30 µg PreF 60 PreF = 60 µg PreF 120 PreF = 120 µg PreF Control = Placebo

GMT = geometric mean antibody titer calculated on subjects with results available at all timepoints **Note:** 

- This graph is provided as an example. For each assay separately, this graph will display the 4 groups and the 4 immuno timepoints PRE, PI(D30), PI(D60) and PI(D90)
- For the kinetic of the estimated GMTs, footnote will be adapted as: GMT = geometric mean antibody titer estimated by the ANOVA model for repeated measures

#### Template 41 Distribution of anti-Neogenin antibody concentration (Exposed set)

| | | | | | <55<br>g/ml | | ≥55<br>g/ml | | :100<br>g/ml | | 150<br>g/ml | | 200<br>g/ml | | 250<br>g/ml | | 300<br>g/ml |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Antibody | Group | Timing | N | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Anti-neogenin antibody | <each<br>group&gt;</each<br> | PRE | | | | | | | | | | | | | | | |
| | , | PI(D30) | | | | | | | | | | | | | | | |
| | | PI(D60) | | | | | | | | | | | | | | | |
| | | PI(D90) | | | | | | | | | | | | | | | |

#### <each group>:

 $30 \text{ PreF} = 30 \mu \text{g PreF}$ 

60 PreF = 60 µg PreF

120 PreF = 120 µg PreF

Control = Placebo

N = number of subjects with available results

n/% = number/percentage of subjects with concentration within the specified range

PRE = Pre-vaccination at Day 0

PI(D30) = Post-vaccination at Day 30

PI(D60) = Post-vaccination at Day 60

PI(D90) = Post-vaccination at Day 90

## Template 42 Distribution of fold of anti-neogenin antibody concentration (Exposed set)

| | | | | < | :1 | > | =1 | >= | 1.5 | > | =2 | >= | 2.5 | > | =3 | >= | 3.5 | > | =4 | >= | 4.5 | >: | =5 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Antibody | Group | Timing | N | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Anti-neogenin antibody | <each group=""></each> | PI(D30) | | | | | | | | | | | | | | | | | | | | | |
| | | PI(D60) | | | | | | | | | | | | | | | | | | | | | |
| | | PI(D90) | | | | | | | | | | | | | | | | | | | | | |

#### <each group>:

30 PreF = 30 µg PreF

60 PreF = 60 µg PreF

120 PreF = 120 µg PreF

Control = Placebo

N = number of subjects with available results

n/% = number/percentage of subjects with concentration within the specified range

PI(D30) = Post-vaccination at Day 30

PI(D60) = Post-vaccination at Day 60

PI(D90) = Post-vaccination at Day 90

204812 (RSV F-021)

Statistical Analysis Plan Amendment 3 Final

## Template 43 Distribution of anti-RSV-A neutralising antibody titer (Per protocol set)

| | | | | | <7<br>og2 | _ | ≥7<br>og2 | | ≥8<br>og2 | _ | ≥9<br>og2 | | ≥10<br>og2 | _ | :11<br>og2 | _ | :12<br>og2 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Antibody | Group | Timing | N | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Anti-RSV A Neutralizing Antibody | <each group=""></each> | PRE | | | | | | | | | | | | | | | |
| | | PI(D30) | | | | | | | | | | | | | | | |
| | | PI(D60) | | | | | | | | | | | | | | | |
| | | PI(D90) | | | | | | | | | | | | | | | |

#### <each group>:

30 PreF = 30 μg PreF

60 PreF = 60 μg PreF

120 PreF = 120 µg PreF

Control = Placebo

N = number of subjects with available results

n/% = number/percentage of subjects with titre within the specified range

PRE = Pre-vaccination at Day 0

PI(D30) = Post-vaccination at Day 30

PI(D60) = Post-vaccination at Day 60

PI(D90) = Post-vaccination at Day 90

204812 (RSV F-021) Statistical Analysis Plan Amendment 3 Final

## Template 44 Distribution of fold of anti-RSV-A neutralising antibody titer by pre-vaccination titer category (Per protocol set)

| A 4!lal | 0 | 0 | Time! | N. | | 1 | | 1 | <u>4</u> | - - | 2.5 | - | .u | ^_ | ′ | <u> '</u> | , : | _U | ŕ | 10 | _ | 1 2 | _ ! |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Antibody | Group | Sub-group | Timing | N | n | % | n º | % | n º | % n | % | n | % | n º | 6 | n ⁰ | 6 n | % | n | % | n | % I | n |
| Anti-RSV A Neutralizing | 30 PreF | <7 | PI (D30) | | | | | | | | | | | | | | | | | | | | |
| Antibody | | | PI (D60) | | | | | | | | | | | | | | | | | | | | |
| | | | PI (D90) | | | | | | | | | | | | | | | | | | | | |
| | | [7-8] | PI (D30) | | | | | | | | | | | | | | | | | | | | |
| | | | PI (D60) | | | | | | | | | | | | | | | | | | | | |
| | | | PI (D90) | | | | | | | | | | | | | | | | | | | | |
| | | ]8-9] | PI (D30) | | | | | | | | | | | | | | | | | | | | |
| | | 1 | PI (D60) | | | | | | | | | | | | | | | | | | | | T |
| | | | PI (D90) | | | | | | | | | | | | | | | | | | | | |
| | | ]9-10] | PI (D30) | | | | | | | | | | | | | | | | | | | | 7 |
| | | 10 101 | PI (D60) | | | | | | | | | | | | | | | T | | | | | |
| | | | PI (D90) | | | | | | T | | | | | | | | | | | | | | T |
| | | ]10-11] | PI (D30) | | | | | | + | | | | | | | | | t | | | | | |
| | | 1.0 | PI (D60) | | | | | | + | | | | | | | | | t | | | | | |
| | | | PI (D90) | | | | | | | | | | | | | | | | | | | | 7 |
| | | ]11-12] | PI (D30) | | | | | | | | | | | | | | | | | | | | 7 |
| | | j <u>-</u> j | PI (D60) | | | | | | | | | | | | | | | | | | | | 7 |
| | | | PI (D90) | | | | | | | | | | | | | | | t | | | | | 7 |
| | | > 12 | PI (D30) | | | | | | | | | | | | | | | | | | | | 1 |
| | | - 12 | PI (D60) | | | | | | - | | | | | | | | | | | | | | _ |
| | | | PI (D90) | | | | | | | | | | | | | + | | + | | | | | - |
| | | Total | PI (D30) | | | | | | | | | | | | | | + | | | | | | - |
| | | TOtal | PI (D60) | | | | | | | | | | | | | - | + | + | | | | | $\dashv$ |
| | | | PI (D00) | | | | | | | | | | | | | | | | | | | | 4 |
| | 60 DroF | <7 | PI (D30) | | | | | | - | | | | | | | | | | | | | | $\dashv$ |
| | 60 PreF | <1 | PI (D30) | | | | | | | | | | | | | | | - | | | | | 4 |
| | | | PI (D00) | | | | | | | | | | | | | _ | | | | | | | |
| | | [7 0] | PI (D30) | | | | | | | | | | | | | _ | | | | | | | |
| | | [7-8] | | | | | | | | | | | | | | | | | | | | | _ |
| | | | PI (D60) | | | | | | | | | | | | | | | | | | | | _ |
| | | 10.01 | PI (D90) | | | | | | | | | | | | | | | | | | | | _ |
| | | ]8-9] | PI (D30) | | | | | | | | | | | | | | _ | | | | | | 4 |
| | | | PI (D60) | | | | | | | | | | | | | | | | | | | | |
| | | | PI (D90) | | | | | | | | | | | | | | | | | | | | |
| | | ]9-10] | PI (D30) | | | | | | | | | | | | | | | | | | | | |
| | | | PI (D60) | | | | | | | | | | | | | | | | | | | | |
| | | | PI (D90) | | | | | | | | | | | | | | | | | | | | |
| | | ]10-11] | PI (D30) | | | | | | | | | | | | | | | | | | | | |
| | | | PI (D60) | | | | | | | | | | | | | | | | | | | | |
| | | | PI (D90) | | | | | | | | | | | | | | | | | | | | |
| | | ]11-12] | PI (D30) | | | | | | | | | | | | | | | | | | | | |
| | | | PI (D60) | | | | | | | | | | | | | | | | | | | | |
| | | | PI (D90) | | | | | | | | | | | | | | | | | | | | |
| | | > 12 | PI (D30) | | | | | | | | | | | | | T | 1 | T | | | | | 7 |
| | | | PI (D60) | | | | | | | | | | | | | | | | | | | | 7 |
| | | | PI (D90) | | | | | | $\dagger$ | | | | | | | | | T | | | П | | Ħ |
| | | Total | PI (D30) | 1 | | | | | | | | 1 | | H | | 1 | $\dagger$ | T | 1 | | | | $\exists$ |
| | | 1 0 101 | PI (D60) | | | | H | | $\dagger$ | | | 1 | | H | | 1 | $\dagger$ | t | | | H | | $\exists$ |
| | | | PI (D90) | | | | $\vdash$ | - | + | + | +- | - | - | H | | | | + | | | | | _ |

#### 204812 (RSV F-021)

Statistical Analysis Plan Amendment 3 Final

| | | | | | | 1 | | :1 | _≥ | 2 | ≥2 | <u></u> 5 | ≥ | 3 | ≥4 | | ≥6 | _ ≥ | 28 | ≥′ | 10 | ≥1 | 1 | ≥′ |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Antibody | Group | Sub-group | Timing | N | n | % | n | % | n | % | n | % | n | % | n % | r | ۱ % | n | % | n | % | n | % | n |
| | 120 PreF | <7 | PI (D30) | | | | | | | | | | | | | | | | | | | | | |
| | | | PI (D60) | | | | | | | | | | | | | | | | | | | | | |
| | | | PI (D90) | | | | | | | | | | | | | | | | | | | | | |
| | | [7-8] | PI (D30) | | | | | | | | | | | | | | | | | | | | | |
| | | | PI (D60) | | | | | | | | | | | | | | | | | | | | | |
| | | | PI (D90) | | | | | | | | | | | | | Ī | | | | | | | | _ |
| | | ]8-9] | PI (D30) | | | | | | | | | | | | | Ī | | | | | | | | _ |
| | | | PI (D60) | | | | | | | | | | | | | | | | | | | | | _ |
| | | | PI (D90) | | | | | | | | | | | | | | | | | | | | | |
| | | ]9-10] | PI (D30) | | | | | | | | | | | | | Ī | | | | | | | | _ |
| | | 10 101 | PI (D60) | | | | | | | | | | | | | Ī | | | | | | | | _ |
| | | | PI (D90) | | | | | | | | | | | | | T | | | | | | | | |
| | | ]10-11] | PI (D30) | | | | | | | | | | | | | T | | | | | | | | |
| | | 1.0 | PI (D60) | | | | | | | | | | | | | T | | | | | | | | |
| | | | PI (D90) | | | | | | | | | | | | | t | | | | | | | | |
| | | ]11-12] | PI (D30) | | | | | | | | | | | | | | | | | | | | | _ |
| | | j <u>-</u> j | PI (D60) | | | | | | | | | | | | | | | | | | | | | _ |
| | | | PI (D90) | | | | | | | | | | | | | | | | | | | | | _ |
| | | > 12 | PI (D30) | | | | | | | | | | | | | t | | | | | | | | |
| | | 12 | PI (D60) | | | | | | | | | | | | | t | | | | | | | | |
| | | | PI (D90) | | | | | | | | | | | | | + | | | | | | | | |
| | | Total | PI (D30) | | | | | | | | | | | | | + | | | | | | | | |
| | | Total | PI (D60) | | | | | | | | | | | | | + | | | | | | | | |
| | | | PI (D90) | | | | | | | | | | | | | t | | | | | | | | |
| | Control | <7 | PI (D30) | | | | | | | | | | | | | t | | | | | | | | |
| | Control | 1 | PI (D60) | | | | | | | | | | | | | t | | | | | | | | |
| | | | PI (D90) | | | | | | | | | | | | | + | | | | | | | | |
| | | [7-8] | PI (D30) | | | | | | | | | | | | | t | | | | | | | | |
| | | [7-0] | PI (D60) | | | | | | | | | | | | | + | | | | | | | | |
| | | | PI (D90) | | | | | | | | | | | | | + | | | | | | | | |
| | | ]8-9] | PI (D30) | | | | | | | | | | | | | + | | | | | | | | |
| | | 10-91 | PI (D60) | | | | | | | | | | | | | | | | | | | | | _ |
| | | | PI (D00) | | | | | | | | | | | | | + | | | | | | | | |
| | | 10.401 | PI (D30) | | | | | | | | | | | | | + | | | | | | | | |
| | | ]9-10] | PI (D30) | | | | | | | | | | | | | + | | | | | | | | |
| | | | | | | | | | | | | | | | | + | | + | | | | | | |
| | | 140 441 | PI (D90) | | | | | | | | | | | | | - | | | | | | | | |
| | | ]10-11] | PI (D30) | | | | | | | | | | | | | - | | | | | | | | |
| | | | PI (D60) | | | | | | | | | | | | | + | | | | | | | | |
| | | 144 401 | PI (D90) | | | | | | | | | | | | | - | | | | | | | | |
| | | ]11-12] | PI (D30) | | | | | | | | | | | | | 1 | | | | | | | | |
| | | | PI (D60) | | | | | | | | | | | | | 1 | | | | | | | | |
| | | | PI (D90) | | | | | | | | | | | | | | | | | | | | | |
| | | > 12 | PI (D30) | - | | | | | $\sqcup$ | | | | | | | 1 | $\perp$ | - | | | | | | _ |
| | | | PI (D60) | - | | | | | Ш | | | | | | | 1 | 1 | | | | | | | |
| | | | PI (D90) | | | | | | Ш | | | | Ш | | | 1 | | | | | | | | |
| | | Total | PI (D30) | | Щ | | | | Ш | | | | | | | 1 | | | | | | | | |
| | | | PI (D60) | | | | | | | | | | | | | | | | | | | | | |
| | | | PI (D90) | | | | | | | | | | | | | | | | | | | | | |

**<each group>:**30 PreF = 30 μg PreF
60 PreF = 60 μg PreF 120 PreF = 120 µg PreF

Control = Placebo

N = number of subjects with available results

204812 (RSV F-021)

Statistical Analysis Plan Amendment 3 Final

n/% = number/percentage of subjects with titer within the specified range PI(D30) = Post-vaccination at Day 30

PI(D60) = Post-vaccination at Day 60 PI(D90) = Post-vaccination at Day 90

204812 (RSV F-021) Statistical Analysis Plan Amendment 3 Final

## Template 45 Distribution of fold of anti-RSV-A neutralising antibody titer by cumulative pre-vaccination titer category (Per protocol set)

| Antibody | Graun | Sub- | Timing | | <1<br>% | | | | | | | | | | ≥6<br>ո <sup>0</sup> / | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Antibouy | Group | | illing | ואו | 70 | | /0 | 11 7 | o U | 70 | 11 | /0 | 11 7 | /0 | 11 70 | u | 70 | 11 | 70 | 11 | o ľ | il [ |
| Anti DOV A Novitralinina | 20 D== F | group | DI/D20\ | | | | | | | | H | | | | | - | - | - | | | $\perp$ | _ |
| Anti-RSV A Neutralizing | 30 PreF | <7 | PI(D30) | | | | | | | | | | | | | | | | | | | |
| Antibody | | | DI/DCO) | | | | | | | | | | | | | | | | | | 4 | $\dashv$ |
| | | | PI(D60) | | | | | | | | | | | | | | | | | | | _ |
| | | . = | PI(D90) | | | | | | | | | | | | | | | | | | 4 | _ |
| | | ≥7 | PI(D30) | | | | | | | | | | | | | | | | | | | _ |
| | | | PI(D60) | | | | | | | | | | | | | | | | | | _ | |
| | | | PI(D90) | | | | | | | | Ш | | | | | | | | | | | |
| | | ≥8 | PI(D30) | | | | | | | | Ш | | | | | | | | | | | |
| | | | PI(D60) | | | | | | | | | | | | | | | | | | | |
| | | | PI(D90) | | | | | | | | Ш | | | | | | | | | | | |
| | | ≥9 | PI(D30) | | | | | | | | | | | | | | | | | | | |
| | | | PI(D60) | | | | | | | | | | | | | | | | | | | |
| | | | PI(D90) | | | | | | | | | | | | | | | | | | | |
| | | ≥10 | PI(D30) | | | | | | | | | | | | | | | | | | | |
| | | | PI(D60) | | | | | | | | | | | | | | | | | | | |
| | | | PI(D90) | | | | | | | | | | | | | | | | | | | |
| | | ≥11 | PI(D30) | | | | | | | | | | | | | | | | | | | |
| | | | PI(D60) | | | | | | | | | | | | | | | | | | | |
| | | | PI(D90) | | | | | | | | | | | | | | | | | | T | ٦ |
| | | Total | PI(D30) | | | | | | | | П | | | | | | | | | | T | |
| | | | PI(D60) | | | | | | | | | | | | | | | | | | T | |
| | | | PI(D90) | | | | | | | | П | | | | | | | | | | T | 7 |
| | 60 PreF | <7 | PI(D30) | | | | | | | | | | | | | | | | | | T | ٦ |
| | | | PI(D60) | | | | | | | | Ħ | | | | | | | | | | T | |
| | | | PI(D90) | | | | | | | | | | | | | | | | | | 7 | T |
| | | ≥7 | PI(D30) | | | | | | | | | | | | | | | | | | T | = |
| | | -' | PI(D60) | | | | | | | | | | | | | | | | | | | $\exists$ |
| | | | PI(D90) | | | | | | | | | | | | | | | | | | $\dashv$ | = |
| | | ≥8 | PI(D30) | | | | | | | | | | | | | | | | | | + | + |
| | | 20 | PI(D60) | | | | | | | | | | | | | | | | | | + | $\dashv$ |
| | | | PI(D90) | | | | | | | | | | | | | | | | | | + | $\dashv$ |
| | | ≥9 | PI(D30) | | | + | | | | | | | | | | | | | | | _ | _ |
| | | ≥9 | PI(D30) | | | | | | | | | | | | | | | | | | 4 | _ |
| | | | PI(D00) | | | | | | | | Н | | | | | - | | | | | $\dashv$ | $\dashv$ |
| | | >10 | | | | | | | | | Н | | | | | - | | | | | $\dashv$ | 4 |
| | | ≥10 | PI(D30) | | | | | | | | | | | | | | | | | | 4 | $\dashv$ |
| | | | PI(D60) | | | | | | | | Н | | | | | | - | - | | | 4 | |
| | | | PI(D90) | | | | | | | | | | | | | | | | | | 4 | _ |
| | | Total | PI(D30) | | | | | | | | | | | | | | | | | | | _ |
| | | | PI(D60) | | | | | | | | | | | | | | | | | | | _ |
| | | <u> </u> | PI(D90) | | | $\perp \downarrow$ | | _ | | | Ш | | | | $\perp$ | 1 | | | | Ш | 4 | 4 |
| | 120 | <7 | PI(D30) | | | | | | | | | | | | | | | | | | | |
| | PreF | | | | | | | | | | Ш | | | | | | | | | Ш | 4 | _ |
| | | | PI(D60) | | | | | | | | Ш | | | | | | | | | | | |
| | | | PI(D90) | | | | | | | | Ш | | | | | | | | | | | |
| | | ≥7 | PI(D30) | | | | | | | | | | | | | | | | | | | |
| | | | PI(D60) | | | | | | | L | | | | | | | | | | | | |
| | | | PI(D90) | | | | T | | | | Π | | ١T | | | | | | | ΙŢ | I | Ī |
| | | ≥8 | PI(D30) | | | | | | | | П | | | | | | | | | | T | |
| | | | PI(D60) | | | | | | | | П | | | | | | | T | | | T | ٦ |
| | | | PI(D90) | | | $\dagger \dagger$ | | | 1 | | Ħ | | | | 1 | t | T | T | | H | $\exists$ | ٦ |

204812 (RSV F-021)

Statistical Analysis Plan Amendment 3 Final

| | | | | | <1 | | ≥1 | | | 1aıy<br>≥ <b>2</b> .5 | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| A náib a du | Cua | Sub- | Timing | NI | | | | | | | | | | | | | | | | | | | |
| Antibody | Group | group | riming | N | n 7 | ′o I | 11 % | n | 70 I | 1 % | n | 70 | n | 70 | n | 70 | n ? | /0 | n 7 | 'o I | 1 % | n | 7 |
| | | ≥9 | PI(D30) | | | | | | | | | | | | | | | | | | | | T |
| | | | PI(D60) | | | | | | | | | | | | H | | | | | | | | T |
| | | | PI(D90) | | | | | | | | t | | | | | | | | | | | | T |
| | | ≥10 | PI(D30) | | | | | | | | | | | | H | | | | | | | | Ť |
| | | | PI(D60) | | | | | | | | | | | | | | | | | | | | + |
| | | | PI(D90) | | | | | | | | t | | | | | | | | | | | | t |
| | | ≥11 | PI(D30) | | | | | | | | | | | | H | | | | | | | | Ť |
| | | | PI(D60) | | | | | | | | | | | | | | | | | | | | Ť |
| | | | PI(D90) | | | | | | | | | | | | | | | | | | | | Ť |
| | | Total | PI(D30) | | | | | | | | | | | | | | | | | | | | Ť |
| | | | PI(D60) | | | | | | | | T | | | | | | | | | | | | 1 |
| | | | PI(D90) | | | | | | | | | | | | H | | | | | | | | Ť |
| | Control | <7 | PI(D30) | | | | | | | | | | | | | | | | | | | | T |
| | | | PI(D60) | | | | | | | | T | | | | | | | | | | | | Ť |
| | | | PI(D90) | | | | | | | | | | | | П | | | | | | | | T |
| | | ≥7 | PI(D30) | | | | | | | | | | | | П | | | | | | | | T |
| | | | PI(D60) | | | | | | | | | | | | П | | | | | | | | T |
| | | | PI(D90) | | | | | | | | T | | | | | | | | | | | | 1 |
| | | ≥8 | PI(D30) | | | | | | | | | | | | П | | | | | | | | Ť |
| | | | PI(D60) | | | | | | | | | | | | П | | | | | | | | Ť |
| | | | PI(D90) | | | | | | | | | | | | | | | | | | | | Ť |
| | | ≥9 | PI(D30) | | | | | | | | | | | | | | | | | | | | Ť |
| | | | PI(D60) | | | | | | | | | | | | | | | | | | | | Ť |
| | | | PI(D90) | | | | | | | | | | | | | | | | | | | | T |
| | | ≥10 | PI(D30) | | | | | | | | | | | | | | | | | | | | T |
| | | | PI(D60) | | | | | | | | | | | | | | П | | | | | | Ť |
| | | | PI(D90) | | | | | | T | | | | | | | | П | | | | | | † |
| | | Total | PI(D30) | | | | | П | 1 | | | | | | П | | П | | | | | | Ť |
| | | | PI(D60) | | | | | | | | | | | | | | П | | | | | | Ť |
| | | | PI(D90) | | | | | | | | | | | | | | | | | | | | T |

30 PreF = 30 μg PreF

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

<7 = Log2 results are less than 7 at pre-vaccination

≥7 = Log2 results are ≥7 at pre-vaccination

≥8 = Log2 results are ≥8 at pre-vaccination

≥9 = Log2 results are ≥9 at pre-vaccination

≥10 = Log2 results are ≥10 at pre-vaccination

≥11 = Log2 results are ≥11 at pre-vaccination

Total = all subjects with pre-vaccination result available

N = number of subjects with available results

n/% = number/percentage of subjects with titre within the specified range

PI(D30) = Post-vaccination at Day 30

PI(D60) = Post-vaccination at Day 60

PI(D90) = Post-vaccination at Day 90

204812 (RSV F-021)

Statistical Analysis Plan Amendment 3 Final

Template 46 Reverse cumulative distribution curves for anti-RSV-A neutralising antibody titers in each group at <each time point> (Per protocol set)



 $30 \text{ PreF} = 30 \mu \text{g PreF}$ 

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

Note: This graph is provided as an example. The same graph will be provided for each time point and each assay comparing the values of the groups:30 PreF, 60 PreF, 120 PreF and Control.

204812 (RSV F-021)

Statistical Analysis Plan Amendment 3 Final

Template 47 Individual results of anti-RSV-A neutralising antibody titer at Day <30/60/90> versus pre-vaccination in <each group> and Control (Per protocol set)



#### <each group>:

30 PreF = 30 μg PreF 60 PreF = 60 μg PreF 120 PreF = 120 μg PreF

Control = Placebo

Note: This graph is provided as an example. The same graph will be generated for each assay and each timepoint separately (Day 30, 60, 90):

204812 (RSV F-021)

Statistical Analysis Plan Amendment 3 Final

## Template 48 Vaccine response for anti-RSV-A neutralising antibody titer at each post-vaccination timepoint (Per protocol set)

| | | | | | | Vaccine | respon | se* |
|---|---|---|---|---|---|---|---|---|
| | | | | | | | 9 | 5% CI |
| Antibody | Group | Post-vaccination timing | Pre-vaccination category (log2) | N | n | % | LL | UL |
| <each<br>antibody&gt;</each<br> | <each group=""></each> | PI(D30) | <7 | | | | | |
| | | | [7-8] | | | | | |
| | | | ]8-10] | | | | | |
| | | | >10 | | | | | |
| | | | Total | | | | | |
| | | PI(D60) | <7 | | | | | |
| | | | [7-8] | | | | | |
| | | | ]8-10] | | | | | |
| | | | >10 | | | | | |
| | | | Total | | | | | |
| | | PI(D90) | <7 | | | | | |
| | | | [7-8] | | | | | |
| | | | ]8-10] | | | | | |
| | | | >10 | | | | | |
| | | | Total | | | | | |

#### <each group>:

30 PreF = 30 µg PreF

60 PreF = 60 µg PreF

120 PreF = 120 µg PreF

Control = Placebo

Total = all subjects with pre-vaccination result available

For subjects with pre-vaccination titer <7 log2: antibody titer at post-vaccination>= 4 fold the pre-vaccination antibody titer For subjects with pre-vaccination titer in [7-8] log2: antibody titer at post-vaccination >= 3 fold the pre-vaccination antibody titer For subjects with pre-vaccination titer in [8-10] log2: antibody titer at post-vaccination >= 2.5 fold the pre-vaccination antibody titer For subjects with pre-vaccination titer >10 log2: antibody titer at post-vaccination >= 1 fold the pre-vaccination antibody titer

N = number of subjects with both pre- and post-vaccination results available

n/% = number/percentage of responders

95% CI = exact 95% confidence interval, LL = Lower Limit, UL = Upper Limit

PI(D30) = Post-vaccination at Day 30

PI(D60) = Post-vaccination at Day 60

PI(D90) = Post-vaccination at Day 90

<sup>\*</sup>Vaccine response defined as :

204812 (RSV F-021)

Statistical Analysis Plan Amendment 3 Final

## Template 49 Estimated GMTs and 95% CIs for anti-RSV-A neutralising antibody titre (Per protocol set)

| | | | | Est | imate | GMT |
|---|---|---|---|---|---|---|
| | | | | | 9 | 5% CI |
| Antibody | Group | Timing | N | value | LL | UL |
| Anti-RSV-A | <each< td=""><td>PRE</td><td></td><td></td><td></td><td></td></each<> | PRE | | | | |
| Neutralizing<br>Antibody | group> | | | | | |
| • | | PI(D30) | | | | |
| | | PI(D60) | | | | |
| | | PI(D90) | | | | |

<each group>:

30 PreF = 30 µg PreF

60 PreF = 60 µg PreF

120 PreF = 120 µg PreF

Control = Placebo

GMT = geometric mean antibody titer estimated by the ANOVA model for repeated measures

N = Number of subjects with available results

95% CI = 95% confidence interval (ANOVA model); LL = lower limit, UL = upper limit

PRE= Pre-vaccination at Day 0

PI(D30) = Post-vaccination at Day 30

PI(D60) = Post-vaccination at Day 60

PI(D90) = Post-vaccination at Day 90

## Template 50 Exploratory comparisons (GMT ratios) between RSV groups with corresponding 95% confidence interval for anti-RSV A neutralizing antibody titre at Day 30 (Per protocol set)

| | | | | | | | | GN | MT rati | 0 | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | | Tukey's | 95% CI |
| Antibody | Timepoint | Group | N | <b>GMT</b> | Group | N | GMT | Ratio order | Value | LL | UL |
| | | description | | | description | | | | | | |
| Anti-RSV A | PI(D30) | 120 PreF | | | 30 PreF | | | 120 PreF/30 PreF | | | |
| Neutralizing | | 120 PreF | | | 60 PreF | | | 120 PreF/60 PreF | | | |
| Antibody | | 60 PreF | | | 30 PreF | | | 60 PreF/30 PreF | | | |

30 PreF = 30 μg PreF

60 PreF = 60 µg PreF

120 PreF = 120 µg PreF

Control = Placebo

antibody titre estimated by the ANCOVA model

N = Number of subjects with pre-vaccination results available

Tukey's 95% CI = 95% confidence interval for the GMT ratio (ANCOVA model, Tukey's adjustment), LL = lower limit, UL = upper limit

Pvalue of ANCOVA model is xxxx

PI(D30) = Post-vaccination at Day 30

204812 (RSV F-021)

Statistical Analysis Plan Amendment 3 Final

Template 51 Individual kinetics of anti-neogenin antibody concentrations by group (Exposed set)



30 PreF = 30 μg PreF

60 PreF = 60 µg PreF

120 PreF = 120 µg PreF

Control = Placebo

Note: This graph is provided as an example. This graph will display the 4 groups and the 4 immuno timepoints: PRE, PI(D30), PI(D60) and PI(D90)

Statistical Analysis Plan Amendment 3 Final

## Template 52 GM of individual ratios (fold increase post over pre) and their 95% Cls for anti-RSV F IgG1 and IgG total antibody assays and each group, at <Day xx> (Per protocol set)



30 PreF = 30 μg PreF 60 PreF = 60 μg PreF

120 PreF = 120 µg PreF

Control = Placebo

Note: this graph is provided as an example. It will be adapted to display IgG total and Ig1 only, and the 4 groups: 30 PreF, 60 PreF, 120 PreF, Control.

204812 (RSV F-021)

Statistical Analysis Plan Amendment 3 Final

## Template 53 Exploratory comparisons (GM ratios of fold increase post/pre) between RSV groups with corresponding 95% confidence interval for anti-RSV F antibody concentrations (IgG Total) at Day 30 (Per protocol set)

| | | | | | | | G | MF rati | 0 | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | | ukey s<br>5% CI |
| Antibody | Timepoint | Group description | N | Group description | N | GMF | Ratio order | Value | LL | UL |
| anti-RSV F antibody<br>(IgG Total) | PI(D30) | 120 PreF | | 60 PreF | | | 120 Pre/60<br>PreF | | | |
| | | 120 PreF | | 30 PreF | | | 120 PreF/30<br>PreF | | | |
| | | 60 PreF | | 30 PreF | | | 60 PreF/30<br>PreF | | | |

30 PreF = 30 µg PreF

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Antibody concentration estimated by the ANOVA model

GMF = Geometric mean of fold increase

N = Number of subjects with pre-vaccination results available

Tukey's 95% CI = 95% confidence interval for the GMF ratio (ANOVA model, Tukey's adjustment), LL = lower limit, UL = upper limit

Pvalue of ANOVA model at PI(D30) is: xxxx

PI(D30) = Post-vaccination at Day 30

204812 (RSV F-021)

Statistical Analysis Plan Amendment 3 Final

# Template 54 Comparisons of GM ratios with corresponding 95% confidence interval between anti-RSV F antibody concentrations (IgG Total) and anti-RSV-A neutralising antibody titers at pre-vaccination (Per protocol set)

| | | | | | | | | | GN | 1 rati | 0 |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | 95% | 95% CI | | 95% CI | | | 95% C | | |
| Timing | Group<br>description | N | IgG Total<br>GMC | LL | UL | RSV-A neut<br>GMT | LL | UL | Value | LL | UL |
| PRE(D0) | <each group=""></each> | | | | | | | | | | |
| PRE(D0) | | | | | | | | | | | |
| PRE(D0) | | | | | | | | | | | |
| PRE(D0) | | | | | | | | | | | |

<each group>:

30 PreF = 30 μg PreF

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 μg PreF

Control = Placebo

N = Number of subjects with available results at Day30 and pre-vaccination for IgG Total and RSV-A neut

GMC = Geometric mean antibody concentration calculated on all subjects for IgG Total

GMT = Geometric mean antibody titre calculated on all subjects for RSV-A neut

GM Ratio=Geometric mean of individual ratio of IgG Total to RSV-A neut for each group

95% CI = 95% confidence interval; LL = lower limit, UL = upper limit

PRE= Pre-vaccination at Day 0

204812 (RSV F-021)

Statistical Analysis Plan Amendment 3 Final

## Template 55 Exploratory comparisons (GM ratios of fold increase post/pre) with corresponding 95% confidence interval between anti-RSV F antibody concentrations (IgG Total) and anti-RSV-A neutralising antibody titers at Day 30 (Per protocol set)

| | | | | | | | | | GN | io | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | 95% | | % CI |
| Timepoint | Group | N IgG Total 95% ( | | CI RSV-A neut | | 95% | | Value | LL | UL | |
| | • | | ĞMF | LL | UL | GMF | LL | UL | 1 | | |
| PI(D30)/PRE | <each group=""></each> | | | | | | | | | | |
| PI(D30)/PRE | | | | | | | | | | | |
| PI(D30)/PRE | | | | | | | | | | | |
| PI(D30)/PRE | | | | | | | | | | | |

<each group>:

30 PreF = 30 μg PreF

60 PreF = 60 μg PreF

120 PreF = 120 μg PreF

Control = Placebo

N = Number of subjects with available results at the two considered time points for IgG Total and anti-RSV-A GMF = Geometric mean of fold increase

GMF Ratio= Geometric mean of individual ratio of fold increase for each group

95% CI = 95% confidence interval; LL = lower limit, UL = upper limit

PRE= Pre-vaccination at Day 0

PI(D30) = Post-vaccination at Day 30

204812 (RSV F-021)

Statistical Analysis Plan Amendment 3 Final

### Template 56 Desirability index of immunogenicity during the 30-day (Days 0-29) post-vaccination period (Per protocol set)

| Group | GMT | LL1 | DI1 | GMC | LL2 | DI2 | DI |
|------------------------|-----|-----|-----|-----|-----|-----|----|
| <each group=""></each> | | | | | | | |
| J. J. J. | | | | | | | |

<each group>:

 $30 \text{ PreF} = 30 \mu \text{g PreF}$ 

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

GMT = estimated log2-scale GMT adjusted for pre-vaccination titres for neutralising anti-RSV-A

GMC = estimated log10-scale GMC adjusted for pre-vaccination concentrations for PCA

LL1 = estimated log2-scale lower limit adjusted for pre-vaccination titres for neutralising anti-RSV-A

LL2 = estimated log10-scale lower limit adjusted for pre-vaccination concentrations for PCA

DI1 = desirability index for neutralising anti-RSV-A

DI2 = desirability index for PCA concentrations

DI = immunogenicity index

### Template 57 Desirability index of reactogenicity during the 7-day (Days 0-6) post-vaccination period (Exposed set)

| Group | Incidence Rate (fR1) | Incidence Rate (fR2) | DR1 | DR2 | DR |
|---|---|---|---|---|---|
| <each group=""></each> | | | | | |

<each group>:

30 PreF = 30 µg PreF

60 PreF = 60 µgPreF

120 PreF = 120 μg PreF

Control = Placebo

IR1 = incidence rate estimated by the model for any Grade 2/3 general AEs and any related SAEs

TR2 = incidence rate estimated by the model for Grade 2/3 fever

DR1 = desirability index for any Grade 2/3 general AEs and any related SAEs

DR2 = desirability index for Grade 2/3 fever

DR = reactogenicity index

204812 (RSV F-021)

Statistical Analysis Plan Amendment 3 Final

## Template 58 Desirability index based on reactogenicity and safety (Exposed set up to Day 7) and immunogenicity (Per protocol set up to Day 30)

| Group | Reactogenicity Index | | | Immuno | genicity | Index | Overall Desirability Index |
|---|---|---|---|---|---|---|---|
| | DR1 | DR2 | DR | DI1 | DI2 | DI | DR <sup>0.4</sup> * DI <sup>0.6</sup> |
| <each group=""></each> | | | | | | | |

<each group>:

30 PreF = 30 μg PreF

60 PreF = 60 μg PreF

120 PreF = 120 μg PreF

Control = Placebo

DR1 = desirability index for any Grade 2/3 general AEs and any related SAEs

DR2 = desirability index for Grade 2/3 fever

DR = reactogenicity index

DI1 = desirability index for neutralising anti-RSV-A

DI2 = desirability index for PCA concentrations

DI = immunogenicity index

204812 (RSV F-021)

Statistical Analysis Plan Amendment 3 Final

Template 59 Percentage of subjects reporting solicited local symptoms (any grade / grade 3) during the 7-day post-vaccination period (Exposed set)



30 PreF = 30 µg PreF 60 PreF = 60 µg PreF 120 PreF = 120 µg PreF Control = Placebo

204812 (RSV F-021) Statistical Analysis Plan Amendment 4 Final

| | Statistical Analysis Plan Amendment 4 Final |
|---|---|
| <b>gsk</b> GlaxoSmithKline | Statistical Analysis Plan |
| Detailed Title: | A Phase II, randomised, observer-blind, controlled, multi-country study to rank different formulations of GSK Biologicals' investigational RSV vaccine (GSK3003891A), based on immunogenicity, reactogenicity and safety, when administered to healthy women, aged 18 – 45 years. |
| eTrack study number and<br>Abbreviated | 204812 (RSV F-021) |
| Scope: | All data pertaining to the above study. |
| Date of Statistical Analysis | Final: Amendment 4 (01-Jun-2018) |
| Plan | Amendment 3 (15-Mar-2018) |
| | Amendment 2 (09-Nov-2017) |
| | Amendment 1 (21-Jul-2017) |
| | Version 2.0 (10-Nov-2016) |
| | Version 1.0 (25-Aug-2016 |
| Co-ordinating author: | PPD (Statistician) |
| 0 01 <b>01.001.001</b> | |
| Reviewed by: | PPD (Clinical and Epidemiology Project Lead) |
| | (Clinical Research and Development Lead) |
| | (Lead statistician) |
| | (Lead statistical analyst) |
| | (Scientific writer) |
| | (Regulatory Affair) |
| | PPD (SERM physician) |
| | (Public disclosure representative) |
| Approved by: | (Clinical Research and Development Lead) |
| | Leuuj |
| | (Lead statistician) |
| | (Lead stat analyst) |
| | (Lead scientific writer) |
| APP 9000058193 | S Statistical Analysis Plan Template (Effective date: 14 April 2017) |

204812 (RSV F-021) Statistical Analysis Plan Amendment 4 Final

#### **TABLE OF CONTENTS**

| LIST OF ABBREVIATIONS | | | | PAGE |
|---|---|---|---|---|
| 2. STUDY DESIGN 18 3. OBJECTIVES 21 3.1. Primary Objective 21 3.2. Secondary objectives 21 3.3. Tertiary objective 21 4. ENDPOINTS 21 4.1. Primary 21 4.2. Secondary 22 4.3. Tertiary 22 5. ANALYSIS SETS 22 5. In Definition 22 5.1.1. Exposed Set (ES) 23 5.1.2. Per-Protocol Set (PPS) for analysis of immunogenicity 23 5.2.1. Elimination from Exposed Set (ES) 23 5.2.2. Elimination from Per-protocol analysis Set (PPS) 24 5.2.2. Elimination from Per-protocol analysis Set (PPS) 24 5.2.2. Right censored Data 26 5.3. Important protocol deviation not leading to elimination from per-protocol analysis set 26 6. STATISTICAL ANALYSES 28 6.1. Demography 28 6.2.1. Analysis of demographics/baseline characteristics planned in the protocol 28 6.2.1. Analysis of immunogenicity planned in the protocol 28 6.2.1.1. Within group analysis 29 6.2.2. Additional considerations 30 | LIS | T OF A | BBREVIATIONS | 10 |
| 3. OBJECTIVES 21 3.1 Primary Objective 21 3.2 Secondary objectives 21 3.3 Tertiary objective 21 4. ENDPOINTS 21 4.1 Primary 21 4.2 Secondary 22 4.3 Tertiary 22 5. ANALYSIS SETS 22 5.1.1 Definition 22 5.1.2 Per-Protocol Set (ES) 23 5.1.2. Per-Protocol Set (PPS) for analysis of immunogenicity 23 5.2. Criteria for eliminating data from Analysis Sets 23 5.2.1 Elimination from Exposed Set (ES) 23 5.2.2. Elimination from Per-protocol analysis Set (PPS) 24 5.2.2.1 Excluded subjects 24 5.2.2.2. Right censored Data 26 5.2.2.3 Visit-specific censored Data 26 5.3. Important protocol deviation not leading to elimination from per-protocol analysis set 26 6. STATISTICAL ANALYSES 28 6.1. Demography 28 6.2.1 Analysis of demographics/baseline characteristics planned in the protocol 28 6.2.1. Analysis of immunogenicity planned in the protocol 28 6.2.1. Between group assessment 3 | 1. | DOCU | JMENT HISTORY | 12 |
| 3.1. Primary Objective 21 3.2. Secondary objectives 21 3.3. Tertiary objective 21 4. ENDPOINTS 21 4.1. Primary 21 4.2. Secondary 22 4.3. Tertiary 22 5. ANALYSIS SETS 22 5.1. Definition 22 5.1.1. Exposed Set (ES) 23 5.1.2. Per-Protocol Set (PPS) for analysis of immunogenicity 23 5.2. Criteria for eliminating data from Analysis Sets 23 5.2.1. Elimination from Per-protocol analysis Set (PPS) 23 5.2.2.1. Excluded subjects 24 5.2.2.2. Right censored Data 26 5.2.2.2. Right censored Data 26 5.3. Important protocol deviation not leading to elimination from perprotocol analysis set 26 6. STATISTICAL ANALYSES 28 6.1. Demography 28 6.2.1. Analysis of demographics/baseline characteristics planned in the protocol 28 6.2.1. | 2. | STUD | Y DESIGN | 18 |
| 3.1. Primary Objective 21 3.2. Secondary objectives 21 3.3. Tertiary objective 21 4. ENDPOINTS 21 4.1. Primary 21 4.2. Secondary 22 4.3. Tertiary 22 5. ANALYSIS SETS 22 5.1. Definition 22 5.1.1. Exposed Set (ES) 23 5.1.2. Per-Protocol Set (PPS) for analysis of immunogenicity 23 5.2. Criteria for eliminating data from Analysis Sets 23 5.2.1. Elimination from Per-protocol analysis Set (PPS) 23 5.2.2.1. Excluded subjects 24 5.2.2.2. Right censored Data 26 5.2.2.2. Right censored Data 26 5.3. Important protocol deviation not leading to elimination from perprotocol analysis set 26 6. STATISTICAL ANALYSES 28 6.1. Demography 28 6.2.1. Analysis of demographics/baseline characteristics planned in the protocol 28 6.2.1. | 2 | 00 IE | OTIVEO | 04 |
| 3.2 Secondary objectives 21 3.3 Tertiary objective 21 4. ENDPOINTS 21 4.1 Primary 21 4.2 Secondary 22 4.3 Tertiary 22 5.1 Definition 22 5.1.1 Exposed Set (ES) 23 5.1.2 Per-Protocol Set (PPS) for analysis of immunogenicity 23 5.2.1 Elimination from Exposed Set (ES) 23 5.2.1 Elimination from Exposed Set (ES) 23 5.2.2 Elimination from Per-protocol analysis Set (PPS) 24 5.2.2.1 Excluded subjects 24 5.2.2.2 Right censored Data 26 5.3. Important protocol deviation not leading to elimination from per-protocol analysis set 26 6. STATISTICAL ANALYSES 28 6.1. Demography 28 6.2.1 Analysis of demographics/baseline characteristics planned in the protocol 28 6.2.1 Avalysis of immunogenicity planned in the protocol 28 6.2.1.1 Within group analysis 29 | 3. | | | |
| 3.3. Tertiary objective 21 4. ENDPOINTS 21 4.1. Primary 21 4.2. Secondary 22 4.3. Tertiary 22 5. ANALYSIS SETS 22 5.1. Definition 22 5.1.2 Per-Protocol Set (PS) for analysis of immunogenicity 23 5.2. Criteria for eliminating data from Analysis Sets 23 5.2.1 Elimination from Exposed Set (ES) 23 5.2.2. Elimination from Per-protocol analysis Set (PPS) 24 5.2.2.1 Excluded subjects 24 5.2.2.2 Right censored Data 26 5.2.2.3 Visit-specific censored Data 26 5.3 Important protocol deviation not leading to elimination from per-protocol analysis set 26 6. STATISTICAL ANALYSES 28 6.1. Demography 28 6.2.1 Analysis of demographics/baseline characteristics planned in the protocol 28 6.2.1. Analysis of immunogenicity planned in the protocol 28 6.2.1. Additional considerations 30 6.2.2. Additional considerations 30 6.3.1 Delimination from per-protocol 31 6.3.1. Analysis of safety 31 6.3.1. De | | _ | | |
| 4.1. Primary 21 4.2. Secondary 22 4.3. Tertiary 22 5. ANALYSIS SETS 22 5.1. Definition 23 5.1.2 Per-Protocol Set (PPS) for analysis of immunogenicity 23 5.2. Criteria for eliminating data from Analysis Sets 23 5.2.1 Elimination from Exposed Set (ES) 23 5.2.2 Eliminiation from Per-protocol analysis Set (PPS) 24 5.2.2.1 Excluded subjects 24 5.2.2.2 Right censored Data 26 5.2.2.3 Visit-specific censored Data 26 5.3. Important protocol deviation not leading to elimination from per-protocol analysis set 26 6. STATISTICAL ANALYSES 28 6.1.1 Analysis of demographics/baseline characteristics planned in the protocol 28 6.2.1 Analysis of immunogenicity planned in the protocol 28 6.2.1. Analysis of immunogenicity planned in the protocol 28 6.2.1.1 Within group analysis 29 6.2.1.2 Between group assessment 30 6.3.3.1 Analysis of safety planned in the protocol 31 6.3.1.1 Within group analysis 31 6.3.1.2 Between group assessment 32 6.4 Ana | | | | |
| 4.1. Primary 21 4.2. Secondary 22 4.3. Tertiary 22 5. ANALYSIS SETS 22 5.1. Definition 23 5.1.2 Per-Protocol Set (PPS) for analysis of immunogenicity 23 5.2. Criteria for eliminating data from Analysis Sets 23 5.2.1 Elimination from Exposed Set (ES) 23 5.2.2 Eliminiation from Per-protocol analysis Set (PPS) 24 5.2.2.1 Excluded subjects 24 5.2.2.2 Right censored Data 26 5.2.2.3 Visit-specific censored Data 26 5.3. Important protocol deviation not leading to elimination from per-protocol analysis set 26 6. STATISTICAL ANALYSES 28 6.1.1 Analysis of demographics/baseline characteristics planned in the protocol 28 6.2.1 Analysis of immunogenicity planned in the protocol 28 6.2.1. Analysis of immunogenicity planned in the protocol 28 6.2.1.1 Within group analysis 29 6.2.1.2 Between group assessment 30 6.3.3.1 Analysis of safety planned in the protocol 31 6.3.1.1 Within group analysis 31 6.3.1.2 Between group assessment 32 6.4 Ana | 4 | FNDF | POINTS | 21 |
| 4.2. Secondary 22 4.3. Tertiary 22 5. ANALYSIS SETS 22 5.1. Definition 22 5.1.1. Exposed Set (ES) 23 5.1.2. Per-Protocol Set (PPS) for analysis of immunogenicity 23 5.2. Criteria for eliminating data from Analysis Sets 23 5.2.1. Elimination from Exposed Set (ES) 23 5.2.2. Elimination from Per-protocol analysis Set (PPS) 24 5.2.2.1. Excluded subjects 24 5.2.2.2. Right censored Data 26 5.2.2.3. Visit-specific censored Data 26 5.3. Important protocol deviation not leading to elimination from per-protocol analysis set 26 6. STATISTICAL ANALYSES 28 6.1. Demography 28 6.1.1. Analysis of demographics/baseline characteristics planned in the protocol 28 6.2. Immunogenicity 28 6.2.1. Analysis of immunogenicity planned in the protocol 28 6.2.1.1. Within group analysis 29 6.2.2. Additional considerations 30 6.3.1. Analysis of safety planned in the protocol 31 6.3.1.1. Within group analysis 31 6.3.1.1. Within group analysis < | • | | | |
| 4.3. Tertiary 22 5. ANALYSIS SETS 22 5.1. Definition 22 5.1.1. Exposed Set (ES) 23 5.1.2. Per-Protocol Set (PPS) for analysis of immunogenicity 23 5.2. Criteria for eliminating data from Analysis Sets 23 5.2.1. Elimination from Exposed Set (ES) 23 5.2.2. Elimination from Per-protocol analysis Set (PPS) 24 5.2.2.1. Excluded subjects 24 5.2.2.2. Right censored Data 26 5.2.2.2. Nisit-specific censored Data 26 5.3. Important protocol deviation not leading to elimination from perprotocol analysis set 26 6. STATISTICAL ANALYSES 28 6.1. Demography 28 6.1.1. Analysis of demographics/baseline characteristics planned in the protocol 28 6.2.1. Analysis of immunogenicity planned in the protocol 28 6.2.1. Analysis of immunogenicity planned in the protocol 28 6.2.1. Additional considerations 30 6.2.2. Additional considerations 30 6.3.1. Analysis of safety 31 6.3.1. Analysis of safety planned in the protocol 31 6.3.1. Definition of desirability in the context of Simulations < | | | | |
| 5.1. Definition 22 5.1.1. Exposed Set (ES) 23 5.1.2. Per-Protocol Set (PPS) for analysis of immunogenicity 23 5.2. Criteria for eliminating data from Analysis Sets 23 5.2.1. Elimination from Exposed Set (ES) 23 5.2.2. Elimination from Per-protocol analysis Set (PPS) 24 5.2.2. Elimination from Per-protocol analysis Set (PPS) 24 5.2.2. Right censored Data 26 5.2.2. Visit-specific censored Data 26 5.3. Important protocol deviation not leading to elimination from per-protocol analysis set 28 6.1. Demography 28 6.1. Analysis of demographics/baseline characteristics planned in the protocol 28 6.2. Immunogenicity 28 6.2.1. Analysis of immunogenicity planned in the protocol 28 6.2.1. Within group analysis 29 6.2.1. Between group assessment 30 6.3.1. Analysis of safety 31 6.3.1. Within group analysis 31 6.3.1.2 Between group assessment 32 6.4. Analysis for ranking RSV formulations 33 6.4.1 Definition of desirability in the context of Simulations 33 6.4.2 Derived endpoints | | 4.3. | | |
| 5.1. Definition 22 5.1.1. Exposed Set (ES) 23 5.1.2. Per-Protocol Set (PPS) for analysis of immunogenicity 23 5.2. Criteria for eliminating data from Analysis Sets 23 5.2.1. Elimination from Exposed Set (ES) 23 5.2.2. Elimination from Per-protocol analysis Set (PPS) 24 5.2.2. Elimination from Per-protocol analysis Set (PPS) 24 5.2.2. Right censored Data 26 5.2.2. Visit-specific censored Data 26 5.3. Important protocol deviation not leading to elimination from per-protocol analysis set 28 6.1. Demography 28 6.1. Analysis of demographics/baseline characteristics planned in the protocol 28 6.2. Immunogenicity 28 6.2.1. Analysis of immunogenicity planned in the protocol 28 6.2.1. Within group analysis 29 6.2.1. Between group assessment 30 6.3.1. Analysis of safety 31 6.3.1. Within group analysis 31 6.3.1.2 Between group assessment 32 6.4. Analysis for ranking RSV formulations 33 6.4.1 Definition of desirability in the context of Simulations 33 6.4.2 Derived endpoints | 5. | ANAL | YSIS SETS | 22 |
| 5.1.2. Per-Protocol Set (PPS) for analysis of immunogenicity 23 5.2. Criteria for eliminating data from Analysis Sets 23 5.2.1. Elimination from Exposed Set (ES) 23 5.2.2. Elimination from Per-protocol analysis Set (PPS) 24 5.2.2.1. Excluded subjects 24 5.2.2.2. Right censored Data 26 5.3. Important protocol deviation not leading to elimination from perprotocol analysis set 26 6. STATISTICAL ANALYSES 28 6.1. Demography 28 6.1.1. Analysis of demographics/baseline characteristics planned in the protocol 28 6.2.1. Analysis of immunogenicity planned in the protocol 28 6.2.1. Within group analysis 29 6.2.1. Within group assessment 30 6.3. Analysis of safety 31 6.3.1. Analysis of safety planned in the protocol 31 6.3.1. Within group analysis 31 6.3.1. Between group assessment 32 6.4. Analysis for ranking RSV formulations 33 6.4.1. Definition | | | | |
| 5.2. Criteria for eliminating data from Analysis Sets 23 5.2.1 Elimination from Exposed Set (ES) 23 5.2.2. Elimination from Per-protocol analysis Set (PPS) 24 5.2.2.1 Excluded subjects 24 5.2.2.2 Right censored Data 26 5.2.2.3 Visit-specific censored Data 26 5.3. Important protocol deviation not leading to elimination from perprotocol analysis set 26 6. STATISTICAL ANALYSES 28 6.1. Demography 28 6.1.1. Analysis of demographics/baseline characteristics planned in the protocol 28 6.2. Immunogenicity 28 6.2.1. Analysis of immunogenicity planned in the protocol 28 6.2.1.1. Within group analysis 29 6.2.2. Additional considerations 30 6.3. Analysis of safety 31 6.3.1. Analysis of safety planned in the protocol 31 6.3.1. Between group assessment 32 6.4. Analysis for ranking RSV formulations 33 6.4.1. Definition of desirability in the context of Simulations 33 6.4.2. Derived endpoints 33 6.5. Analysis of medically attended RTIs 34 | | | 5.1.1. Exposed Set (ES) | 23 |
| 5.2.1. Elimination from Exposed Set (ES) 23 5.2.2. Elimination from Per-protocol analysis Set (PPS) 24 5.2.2.1. Excluded subjects 24 5.2.2.2. Right censored Data 26 5.3. Important protocol deviation not leading to elimination from per-protocol analysis set 26 6. STATISTICAL ANALYSES 28 6.1. Demography 28 6.1.1. Analysis of demographics/baseline characteristics planned in the protocol 28 6.2. Immunogenicity 28 6.2.1. Analysis of immunogenicity planned in the protocol 28 6.2.1. Within group analysis 29 6.2.1. Between group assessment 30 6.3. Analysis of safety 31 6.3.1. Analysis of safety planned in the protocol 31 6.3.1. Within group analysis 31 6.3.1. Within group analysis 31 6.3.1. Between group assessment 32 6.4. Analysis for ranking RSV formulations 33 6.4.1. Definition of desirability in the context of Simulations 33 6.4.2. Derived endpoints 33 6.5. Analysis of medically attended RTIs 34 | | | 5.1.2. Per-Protocol Set (PPS) for analysis of immunogenicity | 23 |
| 5.2.2. Elimination from Per-protocol analysis Set (PPS). 24 5.2.2.1. Excluded subjects. 24 5.2.2.2. Right censored Data 26 5.2.2.3. Visit-specific censored Data 26 5.3. Important protocol deviation not leading to elimination from perprotocol analysis set 26 6. STATISTICAL ANALYSES 28 6.1. Demography 28 6.1.1. Analysis of demographics/baseline characteristics planned in the protocol 28 6.2. Immunogenicity 28 6.2.1. Analysis of immunogenicity planned in the protocol 28 6.2.1. Within group analysis 29 6.2.1.2. Between group assessment 30 6.3. Analysis of safety 31 6.3.1. Within group analysis 31 6.3.1.1. Within group analysis 31 6.3.1.2. Between group assessment 32 6.4. Analysis for ranking RSV formulations 33 6.4.1. Definition of desirability in the context of Simulations 33 6.4.2. Derived endpoints 33 <t< td=""><td></td><td>5.2.</td><td></td><td></td></t<> | | 5.2. | | |
| 5.2.2.1. Excluded subjects. 24 5.2.2.2. Right censored Data 26 5.2.2.3. Visit-specific censored Data 26 5.3. Important protocol deviation not leading to elimination from perprotocol analysis set 26 6. STATISTICAL ANALYSES 28 6.1. Demography 28 6.1.1. Analysis of demographics/baseline characteristics planned in the protocol 28 6.2. Immunogenicity 28 6.2.1. Analysis of immunogenicity planned in the protocol 28 6.2.1. Within group analysis 29 6.2.1.2. Between group assessment 30 6.3. Analysis of safety 31 6.3.1. Analysis of safety planned in the protocol 31 6.3.1.1. Within group analysis 31 6.3.1.2. Between group assessment 32 6.4. Analysis for ranking RSV formulations 33 6.4.1. Definition of desirability in the context of Simulations 33 6.4.2. Derived endpoints 33 6.5. Analysis of medically attended RTIs 34 | | | | |
| 5.2.2.2. Right censored Data 26 5.2.2.3. Visit-specific censored Data 26 5.3. Important protocol deviation not leading to elimination from perprotocol analysis set 26 6. STATISTICAL ANALYSES 28 6.1. Demography 28 6.1.1. Analysis of demographics/baseline characteristics planned in the protocol 28 6.2. Immunogenicity 28 6.2.1. Analysis of immunogenicity planned in the protocol 28 6.2.1. Within group analysis 29 6.2.1.2. Between group assessment 30 6.3. Analysis of safety 31 6.3.1. Analysis of safety planned in the protocol 31 6.3.1. Within group analysis 31 6.3.1. Between group assessment 32 6.4. Analysis for ranking RSV formulations 33 6.4.1. Definition of desirability in the context of Simulations 33 6.4.2. Derived endpoints 33 6.5. Analysis of medically attended RTIs 34 | | | | |
| 5.2.2.3. Visit-specific censored Data | | | 5.2.2.1. Excluded subjects | 24 |
| 5.3. Important protocol deviation not leading to elimination from perprotocol analysis set | | | 5.2.2.2. Right censored Data | 26 |
| 6. STATISTICAL ANALYSES 28 6.1. Demography 28 6.1.1. Analysis of demographics/baseline characteristics planned in the protocol 28 6.2. Immunogenicity 28 6.2.1. Analysis of immunogenicity planned in the protocol 28 6.2.1.1. Within group analysis 29 6.2.1.2. Between group assessment 30 6.3. Analysis of safety 31 6.3.1. Analysis of safety planned in the protocol 31 6.3.1.1. Within group analysis 31 6.3.1.2. Between group assessment 32 6.4. Analysis for ranking RSV formulations 33 6.4.1. Definition of desirability in the context of Simulations 33 6.4.2. Derived endpoints 33 6.5. Analysis of medically attended RTIs 34 | | <b>5</b> 2 | | 20 |
| 6.1. Demography 28 6.1.1. Analysis of demographics/baseline characteristics planned in the protocol 28 6.2. Immunogenicity 28 6.2.1. Analysis of immunogenicity planned in the protocol 28 6.2.1.1. Within group analysis 29 6.2.1.2. Between group assessment 30 6.2.2. Additional considerations 30 6.3.1. Analysis of safety 31 6.3.1. Within group analysis 31 6.3.1.1. Within group analysis 31 6.3.1.2. Between group assessment 32 6.4. Analysis for ranking RSV formulations 33 6.4.1. Definition of desirability in the context of Simulations 33 6.4.2. Derived endpoints 33 6.5. Analysis of medically attended RTIs 34 | | 5.5. | | 26 |
| 6.1. Demography 28 6.1.1. Analysis of demographics/baseline characteristics planned in the protocol 28 6.2. Immunogenicity 28 6.2.1. Analysis of immunogenicity planned in the protocol 28 6.2.1.1. Within group analysis 29 6.2.1.2. Between group assessment 30 6.2.2. Additional considerations 30 6.3.1. Analysis of safety 31 6.3.1. Within group analysis 31 6.3.1.1. Within group analysis 31 6.3.1.2. Between group assessment 32 6.4. Analysis for ranking RSV formulations 33 6.4.1. Definition of desirability in the context of Simulations 33 6.4.2. Derived endpoints 33 6.5. Analysis of medically attended RTIs 34 | 6 | СТАТ | ICTICAL ANALYSES | 20 |
| 6.1.1. Analysis of demographics/baseline characteristics planned in the protocol | 0. | | | |
| in the protocol | | 0.1. | | 20 |
| 6.2. Immunogenicity 28 6.2.1. Analysis of immunogenicity planned in the protocol 28 6.2.1.1. Within group analysis 29 6.2.1.2. Between group assessment 30 6.2.2. Additional considerations 30 6.3. Analysis of safety 31 6.3.1. Analysis of safety planned in the protocol 31 6.3.1.1. Within group analysis 31 6.3.1.2. Between group assessment 32 6.4. Analysis for ranking RSV formulations 33 6.4.1. Definition of desirability in the context of Simulations 33 6.4.2. Derived endpoints 33 6.5. Analysis of medically attended RTIs 34 | | | | 28 |
| 6.2.1.1. Within group analysis 29 6.2.1.2. Between group assessment 30 6.2.2. Additional considerations 30 6.3. Analysis of safety 31 6.3.1. Analysis of safety planned in the protocol 31 6.3.1.1. Within group analysis 31 6.3.1.2. Between group assessment 32 6.4. Analysis for ranking RSV formulations 33 6.4.1. Definition of desirability in the context of Simulations 33 6.4.2. Derived endpoints 33 6.5. Analysis of medically attended RTIs 34 | | 6.2. | · | |
| 6.2.1.2. Between group assessment 30 6.2.2. Additional considerations 30 6.3. Analysis of safety 31 6.3.1. Analysis of safety planned in the protocol 31 6.3.1.1. Within group analysis 31 6.3.1.2. Between group assessment 32 6.4. Analysis for ranking RSV formulations 33 6.4.1. Definition of desirability in the context of Simulations 33 6.4.2. Derived endpoints 33 6.5. Analysis of medically attended RTIs 34 | | | | 28 |
| 6.2.2. Additional considerations | | | <u> </u> | |
| 6.3.Analysis of safety316.3.1.Analysis of safety planned in the protocol316.3.1.1.Within group analysis316.3.1.2.Between group assessment326.4.Analysis for ranking RSV formulations336.4.1.Definition of desirability in the context of Simulations336.4.2.Derived endpoints336.5.Analysis of medically attended RTIs34 | | | • • | |
| 6.3.1. Analysis of safety planned in the protocol 31 6.3.1.1. Within group analysis 31 6.3.1.2. Between group assessment 32 6.4. Analysis for ranking RSV formulations 33 6.4.1. Definition of desirability in the context of Simulations 33 6.4.2. Derived endpoints 33 6.5. Analysis of medically attended RTIs 34 | | | | |
| 6.3.1.1. Within group analysis | | 6.3. | | |
| 6.3.1.2. Between group assessment 32 6.4. Analysis for ranking RSV formulations 33 6.4.1. Definition of desirability in the context of Simulations 33 6.4.2. Derived endpoints 33 6.5. Analysis of medically attended RTIs 34 | | | | |
| 6.4. Analysis for ranking RSV formulations | | | | |
| 6.4.1. Definition of desirability in the context of Simulations 33 6.4.2. Derived endpoints 33 6.5. Analysis of medically attended RTIs 34 | | 6.4 | | |
| 6.4.2. Derived endpoints | | 0.7. | | |
| 6.5. Analysis of medically attended RTIs | | | | |
| 7 ANALYSIS INTERPRETATION 24 | | 6.5. | | |
| | 7 | ٨٨١٨١ | VOIS INTERDRETATION | 24 |

| | 204812 (RSV F-<br>Statistical Analysis Plan Amendment 4 F | |
|---|---|---|
| 8. | CONDUCT OF ANALYSES | |
| | 8.1. Sequence of analyses | |
| | 8.2. Statistical considerations for interim analyses | |
| 9. | CHANGES FROM PLANNED ANALYSES | 36 |
| 10. | LIST OF FINAL REPORT TABLES, LISTINGS AND FIGURES | 40 |
| 11. | ANNEX 1 STANDARD DATA DERIVATION RULE AND STATISTICAL METHODS | 40<br>40<br>41<br>41<br>42 |
| 12. | ANNEX 2: SUMMARY ON ELIMINATION CODES | 46 |
| 13. | ANNEX 3 CALCULATION OF INDIVIDUAL AND OVERALL DESIRABILITY INDEX | 46 |

14. ANNEX 4: STUDY SPECIFIC MOCK TFL 51

#### 204812 (RSV F-021) Statistical Analysis Plan Amendment 4 Final

#### **LIST OF TABLES**

| | | PAGE |
|---------|--------------------------------------------------|------|
| Table 1 | Study groups and epochs foreseen in the study | 19 |
| Table 2 | Study groups and treatment foreseen in the study | 19 |
| Table 3 | Blinding of study epochs | 19 |

204812 (RSV F-021) Statistical Analysis Plan Amendment 4 Final

#### **LIST OF FIGURES**

| | | PAGE |
|---|---|---|
| Figure 1. | Study design overview | 18 |
| Figure 2 | Desirability function for the incidence rate of Grade 2/3 general AEs and related SAEs - for each investigational RSV vaccine formulation | 47 |
| Figure 3 | Desirability function for the incidence rate of Grade 2/3 fever - for each investigational RSV vaccine formulation | 48 |
| Figure 4 | Desirability function for neutralising anti-RSV-A GMTs - for each investigational RSV vaccine formulation | 49 |
| Figure 5 | Desirability function for PCA concentrations - for each investigational RSV vaccine formulation | 50 |

204812 (RSV F-021) Statistical Analysis Plan Amendment 4 Final

#### **LIST OF TEMPLATE**

| | | PAGE |
|---|---|---|
| Template 1 | Number of subjects enrolled into the study as well as the number of subjects excluded from the PPS analyses with reasons for exclusion | 54 |
| Template 2 | Number of subjects vaccinated, completed and withdrawn with reason for withdrawal (Exposed set) | 54 |
| Template 3 | Number of subjects vaccinated, completed and withdrawn with reason for withdrawal (Exposed set) | 55 |
| Template 4 | Number of subjects at each visit and list of withdrawn subjects (Exposed set) | 55 |
| Template 5 | Summary of demographic characteristics (Per Protocol Set) | 56 |
| Template 6 | Summary of demographic characteristics by age category (Exposed set) | 57 |
| Template 7 | Number of subjects by center (Exposed set) | 58 |
| Template 8 | Number of subjects by center for each age category (Exposset) | |
| Template 9 | Number of subjects by country and center (Exposed set) | 58 |
| Template 10 | Deviations from specifications for age and intervals between study visits (Exposed set) | 59 |
| Template 11 | Summary of vital signs characteristics at VISIT 1 (Day 0) (Exposed set) | 60 |
| Template 12 | Study Population (Exposed set) | 61 |
| Template 13 | Number of enrolled subjects by country | 62 |
| Template 14 | Number of enrolled subjects by age category | 62 |
| Template 15 | Minimum and maximum activity dates (Exposed set) | 62 |
| Template 16 | Incidence and nature of symptoms (solicited and unsolicited reported during the 7-day (Days 0-6) post-vaccination period (Exposed set). | 63 |
| Template 17 | Daily prevalence of any fever during the 7-day (Days 0-6) post-vaccination period (Exposed set) | 63 |
| Template 18 | Incidence of solicited local symptoms reported during the 7-day (Days 0-6) post-vaccination period (Exposed set) | 64 |

204812 (RSV F-021)

| Template 19 | Statistical Analysis Plan Amendment 4 Incidence of solicited local symptoms reported during the 7-day (Days 0-6) post-vaccination period by maximum intensity | l Final |
|---|---|---|
| | (Exposed set) | 65 |
| Template 20 | Incidence of solicited general symptoms reported during the 7-day (Days 0-6) post-vaccination period (Exposed set) | 66 |
| Template 21 | Incidence of solicited general symptoms reported during the 7-day (Days 0-6) post-vaccination period by maximum intensity (Exposed set) | 67 |
| Template 22 | Percentage of subjects reporting the occurrence of unsolicited symptoms classified by MedDRA Primary System Organ Class and Preferred Term within the 30-day (Days 0-29) post-vaccination period (Exposed set). | 69 |
| Template 23 | Percentage of subjects reporting the occurrence of unsolicited symptoms classified by MedDRA Primary System Organ Class and Preferred Term within the 30-day (Days 0-29) post-vaccination period (Exposed set) | 69 |
| Template 24 | Listing of SAEs reported up to study end (Exposed set) | 70 |
| Template 25 | Number (%) of subjects with serious adverse events up to study end (Exposed set) | 71 |
| Template 26 | Compliance in returning symptom information (Exposed set) | 71 |
| Template 27 | Number and percentage of subjects taking a concomitant medication during the 7- day (Days 0-6) post -vaccination period (Exposed set) | 72 |
| Template 28 I | Exploratory comparisons between groups in terms of percentage of subjects reported any Grade 2/3 AE and/or any fever >38.5°C and/or any vaccine-related SAE during the 7-day (Days 0-6) post-vaccination period (Exposed set) | 72 |
| Template 29 | Solicited and unsolicited symptoms experienced by at least 5 % of subjects, classified by MedDRA Primary System Organ Class and Preferred Term within the 30-day (Days 0-29) post-vaccination period including number of events - SAE excluded (Exposed set). | 73 |
| Template 30 | Distribution of change from baseline in haematology and biochemistry with respect to normal laboratory ranges (Exposed set) | 73 |
| Template 31 | | |

204812 (RSV F-021)

| Template 32 | Statistical Analysis Plan Amendment 4 Fin Summary of haematology and biochemistry results by maximum | naĺ |
|---|---|---|
| | grade in the specified category from VISIT 2 (D7) up to VISIT 3 (D30) (Exposed set) | 76 |
| Template 33 | Summary of haematology change from baseline by maximum grade from VISIT2 (D7) up to VISIT3 (D30) (Exposed set) | 77 |
| Template 34 | Summary of haematology change from baseline by maximum grade in the specified category from VISIT2 (D7) up to VISIT3 (D30) (Exposed set) | <b>7</b> 8 |
| Template 35 | Individual results of hemoglobin levels outside of the normal ranges in < group> (Exposed set) | 79 |
| Template 36 | Number and percentage of subjects with anti-RSV-A neutralising antibody titer equal to or above <cut-off> and GMTs (Per protocol set)</cut-off> | 80 |
| Template 37 | Number and percentage of subjects with anti-RSV-A neutralising antibody titer equal to or above <cut-off> and GMTs - by age category (Per protocol set)</cut-off> | 81 |
| Template 38 | Geometric mean of the individual ratio of anti-RSV-A neutralising antibody titers at each post-vaccination timepoint compared to pre-vaccination with 95% CI (Per protocol set) | 82 |
| Template 39 | GMTs and their 95% CIs for anti-RSV-A neutralising antibody at each timepoint (Per protocol set) | 83 |
| Template 40 | Kinetics of GMTs for anti-RSV-A neutralising antibody on subjects with results available at all timepoints (Per protocol set) | 84 |
| Template 41 | Distribution of anti-Neogenin antibody concentration (Exposed set) | 85 |
| Template 42 | Distribution of fold of anti-neogenin antibody concentration (Exposed set) | 85 |
| Template 43 | Distribution of anti-RSV-A neutralising antibody titer (Per protocol set) | 86 |
| Template 44 | Distribution of fold of anti-RSV-A neutralising antibody titer by pre-vaccination titer category (Per protocol set) | 87 |
| Template 45 | Distribution of fold of anti-RSV-A neutralising antibody titer by cumulative pre-vaccination titer category (Per protocol set) | 90 |
| Template 46 | Reverse cumulative distribution curves for anti-RSV-A neutralising antibody titers in each group at <each point="" time=""> (Per protocol set)</each> | 92 |

204812 (RSV F-021)

| Template 47 | Statistical Analysis Plan Amendment 4 Individual results of anti-RSV-A neutralising antibody titer at Day <30/60/90> versus pre-vaccination in <each group=""> and Control</each> | Final |
|---|---|---|
| | (Per protocol set) | 93 |
| Template 48 | Vaccine response for anti-RSV-A neutralising antibody titer at each post-vaccination timepoint (Per protocol set) | 94 |
| Template 49 | Estimated GMTs and 95% CIs for anti-RSV-A neutralising antibody titre (Per protocol set) | 95 |
| Template 50 | Exploratory comparisons (GMT ratios) between RSV groups with corresponding 95% confidence interval for anti-RSV A neutralizing antibody titre at Day 30 (Per protocol set) | 95 |
| Template 51 | Individual kinetics of anti-neogenin antibody concentrations by group (Exposed set) | 96 |
| Template 52 | GM of individual ratios (fold increase post over pre) and their 95% CIs for anti-RSV F IgG1 and IgG total antibody assays and each group, at <day xx=""> (Per protocol set)</day> | 97 |
| Template 53 | Exploratory comparisons (GM ratios of fold increase post/pre) between RSV groups with corresponding 95% confidence interval for anti-RSV F antibody concentrations (IgG Total) at Day 30 (Per protocol set). | 98 |
| Template 54 | Comparisons of GM ratios with corresponding 95% confidence interval between anti-RSV F antibody concentrations (IgG Total) and anti-RSV-A neutralising antibody titers at pre-vaccination (Per protocol set) | 99 |
| Template 55 | Exploratory comparisons (GM ratios of fold increase post/pre) with corresponding 95% confidence interval between anti-RSV F antibody concentrations (IgG Total) and anti-RSV-A neutralising antibody titers at Day 30 (Per protocol set) | . 100 |
| Template 56 | Desirability index of immunogenicity during the 30-day (Days 0-29) post-vaccination period (Per protocol set) | . 101 |
| Template 57 | Desirability index of reactogenicity during the 7-day (Days 0-6) post-vaccination period (Exposed set) | . 101 |
| Template 58 | Desirability index based on reactogenicity and safety (Exposed set up to Day 7) and immunogenicity (Per protocol set up to Day 30) | 102 |
| Template 59 | Percentage of subjects reporting solicited local symptoms (any grade / grade 3) during the 7-day post-vaccination period (Exposed set) | . 103 |

204812 (RSV F-021)

#### Statistical Analysis Plan Amendment 4 Final

#### LIST OF ABBREVIATIONS

AE Adverse Event

AIDS Acquired Immunodeficiency Syndrome

ANCOVA Analysis of Covariance
ANOVA Analysis of Variance

ALT Alanine Aminotransferase AST Aspartate Aminotransferase

ATP According-to-Protocol

CDISC Clinical Data Interchange Standards Consortium

CI Confidence Interval

eCRF Electronic Case Report Form

Eli Type Internal GSK database code for type of elimination code

ES Exposed Set

FAS Full Analysis Set

GMC Geometric mean antibody concentration

GMT Geometric mean antibody titer

GSK GlaxoSmithKline

ICH International Conference on Harmonisation
IDMC Independent Data Monitoring Committee

IND Investigational New Drug

iSRC Internal Safety Review Committee

LL Lower Limit of the confidence interval

LLOQ Lower Limit of Quantification

MA-RTI Medically Attended Respiratory Tract Infection

MedDRA Medical Dictionary for Regulatory Activities

NEO Neogenin

PCA Palivizumab Competing Antibodies

PCD Primary completion Date
PCR Polymerase Chain Reaction

PPS Per Protocol Set

PreF Purified recombinant RSV F protein, engineered to preferentially

maintain the pre-fusion conformation

RSV Respiratory syncytial virus

#### 204812 (RSV F-021)

Statistical Analysis Plan Amendment 4 Final

RTI Respiratory Track Infection

SAE Serious adverse event

SAP Statistical Analysis Plan

SAS Statistical Analysis System

SBIR (GSK) Biological's Internet Randomization System

SD Standard Deviation

SRT Safety Review Team

TFL Tables Figures and Listings

TOC Table of Content

TVC Total Vaccinated Cohort

UL Upper Limit of the confidence interval

WBC White Blood Cells

### 1. DOCUMENT HISTORY

| Date | Description | Protocol Version |
|---|---|---|
| 25-AUG-2016 | Version1: first version | RSV F-021 (204812)<br>Protocol (20-Jul-2016) |
| 10-NOV-2016 | Version2.0: Description of changes from Version 1.0 are as below 1. The table of elimination code has been modified 2. Algorithm for handling of data of PCA neutralising antibody concentrations between the LOB and LLOQ was added | Final - 20-Jul-2016 |
| 21-JUL-2017 | Amendment 1: Description of changes from Version 2.0 are as below: - Use of new template for SAP (Default-APP 9000058193 Statistical Analysis Plan_v1) - In section 6. Statistical Analyses, immunogenicity was moved before safety - For the sequence of analysis, IDMC analysis up to at least Day 30 including haematology and biochemistry parameters was newly-added - The table of elimination code has been modified for more clarity - In the analysis of immunogenicity section, the distribution of fold increase of the antibody titres against RSV-A/B and concentrations against NEO have been added - In the analysis of safety section, the percentage of subjects reporting each individual solicited local/general AE during the 7-day follow-up period post vaccination based on maximum intensity per subject has been added - Evaluation of last secondary objective 'To estimate the incidence of medically attended RSV-associated RTIs up to study conclusion' will be performed based on MA-RTIs rather than MA-RSV associated RTIs - The cut-off for the updated (qualified) version of the PCA assay will be set at the level of the assay LLOQ (9.60 µg/mL). | Final - 20-Jul-2016 |

Statistical Analysis Plan Amendment 4 Final

- Algorithm for handling of data of RSV-B neutralising antibody tires between the LOB and LLOQ is defined as similar as for RSV A by considering the LOB for RSV-B is 6
- Addition of analysis of the IgG total and IgG1 subclass
- Addition of analysis of anti-RSV A and anti-PCA in the subset of subjects with IgG/IgG1 data available
- Changes of TFL/TOC
  - In the analysis of safety section, analysis on 'Individuals results of haematological and biochemical parameters outside of the normal ranges in each group' will be reported
  - In the analysis of safety section, the titles in all tables reporting 'incidence and nature of solicited and unsolicited symptoms' have been changed from 'with causal relationship to' to 'considered related to vaccination'
  - In the analysis of safety section, analysis on 'Incidence of solicited local/general symptoms reported during the 7-day post-vaccination period' will also be reported based on maximum intensity per subject for each grade
  - In the analysis of safety section, analysis on 'Number (%) of subjects reporting the occurrence of adverse events within the 7-day and 30-day postvaccination period' will be added
  - In the analysis of safety section, analysis on 'Number (%) of subjects with SAE or SAE considered related to vaccination during the study period' will not be reported
  - In the analysis of safety section, analysis on 'Number and percentage of subjects reporting the occurrence of medically attended respiration tract infections (MA-RTIs), during the 30/60/90-day post-vaccination period and up to study end' will be reported

204812 (RSV F-021) Statistical Analysis Plan Amendment 4 Final

| In the analysis of medically attended RTIs, analysis on 'viral load assessed by the quantitative PCR (RSV-A/B) of RSV-RTI cases' will be only listed in the individual listings In the analysis of immunogenicity section, tables/figures related to the analysis of RSV-B will be added In the analysis of immunogenicity section, tables/figures related to the analysis of the lgG total and lgG1 subclass will be added In the analysis of immunogenicity section, tables/figures related to the analysis of anti-RSV A and anti-PCA in the subset of subjects with lgG/lgG1 data available will be added Amendment 2: Description of changes from Amendment 2: Description of changes from Amendment 2: Description of changes from Amendment 1 are as below: Clinical Research and Development Lead) was added In the analysis of immunogenicity section, the analysis on GM ratios between anti-RSV F antibody concentrations (lgG Total) and anti-RSV-A neutralising antibody titers at pre-vaccination has been added In the analysis of immunogenicity section, the analysis on GM ratios of fold increase post/pre (Day 30/Day 0) between anti-RSV F antibody concentrations (lgG Total) and anti-RSV-A neutralising antibody titers has been added Changes of TFL/TOC In the analysis of safety section, analysis on 'individual results of hemoglobin levels beyond grade 2' have been added In the analysis of safety section, analysis on 'individual results of white |
|---|
| blood cells counts levels lower than LL' and the figures of 'Individual results of white blood cells counts levels higher |
204812 (RSV F-021)

Statistical Analysis Plan Amendment 4 Final

- In the analysis of immunogenicity section, one new template of "Comparisons of GM ratios with corresponding 95% confidence interval between anti-RSV F antibody concentrations (IgG Total) and anti-RSV-A neutralising antibody titers at prevaccination (Per protocol set)"has been added
- In the analysis of immunogenicity section, one new template of "Exploratory comparisons (GM ratios of fold increase post/pre) with corresponding 95% confidence interval between anti-RSV F antibody concentrations (IgG Total) and anti-RSV-A neutralising antibody titers at Day 30 (Per protocol set)" has been added

204812 (RSV F-021) Statistical Analysis Plan Amendment 4 Final

| | Statistical Analysis Plan Amendment 4 Final | |
|---|---|---|
| 15-Mar-2018 | Amendment 3: Description of changes from | Amendment 1 - 21- |
| | Amendment 2 are as below: | Aug-2017 |
| | For final analysis, | |
| | Some tables have been updated including | |
| | removing to Annex, creating new | |
| | corresponding in-text table by deleting or | |
| | collapsing some columns/rows; | |
| | Two figures of 'percentage of subjects | |
| | reporting solicited local/general symptoms | |
| | (any grade / grade 3) during the 7-day post- | |
| | vaccination period' have been newly | |
| | generated for the final analysis, respectively; | |
| | The table of 'Distribution of change from | |
| | baseline in haematology and biochemistry | |
| | with respect to normal laboratory ranges' | |
| | has been splitted and modified into three in- | |
| | text tables for Alanine Aminotransferase | |
| | (ALT)/ Aspartate Aminotransferase | |
| | (AST)/Eosinophils, Creatinine/Lymphocytes/ | |
| | White Blood Cells (WBC), | |
| | Haemoglobin/platelet count/Neutrophils, | |
| | separately; | |
| | Two new in-text tables of 'Summary of | |
| | haematology and biochemistry results by | |
| | maximum grade in the specified category' | |
| | and 'Summary of haematology change from | |
| | baseline by maximum grade in the specified | |
| | category' have been generated; | |
| | Some figures of Individual results for each | |
| | parameter have been modified. | |

204812 (RSV F-021) Statistical Analysis Plan Amendment 4 Final

| 01-Jun-2018 | Amendment 4: Description of changes from | Amendment 1 - 21- |
|---|---|---|
| | Amendment 3 are as below: | Aug-2017 |
| | For final analysis | |
| | Many tables and figures have been moved | |
| | between in-text and post-text; | |
| | Two figures of 'percentage of subjects | |
| | reporting solicited local/general symptoms | |
| | (any grade / grade 3) during the 7-day post- | |
| | vaccination period' will be updated to | |
| | include grade 2, respectively; | |
| | The parameter of BMI has been added in the | |
| | table of 'Summary of vital signs | |
| | characteristics (Exposed set)' and report at | |
| | VISIT 1 (D0), MA-RTI VISIT 1 and MA-RTI | |
| | VISIT 2; | |
| | <ul> <li>This table of 'Summary of haematology and</li> </ul> | |
| | biochemistry results by maximum grade in | |
| | the specified category from <u>VISIT 1 (D0) up</u> | |
| | to VISIT 2 (D7) (Exposed set)' will be newly | |
| | added for the final analysis in in-text; | |
| | Please check the dry run meeting minutes | |
| | for the details | |

#### 2. STUDY DESIGN

#### Study design overview Figure 1.



- V = Visit; D = Day; VACC = vaccination; BS = blood sample; h/b = blood sample for haematology/biochemistry; lmm = blood sample for immunogenicity; C = contact; RSV = Respiratory Syncytial Virus; PCR = Polymerase Chain Reaction.
- 1 Safety data up to (minimum) 7 days post-vaccination (including Day 7 haematology and biochemistry parameters) of the first 25% of subjects vaccinated in the study will be reviewed by iSRC.
- 2 In case of a MA-RTI (e.g. visit to the GP for respiratory symptoms including but not limited to cough, sputum production, difficulty breathing), the subject will be asked to contact the Investigator to enable completion of an event related eCRF and the collection of a nasal swab within 72h after the medical attendance.

Vertical lines stand for analysis on all subjects.

- **Experimental design**: Phase II, observer-blind, randomised, controlled, multicountry, study with four parallel groups.
  - **Duration of the study**: the intended duration of the study will be approximately 1 year from Visit 1 to study conclusion (Day 360).
  - Epoch 001: Primary starting at Visit 1 (Day 0) and ending at Visit 5 (Day 90).
  - Epoch 002: Follow-up phase starting one day after Day 90 and ending at Day 360 contact.
- **Primary Completion Date (PCD)**: Visit 3 (Day 30).
- End of Study (EoS): Last testing results released of samples collected at Visit 5 (i.e. last testing results released for the assays related to the primary and secondary endpoints).
- **Study groups:**

Table 1 Study groups and epochs foreseen in the study

| Study groups | Number of aubicate | and of subjects Are (Min/May) | | ochs |
|---|---|---|---|---|
| Study groups | Number of subjects | Age (Min/Max) | Epoch 001 | Epoch 002 |
| 30 PreF | ~100 | 18 - 45 years | Х | Х |
| 60 PreF | ~100 | 18 - 45 years | Х | Х |
| 120 PreF | ~100 | 18 - 45 years | Х | Х |
| Control | ~100 | 18 - 45 years | Х | Х |

Table 2 Study groups and treatment foreseen in the study

| Tractment name | Vaccina/ Draduct name | Study Groups | | | |
|---|---|---|---|---|---|
| Treatment name | Vaccine/ Product name | 30 PreF | 60 PreF | 120 PreF | Control |
| 20 ug ProE | PreF-30 | Х | | | |
| 30 µg PreF | NaCl | ۸ | ^ | | |
| 60 ug DroE | PreF-60 | | Х | | |
| 60 µg PreF | NaCl | | ^ | | |
| 120 ug DroE | PreF-120 | | | Х | |
| 120 µg PreF | NaCl | | | ^ | |
| Placebo | Formulation buffer S9b | | | | Х |

- **Control**: Placebo control
- **Vaccination schedule**: One intramuscular vaccination at Day 0.
- Treatment allocation: Subjects will be randomised using a centralised randomisation system on internet (SBIR) at Day 0. The randomisation algorithm will use a minimisation procedure accounting for age (18 32 years or 33 45 years) and centre.

The following group and sub-group names will be used for the statistical analyses:

| Group order in tables | Group label in tables | Group definition for footnote |
|---|---|---|
| 1 | 30 PreF | 30 µg PreF |
| 2 | 60 PreF | 60 µg PreF |
| 3 | 120 PreF | 120 µg PreF |
| 4 | Control | Placebo |

Some tables might be presented by age category according to the following description:

| Sub-group | Sub-group order in tables | Sub-group label in tables | Sub-group definition for footnote |
|---|---|---|---|
| Age | 1 18-32 | | 18-32 years old subjects |
| | 2 | 33-45Y | 33-45 years old subjects |

• **Blinding**: Observer-blind in Epoch 001 and single-blind in Epoch 002.

Table 3 Blinding of study epochs

| Study Epochs | Blinding |
|--------------|----------------|
| Epoch 001 | observer-blind |
| Epoch 002 | single-blind |

204812 (RSV F-021) Statistical Analysis Plan Amendment 4 Final

#### • Sampling schedule:

- O Blood samples for haematology/biochemistry will be collected (~10 mL) from all subjects at Visit 1 (Day 0), Visit 2 (Day 7), Visit 3 (Day 30), Visit 4 (Day 60) and Visit 5 (Day 90).
- O Blood samples for humoral immune response evaluation will be collected (~17 mL) from all subjects at Visit 1 (Day 0), Visit 3 (Day 30), Visit 4 (Day 60) and at Visit 5 (Day 90).
- Nasal swabs will be collected from subjects in case of a medically attended respiratory tract infection from enrolment (Visit 1) until study end (Contact 3).
- Type of study: self-contained
- **Data collection:** Electronic Case Report Form (eCRF).

#### • Safety monitoring:

- When the first 25% of subjects (i.e. ~100 subjects; ~25 subjects per study group) have been vaccinated, enrolment will be paused until completion of an unblinded review by a GSK internal Safety Review Committee (iSRC). Continuation of study enrolment will be conditional to a favourable outcome of the iSRC evaluation of all available safety and reactogenicity data collected up to at least 7 days post-vaccination (including Day 7 haematology and biochemistry parameters). In addition, the blinded safety data will be reviewed by GSK Biologicals' Safety Review Team (SRT) on a regular basis throughout the study. Analyses related to iSRC evaluation will be described in a separate document (SAP/TFL for iSRC).
- When all subjects have been vaccinated, IDMC will review all available safety and reactogenicity data (including haematology/biochemistry parameters) of all enrolled subjects up to at least 30 days post administration of the study vaccine or placebo. The blinded safety data will be reviewed by the GSK Biologicals' SRT. Analyses related to IDMC evaluation will be described in a separate document (SAP/TFL for IDMC).
- In case of a MA-RTI (e.g. visit to the GP for respiratory symptoms including but not limited to cough, sputum production, difficulty breathing), the subject will be asked to contact the investigator to enable the collection of a nasal swab within 72 hours after the medical attendance.

#### 3. OBJECTIVES

### 3.1. Primary Objective

• To rank different formulations of the investigational RSV vaccine based on safety/reactogenicity and immunogenicity data up to 1 month post-vaccination (Day 30).

### 3.2. Secondary objectives

- To evaluate the reactogenicity and safety of a single intramuscular dose of the RSV investigational vaccines up to study conclusion.
- To evaluate the immunogenicity of a single intramuscular dose of the RSV investigational vaccines up to 90 days after vaccination (Day 90).
- To further assess the safety of the investigational RSV vaccines by evaluating whether a single dose of the vaccines induces antibodies against the residual host cell protein neogenin (NEO) up to 1 month post-vaccination (Day 30).
- To estimate the incidence of medically attended RSV-associated RTIs up to study conclusion.

### 3.3. Tertiary objective

• If deemed necessary, to further characterize the immune response of a single intramuscular dose of the RSV investigational vaccines.

Refer to Section 5.7.3 Laboratory assays of the Protocol for additional testing proposed to further characterize the immune response to the investigational RSV vaccine.

#### 4. ENDPOINTS

# 4.1. Primary

- Occurrence of AEs from vaccination up to Day 7, for all subjects in each investigational RSV vaccine group:
  - Occurrence of any Grade 2 and Grade 3 general AE (solicited and unsolicited);
  - o Occurrence of Grade 2 and Grade 3 fever;
  - Occurrence of any vaccine-related SAE.
- Functional antibody titres against RSV at Day 0 and Day 30, for all subjects in each investigational RSV vaccine group.
  - Neutralising antibody titres against RSV-A
- PCA concentrations at Day 0 and Day 30 for all subjects in each investigational RSV vaccine group

#### 4.2. Secondary

- Occurrence of AEs from vaccination up to study conclusion:
  - Occurrence of each solicited local and general AE, during a 7-day follow-up period after vaccination (i.e. the day of vaccination and 6 subsequent days), for all subjects in all groups;
  - Occurrence of any unsolicited AE, during a 30-day follow-up period after vaccination (i.e. the day of vaccination and 29 subsequent days), for all subjects in all groups;
  - Occurrence of any haematological (haemoglobin level, White Blood Cells [WBC], lymphocyte, neutrophil, eosinophil and platelet count) and biochemical (alanine amino-transferase [ALT], aspartate amino-transferase [AST] and creatinine) laboratory abnormality at Day 0, Day 7, Day 30, Day 60 and Day 90 for all subjects in all groups;
  - Occurrence of any SAE, for all subjects in all groups.
- Functional antibody titres against RSV for all subjects in all groups:
  - Neutralising antibody titres against RSV-A at Day 0, Day 30, Day 60 and Day 90;
  - Neutralising antibody titres against RSV-B at Day 0, Day 30, Day 60 and Day 90
- PCA concentration at Day 0, Day 30, Day 60 and Day 90 for all subjects in all groups.
- Humoral immune response to the residual host cell protein NEO in the investigational RSV vaccine at pre-vaccination (Day 0), and 1 month post-vaccination (Day 30) for all subjects in all groups.
  - Antibody concentrations against NEO
- Occurrence of medically attended RSV-associated RTIs up to study conclusion

### 4.3. Tertiary

See section 5.7.3 of the Protocol for additional testing proposed to further characterize the immune response to the investigational RSV vaccine.

#### 5. ANALYSIS SETS

#### 5.1. Definition

In order to align to ICH and CDISC terminology, the Total Vaccinated Cohort (TVC) and the According To Protocol cohort (ATP) have been renamed Exposed Set (ES) and Per-Protocol Set (PPS) respectively. Two cohorts will be defined for the purpose of the analysis: the Exposed Set (ES) and the Per-Protocol Set (PPS) for analysis of immunogenicity. All analyses will be performed per treatment actually administered.

#### 5.1.1. Exposed Set (ES)

The ES will include all subjects with study vaccine administration documented:

- A **safety** analysis based on the ES will include all vaccinated subjects
- An **immunogenicity** analysis based on the ES will include all vaccinated subjects for whom immunogenicity data are available.

#### 5.1.2. Per-Protocol Set (PPS) for analysis of immunogenicity

The PPS for immunogenicity will be defined by time point and will include all vaccinated subjects.

- Meeting all eligibility criteria (i.e. no protocol violation linked to the inclusion/exclusion criteria, including age).
- Who received the study vaccine according to protocol procedures.
- Who did not receive a concomitant vaccination/medication/product leading to exclusion from the PPS analysis up to the corresponding timepoint as described in Section 6.6.2 of the Protocol.
- Who did not present with an intercurrent medical condition leading to exclusion from the PPS analysis up to the corresponding timepoint, as described in Section 6.7 of the Protocol.
- Who complied with the post-vaccination blood sampling schedule at the corresponding timepoint, as specified in Table 5 of the Protocol.
- For whom post-vaccination immunogenicity results are available for at least 1 assay at the corresponding timepoint.

When presenting different timepoints, the PPS for immunogenicity will be adapted for each timepoint (up to D30 and up to D90).

# 5.2. Criteria for eliminating data from Analysis Sets

Elimination codes are used to identify subjects to be eliminated from analysis. Detail is provided below for each sets.

#### 5.2.1. Elimination from Exposed Set (ES)

Code 1030 (Study vaccine not administered at all) and code 900 (invalid informed consent or fraud data) will be used for identifying subjects eliminated from ES.

#### 5.2.2. **Elimination from Per-protocol analysis Set (PPS)**

#### 5.2.2.1. **Excluded subjects**

A subject will be excluded from the PPS analysis under the following conditions.

| | | Applicable Eli Type | |
|---|---|---|---|
| Code | Condition under which the code is used | 'M1' (Applicable<br>up to Visit 3 - Day<br>30) | 'M2' (Applicable<br>up to Visit 5 - Day<br>90) |
| 900 | Invalid informed consent or fraud data (Subjects receiving a code 900 should not receive any other elimination codes) | Applicable | Applicable |
| 1030 | Study vaccine not<br>administered at all<br>(Subjects receiving a code<br>1030 should not receive any<br>other elimination codes) | Applicable | Applicable |
| 1040* | Administration of concomitant vaccine(s) forbidden in the protocol | Applicable<br>(To check up to<br>Visit 3 – Day 30) | Applicable<br>(To check up to<br>Visit 5 – Day 90) |
| 1050 | Randomization failure (subject not randomized in the correct group) | Applicable | Applicable |
| 1060 | Randomization code was broken | Applicable | Applicable |
| 1070** | Subjects got vaccinated with the correct vaccine but containing a lower volume | Applicable | Applicable |
| 1070** | Administration not according to protocol for reason specified by the investigator other than site and route | Applicable | Applicable |
| 1070** | Site or route of study vaccine administration wrong or unknown | Applicable | Applicable |
| 1070** | Wrong replacement or study vaccine administered (not compatible with the vaccine regimen associated to the treatment number) | Applicable | Applicable |

204812 (RSV F-021) Statistical Analysis Plan Amendment 4 Final

| | | Statistical An | alysis Plan Amendm |
|---|---|---|---|
| | | Applicable Eli Type | |
| Code | Condition under which the code is used | 'M1' (Applicable<br>up to Visit 3 - Day<br>30) | 'M2' (Applicable<br>up to Visit 5 - Day<br>90) |
| 1070** | Administered study vaccine reported as being the correct one but is not compatible with the vaccine regimen associated to the treatment number | Applicable | Applicable |
| 1080 | Vaccine temperature deviation | Applicable | Applicable |
| 1090 | Expired vaccine administered | Applicable | Applicable |
| 2010 | Protocol violation<br>(inclusion/exclusion<br>criteria) | Applicable DOB-VAC=18-45 years | Applicable DOB-VAC=18-45 years |
| 2040* | Administration of any medication forbidden by the protocol | Applicable<br>(To check up to<br>Visit 3 – Day 30) | Applicable<br>(To check up to<br>Visit 5 – Day 90) |
| 2050* | Underlying medical condition forbidden by the protocol | Applicable<br>(To check up to<br>Visit 3 – Day 30) | Applicable<br>(To check up to<br>Visit 5 – Day 90) |
| 2060* | Concomitant infection related to the vaccine which may influence the immune response | Applicable<br>(To check up to<br>Visit 3 – Day 30) | Applicable<br>(To check up to<br>Visit 5 – Day 90) |
| 2070* | Concomitant infection not related to the vaccine which may influence the immune response | Applicable<br>(To check up to<br>Visit 3 – Day 30) | Applicable<br>(To check up to<br>Visit 5 – Day 90) |
| 2090 | Subjects did not comply<br>with blood sample<br>schedule | Applicable VAC_1 to SER_2 = 30-44 (days) | Applicable VAC_1 to SER_3 = 56-70 (days) VAC_1 to SER_4 = 86-100 (days) |
| 2100 | Serological results not available post-vaccination | All assay for Day 30 elimination code | All assay for Day60 and Day90 elimination code |
| | | if ALL are<br>missing | if ALL are<br>missing |

| | | Applicable Eli Type | |
|---|---|---|---|
| Code | Condition under which the code is used | 'M1' (Applicable<br>up to Visit 3 - Day<br>30) | 'M2' (Applicable<br>up to Visit 5 - Day<br>90) |
| | | v_ID for Neutra<br>RSV-A=3240.001 | v_ID for Neutra<br>RSV-A=3240.001 |
| | | v_ID for Neutra<br>RSV-B=3240.002 | v_ID for Neutra<br>RSV-B=3240.002 |
| | | v_ID for Neutra<br>PCA=3241.009 | v_ID for Neutra<br>PCA=3241.009 |
| | | v_ID for IgG<br>total=3241.002 | v_ID for IgG<br>total=3241.002 |
| | | v_ID for IgG<br>1=3241.005 | v_ID for IgG<br>1=3241.005 |
| 2120* | Obvious incoherence or abnormality or error in data*** | All assay for Day<br>30 | All assay for Day<br>60 and Day90 |

<sup>\*</sup> Attribution of these elimcodes to subject need CRDL review of individual data listings

Eli type is Internal GSK database code for type of elimination code M1 for Visit 3 (Day30) analysis; M2 for Visit 5 (Day 90) analysis;

#### 5.2.2.2. Right censored Data

Not applicable

#### 5.2.2.3. Visit-specific censored Data

Not applicable

# 5.3. Important protocol deviation not leading to elimination from per-protocol analysis set

The following important protocol deviations will be reported by groups:

Forced randomization: In case of supplies shortage for the next assigned vaccine according to the randomization schedule at the clinical site, the randomization system will use the forced randomization procedure in order to continue to enrol and vaccinate subjects. The system moves seamlessly to the next treatment/randomization number for which vaccine supplies are available. The site will not be aware of the forced randomization event.

<sup>\*\*</sup> Attribution of code 1070 to a subject requires CRDL confirmation

<sup>\*\*\*</sup> Elimination criteria for implausible RSV serum immune responses (neut and/or ELISA): More than 4 fold decrease from pre-vaccination to Day 30; After Day 30, more than 4 fold increase or more than 8 fold decrease within a 30 day period

204812 (RSV F-021)

Statistical Analysis Plan Amendment 4 Final

Manual randomization: In case of the randomization system is unavailable, the investigator has the option to perform randomization by selecting supplies available at the site according to a pre-defined rule.

Short follow-up: subjects who completed the last study contact before the minimum length of follow-up requirement.

#### 6. STATISTICAL ANALYSES

Note that standard data derivation rule and stat methods are described in Annex 1 standard data derivation rule and statistical methods and will not be repeated below.

## 6.1. Demography

# 6.1.1. Analysis of demographics/baseline characteristics planned in the protocol

The analysis of demography will be performed on the ES and on the PPS for immunogenicity.

Demographic characteristics such as age at vaccination in years, race, ethnicity, vital signs and cohort description will be summarised by group using descriptive statistics:

- Frequency tables will be generated for categorical variable such as race.
- Mean, median, standard error and range will be provided for continuous data such as age.

The distribution of subjects will be tabulated as a whole and per group and for each age category (18 - 32 years and 33 - 45 years).

Withdrawal status will be summarised by group using descriptive statistics:

- The number of subjects enrolled into the study as well as the number of subjects excluded from PPS analyses will be tabulated.
- The number of withdrawn subjects will be tabulated according to the reason for withdrawal.

# 6.2. Immunogenicity

#### 6.2.1. Analysis of immunogenicity planned in the protocol

The analysis will be performed on the applicable PPS cohort for immunogenicity and, if in any group the percentage of vaccinated subjects with serological results excluded from the PPS for analysis of immunogenicity is  $\geq 5\%$ , a second analysis will be performed on the ES.

#### 6.2.1.1. Within group analysis

Humoral Immune response to RSV vaccine

For each group, at each timepoint that blood samples are collected and for each assay (unless specified otherwise):

- GMTs/GMCs will be tabulated with 95% CI based on log-transformed values and represented graphically.
- Percentage of subjects above the seropositivity threshold will be tabulated with exact 95% CI.
  - Percentage of subjects above the seropositivity threshold and GMTs/GMCs will also be tabulated by group for each age category (18 32 years and 33 45 years).
- Pre- and post-vaccination antibody titres/concentrations will be displayed using reverse cumulative curves.
- The distributions of **neutralising** antibody titres will be tabulated in the tables with log2 scale (< 7, 7-8, > 8-9, > 9-10, > 10-11, > 11-12, > 12 log2).
- Percentage of responders in terms of **neutralising** antibody titres will be tabulated with exact 95% CI.
- Individual post-vaccination *versus* pre-vaccination results will be plotted using scatter plots. Results of the control group will be used as a reference.
- Geometric mean of ratios of antibody titres/concentrations at each post-vaccination timepoint over pre-vaccination will be tabulated with 95% CI.
- Distribution of the fold increase of the antibody titres/concentrations will be tabulated:
  - For neutralising antibody titres against RSV-A and RSV-B: percentage of subjects with a fold increase equal to or above 1, 2, 2.5, 3, 4, 6, 8 10, 11 and 12 by pre-vaccination titre category: <7, 7-8, ]8-9, ]9-10, ]10-11, ]11-12, >12 log2, and cumulative: <7,  $\ge 7$ ,  $\ge 8$ ,  $\ge 9$ ,  $\ge 10$ ,  $\ge 11$ ,  $\ge 12 log2$ .
  - For antibody concentrations against NEO: percentage of subjects with a fold increase equal to or above 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5 and 5.

The kinetics of individual antibody titres/concentrations will be plotted as a function of time for subjects with results available at all timepoints.

 An analysis of variance model for repeated measures will be fitted to calculate GMTs/GMCs with treatment group, visit and their interaction as fixed effects if necessary.

If deemed necessary, the same analyses may be done by age category (18 - 32 years and 33 - 45 years).

#### 6.2.1.2. Between group assessment

Exploratory comparisons will be performed for RSV neutralising antibody titres and PCA concentrations post-vaccination (Day 30, Day 60 and Day 90) between the different RSV vaccine groups.

- Estimation of GMT/GMC ratios between groups with corresponding 95% CI using an ANCOVA model on the logarithm10 transformation of the titres/concentrations. If a statistically significant difference is found (p <0.05), pairwise comparisons will be made using Tukey's multiple comparison adjustment. This model includes:
  - o The vaccine group as the fixed effect
  - o The pre-vaccination titre/concentration as the covariate
  - Age groups (18-32 years and 33-45 years) and center as the categorical covariate if deemed necessary
- GMT/GMC ratios with corresponding 95% CI will be computed between the RSV vaccine groups
  - o PreF-120 minus PreF-30
  - o PreF-120 minus PreF-60
  - o PreF-60 minus PreF-30

#### 6.2.2. Additional considerations

In order to add the analysis of the <u>anti-RSV F IgG Total and IgG1 subclass</u> tested at Day 0 and Day 30 in a random subset of 50 subjects per group. The following analysis will be performed on the Per-Protocol Set (PPS) for analysis of immunogenicity for each group and for both assays:

- GMCs with 95% CI will be tabulated.
- Percentage of subjects above the seropositivity threshold will be tabulated with exact 95% CI.
- Geometric mean of ratios of antibody concentrations at each post-vaccination timepoint over pre-vaccination (fold increase) will be tabulated with 95% CI, and represented graphically.
- Individual ratios of antibody concentrations will be displayed using reverse cumulative curves.
- Exploratory comparisons between groups: geometric mean ratios and 95% CIs of fold increase post/pre between the RSV groups:
  - o 120 PreF versus 60 PreF
  - 120 PreF versus 30 PreF
  - o 60 PreF versus 30 PreF

204812 (RSV F-021)

Statistical Analysis Plan Amendment 4 Final

This will be performed using an ANOVA model on the logarithm10 transformation of the concentrations including the vaccine group as covariates. If a statistically significant difference is found (p < 0.05), pairwise comparisons will be made using Tukey's multiple comparison adjustment.

In addition, the following immunogenicity analysis will be performed in the subset of subjects with IgG/IgG1data available:

- GMCs will be tabulated with 95% CI for anti-RSV A and anti-PCA
- Percentage of subjects above the seropositivity threshold will be tabulated with exact 95% CI for anti-RSV A and anti-PCA.

# 6.3. Analysis of safety

#### 6.3.1. Analysis of safety planned in the protocol

The analysis of safety will be performed on the ES.

#### 6.3.1.1. Within group analysis

The percentage of subjects with at least one **local AE** (solicited and unsolicited), with at least one **general AE** (solicited and unsolicited) and with any AE during the 7-day or 30-day follow-up period after vaccination will be tabulated with exact 95% CI. The same computations will be done for ≥ Grade 2 and Grade 3 AEs, for any AEs considered related to vaccination, for any Grade 3 AEs considered related to vaccination and for AEs resulting in medically attended visit.

The percentage of subjects reporting each individual **solicited local AE** (any grade,  $\geq$  Grade 2, Grade 3, resulting in medically attended visit) during the 7-day follow-up period after vaccination will be tabulated for each study vaccine for each group. The percentage of subjects reporting each individual **solicited general AE** (any grade,  $\geq$  Grade 2, Grade 3, any related,  $\geq$  Grade 2 related, Grade 3 related, resulting in medically attended visit) during the 7-day follow-up period after vaccination will be tabulated for each group.

For fever during the 7-day follow-up period after vaccination, the number and percentage of subjects reporting fever will be reported by half degree (°C) cumulative increments. Similar tabulations will be performed for causally related fever, Grade 3 (> 39.5°C) causally related fever and fever resulting in a medically attended visit. In addition, the prevalence of any and Grade 3 fever will be presented graphically over time after vaccination

The percentage of subjects with any **unsolicited** symptoms within 30 days after vaccination with its exact 95% CI will be tabulated by group and by Medical Dictionary for Regulatory Activities (MedDRA) preferred term. Similar tabulation will be done for Grade 3 unsolicited symptoms, for any causally related unsolicited symptoms, for Grade 3 causally related unsolicited symptoms and for unsolicited symptoms resulting in a medically attended visit (The verbatim reports of unsolicited symptoms will be reviewed by a physician and the signs and symptoms will be coded according to the MedDRA

204812 (RSV F-021)

Statistical Analysis Plan Amendment 4 Final

Dictionary for Adverse Reaction Terminology. Every verbatim term will be matched with the appropriate Preferred Term).

**SAEs** reported throughout the study will be described in detail.

**Pregnancy** exposures throughout the study and pregnancy outcomes will be described in detail (if applicable).

The percentage of subjects using **concomitant medication** (any medication, any antipyretic and any antipyretic taken prophylactically) during the 7-day (Day 0 to Day 6) or 30-day (Day 0 to Day 29) follow-up period after vaccination will be summarised by group.

For all subjects in each group and each **haematology and biochemistry** parameter:

- The percentage of subjects having haematology and biochemistry results below or above the local laboratory normal ranges will be tabulated for each timepoint.
- The maximum grading post-vaccination (from Day 7 to Day 90) versus baseline (Day 0) and the percentage of subjects with laboratory parameters above or equal to Grade 1, Grade 2, Grade 3 and Grade 4 will be tabulated (Grades will be based on the FDA Guidance for Industry "Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials", see APPENDIX D of the Protocol: FDA toxicity grading scale. Those laboratory parameters not included on FDA Toxicity Grading Scale will not be graded).

Assessment of anti-NEO immune response at Day 30 post-vaccination for each group:

- GMCs pre-and post-vaccination will be tabulated with 95% CI and represented graphically.
- Individual post-vaccination *versus* pre-vaccination results will be plotted using scatter plots. Results of the control group will be used as a reference.
- Geometric mean of ratios of antibody concentrations at Day 30 over pre-vaccination will be tabulated with 95% CI.
- Distribution of the antibody concentrations pre-and post-vaccination and of fold increase after vaccination will be tabulated.

#### 6.3.1.2. Between group assessment

Exploratory comparisons between each investigational RSV vaccine group and (minus) the control group (*placebo*), and between the RSV vaccine groups will be done in terms of the percentage of subjects reporting any ≥ Grade 2, Grade 3 AE (solicited and unsolicited), and/or any fever > 38.5°C, and/or any vaccine-related SAE during the 7-day follow-up period after vaccination.

- o PreF-30 minus placebo
- o PreF-60 *minus* placebo
- o PreF-120 *minus* placebo

- Statistical Analysis Plan Amendment 4 Final
- o PreF-120 minus PreF-30
- o PreF-120 minus PreF-60
- o PreF-60 minus PreF-30

The standardised asymptotic 95% CI for the difference between the investigational RSV vaccine groups as well as between the investigational RSV groups and (minus) the control group will be computed.

#### 6.4. Analysis for ranking RSV formulations

The totality of data and sum total of evidence for particular dose(s) in terms of safety and immunogenicity will be evaluated by study team in addition to the analyses described in section 6.1 and 6.3 on formulation selection. The desirability index approach described in the section below will be used as a descriptive tool to guide the formulation selection. In addition, any pertinent information from outside this study will be evaluated and may be used by the study team to help to make the final decision on a dose/formulation.

#### 6.4.1. Definition of desirability in the context of Simulations

A desirability approach will be based on safety/reactogenicity and immunogenicity data up to 1 month post-vaccination.

This method is a multi-criteria decision making approach based on desirability functions. The main idea is to identify for each endpoint a desirability function that associates any value to another one between 0 and 1 depending on its desirability ('0' being considered as not desirable at all and '1' as the most desirable). An index with values between 0 and 1 will be created for each endpoint. An overall desirability index can be calculated by computing a weighted geometric mean of the endpoint indexes. By definition, this overall index also takes values between 0 and 1 and characterises the level of desirability of any candidate formulation by a single value [Dewé, 2015].

The desirability index calculations will include reactogenicity and safety data up to Day 7 post vaccination (on the TVC) and immunogenicity data at 30 days post-vaccination (on the ATP cohort for immunogenicity up to Day 30). The formulations will be ranked based on the values obtained with this overall desirability index.

# 6.4.2. Derived endpoints

The following endpoints will be computed and taken into account in the desirability analysis:

- 1. Incidence rate of any Grade 2 and any Grade 3 general AE (solicited and unsolicited) and any vaccine-related SAE during the 7-day follow-up period after vaccination for each investigational RSV vaccine formulation.
- 2. Incidence rate of Grade 2 and Grade 3 fever during the 7-day follow-up period after vaccination for each investigational RSV vaccine formulation.

- 3. Geometric mean of neutralising antibody titres against RSV-A at Day 30 adjusted for pre-vaccination titres.
- 4. Geometric mean of PCA concentrations at Day 30 adjusted for pre-vaccination titres.

Each individual desirability index will be calculated based on data and tabulated by the treatment group and endpoints above. The details on how to calculate individual desirability index in terms of reactogenicity and immunogenicity and overall desirability index are elaborated in Annex 2.

### 6.5. Analysis of medically attended RTIs

The analysis will be performed on the ES by study group.

The proportion of subjects (with 95% CI) with at least one medically attended RTI (all causes) will be calculated by group.

Viral load assessed by the quantitative PCR (RSV-A/B) of RSV-RTI cases will be listed for any cases where this assay is performed.

Medically attended RSV-associated RTI co-infected or colonisation with another viral etiology identified by multiplex PCR will be described.

Medically attended RTI with any viral etiology identified by multiplex PCR will be described

#### 7. ANALYSIS INTERPRETATION

All comparative analyses will be descriptive with the aim to characterise the difference in reactogenicity/immunogenicity between groups. These descriptive analyses should be interpreted with caution considering that there is no adjustment for multiplicity for these comparisons.

#### 8. CONDUCT OF ANALYSES

Any deviation(s) or change(s) from the original statistical plan outlined in this protocol will be described and justified in the final study report.

#### 8.1. Sequence of analyses

The statistical analyses will be performed in several steps:

- In preparation of the planned iSRC evaluation, analysis of safety and reactogenicity data up to at least 7 days post-vaccination of the first 25% of all subjects will be performed (see Section 8.10.2 of the Protocol for more information).
- In preparation of the planned IDMC evaluation, analysis of safety and reactogenicity data (including haematology/ biochemistry parameters) up to at least 30 days post-vaccination of all enrolled subjects will be performed.

204812 (RSV F-021)

Statistical Analysis Plan Amendment 4 Final

- The first main analysis on all subjects will be performed when all data up to 30 days post-vaccination are available (primary endpoints). In order to maintain the blind, this analysis by group will be performed by an independent statistician and the results which would lead to the unblinding of some subjects (e.g. a specific AE reported by one subject only) will be blinded (i.e. the group in which this event occurred will not be identified). No individual data listings will be provided.
- A second analysis will be performed when all data up to 90 days post-vaccination are available (secondary endpoints). At this point, the GSK statistician will be unblinded (i.e. will have access to the individual subject treatment assignments), but no individual listings will be provided. Given that summary results may unblind some specific subjects, the study will be conducted in a single-blind manner from this point onwards, with subjects remaining blinded up to study conclusion and the investigators will not have access to the treatment allocation up to study conclusion.
- The final analysis will be performed when all data up to study conclusion are available. All available tertiary endpoints will also be analysed in this step. Individual listings will only be provided at this stage.
- An integrated study report presenting all analyses will be written and made available to the investigators at the time of final analysis.
- If data for tertiary endpoints become available at a later stage, (an) additional analysis/analyses will be performed. These data will be documented in Annex(es) to the study report and will be made available to the investigators at that time.

| Description | Analysis ID | Disclosure Purpose<br>(CTRS=web posting,<br>SR=study report,<br>internal) | Dry run review<br>needed (Y/N) | Study Headline Summary (SHS)requiring expedited communication to upper management (Yes/No) | Reference<br>for TFL |
|---|---|---|---|---|---|
| Final<br>Analysis | E1_01 | Study report<br>CTRS | N | Yes | All tables<br>from TFL<br>dated<br>01JUN2018 |
| Analysis of<br>Day 30 | E1_04 | Internal<br>CTRS | N | Yes | All tables<br>from TFL<br>dated<br>13NOV2017 |
| Analysis of<br>Day 90 | E1_05 | Internal<br>CTRS | N | Yes | All tables<br>from TFL<br>dated<br>13NOV2017 |

# 8.2. Statistical considerations for interim analyses

No interim analysis will be performed.

#### 9. CHANGES FROM PLANNED ANALYSES

In order to align to ICH and CDISC terminology the Total Vaccinated Cohort and the According To Protocol cohort have been renamed Exposed Set (ES) and Per-Protocol Set (PPS) respectively.

#### Changes in Amendment 1 mainly include the following.

For the sequence of analysis, the IDMC evaluation was newly added to review all available safety and reactogenicity data (including Day 30 haematology and biochemistry parameters) of all enrolled subjects up to at least 30 days post administration of the study vaccine or placebo.

Since the document of criteria for eliminating subjects from analysis will not be used anymore, the table of Elimination codes has been modified for more clarity. Attribution of code 1070 to a subject requires CRDL confirmation. Attribution of these elimcodes including 1040, 2040, 2050, 2060, 2070 and 2120 to subject need CRDL review of individual data listings.

In the analysis of immunogenicity section, the distribution of fold increase of the antibody titres against RSV-A and RSV-B and concentrations against NEO have been added.

For the analysis of safety, the percentage of subjects reporting each individual solicited local AE (any, each grade, resulting in medically attended visit) during the 7-day follow-up period after vaccination will also be tabulated based on maximum intensity per subject for each study vaccine group; the percentage of subjects reporting each individual solicited general AE (any, each grade, any related, any Grade 2 related, any Grade 3 related, resulting in medically attended visit) during the 7-day follow-up period after vaccination will also be based on maximum intensity per subject for each study vaccine group.

Evaluation of last secondary objective 'To estimate the incidence of medically attended RSV-associated RTIs up to study conclusion' will be performed based on MA-RTIs rather than MA-RSV associated RTIs.

The cut-off for the updated (qualified) version of the PCA assay will be set at the level of the assay LLOQ (9.60 µg/mL). Hence the SAP does not need to define handling of data between the LOD and LLOQ anymore, as results will only be provided as of the LLOQ. It only needs to be defined that for results below the cut-off (LLOQ), an arbitrary value of half of the cut-off will be considered for calculation of GMC and fold increase.

Algorithm for handling of data of RSV-B neutralising antibody tires between the LOB and LLOQ is defined as similar as for RSV-A by considering the LOB for RSV-B is 6.

Additional analysis of the IgG total and IgG1 subclass and analysis of anti-RSV A and anti-PCA in the subset of subjects with IgG/IgG1 data have been added.

#### **Changes of TFL/TOC**

- In the analysis of safety section, figures of 'Individuals results of haematological (haemoglobin level, white blood cells and platelet count) and biochemical (ALT, AST and creatinine) parameters outside of the normal ranges in each group' has been added to replace the figures of 'Mean profile of haematological and biochemical parameters change from baseline (Day 0)';
- In the analysis of safety section, the titles in all tables reporting 'Incidence and nature of symptoms (solicited and unsolicited) during the 7-day and 30-day post-vaccination period' have been changed from 'with causal relationship to' to 'considered related to vaccination';
- In the analysis of safety section, analysis on 'Incidence of solicited local/general symptoms reported during the 7-day post-vaccination period' will be summarized based on maximum intensity for each grade per subject for each group; therefore, analysis on 'incidence of solicited local/general symptoms reported during the 7-day post-vaccination period, including >=grade 2 category' will not be generated.
- In the analysis of safety section, analysis on 'Number (%) of subjects reporting the occurrence of adverse events within the 7-day and 30-day post-vaccination period' will be added.
- In the analysis of safety section, analysis on 'Number (%) of subjects with serious adverse events during the study period including number of events reported' and 'Number (%) of subjects with serious adverse events considered related to vaccination during the study period including number of events reported' by %UNSOL (EVENT=1) will not be reported because %CTR\_SAE macro has been adapted to generate SAE, related SAE, fatal SAE and related fatal SAE.
- In the analysis of safety section, analysis on 'Number and percentage of subjects reporting the occurrence of medically attended respiration tract infections (MA-RTIs), during the 30-day, 60-day or 90-day post-vaccination period and up to study end' will be reported; Therefore, 'Number and percentage of subjects reporting one medically attended RSV-associated RTI and medically attended RTI (all causes) within the 30-day post-vaccination period or throughout the study period' will not be generated;
- In the analysis of medically attended RTIs, viral load assessed by the quantitative PCR (RSV-A/B) of RSV-RTI cases will be only listed in the individual listings; therefore, analysis on 'Descriptive statistics of the viral load assessed by the quantitative PCR (RSV-A/B) of RSV-RTI cases (All vaccinated subjects)' will not be reported;
- In the analysis of immunogenicity section, tables/figures related to the analysis of RSV-B will be added;
- In the analysis of immunogenicity section, tables/figures related to the analysis of the IgG total and IgG1 subclass will be added;
- In the analysis of immunogenicity section, tables related to the analysis of anti-RSV A and anti-PCA in the subset of subjects with IgG/IgG1 data available will be added.

204812 (RSV F-021)

Statistical Analysis Plan Amendment 4 Final

#### Changes in Amendment 2 mainly include the following.

- In the analysis of immunogenicity section, the analysis on GM ratios between anti-RSV F antibody concentrations (IgG Total) and anti-RSV-A neutralising antibody titers at pre-vaccination has been added for Day 90 and final analysis;
- In the analysis of immunogenicity section, the analysis on GM ratios of fold increase post/pre (Day 30/Day 0) between anti-RSV F antibody concentrations (IgG Total) and anti-RSV-A neutralising antibody titers has been added for Day 90 and final analysis.

#### Changes of TFL/TOC

- In the analysis of safety section, figures of "Individual results of hemoglobin levels beyond grade 2" will be reported for Day 90 and final analysis to replace the figures of "Individual results of hemoglobin levels outside of normal range";
- In the analysis of safety section, figures of "Individual results of white blood cells counts levels lower than LL" and figures of "Individual results of white blood cells counts levels higher than UL" will be reported for Day 90 and final analysis to replace the figures of "Individual results of white blood cells counts levels outside of normal range".
- In the analysis of immunogenicity section, one new template (Template 54) for "Comparisons of GM ratios with corresponding 95% confidence interval between anti-RSV F antibody concentrations (IgG Total) and anti-RSV-A neutralising antibody titers at pre-vaccination (Per protocol set)" has been added for Day 90 and final analysis;
- In the analysis of immunogenicity section, one new template (Template 55) for "Exploratory comparisons (GM ratios of fold increase post/pre) with corresponding 95% confidence interval between anti-RSV F antibody concentrations (IgG Total) and anti-RSV-A neutralising antibody titers at Day 30 (Per protocol set)" has been added for Day 90 and final analysis;

#### Changes in Amendment 3 mainly include the following.

#### Changes of TFL/TOC for final analysis

- All tables concerned with 'Incidence and nature of symptoms (solicited and unsolicited)' have been moved to Annex; such tables for Grade 3 are kept as intext tables;
- Tables of 'Incidence of solicited local/general symptoms reported during the 7-day (Days 0-6) post-vaccination period' have been moved to Annex; such tables by maximum intensity are kept as in-text tables and corresponding figures have been newly generated for the final analysis, that is, 'Percentage of subjects reporting solicited local/general symptoms (any grade / grade 3) during the 7-day post-vaccination period';
- All tables concerned with 'Percentage of subjects reporting the occurrence of unsolicited symptoms' have been moved to Annex; Such tables for Grade 3 and/or considered related to vaccination are kept as in-text tables with the simplification by removing the columns of LL and UL;

204812 (RSV F-021)

Statistical Analysis Plan Amendment 4 Final

- Tables of 'Percentage of subjects reporting the occurrence of SAE within the 30-day (Days 0-29) post-vaccination period/throughout the study period' are kept as in-text tables with the simplification by removing the columns of LL and UL;
- All tables concerned with 'Number (%) of subjects reporting the occurrence of adverse events' have been moved to Annex;
- All tables of 'Number and percentage of subjects reporting the occurrence of medically attended respiration tract infections (MA-RTIs)' have been moved to Annex; MA-RTIs reported up to DBF of final analysis is kept as one in-text table with the simplification by removing the columns of LL and UL;
- The table of 'Compliance in returning symptom information' and all tables concerned with 'Number and percentage of subjects taking a concomitant medication' have been moved to Annex;
- The table of 'Exploratory comparisons between groups in terms of percentage of subjects reported any Grade 2/3 AE and/or any fever >38.5°C and/or any vaccine-related SAE during the 7 day (Days 0-6) Post-vaccination period' will not be reported in the final analysis;
- The table of 'Distribution of change from baseline in haematology and biochemistry with respect to normal laboratory ranges' has been moved to Annex; Three splitted in-text tables for ALT/AST /Eosinophils, Creatinine/Lymphocytes/White Blood Cells and Haemoglobin/ platelet count/ Neutrophils have been generated, separately;
- The table of 'Summary of haematology and biochemistry results by maximum grade' has been moved to Annex; One newly formatted in-text table of 'Summary of haematology and biochemistry results by maximum grade in the specified category' has been generated by collapsing the categories of unknown/grade 0 and grade 1 then renaming the new category of 'other', keeping grade 2, 3 and 4 column, and removing the column of n;
- The table of 'Summary of haematology change from baseline by maximum grade' has been moved to Annex; One newly formatted in-text table of 'Summary of haematology change from baseline by maximum grade in the specified category' has been generated by collapsing the categories of unknown/grade 0 and grade 1 then renaming the new category of 'other', keeping grade 2, 3 and 4 column, and removing the column of n;

#### Changes in Amendment 4 mainly include the following.

Please check the dry run meeting minutes for details.

C.A.R.S./Clinical R&D/RSV F/Studies/021 (204812)/11 Statistics/11.05 General/11.05.03 Meeting Material/Analysis E01\_01/RSV F-021 (204812) Dry Run Minutes E01\_01.

# 10. LIST OF FINAL REPORT TABLES, LISTINGS AND FIGURES

The TFL TOC provides the list of tables/listings and figures needed for the study report. It also identifies the tables eligible for each analyses and their role (synopsis, in-text, post-text, SHS, CTRS,...).

# 11. ANNEX 1 STANDARD DATA DERIVATION RULE AND STATISTICAL METHODS

#### 11.1. Statistical Method References

The exact two-sided 95% CIs for a proportion within a group will be the Clopper-Pearson exact CI [Clopper CJ, Pearson ES. The use of confidence or fiducial limits illustrated in the case of binomial. *Biometrika*. 1934;26:404-413].

The standardised asymptotic two-sided 95% CI for the group difference in proportions is based on the method described in the following paper:Robert G. Newcombe, interval estimation for the difference between independent proportions: comparison of eleven methods, *Statist Med.* 1998; 17, 873-890]. The standardised asymptotic method used is the method six.

Dewé W, Durand Ch, Marion S *et al*. A multi-criteria decision making approach to identify a vaccine formulation. *Journal of Biopharmaceutical Statistics*, 2015; epublication ahead of print: DOI: 10.1080/10543406.2015.1008517.

#### 11.2. Standard data derivation

#### 11.2.1. Date derivation

- SAS date derived from a character date: In case day is missing, 15 is used. In case day and month are missing, 30 June is used.
- Onset day for an event (ae, medication, vaccination, ...): The onset day is the number of days between the last study vaccination & the start date of the event. This is 0 for an event starting on the same day as a vaccination. See SAS date derived in case the start date of the event is incomplete.
- Duration: Duration of an event is expressed in days. It is the number of days between the start & the stop dates + 1. Therefore duration is 1 day for an event starting & ending on the same day.
- Association of an event to the primary epoch: An adverse event belongs to the primary epoch, if the onset date is before and excluding Visit 5 or the last contact date, whichever is coming first.

#### 11.2.2. Dose number

- The study dose number is defined in reference to the number of study visits at which vaccination occurred.
- Relative dose: the relative dose for an event (AE, medication, vaccination) is the most recent study dose given before an event. In case the event takes place on the day a study dose is given, the related dose will be that of the study dose, even if the event actually took place before vaccination. For instance, if an adverse event begins on the day of the study vaccination but prior to administration of the vaccine, it will be assigned to this dose.

#### 11.2.3. Demography

- Age: Age at the reference activity, computed as the number of units between the date of birth and the reference activity. Note that due to incomplete date, the derived age may be incorrect by 1 month when month is missing from the birthdate. This may lead to apparent inconsistency between the derived age and the eligibility criteria/the age category used for randomization.
- Conversion of weight to kg

The following conversation rule is used:

- O Weight in Kilogram = weight in Pounds / 2.2
- Weight in Kilogram = weight in ounces / 35.2

The result is rounded to 2 decimals.

• Conversion of height to cm

The following conversation rule is used:

- Height in Centimetres = Height in Feet \* 30.48
- Height in Centimetres = Height in Inch \* 2.54

The result is rounded to the unit (ie no decimal).

• Conversion of temperature to °C

The following conversion rule is used:

o Temperature in °Celsius = ((Temperature in °Fahrenheit -32) \*5)/9

The result is rounded to 1 decimal.

#### 11.2.4. **Immunogenicity**

- For a given subject and given immunogenicity measurement, missing or nonevaluable measurements will not be replaced. Therefore, an analysis will exclude subjects with missing or non-evaluable measurements.
- A seronegative subject is a subject whose antibody titre/concentration is below the cut-off value of the assay. A seropositive subject is a subject whose antibody titre/concentration is greater than or equal to the cut-off value of the assay.
- The Geometric Mean Concentrations/Titres (GMC/Ts) calculations are performed by taking the anti-log of the mean of the log titre transformations. Antibody titres below the cut-off of the assay will be given an arbitrary value of half the cut-off of the assay for the purpose of GMT calculation. The cut-off value is defined by the laboratory before the analysis and is described in the protocol.
- In order to compute fold increase of antibody titres/concentrations (ratio) between post-vaccination and pre-vaccination titres/concentrations and for GMC/GMT calculation, antibody titres/concentrations below the assay cut-off will be given an arbitrary value of half the cut-off.
- The cut-off for the updated (qualified) version of the PCA assay will be set at the level of the assay LLOO (9.60 µg/mL). For results below the cut-off (LLOO), an arbitrary value of half of the cut-off will be considered for calculation of GMC and fold increase.
- Considering cut-offs or neutralising antibody against RSV-A and RSV-B are below the assays' LLOQ, the following rules will be applied:

| Assay | Raw result | Derivation for<br>seropositivity<br>status | Derivation for<br>GMT<br>calculation | Derivation for fold-<br>increase between Post<br>and Pre-vaccination<br>titres |
|---|---|---|---|---|
| Neutra<br>RSV-A | <8 | NEG | 4 | LLOQ/2 |
| | [8-LLOQ[ | POS | 8 | LLOQ/2 |
| | ≥LLOQ | POS | Exact value | Exact value |
| Neutra | <6 | NEG | 3 | LLOQ/2 |
| RSV-B | [6-LLOQ[ | POS | 6 | LLOQ/2 |
| | ≥LLOQ | POS | Exact value | Exact value |

- Vaccine response to the RSV neutralising antibodies (anti-RSV-A and anti-RSV-B) will be defined as:
  - At least a 4-fold increase from pre-vaccination if pre-vaccination neutralising *antibody titre* < 7 *log2* (< 128).
  - At least a 3-fold increase from pre-vaccination if pre-vaccination neutralising antibody titre in [7-8] log2 ([128-256]).
  - At least a 2.5-fold increase from pre-vaccination if pre-vaccination neutralising antibody titre in >8-10 log2 (>256-1024).

204812 (RSV F-021)

Statistical Analysis Plan Amendment 4 Final

- At least 1-fold from pre-vaccination if pre-vaccination neutralising antibody titre >10 log2 (>1024).
- All CI computed will be two-sided 95% CI.

#### 11.2.5. Safety

- For a given subject and the analysis of solicited symptoms within 7 days post-vaccination, missing or non-evaluable measurements will not be replaced. Therefore the analysis of the solicited symptoms based on the Total Vaccinated Cohort will include only vaccinated subjects for doses with documented safety data (i.e., symptom screen completed). More specifically the following rules will be used:
  - Subjects who documented the absence of a solicited symptom after one dose will be considered not having that symptom after that dose.
  - Subjects who documented the presence of a solicited symptom and fully or
    partially recorded daily measurement over the solicited period will be included
    in the summaries at that dose and classified according to their maximum
    observed daily recording over the solicited period.
  - Subjects who documented the presence of a solicited symptom after one dose without having recorded any daily measurement will be assigned to the lowest intensity category at that dose (i.e., 37.5°C for fever or grade 1 for other symptoms).
  - Doses without symptom sheets documented will be excluded.
- For analysis of unsolicited adverse events, such as serious adverse events or adverse
  events by primary MedDRA term, and for the analysis of concomitant medications,
  all vaccinated subjects will be considered. Subjects who did not report the event or
  the concomitant medication will be considered as subjects without the event or the
  concomitant medication respectively.
- The preferred route for recording temperature in this study will be oral. For the analysis, temperatures will be coded as follows:

| Grade | Temperature for oral, axillary or tympanic route | Temperature for rectal route |
|---|---|---|
| 0 | < 37.5°C | < 38.0°C |
| 1 | ≥ 37.5°C - ≤ 38.5°C | ≥ 38.0°C - ≤ 39.0°C |
| 2 | > 38.5°C - ≤ 39.5°C | > 39.0°C - ≤ 40.0°C |
| 3 | > 39.5°C | > 40.0°C |

204812 (RSV F-021) Statistical Analysis Plan Amendment 4 Final

Note that for all tables described in this section, the way the percentage of subjects will be derived will depend on the event analysed (see table below for details). As a result, the N value will differ from one table to another.

| Event | N used for deriving % per subject for Vaccination phase |
|---|---|
| Concomitant vaccination | All subjects with study vaccine administered |
| Solicited general symptom | All subjects with at least one solicited general symptom documented as either present or absent (i.e., symptom screen completed) |
| Solicited local symptom | All subjects with at least one solicited local symptom documented as either present or absent (i.e., symptom screen completed) |
| Unsolicited symptom | All subjects with study vaccine administered |
| Concomitant medication | All subjects with study vaccine administered |

The intensity scale of the following solicited AEs will be assessed as described:

| Adverse Event | Intensity<br>grade | Parameter |
|---|---|---|
| Pain at injection site | 0 | None |
| | 1 | Mild: Any pain neither interfering with nor preventing normal every day activities. |
| | 2 | Moderate: Painful when limb is moved and interferes with every day activities. |
| | 3 | Severe: Significant pain at rest. Prevents normal every day activities. |
| Redness at injection site | | Record greatest surface diameter in mm |
| Swelling at injection site | | Record greatest surface diameter in mm |
| Fever* | | Record temperature in °C |
| Headache | 0 | Normal |
| | 1 | Mild: Headache that is easily tolerated |
| | 2 | Moderate: Headache that interferes with normal activity |
| | 3 | Severe: Headache that prevents normal activity |
| Fatigue | 0 | Normal |
| | 1 | Mild: Fatigue that is easily tolerated |
| | 2 | Moderate: Fatigue that interferes with normal activity |
| | 3 | Severe: Fatigue that prevents normal activity |
| Gastrointestinal | 0 | Normal |
| symptoms (nausea, | 1 | Mild: Gastrointestinal symptoms that are easily tolerated |
| vomiting, diarrhoea 2 Moderate: Gastrointestinal symptoms that interfere with normal ac | | Moderate: Gastrointestinal symptoms that interfere with normal activity |
| and/or abdominal pain) | 3 | Severe: Gastrointestinal symptoms that prevent normal activity |

<sup>\*</sup>Fever is defined as temperature  $\geq$  37.5°C for oral, axillary or tympanic route, or  $\geq$  38.0°C for rectal route. The preferred route for recording temperature in this study will be oral.

The maximum intensity of local injection site redness/swelling will be scored at GSK Biologicals according to the standard GSK Biologicals' scoring system for adults:

0:  $\leq 20 \text{ mm}$ 

1:  $> 20 \text{ mm to} \le 50 \text{ mm}$ 

2:  $> 50 \text{ mm to} \le 100 \text{ mm}$ 

3: > 100 mm

The maximum intensity of fever will be scored at GSK Biologicals according to the standard GSK Biologicals' scoring system for adults (via the preferred route for recording temperature in this study which is oral):

0:  $< 37.5 \, ^{\circ}\text{C}$ 

1:  $\geq 37.5 \,^{\circ}\text{C} \text{ to} \leq 38.5 \,^{\circ}\text{C}$ 

2:  $> 38.5 \, ^{\circ}\text{C} \text{ to} \le 39.5 \, ^{\circ}\text{C}$ 

3: > 39.5°C

The investigator assessed the maximum intensity that occurred over the duration of the event for all unsolicited AEs (including SAEs) recorded during the study. The assessment was based on the investigator's clinical judgement.

For clintrial gov and EudraCT posting purposes, a summary of subjects with all combined solicited (regardless of their duration) and unsolicited adverse events will be provided. Solicited adverse events will be coded by MedDRA as per the following codes.

204812 (RSV F-021)

Statistical Analysis Plan Amendment 4 Final

| Solicited symptom | Lower level term name | Lower level term code | Corresponding Primary<br>Term code |
|---|---|---|---|
| Pain | Pain | 10033371 | 10033371 |
| Redness | Erythema | 10015150 | 10015150 |
| Swelling | Swelling | 10042674 | 10042674 |
| Fatigue | Fatigue | 10016256 | 10016256 |
| Fever | Fever | 10016558 | 10037660 |
| Gastroinstestinal symptoms | Gastroinstestinal disorder | 10017944 | 10017944 |
| Headache | Headache | 10019211 | 10019211 |

#### 11.2.6. Number of decimals displayed

The following decimal description from the decision rules will be used for the demography, immunogenicity and safety/reactogenicity.

| Display Table | Parameters | Number of decimal digits |
|---|---|---|
| All summaries | % of count, including LL & UL of CI | 1 |
| All summaries | % of difference, including LL & UL of CI | 2 |
| Demographic characteristics | Mean, median age, SD (age) | 1 |
| Reactogenicity | Mean, Min, Q1, Median, Q3, Max for duration | 1 |
| Immunogenicity | Ratio of GMT/GMC | 2 |

#### 12. ANNEX 2: SUMMARY ON ELIMINATION CODES

Refer to section 5.2

# 13. ANNEX 3 CALCULATION OF INDIVIDUAL AND OVERALL DESIRABILITY INDEX

The section below provide the details on how to calculate individual desirability index and overall desirability index score based on Annex E in the Protocol.

#### Reactogenicity

A logistic regression model will be fitted on each reactogenicity endpoint (any Grade 2/3 general AE and any related SAE, Grade 2/3 fever) reported during the 7-day follow-up period after vaccination, including all RSV formulations.

- The vaccine group as the fixed effect
- The age groups (18-32 years and 33-45 years) as the categorical covariant if deemed necessary.

The estimation of indication rate will be tabulated by treatment group. The SAS codes can be used as reference:

proc logistic data=React;

class Treatment AgeGroup / param=glm;

model response (event='AE')= Treatment | AgeGroup;

lsmeans Treatment / ILINK e diff oddsratio adjust=bon cl; run;

For any Grade 2/3 general AEs and any related SAEs, the incidence rate estimate (IR) will be transformed in a [0,1] desirability index using the following function:

DR1 = 
$$\begin{cases} \frac{1}{1 + \exp(-50 * (0.25 - H))}, & \text{if } HR \le 0.25 \\ \frac{1}{1 + \exp(-25 * (0.25 - HR))}, & \text{if } IR \ge 0.25 \end{cases}$$

where IR is the incidence rate estimated by the model. This function will allocate a desirability value of 1, 0.5 and 0 to incidence rate equal to 0.1, 0.25 and 0.5 respectively (see Figure 2). But the calculation equally weights Grade 2/3 general AEs and any related SAEs.

Figure 2 Desirability function for the incidence rate of Grade 2/3 general AEs and related SAEs - for each investigational RSV vaccine formulation



For Grade 2/3 fever, the incidence rate estimate (IR) will be transformed in a [0,1] desirability index using the following function:

$$DR2 = \frac{1}{1 + \exp(-120 * (0.05 - IR))}$$

where IR is the incidence rate estimated by the model. As illustrated in Figure 3, the function will allocate desirability values of 1, 0.5 and 0 to incidence rate equal to 0, 0.05 and 0.1 respectively.

Figure 3 Desirability function for the incidence rate of Grade 2/3 fever - for each investigational RSV vaccine formulation



Finally, the reactogenicity index will be computed by taking the geometric mean of the 2 indexes:

$$DR = \sqrt{DR1 * DR2}$$

#### **Immunogenicity**

The ANCOVA model will be fitted on the log-transformed titre for each immune response of neutralising anti-RSV-A and PCA separately including

- The vaccine group as the fixed effect
- o The pre-vaccination titre/concentration and age groups (18-32 years and 33-45 years) as the covariates if deemed necessary

The mean estimations of GMTs/GMCs for each treatment group at Day 30 and its 95% CI will be provided for immunogenicity desirability calculation. The estimated GMT and LL will be tabulated by treatment group.

As formulations inducing a high immune response will be considered suitable, the lower limit (LL) of the estimated GMT/C adjusted for pre-vaccination titres will be the statistical criterion considered for decision making.

Neutralising anti-RSV-A titres

The LL of the GMT estimate will be transformed into a [0, 1] desirability index using the function:

DI1 = 
$$\frac{1}{1 + \exp(1.5 * (9.5 - LL))}$$

where LL is the lower limit of the 95% confidence interval of the GMT adjusted for prevaccination titres in log base 2. The function was chosen to have a desirability of 0 at LL value  $\leq$  6 log2 (=128), and a desirability of 1 at LL value  $\geq$  13 log2. This function is illustrated in Figure 4.

Figure 4 Desirability function for neutralising anti-RSV-A GMTs - for each investigational RSV vaccine formulation



#### PCA concentrations

The LL of the GMC adjusted for pre-vaccination titres estimate will be transformed using the following function:

DI2 = 
$$\frac{\frac{1}{1 + \exp(0.05 * (150 - LL))}}, \quad \text{if LL} \le 150$$
$$\frac{1}{1 + \exp(0.025 * (150 - LL))}, \quad \text{if LL} \ge 150$$

As illustrated in Figure 5, a PCA response of 25, 150 and 400 μg/mL will have a desirability value of 0, 0.5 and 1 respectively.

Figure 5 Desirability function for PCA concentrations - for each investigational RSV vaccine formulation



Finally, the immunogenicity index will be computed by taking the geometric mean of the 2 indexes:

$$DI = \sqrt{DI1 * DI2}$$

# Overall desirability index

The overall desirability index for each formulation will be obtained by computing the following weighted geometric mean:  $D = DR^{0.4} * DI^{0.6}$ .
#### 14. ANNEX 4: STUDY SPECIFIC MOCK TFL

The following draft study specific mock TFLs will be used. The data display, title and footnote are for illustration purpose and will be adapted to the study specificity as indicated in the TFL TOC.

Note that there may be few changes between the study specific SAP mock TFL and the final TFLs. These editorial/minor changes will not lead to a SAP amendment.

| Template # | Table Title | Macro |
|---|---|---|
| Template 1 | Number of subjects enrolled into the study as well as the number of subject excluded from PPS analysis with reasons for exclusion | %ELIMLIST |
| Template 2 | Number of subjects vaccinated, completed and withdrawn with reason for withdrawal (Exposed set) | %DROP_SUM (OTH=1) |
| Template 3 | Number of subjects vaccinated, completed and withdrawn with reason for withdrawal (Exposed set) | %DROP_SUM (OTH=0) |
| Template 4 | Number of subjects at each visit and list of withdrawn subjects (Exposed set) | %DROPOUT |
| Template 5 | Summary of demographic characteristics (Exposed set) | %DEMOGRA |
| Template 6 | Summary of demographic characteristics by age category (Exposed set) | %DEMOGRA |
| Template 7 | Number of subjects by center (Exposed set) | %CENTER |
| Template 8 | Number of subjects by center for each age category (Exposed set) | %CENTER |
| Template 9 | Number of subjects by country and center (Exposed set) | %CENTER |
| Template 10 | Deviations from specifications for age and intervals between study visits (Exposed set) | %INT_VAL |
| Template 11 | Summary of vital signs characteristics (Exposed set) | %VITAL_SIGNS |
| Template 12 | Study Population (Exposed set) | %CTR_DEMOG |
| Template 13 | Number of enrolled subjects by country | %FREQ_DIS |
| Template 14 | Number of enrolled subjects by age category | %FREQ_DIS |
| Template 15 | Minimum and maximum activity dates (Exposed set) | %DATE |
| Template 16 | Incidence and nature of symptoms (solicited and unsolicited) reported during the <b>7-day</b> (Days 0-6) post-vaccination period (Exposed set) | %LOCGEN |
| Template 17 | Daily prevalence of <b>any fever</b> during the 7-day (Days 0-6) post-vaccination period (Exposed set) | %SYMPLOT |
| Template 18 | Incidence of solicited <b>local</b> symptoms reported during the 7-day (Days 0-6) post-vaccination period (Exposed set) | %FREQ |
| Template 19 | Incidence of solicited <b>local</b> symptoms reported during the 7-day (Days 0-6) post-vaccination period by <b>maximum intensity</b> (Exposed set) | %FREQ |
| Template 20 | Incidence of solicited <b>general</b> symptoms reported during the 7-day (Days 0-6) post-vaccination period (Exposed set) | %FREQ |
| Template 21 | Incidence of solicited <b>general</b> symptoms reported during the 7-day (Days 0-6) post-vaccination period <b>by maximum intensity</b> (Exposed set) | %FREQ |
| Template 22 | Percentage of subjects reporting the occurrence of unsolicited symptoms classified by MedDRA Primary System Organ Class | %UNSOL |

### 204812 (RSV F-021) Statistical Analysis Plan Amendment 4 Final

| | | alysis Plan Amendment 4 Final |
|---|---|---|
| | and Preferred Term, during the <b>30-day</b> (Days 0-29) post-vaccination period (Exposed set) | |
| Template 23 | Percentage of subjects reporting the occurrence of unsolicited symptoms classified by MedDRA Primary System Organ Class and Preferred Term, during the 30-day (Days 0-29) post-vaccination period (Exposed set) | %UNSOL |
| Template 24 | Listing of <b>SAEs</b> reported up to study end (Exposed set) | %SAE |
| Template 25 | Number (%) of subjects with serious adverse events up <b>Day 7</b> (Exposed set) | %CTR_SAE |
| Template 26 | Compliance in returning symptom information (Exposed set) | % COMPLI |
| Template 27 | Number and percentage of subjects taking a <b>concomitant medication</b> during the <b>7- day</b> (Days 0-6) post -vaccination period (Exposed set) | %CMED_INC |
| Template 28 | Exploratory comparisons between groups in terms of percentage of subjects reported any Grade 2/3 AE and/or any fever >38.5°C and/or any vaccine-related SAE during the 7 day (Days 0-6) Post- vaccination period (Exposed set) | %COMP_FQ_AE |
| Template 29 | Solicited and unsolicited symptoms experienced by at least 5 % of subjects, classified by MedDRA Primary System Organ Class and Preferred Term within the 30-day (Days 0-29) post-vaccination period including number of events - SAE excluded (Exposed set) | %UNSOL (NIH=5, EVENT=1) |
| Template 30 | Distribution of change from baseline in haematology and biochemistry with respect to normal laboratory ranges (Exposed set) | %HAEMATO_BIOCH |
| Template 31 | Summary of haematology and biochemistry results by maximum grade from VISIT 2 (D7) up to VISIT 3 (D30) versus baseline (Exposed set) | %HAEMATO_BIOCH_GR_CHAN<br>GE |
| Template 32 | Summary of haematology and biochemistry results by maximum grade in the specified category from VISIT 2 (D7) up to VISIT 3 (D30) versus baseline (Exposed set) | %freq_dis |
| Tomplete 22 | Summary of <b>haematology</b> change from baseline by maximum | %HAEMATO_BIOCH_GR_CHAN |
| Template 33 | grade from VISIT2 (D7) up to VISIT 3 (D30) (Exposed set) | GE |
| Template 34 | | |
| • | grade from VISIT2 (D7) up to VISIT 3 (D30) (Exposed set) Summary of haematology change from baseline by maximum grade in the specified category from VISIT2 (D7) | GE |
| Template 34 Template 35 Template 36 | grade from VISIT2 (D7) up to VISIT 3 (D30) (Exposed set) Summary of haematology change from baseline by maximum grade in the specified category from VISIT2 (D7) up to VISIT3 (D30) (Exposed set) Individual results of hemoglobin levels outside of the normal ranges in <group> (Exposed set) Number and percentage of subjects with anti-RSV-A neutralising antibody titer equal to or above <cut-off> and GMTs (Per protocol set)</cut-off></group> | GE %freq_dis %HB_PROFIL %GMT |
| Template 35 Template 36 Template 37 | grade from VISIT2 (D7) up to VISIT 3 (D30) (Exposed set) Summary of haematology change from baseline by maximum grade in the specified category from VISIT2 (D7) up to VISIT3 (D30) (Exposed set) Individual results of hemoglobin levels outside of the normal ranges in <group> (Exposed set) Number and percentage of subjects with anti-RSV-A neutralising antibody titer equal to or above <cut-off> and GMTs (Per protocol set) Number and percentage of subjects with anti-RSV-A neutralising antibody titer equal to or above <cut-off> and GMTs - by age category (Per protocol set)</cut-off></cut-off></group> | GE %freq_dis %HB_PROFIL |
| Template 35 Template 36 Template 37 Template 38 | grade from VISIT2 (D7) up to VISIT 3 (D30) (Exposed set) Summary of haematology change from baseline by maximum grade in the specified category from VISIT2 (D7) up to VISIT3 (D30) (Exposed set) Individual results of hemoglobin levels outside of the normal ranges in <group> (Exposed set) Number and percentage of subjects with anti-RSV-A neutralising antibody titer equal to or above <cut-off> and GMTs (Per protocol set) Number and percentage of subjects with anti-RSV-A neutralising antibody titer equal to or above <cut-off> and GMTs - by age category (Per protocol set) Geometric mean of the individual ratio of anti-RSV-A neutralising antibody titers at each post-vaccination timepoint compared to pre-vaccination with 95% CI (Per protocol set)</cut-off></cut-off></group> | GE %freq_dis %HB_PROFIL %GMT %GMT |
| Template 34 Template 35 Template 36 Template 37 Template 38 Template 39 | grade from VISIT2 (D7) up to VISIT 3 (D30) (Exposed set) Summary of haematology change from baseline by maximum grade in the specified category from VISIT2 (D7) up to VISIT3 (D30) (Exposed set) Individual results of hemoglobin levels outside of the normal ranges in <group> (Exposed set) Number and percentage of subjects with anti-RSV-A neutralising antibody titer equal to or above <cut-off> and GMTs (Per protocol set) Number and percentage of subjects with anti-RSV-A neutralising antibody titer equal to or above <cut-off> and GMTs - by age category (Per protocol set) Geometric mean of the individual ratio of anti-RSV-A neutralising antibody titers at each post-vaccination timepoint compared to pre-vaccination with 95% CI (Per protocol set) GMTs and their 95% CIs for anti-RSV-A neutralising antibody at each timepoint (Per protocol set)</cut-off></cut-off></group> | GE %freq_dis %HB_PROFIL %GMT %GMT %GMRACT %GMTPLOT* |
| Template 34 Template 35 Template 36 Template 37 Template 38 Template 39 Template 40 | grade from VISIT2 (D7) up to VISIT 3 (D30) (Exposed set) Summary of haematology change from baseline by maximum grade in the specified category from VISIT2 (D7) up to VISIT3 (D30) (Exposed set) Individual results of hemoglobin levels outside of the normal ranges in <gravesyselses <cut-off="" above="" anti-rsv-a="" antibody="" equal="" neutralising="" of="" or="" subjects="" titer="" to="" with=""> and GMTs (Per protocol set) Number and percentage of subjects with anti-RSV-A neutralising antibody titer equal to or above <cut-off> and GMTs - by age category (Per protocol set) Geometric mean of the individual ratio of anti-RSV-A neutralising antibody titers at each post-vaccination timepoint compared to pre-vaccination with 95% CI (Per protocol set) GMTs and their 95% CIs for anti-RSV-A neutralising antibody at each timepoint (Per protocol set) Kinetics of GMTs for anti-RSV-A neutralising antibody on subjects with results available at all timepoints (Per protocol set)</cut-off></gravesyselses> | GE %freq_dis %HB_PROFIL %GMT %GMRACT %GMTPLOT* %KIN_GM* |
| Template 34 Template 35 Template 36 Template 37 Template 38 Template 39 Template 40 Template 41 | grade from VISIT2 (D7) up to VISIT 3 (D30) (Exposed set) Summary of haematology change from baseline by maximum grade in the specified category from VISIT2 (D7) up to VISIT3 (D30) (Exposed set) Individual results of hemoglobin levels outside of the normal ranges in <group> (Exposed set) Number and percentage of subjects with anti-RSV-A neutralising antibody titer equal to or above <cut-off> and GMTs (Per protocol set) Number and percentage of subjects with anti-RSV-A neutralising antibody titer equal to or above <cut-off> and GMTs - by age category (Per protocol set) Geometric mean of the individual ratio of anti-RSV-A neutralising antibody titers at each post-vaccination timepoint compared to pre-vaccination with 95% CI (Per protocol set) GMTs and their 95% CIs for anti-RSV-A neutralising antibody at each timepoint (Per protocol set) Kinetics of GMTs for anti-RSV-A neutralising antibody on subjects with results available at all timepoints (Per protocol set) Distribution of anti-neogenin antibody concentration (Exposed set)</cut-off></cut-off></group> | GE %freq_dis %HB_PROFIL %GMT %GMT %GMRACT %GMTPLOT* %KIN_GM* |
| Template 34 Template 35 Template 36 Template 37 Template 38 Template 39 Template 40 Template 41 Template 41 | grade from VISIT2 (D7) up to VISIT 3 (D30) (Exposed set) Summary of haematology change from baseline by maximum grade in the specified category from VISIT2 (D7) up to VISIT3 (D30) (Exposed set) Individual results of hemoglobin levels outside of the normal ranges in <group> (Exposed set) Number and percentage of subjects with anti-RSV-A neutralising antibody titer equal to or above <cut-off> and GMTs (Per protocol set) Number and percentage of subjects with anti-RSV-A neutralising antibody titer equal to or above <cut-off> and GMTs - by age category (Per protocol set) Geometric mean of the individual ratio of anti-RSV-A neutralising antibody titers at each post-vaccination timepoint compared to pre-vaccination with 95% CI (Per protocol set) GMTs and their 95% CIs for anti-RSV-A neutralising antibody at each timepoint (Per protocol set) Kinetics of GMTs for anti-RSV-A neutralising antibody on subjects with results available at all timepoints (Per protocol set) Distribution of fold of anti-neogenin antibody concentration (Exposed set) Distribution of fold of anti-neogenin antibody concentration (Exposed set)</cut-off></cut-off></group> | GE %freq_dis %HB_PROFIL %GMT %GMT %GMRACT %GMTPLOT* %KIN_GM* %DIS %DIS |
| Template 34 Template 35 Template 36 Template 37 Template 38 Template 39 Template 40 Template 41 | grade from VISIT2 (D7) up to VISIT 3 (D30) (Exposed set) Summary of haematology change from baseline by maximum grade in the specified category from VISIT2 (D7) up to VISIT3 (D30) (Exposed set) Individual results of hemoglobin levels outside of the normal ranges in <group> (Exposed set) Number and percentage of subjects with anti-RSV-A neutralising antibody titer equal to or above <cut-off> and GMTs (Per protocol set) Number and percentage of subjects with anti-RSV-A neutralising antibody titer equal to or above <cut-off> and GMTs - by age category (Per protocol set) Geometric mean of the individual ratio of anti-RSV-A neutralising antibody titers at each post-vaccination timepoint compared to pre-vaccination with 95% CI (Per protocol set) GMTs and their 95% CIs for anti-RSV-A neutralising antibody at each timepoint (Per protocol set) Kinetics of GMTs for anti-RSV-A neutralising antibody on subjects with results available at all timepoints (Per protocol set) Distribution of anti-neogenin antibody concentration (Exposed set) Distribution of fold of anti-neogenin antibody concentration</cut-off></cut-off></group> | GE %freq_dis %HB_PROFIL %GMT %GMT %GMRACT %GMTPLOT* %KIN_GM* |

## 204812 (RSV F-021) Statistical Analysis Plan Amendment 4 Final

| | protocol set) | |
|---|---|---|
| Template 45 | Distribution of fold of anti-RSV-A neutralising antibody titer by cumulative pre-vaccination titer category (Per protocol set) | %DIS |
| Template 46 | Reverse cumulative distribution curves for <b>anti-RSV-A</b> neutralising antibody titers in each group at pre-vaccination (Per protocol set) | %REVCUM |
| Template 47 | Individual results of <b>anti-RSV-A</b> neutralising antibody titer at Day <30/60/90> versus pre-vaccination in <each group=""> and Control (Per protocol set)</each> | %SCATTERPLOT* |
| Template 48 | Vaccine response for <b>anti-RSV-A</b> neutralising antibody titer at each post-vaccination timepoint (Per protocol set) | %HUM_RESP* |
| Template 49 | Estimated GMTs and 95% CIs for <b>anti-RSV-A</b> neutralising antibody titre (Per protocol set) | %GMT_ANOVA |
| Template 50 | Exploratory comparisons (GMT ratios) between RSV groups with corresponding 95% confidence interval for <b>anti-RSV A</b> neutralizing antibody titre at <b>Day 30</b> (Per protocol set) | %GMT_RATIO |
| Template 51 | Individual kinetics of <b>anti-neogenin</b> antibody concentrations by group (Exposed set) | %NEO_INDKIN* |
| Template 52 | GM of individual ratios (fold increase post over pre) and their 95% CIs for <b>anti-RSV F IgG1 and IgG total</b> antibody assays and each group, at <b>Day 30</b> (Per protocol set) | %GMRPLOT* |
| Template 53 | Exploratory comparisons (GM ratios of fold increase post/pre) between RSV groups with corresponding 95% confidence interval for anti-RSV F lgG1 antibody concentrations at Day 30 (Per protocol set) | %GMF_RATIO* |
| Template 54 | Comparisons of GM ratios with corresponding 95% confidence interval between anti-RSV F antibody concentrations (IgG Total) and anti-RSV-A neutralising antibody titers at pre-vaccination (Per protocol set) | %GM_RATIO_PRE.SAS** |
| Template 55 | Exploratory comparisons (GM ratios of fold increase post/pre) with corresponding 95% confidence interval between anti-RSV F antibody concentrations (IgG Total) and anti-RSV-A neutralising antibody titers at Day 30 (Per protocol set) | %GM_RATIO_FI.SAS** |
| Template 56 | Desirability index of immunogenicity during the 30-day (Days 0-29) post-vaccination period (Per protocol set) | %Immuno_DI** |
| Template 57 | Desirability index of reactogenicity during the 7-day (Days 0-6) post-vaccination period (Exposed set) | %Reacto_DI** |
| Template 58 | Desirability index based on reactogenicity and safety (Exposed set up to Day 7) and immunogenicity (Per protocol set up to Day 30) | %Overall_DI** |
| Template 59 | Percentage of subjects reporting solicited local symptoms (any grade / grade 3) during the 7-day post-vaccination period (Exposed set) | %GFREQ |

<sup>\*</sup> Name of specific macros created in study RSV F-001 (116969), RSV F-020 (201510)

<sup>\*\*</sup> Name of specific macros created in study RSV F-021 (204812)
\*\*\* It is the simplified version of Template 22 without UL and LL added for the final analysis

204812 (RSV F-021)

Statistical Analysis Plan Amendment 4 Final

### Template 1 Number of subjects enrolled into the study as well as the number of subjects excluded from the PPS analyses with reasons for exclusion

| | Total | | | <each group=""></each> | |
|---|---|---|---|---|---|
| Title | n | s | % | n | s |
| Total enrolled cohort | | | | | |
| Study vaccine dose not administered at all but subject number allocated (code 1030) | | | | | |
| Exposed set | | | | | |
| <reason &="" code="" elimination="" for=""></reason> | | | | | |
| <reason &="" code="" elimination="" for=""></reason> | | | | | |
| Per protocol set for immunogenicity | | | | | |

#### <each group>:

30 PreF = 30 µg PreF

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

Note: Subjects may have more than one elimination code assigned

n = number of subjects with the elimination code assigned excluding subjects who have been assigned a lower elimination code number

s = number of subjects with the elimination code assigned

% = percentage of subjects in the considered Per protocol set relative to the Exposed set

### Template 2 Number of subjects vaccinated, completed and withdrawn with reason for withdrawal (Exposed set)

| | <each group=""></each> | Total |
|---|---|---|
| Number of subjects vaccinated | | |
| Number of subjects completed | | |
| Number of subjects withdrawn | | |
| Reasons for withdraw: | | |
| Serious Adverse Event | | |
| Non-serious adverse event | | |
| Protocol violation | | |
| Consent withdrawal (not due to an adverse event) | | |
| Migrated/moved from study area | | |
| Lost to follow-up (subjects with incomplete vaccination course) | | |
| Lost to follow-up (subjects with complete vaccination course) | | |
| Others | | |

#### <each group>:

30 PreF = 30 µg PreF

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

Vaccinated = number of subjects who were vaccinated in the study

Completed = number of subjects who completed last study visit

withdrawn = number of subjects who did not come for the last study visit

204812 (RSV F-021)

Statistical Analysis Plan Amendment 4 Final

### Template 3 Number of subjects vaccinated, completed and withdrawn with reason for withdrawal (Exposed set)

| | <each group=""></each> | Total |
|---|---|---|
| Number of subjects vaccinated | | |
| Number of subjects completed | | |
| Number of subjects withdrawn | | |
| Reasons for withdrawal : | | |
| Serious Adverse Event | | |
| Non-Serious Adverse Event | | |
| Protocol violation | | |
| Consent withdrawal (not due to an adverse event) | | |
| Migrated/moved from study area | | |
| Lost to follow-up (subjects with incomplete vaccination course) | | |
| Lost to follow-up (subjects with complete vaccination course) | | |
| Sponsor study termination | | |
| Other - <reason></reason> | | |
| Other - <reason></reason> | | |

#### <each group>:

30 PreF = 30  $\mu$ g PreF

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

Vaccinated = number of subjects who were vaccinated in the study

Completed = number of subjects who completed last study visit

Withdrawn = number of subjects who did not come for the last study visit

Template 4 Number of subjects at each visit and list of withdrawn subjects (Exposed set)

| Group | Visit | N | Withdrawn Subject number | Reason for withdrawal |
|---|---|---|---|---|
| <each group=""></each> | VISIT 1 (D0) | | | |
| , | VISIT 2 (D7) | | | |
| | VISIT 3 (D30) | | | |
| | VISIT 4 (D60) | | | |
| | VISIT 5 (D90) | | | |

#### <each group>:

 $30 \text{ PreF} = 30 \mu \text{g PreF}$ 

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

N = Number of subjects who are still in the study up to the visit

Withdrawn = Subject who did not return after the visit

204812 (RSV F-021)

Statistical Analysis Plan Amendment 4 Final

#### Template 5 Summary of demographic characteristics (Per Protocol Set)

| | | | n group><br>N= ) | Total<br>(N= ) | |
|---|---|---|---|---|---|
| Characteristics | Parameters or | Value or n | % | Value<br>or n | % |
| Age (years) at vaccination | Categories Mean | | | | |
| | SD<br>Median | | | | |
| | Minimum<br>Maximum | | | | |
| Ethnicity | American Hispanic or Latino Not American Hispanic or Latino | | | | |
| Geographic Ancestry | African Heritage / African American American Indian or Alaskan Native | | | | |
| | Asian - Central/South Asian Heritage | | | | |
| | Asian - East Asian Heritage Asian - Japanese Heritage | | | | |
| | Asian - South East Asian Heritage Native Hawaiian or Other Pacific Islander | | | | |
| | White - Arabic / North African Heritage<br>White - Caucasian / European Heritage | | | | |
| | Other | | | | |

#### <each group>:

30 PreF = 30 μg PreF

60 PreF = 60 μg PreF

120 PreF = 120 µg PreF

Control = Placebo

N = total number of subjects

n/% = number / percentage of subjects in a given category

Value = value of the considered parameter

SD = standard deviation

204812 (RSV F-021)

Statistical Analysis Plan Amendment 4 Final

## Template 6 Summary of demographic characteristics by age category (Exposed set)

| | | <each group=""><br/>(N=)</each> | | | | Total<br>(N= ) | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | <subgroup></subgroup> | | <subgroup></subgroup> | | <subgroup></subgroup> | | <subgroup< th=""></subgroup<> | |
| Characteristics | Parameters or<br>Categories | Value<br>or n | % | Value<br>or n | % | Value<br>or n | % | Value<br>or n | % |
| Age (years) at | Mean<br>SD | | | | | | | | |
| vaccination | Median | | | | | | | | |
| | Minimum<br>Maximum | | | | | | | | |
| Ethnicity | American Hispanic or Latino | | | | | | | | |
| Geographic<br>Ancestry | Not American Hispanic or Latino African Heritage / African American | | | | | | | | |
| , | American Indian or Alaskan Native Asian - Central/South Asian Heritage | | | | | | | | |
| | Asian - East Asian Heritage | | | | | | | | |
| | Asian - Japanese Heritage Asian - South East Asian Heritage | | | | | | | | |
| | Native Hawaiian or Other Pacific Islander | | | | | | | | |
| | White - Arabic / North African<br>Heritage | | | | | | | | |
| | White - Caucasian / European<br>Heritage | | | | | | | | |
| | Other | | | | | | | | |

#### <each group>:

30 PreF = 30 μg PreF

60 PreF = 60 µg PreF

120 PreF = 120 µg PreF

Control = Placebo

N = total number of subjects

n/% = number / percentage of subjects in a given category

Value = value of the considered parameter

SD = standard deviation

#### <subgroup> by age category:

18-32Y = 18-32 years old subjects

33-45Y = 33-45 years old subjects

204812 (RSV F-021)

Statistical Analysis Plan Amendment 4 Final

#### Template 7 Number of subjects by center (Exposed set)

| | | <each group=""></each> | То | tal |
|--------|---|------------------------|----|-----|
| Center | • | n | n | % |
| PPD | | | | |
| PPD | | | | |
| All | | | | |

#### <each group>:

30 PreF = 30 µg PreF

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

n = number of subjects included in each group or in total for a given center or for all centers

All = sum of all subjects in each group or in total (sum of all groups)

 $% = n/AII \times 100$ 

Center = GSK Biologicals assigned center number

#### Template 8 Number of subjects by center for each age category (Exposed set)

| | 30 F | 30 PreF | | 60 PreF | | 120 PreF | | Control | | Total | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 18-32Y | 33-45Y | 18-32Y | 33-45Y | 18-32Y | 33-45Y | 18-32Y | 33-45Y | 18-3 | 2Y | 33-4 | 5Y |
| Center | n | n | n | n | n | n | n | n | n | % | n | % |

 $30 \text{ PreF} = 30 \mu \text{g PreF}$ 

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

18-32Y = 18-32 years old subjects

33-45Y = 33-45 years old subjects

n = number of subjects included in each group or in total for a given center or for all centers

All = sum of all subjects in each group or in total (sum of all groups)

 $% = n/AII \times 100$ 

Center = GSK Biologicals assigned center number

#### Template 9 Number of subjects by country and center (Exposed set)

| | | <each group=""></each> | | Total |
|---------|--------|------------------------|---|-------|
| Country | Center | n | n | % |
| | All | | | |
| All | All | | | |

#### <each group>:

30 PreF = 30 µg PreF

60 PreF = 60 µg PreF

120 PreF = 120 µg PreF

Control = Placebo

n = number of subjects included in each group or in total for a given center or for all centers

All = sum of all subjects in each group or in total (sum of all groups)

 $% = n/AII \times 100$ 

Center = GSK Biologicals assigned center number

204812 (RSV F-021)

Statistical Analysis Plan Amendment 4 Final

## Template 10 Deviations from specifications for age and intervals between study visits (Exposed set)

| | | Age | Dose:1-PI (D30) | Dose:1-PI (D60) | Dose:1-PI (D90) | Dose:1-<br>CONCLUSION |
|---|---|---|---|---|---|---|
| Group | | Protocol | Protocol | Protocol | Protocol | Protocol |
| | | from 18 to 45 years | from 30 to 44 days | from 56 to 70 days | from 86 to 100 days | from 330 to 390<br>days |
| <each<br>group&gt;</each<br> | n | | | | | |
| | N | | | | | |
| | % | | | | | |
| | range | | | | | |

#### <each group>:

30 PreF = 30 μg PreF

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

N = total number of subjects with available results

n/% = number / percentage of subjects with results outside of the interval

range = minimum-maximum for age and intervals

PI(D30) = Post-vaccination at Day 30

PI(D60) = Post-vaccination at Day 60

204812 (RSV F-021)

Statistical Analysis Plan Amendment 4 Final

## Template 11 Summary of vital signs characteristics at VISIT 1 (Day 0) (Exposed set)

| | | <each group=""><br/>N =</each> | Total<br>N = |
|---|---|---|---|
| Characteristics | Parameters | Value | Value |
| Height (Cm) | Mean | | |
| | SD | | |
| | Median | | |
| | Minimum | | |
| | Maximum | | |
| | Unknown | | |
| Weight (Kg) | Mean | | |
| | SD | | |
| | Median | | |
| | Minimum | | |
| | Maximum | | |
| | Unknown | | |
| Heart rate (Beats per minute) | Mean | | |
| , , | SD | | |
| | Median | | |
| | Minimum | | |
| | Maximum | | |
| | Unknown | | |
| Respiratory rate (Breadth per minute) | Mean | | |
| | SD | | |
| | Median | | |
| | Minimum | | |
| | Maximum | | |
| | Unknown | | |
| Systolic blood pressure (Mmhg) | Mean | | |
| | SD | | |
| | Median | | |
| | Minimum | | |
| | Maximum | | |
| | Unknown | | |
| Diastolic blood pressure (Mmhg) | Mean | | |
| | SD | | |
| | Median | | |
| | Minimum | | |
| | Maximum | | |
| | Unknown | | |

#### <each group>:

 $30 \text{ PreF} = 30 \mu \text{g PreF}$ 

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 μg PreF

Control = Placebo

N = total number of subjects

Value = value of the considered parameter

SD = standard deviation

204812 (RSV F-021)

#### Statistical Analysis Plan Amendment 4 Final

#### **Template 12 Study Population (Exposed set)**

| Number of subjects | <each group=""></each> | Total |
|---|---|---|
| Planned, N | | |
| Randomised, N (Exposed set) | | |
| Completed, n (%) | | |
| Demographics | <each group=""></each> | Total |
| N (Exposed set) | | |
| Females:Males | | |
| Mean Age, years (SD) | | |
| Median Age, years (minimum, maximum) | | |
| White - caucasian / european heritage, n (%) | | |
| Asian – South East Asian heritage, n (%) | | |

<each group>: 30 PreF = 30 μg PreF

60 PreF = 60 µg PreF 120 PreF = 120 µg PreF Control = Placebo

204812 (RSV F-021)

Statistical Analysis Plan Amendment 4 Final

#### Template 13 Number of enrolled subjects by country

| | | <each group=""><br/>N =</each> | Total<br>N = |
|---|---|---|---|
| Characteristics | Categories | n | n |
| Country | Czech Republic | | |
| | Australia | | |

<each group>:

 $30 \text{ PreF} = 30 \mu \text{g PreF}$ 

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

N = Number of enrolled subjects

n= number of enrolled subjects included in each group or in total for a given country or for all countries

#### Template 14 Number of enrolled subjects by age category

| | | <each group=""><br/>N =</each> | Total<br>N = |
|---|---|---|---|
| Characteristics | Categories | n | n |
| Age category | Adults (18-45 years) | | |
| | Missing | | |

<each group>:

 $30 \text{ PreF} = 30 \mu \text{g PreF}$ 

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

N = Number of enrolled subjects

n= number of enrolled subjects included in each group or in total for a given age category or for all age categories Missing = age at dose 1 unknown

#### Template 15 Minimum and maximum activity dates (Exposed set)

| Group | Activity | <b>Activity Description</b> | Minimum date | Maximum date |
|---|---|---|---|---|
| | number | | | |
| <each group=""></each> | 10 | VISIT 1 (DAY 0) | | |
| | 20 | VISIT 2 (M 1) | | |
| | 30 | VISIT 3 (M 2) | | |
| | 40 | VISIT 4 (M 3) | | |

<each group>:

 $30 \text{ PreF} = 30 \mu \text{g PreF}$ 

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

204812 (RSV F-021)

Statistical Analysis Plan Amendment 4 Final

## Template 16 Incidence and nature of symptoms (solicited and unsolicited reported during the 7-day (Days 0-6) post-vaccination period (Exposed set)

| | Any sy | mptom | | | | Genera | l sympt | oms | | | Local s | ymptor | ns | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | 95% ( | CI | | | | 95% C | Cl | | | | 95% | CI |
| Group | N | n | % | LL | UL | N | n | % | LL | UL | N | n | % | LL | UL |
| <each group=""></each> | | | | | | | | | | | | | | | |

#### <each group>:

30 PreF = 30 µg PreF

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

N = number of subjects with the administered dose

n/% = number/percentage of subjects presenting at least one type of symptom whatever the study vaccine administered

95% CI = exact 95% confidence interval, LL = Lower Limit, UL = Upper Limit

Note: the same table will be generated by group/sub-group, with sub-group= age category (see SAP).

Template 17 Daily prevalence of any fever during the 7-day (Days 0-6) post-vaccination period (Exposed set)



30 PreF = 30 µg PreF 60 PreF = 60 µg PreF 120 PreF = 120 µg PreF Control = Placebo

204812 (RSV F-021)

Statistical Analysis Plan Amendment 4 Final

### Template 18 Incidence of solicited local symptoms reported during the 7-day (Days 0-6) post-vaccination period (Exposed set)

| | | | | <each gro<="" th=""><th>up&gt;</th><th></th></each> | up> | |
|---|---|---|---|---|---|---|
| | | | | | | 95 % CI |
| Symptom | Туре | N | n | % | LL | UL |
| edness (mm) | All | | | | | |
| Pain<br>Redness (mm) | Grade 1 | | | | | |
| | Grade 2 | | | | | |
| | Grade 3 | | | | | |
| | Onset ≤48h | | | | | |
| | Medical advice | | | | | |
| Redness (mm) | All | | | | | |
| , , | >20 and ≤ 50 | | | | | |
| | >50 and ≤ 100 | | | | | |
| | >100 | | | | | |
| | Onset ≤48h | | | | | |
| | Medical advice | | | | | |
| Swelling (mm) | All | | | | | |
| | >20 and ≤ 50 | | | | | |
| | >50 and ≤ 100 | | | | | |
| | >100 | | | | | |
| | Onset ≤48h | | | | | |
| | Medical advice | | | | | |

#### <each group>:

 $30 \text{ PreF} = 30 \mu \text{g PreF}$ 

60 PreF = 60 µg PreF

120 PreF =120 µg PreF

Control = Placebo

N= number of subjects with the documented dose

n/%= number/percentage of subjects reporting at least once the symptom

95%CI= Exact 95% confidence interval; LL = lower limit, UL = upper limit

The maximum intensity of local injection site redness/swelling was coded as follows for adults:

- 0: ≤ 20 mm
- 1:  $> 20 \text{ mm to} \le 50 \text{ mm}$
- 2:  $> 50 \text{ mm to} \le 100 \text{ mm}$
- 3: > 100 mm

204812 (RSV F-021)

Statistical Analysis Plan Amendment 4 Final

## Template 19 Incidence of solicited local symptoms reported during the 7-day (Days 0-6) post-vaccination period by maximum intensity (Exposed set)

| | | | < | each gro | oup> | |
|---------------|----------------|---|---|----------|------|--------|
| | | | | | | 5 % CI |
| Symptom | Туре | N | n | % | LL | UL |
| Pain | All | | | | | |
| | Grade 1 | | | | | |
| | Grade 2 | | | | | |
| | Grade 3 | | | | | |
| | Onset ≤48h | | | | | |
| | Medical advice | | | | | |
| Redness (mm) | All | | | | | |
| , , | >20 and ≤50 | | | | | |
| | >50 and ≤100 | | | | | |
| | >100 | | | | | |
| | Onset ≤48h | | | | | |
| | Medical advice | | | | | |
| Swelling (mm) | All | | | | | |
| | >20 and ≤50 | | | | | |
| | >50 and ≤100 | | | | | |
| | >100 | | | | | |
| | Onset ≤48h | | | | | |
| | Medical advice | | | | | |

#### <each group>:

30 PreF = 30 μg PreF

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

Type=Max grade & onset

All=any severity >Grade 0 for pain and any diameter >20mm for redness and swelling

N=number of vaccinated subjects who returned the diary card

n/% = number/percentage of subjects reporting the AE at least once. Maximum intensity only

95%CI = Exact 95% confidence interval; LL = lower limit, UL = upper limit

The maximum intensity of local injection site redness/swelling was coded as follows for adults:

0: ≤ 20 mm

1:  $> 20 \text{ mm to} \le 50 \text{ mm}$ 

 $2: > 50 \text{ mm to} \le 100 \text{ mm}$ 

3: > 100 mm

204812 (RSV F-021)

Statistical Analysis Plan Amendment 4 Final

### Template 20 Incidence of solicited general symptoms reported during the 7-day (Days 0-6) post-vaccination period (Exposed set)

| | | | | <each gi<="" th=""><th>roup&gt;</th><th></th></each> | roup> | |
|---|---|---|---|---|---|---|
| | | | | | 9: | 5 % CI |
| Symptom | Туре | N | n | % | LL | UL |
| Fatigue | All | | | | | |
| - | Grade 1 | | | | | |
| | Grade 2 | | | | | |
| | Grade 3 | | | | | |
| | Related | | | | | |
| | Grade 2 Related | | | | | |
| | Grade 3 Related | | | | | |
| | Onset ≤48h | | | | | |
| | Medical advice | | | | | |
| Temperature (Oral)<br>(°C) | All (≥37.5) | | | | | |
| ( ) | >38.0 | | | | | |
| | >38.5 | | | | | |
| | >39.0 | | | | | |
| | >39.5 | | | | | |
| | Related | | | | | |
| | >38.5 Related | | | | | |
| | >39.5 Related | | | | | |
| | Onset ≤48h | | | | | |
| | Medical advice | | | | | |
| Gastrointestinal | All | | | | | |
| symptoms | Grade 1 | | | | | |
| -, | Grade 2 | | | | | |
| | Grade 3 | | | | | |
| | Related | | | | | |
| | Grade 2 Related | | | | | |
| | Grade 3 Related | | | | | |
| | Onset ≤48h | | | | | |
| | Medical advice | | | | | |
| Headache | All | | | | | |
| | Grade 1 | | | | | |
| | Grade 2 | | | | | |
| | Grade 3 | | | | | |
| | Related | | | | | |
| | Grade 2 Related | | | | | |
| | Grade 3 Related | | | | | |
| | Onset ≤48h | | | | | |
| | Medical advice | | | | | |

#### <each group>:

30 PreF = 30 μg PreF

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF =120 µg PreF

Control = Placebo

N = number of subjects with the documented dose

n/% = number/percentage of subjects reporting the symptom at least once 95%CI = Exact 95% confidence interval; LL = lower limit, UL = upper limit

Temperatures were coded as follows for adults:

0: < 37.5 °C

1:  $\geq 37.5 \,^{\circ}\text{C} \text{ to} \leq 38.5 \,^{\circ}\text{C}$ 

2: > 38.5 °C to  $\le 39.5$  °C

3: > 39.5°C

204812 (RSV F-021)

Statistical Analysis Plan Amendment 4 Final

## Template 21 Incidence of solicited general symptoms reported during the 7-day (Days 0-6) post-vaccination period by maximum intensity (Exposed set)

| | | | < | each gro | oup> | |
|-------------------|-----------------|---|---|----------|------|--------|
| | | | | | | 5 % CI |
| Symptom | Туре | N | n | % | LL | UL |
| Fatigue | All | | | | | |
| · · | Grade 1 | | | | | |
| | Grade 2 | | | | | |
| | Grade 3 | | | | | |
| | Related* | | | | | |
| | Grade 2 Related | | | | | |
| | Grade 3 Related | | | | | |
| | Onset ≤48h | | | | | |
| | Medical advice | | | | | |
| Gastrointestinal | All | | | | | |
| symptoms | | | | | | |
| • | Grade 1 | | | | | |
| | Grade 2 | | | | | |
| | Grade 3 | | | | | |
| | Related* | | | | | |
| | Grade 2 Related | | | | | |
| | Grade 3 Related | | | | | |
| | Onset ≤48h | | | | | |
| | Medical advice | | | | | |
| Headache | All | | | | | |
| | Grade 1 | | | | | |
| | Grade 2 | | | | | |
| | Grade 3 | | | | | |
| | Related* | | | | | |
| | Grade 2 Related | | | | | |
| | Grade 3 Related | | | | | |
| | Onset ≤48h | | | | | |
| | Medical advice | | | | | |
| Fever/(Oral) (°C) | All | | | | | |
| , , , , | >38.0 | | | | | |
| | >38.5 | | | | | |
| | >39.0 | | | | | |
| | >39.5 | | | | | |
| | Related* | | | | | |
| | >38.5 Related | | | | | |
| | >39.5 Related | | | | | |
| | Medical advice | | | | | |

#### <each group>:

 $30 \text{ PreF} = 30 \mu \text{g PreF}$ 

60 PreF = 60 µg PreF

120 PreF = 120 µg PreF

Control = Placebo

 $All = any\ grade > 0\ for\ Fatigue,\ Gastrointestinal\ symptoms,\ Headache\ and\ any\ > 37.5^{\circ}C\ for\ Temperature/(Oral)$ 

Related\*= any grade>0 for Fatigue, Gastrointestinal symptoms, Headache and any >37.5°C for Temperature/(Oral) considered related to vaccination by the investigator

N=number of vaccinated subjects who returned the diary card

n/% = number/percentage of subjects reporting the AE at least once. Maximum intensity only

95%CI = Exact 95% confidence interval; LL = lower limit, UL = upper limit

Temperatures were coded as follows for adults:

204812 (RSV F-021) Statistical Analysis Plan Amendment 4 Final

0: < 37.5 °C

1: ≥ 37.5 °C to ≤ 38.5 °C

2: > 38.5 °C to ≤ 39.5°C

3: > 39.5°C

204812 (RSV F-021)

Statistical Analysis Plan Amendment 4 Final

# Template 22 Percentage of subjects reporting the occurrence of unsolicited symptoms classified by MedDRA Primary System Organ Class and Preferred Term within the 30-day (Days 0-29) post-vaccination period (Exposed set)

| | | | <eac< th=""><th>h group<br/>N =</th><th>&gt;</th></eac<> | h group<br>N = | > |
|---|---|---|---|---|---|
| | | | | 95% | CI |
| Primary System Organ Class (CODE) | Preferred Term (CODE) | n | % | LL | UL |
| At least one symptom | | | | | |
| <each (code)="" soc=""></each> | <each (code)="" pt=""></each> | | | | |

#### <each group>:

 $30 \text{ PreF} = 30 \mu \text{g PreF}$ 

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

At least one symptom = at least one symptom experienced (regardless of the MedDRA Preferred Term)

N = number of subjects with at least one administered dose

n/% = number/percentage of subjects reporting at least once the symptom

95% CI= exact 95% confidence interval; LL = Lower Limit, UL = Upper Limit

Template 23 Percentage of subjects reporting the occurrence of unsolicited symptoms classified by MedDRA Primary System Organ Class and Preferred Term within the 30-day (Days 0-29) post-vaccination period (Exposed set)

| | | <ea< th=""><th>ch group&gt;<br/>N =</th></ea<> | ch group><br>N = |
|---|---|---|---|
| Primary System Organ Class (CODE) | Preferred Term (CODE) | n | % |
| At least one symptom | | | |
| <each (code)="" soc=""></each> | <each (code)="" pt=""></each> | | |

#### <each group>:

 $30 \text{ PreF} = 30 \mu \text{g PreF}$ 

60 PreF = 60 µg PreF

120 PreF = 120 μg PreF

Control = Placebo

At least one symptom = at least one symptom experienced (regardless of the MedDRA Preferred Term)

N = number of subjects with at least one administered dose

n/% = number/percentage of subjects reporting at least once the symptom

Note: It is the simplified version of Template 22 without UL and LL added for final analysis

204812 (RSV F-021) Statistical Analysis Plan Amendment 4 Final

#### Template 24 Listing of SAEs reported up to study end (Exposed set)

| Group | Sub.<br>No. | Sex | Country | Race | Age at onset (Year) | Verbatim | Preferred<br>term | Primary<br>System<br>Organ<br>Class | MED<br>type | Dose | Day of onset | Duration | Intensity | Causality | Outcome |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| <each< td=""><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td></each<> | | | | | | | | | | | | | | | |
| group> | | | | | | | | | | | | | | | |

#### <each group>:

30 PreF = 30 μg PreF 60 PreF = 60 μg PreF 120 PreF = 120 μg PreF Control = Placebo

01-JUN-2018 Page 70 of 103

204812 (RSV F-021)

Statistical Analysis Plan Amendment 4 Final

### Template 25 Number (%) of subjects with serious adverse events up to study end (Exposed set)

| | | | <each group=""><br/>N =</each> | | |
|---|---|---|---|---|---|
| Type of Event | Primary System Organ Class | Preferred Term (CODE) | n* | n | % |
| SAE | At least one symptom | | | | |
| | <each soc=""></each> | <each pt="" term=""></each> | | | |
| Related SAE | At least one symptom | | | | |
| | <each soc=""></each> | <each pt="" term=""></each> | | | |
| Fatal SAE | At least one symptom | | | | |
| | <each soc=""></each> | <each pt="" term=""></each> | | | |
| Related fatal SAE | At least one symptom | | | | |
| | <each soc=""></each> | <each pt="" term=""></each> | | | |

#### <each group>:

 $30 \text{ PreF} = 30 \mu \text{g PreF}$ 

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

N = number of subjects with the administered dose

n\* = number of events reported

n/% = number/percentage of subjects reporting the symptom at least once

#### Template 26 Compliance in returning symptom information (Exposed set)

| Group | Number | Doses | Number | Compliance | Number | Compliance |
|---|---|---|---|---|---|---|
| | of | NOT | of | % | of | % |
| | doses | according to | general SS | general SS | local SS | local SS |
| | | protocol | | | | |
| <each group=""></each> | | | | | | |

#### <each group>:

 $30 \text{ PreF} = 30 \mu \text{g PreF}$ 

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

SS = Symptom screens/sheets used for the collection of local and general solicited AEs

Compliance % = (number of doses with symptom screen/sheet return / number of administered doses) X 100

204812 (RSV F-021)

Statistical Analysis Plan Amendment 4 Final

## Template 27 Number and percentage of subjects taking a concomitant medication during the 7- day (Days 0-6) post -vaccination period (Exposed set)

| | <each group=""></each> | | | | |
|---|---|---|---|---|---|
| | | | 95% | CI | |
| | N | n | % | LL | UL |
| Any | | | | | |
| Any antipyretics | | | | | |
| Prophylactic antipyretics | | | | | |

#### <each group>:

30 PreF = 30 µg PreF

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

N= number of administered doses

n/%= number/percentage of subjects who took the specified concomitant medication at least once during the mentioned period

95% CI = exact 95% confidence interval, LL = Lower Limit, UL = Upper Limit

# Template 28 Exploratory comparisons between groups in terms of percentage of subjects reported any Grade 2/3 AE and/or any fever >38.5°C and/or any vaccine-related SAE during the 7-day (Days 0-6) post-vaccination period (Exposed set)

| | | | | | | | | Difference in<br>(Group 1 min | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | | 95 | % CI |
| Group 1 | N | n | % | Group 2 | N | n | % | Difference | % | LL | UL |
| 30 PreF | | | | Control | | | | 30 PreF - Control | | | |
| 60 PreF | | | | Control | | | | 60 PreF - Control | | | |
| 120 PreF | | | | Control | | | | 120 PreF - Control | | | |
| 60 PreF | | | | 30 PreF | | | | 60 PreF - 30 PreF | | | |
| 120 PreF | | | | 30 PreF | | | | 120 PreF - 30 PreF | | | |
| 120 PreF | | | | 60 PreF | | | | 120 PreF - 60 PreF | | | |

#### <each group>:

30 PreF = 30 µg PreF

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 μg PreF

Control = Placebo

N = Number of subjects with the administered dose

n/% = number/percentage of subjects reporting a specified symptom

95% CI = Standardized asymptotic 95% confidence interval, LL = Lower Limit, UL = Upper Limit

204812 (RSV F-021)

Statistical Analysis Plan Amendment 4 Final

# Template 29 Solicited and unsolicited symptoms experienced by at least 5 % of subjects, classified by MedDRA Primary System Organ Class and Preferred Term within the 30-day (Days 0-29) post-vaccination period including number of events - SAE excluded (Exposed set)

| | | <e< th=""><th>ach gi<br/>N =</th><th></th></e<> | ach gi<br>N = | |
|---|---|---|---|---|
| Primary System<br>Organ Class<br>(CODE) | Preferred Term<br>(CODE) | n* | n | % |
| At least one symptom | | | | |
| <each soc=""></each> | <each pt="" term=""></each> | | | |

#### <each group>:

30 PreF = 30 µg PreF

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

At least one symptom = at least one symptom experienced (regardless of the MedDRA Preferred Term)

N = number of subjects with the administered dose

n\* = number of events reported

n/% = number/percentage of subjects reporting the symptom at least once

Template 30 Distribution of change from baseline in haematology and biochemistry with respect to normal laboratory ranges (Exposed set)

| | | | | | <e< th=""><th>ac</th><th>h gro</th><th>ир</th><th>&gt;</th><th></th><th></th></e<> | ac | h gro | ир | > | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | Ur | known | В | elow | W | ithin | Α | bove |
| Laboratory parameter | Timing | Baseline PRE(D0) | N | | % | | | | % | | % |
| Alanine Aminotransferase | PI(D7) | Unknown | | | | | | | | | |
| (ALT) | , , | Below | | | | | | | | | |
| , | | Within | | | | | | | | | |
| | | Above | | | | | | | | | |
| | PI(D30) | | | | | | | | | | |
| | PI(D60) | | | | | | | | | | |
| | PI(D90) | | | | | | | | | | |
| Aspartate Aminotransferase | PI(D7) | Unknown | | | | | | | | | |
| (AST) | | Below | | | | | | | | | |
| | | Within | | | | | | | | | |
| | | Above | | | | | | | | | |
| | PI(D30) | | | | | | | | | | |
| | PI(D60) | | | | | | | | | | |
| | PI(D90) | | | | | | | | | | |
| Creatinine | | | | | | | | | | | |
| Eosinophils | | | | | | | | | | | |
| Haemoglobin | | | | | | | | | | | |
| Lymphocytes | | | | | | | | | | | |
| Neutrophils | | | | | | | | | | | |
| Platelet count | | | | | | | | | | | |
| White Blood Cells (WBC) | | | | | | | | | | | - |

#### <each group>:

30 PreF = 30 μg PreF

60 PreF = 60 µg PreF

120 PreF = 120 µg PreF

Control = Placebo

204812 (RSV F-021)

Statistical Analysis Plan Amendment 4 Final

N = number of subjects with available results for the specified laboratory parameter and timing in a given baseline category

n/% = number/percentage of subjects in the specified category

Below = below the normal laboratory range defined for the specified laboratory parameter

Within = within the normal laboratory range defined for the specified laboratory parameter

Above = above the normal laboratory range defined for the specified laboratory parameter

PI(D7) = Post-vaccination at Day 7

PI(D30) = Post-vaccination at Day 30

PI(D60) = Post-vaccination at Day 60

PI(D90) = Post-vaccination at Day 90

Note: For the final analysis, three newly added in-text tables of 'Distribution of change from baseline in ALT, AST and Eosinophil's with respect to normal laboratory ranges (Exposed set)', 'Distribution of change from baseline in Creatinine, Lymphocytes and White Blood Cells (WBC) with respect to normal laboratory ranges (Exposed set)' and 'Distribution of change from baseline in Hemoglobin, Neutrophils and Platelet count with respect to normal laboratory ranges (Exposed set)' will use Template 30.

204812 (RSV F-021)

Statistical Analysis Plan Amendment 4 Final

## Template 31 Summary of haematology and biochemistry results by maximum grade from VISIT 2 (D7) up to VISIT 3 (D30) versus baseline (Exposed set)

| | | | | | VIS | | (D7) u<br><eac< th=""><th></th><th></th><th></th><th>30)</th><th></th><th></th><th></th></eac<> | | | | 30) | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | Hakı | nown | Cro | | | | | | Cro | de 3 | Cro | do 1 |
| | I= | | | | | | | | | | | | | |
| Laboratory parameter | Baseline PRE(D0) | N | n | % | n | % | n | % | n | % | n | % | n | % |
| Alanine Aminotransferase (ALT) increase by factor | Unknown | | | | | | | | | | | | | |
| • | Grade 0 | | | | | | | | | | | | | |
| | Grade 1 | | | | | | | | | | | | | |
| | Grade 2 | | | | | | | | | | | | | |
| | Grade 3 | | | | | | | | | | | | | |
| | Grade 4 | | | | | | | | | | | | | |
| | Total | | | | | | | | | | | | | |
| Aspartate Aminotransferase (AST) increase by factor | | | | | | | | | | | | | | |
| Creatinine | | | | | | | | | | | | | | |
| Eosinophils increase | | | | | | | | | | | | | | |
| Hemoglobin decrease | | | | | | | | | | | | | | |
| Lymphocytes decrease | | | | | | | | | | | | | | |
| Neutrophils decrease | | | | | | | | | | | | | | |
| Platelet count decrease | | | | | | | | | | | | | | |
| White Blood Cells (WBC) decrease | | | | | | | | | | | | | | |
| White Blood Cells (WBC) increase | | | | | | | | | | | | | | |

#### <each group>:

 $30 \text{ PreF} = 30 \mu \text{g PreF}$ 

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

N = number of subjects with at least one available result for the specified laboratory parameter and follow-up period n/% = number/percentage of patients reporting at least once the laboratory event when the maximum grading over the follow-up period is considered

ALT/AST increase by factor: Grade 1 is 1.1-2.5xULN, Grade 2 is 2.6-5.0xULN, Grade 3 is 5.1-10xULN, Grade 4 is >10ULN; ULN is upper limit of the normal range.

204812 (RSV F-021)

Statistical Analysis Plan Amendment 4 Final

## Template 32 Summary of haematology and biochemistry results by maximum grade in the specified category from VISIT 2 (D7) up to VISIT 3 (D30) (Exposed set)

| | | <ea< th=""><th>ch group &gt;<br/>N =</th></ea<> | ch group ><br>N = |
|---|---|---|---|
| Laboratory parameter | Maximum grade | n | % |
| Alanine Aminotransferase(ALT) increase by factor | Other | | |
| , , | Grade 2 | | |
| | Grade 3 | | |
| | Grade 4 | | |
| Aspartate Aminotransferase(AST) increase by factor | Other | | |
| | Grade 2 | | |
| | Grade 3 | | |
| | Grade 4 | | |
| Creatinine | Other | | |
| | Grade 2 | | |
| | Grade 3 | | |
| | Grade 4 | | |
| Eosinophils increase | Other | | |
| • | Grade 2 | | |
| | Grade 3 | | |
| | Grade 4 | | |
| Hemoglobin decrease | Other | | |
| <b>G</b> | Grade 2 | | |
| | Grade 3 | | |
| | Grade 4 | | |
| Lymphocytes decrease | Other | | |
| | Grade 2 | | |
| | Grade 3 | | |
| | Grade 4 | | |
| Neutrophils decrease | Other | | |
| | Grade 2 | | |
| | Grade 3 | | |
| | Grade 4 | | |
| Platelet count decrease | Other | | |
| | Grade 2 | | |
| | Grade 3 | | |
| | Grade 4 | | |
| White Blood Cells (WBC) decrease | Other | | |
| 2.000 00.10 (1.20) 00010000 | Grade 2 | | |
| | Grade 3 | | |
| | Grade 4 | | |
| White Blood Cells (WBC) increase | Other | | |
| Times 2.300 come (1120) moreuse | Grade 2 | | |
| | Grade 3 | | |
| | Grade 4 | | |

<each group>:

30 PreF = 30 μg PreF

60 PreF = 60 μg PreF

120 PreF = 120 μg PreF

Control = Placebo

*N* = number of subjects with the administered dose

n = number of subjects in the specified category

% = n / Number of subjects with available results x 100

Other=all Unknown, Grade 0 and Grade 1

204812 (RSV F-021)

Statistical Analysis Plan Amendment 4 Final

ALT/AST increase by factor: Grade 1 is 1.1-2.5xULN, Grade 2 is 2.6-5.0xULN, Grade 3 is 5.1-10xULN, Grade 4 is >10ULN; ULN is upper limit of the normal range.

### Template 33 Summary of haematology change from baseline by maximum grade from VISIT2 (D7) up to VISIT3 (D30) (Exposed set)

| | | | | VIS | IT2 ( | D7) u | p to | VISI | T3 (D | 30) | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | <each group=""></each> | | | | | | | | | | | | |
| | | Unkr | nown | Grad | de 0 | Grad | de 1 | Gra | de 2 | Grade 3 | | Grade 4 | |
| Laboratory parameter | N | N n % n % n | | | | n | % | n | % | n | % | n | % |
| Hemoglobin (Change from baseline) | | | | | | | | | | | | | |

#### <each group>:

 $30 \text{ PreF} = 30 \mu \text{g PreF}$ 

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 μg PreF

Control = Placebo

N = number of subjects with at least one available result for the specified laboratory parameter and follow-up period n/% = number/percentage of subjects reporting at least once the laboratory event when the maximum grading over the follow-up period is considered

Hemoglobin (Female) change from baseline value (gm/dL): Grade 1 is any decrease-1.5, Grade 2 is 1.6-2.0, Grade 3 is 2.1-5.0 and Grade 4 is >5.0.

204812 (RSV F-021)

Statistical Analysis Plan Amendment 4 Final

## Template 34 Summary of haematology change from baseline by maximum grade in the specified category from VISIT2 (D7) up to VISIT3 (D30) (Exposed set)

| | | <eac< th=""><th>ch group &gt;<br/>N =</th></eac<> | ch group ><br>N = |
|---|---|---|---|
| Laboratory parameter | Maximum grade | n | % |
| Hemoglobin (Change from baseline) | Other | | |
| , | Grade 2 | | |
| | Grade 3 | | |
| | Grade 4 | | |

<each group>:

30 PreF = 30 μg PreF

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 μg PreF

Control = Placebo

N = number of subjects with the administered dose

n= number of subjects in the specified category

% = n / Number of subjects with available results x 100

Other=all Unknown, Grade 0 and Grade 1

 $Hemoglobin \ (Female) \ change \ from \ baseline \ value \ (gm/dL): \ Grade \ 1 \ is \ any \ decrease -1.5, \ Grade \ 2 \ is \ 1.6-2.0,$ 

Grade 3 is 2.1-5.0 and Grade 4 is >5.0.

204812 (RSV F-021)

Statistical Analysis Plan Amendment 4 Final





**Note:** This figure is shown as an example. For the unblinded report, one figure per group will be performed. For the blinded report, 4 graphs will be performed each of them presenting probable subjects regardless of treatment (the first probable subjects, from the probable the subject...). The X axis will include Day 0, Day 7 and Day 30. The Y axis will be adapted according to each parameter.

204812 (RSV F-021)

Statistical Analysis Plan Amendment 4 Final

## Template 36 Number and percentage of subjects with anti-RSV-A neutralising antibody titer equal to or above <cut-off> and GMTs (Per protocol set)

| | | | | | ≥cı | ıt-off | | | GMT | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | 959 | % CI | | 95% CI | | | |
| Antibody | Group | Timing | N | n | % | LL | UL | value | LL | UL | Min | Max |
| Anti-RSV-A | <each< td=""><td>PRE</td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td></each<> | PRE | | | | | | | | | | |
| Neutralizing<br>Antibody | group> | | | | | | | | | | | |
| , | | PI(D30) | | | | | | | | | | |
| | | PI(D60) | | | | | | | | | | |
| | | PI(D90) | | | | | | | | | | |

#### <each group>:

 $30 \text{ PreF} = 30 \mu \text{g PreF}$ 

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

GMT = geometric mean antibody titer calculated on all subjects

N = Number of subjects with available results

95% CI = 95% confidence interval; LL = lower limit, UL = upper limit

n/% = number/percentage of subjects with titer equal to or above specified value

MIN/MAX = Minimum/Maximum

PRE= Pre-vaccination at Day 0

PI(D30) = Post-vaccination at Day 30

PI(D60) = Post-vaccination at Day 60

204812 (RSV F-021)

Statistical Analysis Plan Amendment 4 Final

## Template 37 Number and percentage of subjects with anti-RSV-A neutralising antibody titer equal to or above <cut-off> and GMTs - by age category (Per protocol set)

| | | | | | | ≥cı | ıt-off | | GMT | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | 95% CI | | | 95 | % CI | | |
| Antibody | Group | Sub-<br>Group | Timing | N | n | % | LL | UL | value | LL | UL | Min | Max |
| Anti-RSV-A<br>Neutralizing<br>Antibody | <each<br>group&gt;</each<br> | 18-32Y | PRE PI(D30) PI(D60) PI(D90) | | | | | | | | | | |
| | | 33-45Y | PRE<br>PI(D30)<br>PI(D60) | | | | | | | | | | |
| | | | PI(D90) | | | | | | | | | | |

#### <each group>:

 $30 \text{ PreF} = 30 \mu \text{g PreF}$ 

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

18-32Y = 18-32 years old subjects

33-45Y = 33-45 years old subjects

GMT = geometric mean antibody titer calculated on all subjects

N = Number of subjects with available results

95% CI = 95% confidence interval; LL = lower limit, UL = upper limit

n/% = number/percentage of subjects with titer equal to or above specified value

MIN/MAX = Minimum/Maximum

PRE= Pre-vaccination at Day 0

PI(D30) = Post-vaccination at Day 30

PI(D60) = Post-vaccination at Day 60

204812 (RSV F-021)

Statistical Analysis Plan Amendment 4 Final

## Template 38 Geometric mean of the individual ratio of anti-RSV-A neutralising antibody titers at each post-vaccination timepoint compared to prevaccination with 95% CI (Per protocol set)

| | | | | | GMT ratio | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | 9 | 5% CI |
| Group | N | Time point description | GMT | Time point description | GMT | Ratio order | Value | LL | UL |
| <each group=""></each> | | PI(D30) | | PRE | | PI(D30) / PRE | | | |
| | | PI(D60) | | PRE | | PI(D60) / PRE | | | |
| | | PI(D90) | | PRE | | PI(D90) / PRE | | | |

#### <each group>:

 $30 \text{ PreF} = 30 \mu \text{g PreF}$ 

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 μg PreF

Control = Placebo

GMT = geometric mean antibody titer

N = Number of subjects with available results at the two considered time points

95% CI = 95% confidence interval; LL = Lower Limit, UL = Upper Limit

PRE= Pre-vaccination at Day 0

PI(D30) = Post-vaccination at Day 30

PI(D60) = Post-vaccination at Day 60

Statistical Analysis Plan Amendment 4 Final

Template 39 GMTs and their 95% Cls for anti-RSV-A neutralising antibody at each timepoint (Per protocol set)



 $30 \text{ PreF} = 30 \mu \text{g PreF}$ 

60 PreF = 60 µg PreF

120 PreF = 120 µg PreF

Control = Placebo

GMT = geometric mean antibody titer calculated on all subjects

95% CI = 95% confidence interval

Note: This graph is provided as an example. For each assay separately, this graph will display the 4 groups and the 4 immuno timepoints: PRE, PI(D30), PI(D60) and PI(D90)

Statistical Analysis Plan Amendment 4 Final

### Template 40 Kinetics of GMTs for anti-RSV-A neutralising antibody on subjects with results available at all timepoints (Per protocol set)



30 PreF = 30 µg PreF 60 PreF = 60 µg PreF 120 PreF = 120 µg PreF Control = Placebo

GMT = geometric mean antibody titer calculated on subjects with results available at all timepoints **Note:** 

- This graph is provided as an example. For each assay separately, this graph will display the 4 groups and the 4 immuno timepoints PRE, PI(D30), PI(D60) and PI(D90)
- For the kinetic of the estimated GMTs, footnote will be adapted as: GMT = geometric mean antibody titer estimated by the ANOVA model for repeated measures

204812 (RSV F-021)

Statistical Analysis Plan Amendment 4 Final

#### Template 41 Distribution of anti-Neogenin antibody concentration (Exposed set)

| | | | | | <55<br>g/ml | ≥55<br>ng/ml | | ≥100<br>ng/ml | | | 150<br>g/ml | | 200<br>g/ml | | 250<br>g/ml | | 300<br>g/ml |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Antibody | Group | Timing | N | n % | | n | % | n | % | n | % | n | % | n | % | n | % |
| Anti-neogenin antibody | <each<br>group&gt;</each<br> | PRE | | | | | | | | | | | | | | | |
| - | | PI(D30) | | | | | | | | | | | | | | | |
| | | PI(D60) | | | | | | | | | | | | | | | |
| | | PI(D90) | | | | | | | | | | | | | | | |

#### <each group>:

 $30 \text{ PreF} = 30 \mu \text{g PreF}$ 

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

N = number of subjects with available results

n/% = number/percentage of subjects with concentration within the specified range

PRE = Pre-vaccination at Day 0

PI(D30) = Post-vaccination at Day 30

PI(D60) = Post-vaccination at Day 60

PI(D90) = Post-vaccination at Day 90

### Template 42 Distribution of fold of anti-neogenin antibody concentration (Exposed set)

| | | | | < | <1 | | >=1 | | >=1.5 | | >=2 | | 2.5 | >=3 | | >=3.5 | | >=4 | | >=4.5 | | >: | =5 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Antibody | Group | Timing | N | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Anti-neogenin antibody | <each group=""></each> | PI(D30) | | | | | | | | | | | | | | | | | | | | | |
| • | | PI(D60) | | | | | | | | | | | | | | | | | | | | | |
| | | PI(D90) | | | | | | | | | | | | | | | | | | | | | |

#### <each group>:

 $30 \text{ PreF} = 30 \mu \text{g PreF}$ 

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

N = number of subjects with available results

n/% = number/percentage of subjects with concentration within the specified range

PI(D30) = Post-vaccination at Day 30

PI(D60) = Post-vaccination at Day 60

204812 (RSV F-021)

Statistical Analysis Plan Amendment 4 Final

## Template 43 Distribution of anti-RSV-A neutralising antibody titer (Per protocol set)

| | | | | <7<br>og2 | ≥7<br>Log2 | | ≥8<br>Log2 | | ≥9<br>Log2 | | | 10 ≥11<br>og2 Log | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Antibody | Group | Timing | Timing N r | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Anti-RSV A Neutralizing Antibody | <each group=""></each> | PRE | | | | | | | | | | | | | | |
| | | PI(D30) | | | | | | | | | | | | | | |
| | | PI(D60) | | | | | | | | | | | | | | |
| | | PI(D90) | | | | | | | | | | | | | | |

#### <each group>:

30 PreF = 30 μg PreF

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

N = number of subjects with available results

n/% = number/percentage of subjects with titre within the specified range

PRE = Pre-vaccination at Day 0

PI(D30) = Post-vaccination at Day 30

PI(D60) = Post-vaccination at Day 60
204812 (RSV F-021) Statistical Analysis Plan Amendment 4 Final

## Template 44 Distribution of fold of anti-RSV-A neutralising antibody titer by pre-vaccination titer category (Per protocol set)

| A (!! ! | | | - · | | <1 | | ≥1 | , | 22 | ≥ | 2.5 | 2 | 3 | ≥4 | 4 | ≥6 | <u> </u> | <b>∠</b> ୪ | 2 | IU | 21 | 1 | 21 | 2 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Antibody | Group | Sub-group | Timing | N | n S | % I | n የ | / <sub>0</sub> | n 🏸 | n | % | n | % | 'n | % | n % | r | ۱ % | n | % | n ' | % | n ' | % |
| Anti-RSV A Neutralizing | 30 PreF | <7 | PI (D30) | | | | | | | | | | | | | | | | | | | | Ш | |
| Antibody | | | PI (D60) | | | | | | | | | | | | | | | | | | | | Ш | |
| | | | PI (D90) | | | | | | | | | | | | | | | | | | | | Ш | _ |
| | | [7-8] | PI (D30) | | | | | | | | | | | | | | | | | | | | Ш | |
| | | | PI (D60) | | | | | | | | | | | | | | | | | | | | Ш | |
| | | | PI (D90) | | | | | | | | | | | | | | | | | | | | Ш | |
| | | ]8-9] | PI (D30) | | | | | | | | | | | | | | | | | | | | Ш | |
| | | | PI (D60) | | | | | | | | | | | | | | | | | | | | lacksquare | |
| | | 10.401 | PI (D90) | | | | | | | | | | | | | | | | | | | | $\vdash$ | |
| | | ]9-10] | PI (D30) | | | | | | | | | | | | | | | | | | | | $\vdash$ | |
| | | | PI (D60) | | | | | | | | | | | | | | | | | | | | H | |
| | | 140 441 | PI (D90) | | | | | | | | | | | | | | | | | | | | lacksquare | _ |
| | | ]10-11] | PI (D30) | | | | | | | | | | | | | | | | | | | | H | |
| | | | PI (D60) | | | | | | | | | | | | | | | | | | | | H | |
| | | 144 401 | PI (D90) | | | | | | | | | | | | | | | | | | | | H | |
| | | ]11-12] | PI (D30) | | | | | | | | | | | | | | | | | | | | $\vdash$ | |
| | | | PI (D60) | | | | | | | | | | | | | | | | | | | | $\vdash$ | |
| | | . 40 | PI (D90) | | | | | | | | | | | | | | | | | | | | H | |
| | | > 12 | PI (D30) | | | | | | | | | | | | | | | | | | | | H | |
| | | | PI (D60)<br>PI (D90) | | | | | | | | | | | | | | | | | | | | H | |
| | | Tatal | | | | | | | | | | | | | | | | | | | | | H | |
| | | Total | PI (D30) | | | | | | | | | | | | | | | | | | | | H | |
| | | | PI (D60) | | | | | | | | | | | | | | | | | | | | H | |
| | 60 D==E | 47 | PI (D90)<br>PI (D30) | | | | | | | | | | | | | | | - | | | | | H | |
| | 60 PreF | <7 | PI (D30) | | | | | | | | | | | | | | | - | | | | | H | |
| | | | | | | | | | | | | | | | | | | - | | | | | H | |
| | | [7 0] | PI (D90) | | | | | | | | | | | | | | | | | | | | H | |
| | | [7-8] | PI (D30) | | | | | | | | | | | | | | | | | | | | H | |
| | | | PI (D60) | | | | | | | | | | | | | | | - | | | | | H | |
| | | 10.01 | PI (D90) | | | | | | | | | | | | | | | - | | | | | H | |
| | | ]8-9] | PI (D30)<br>PI (D60) | | | | | | | | | | | | | | | - | | | | | H | |
| | | | | | | | | | | | | | | | | | | | | | | | H | |
| | | 10.401 | PI (D90) | | | | | | | | | | | | | | | | | | | | H | |
| | | ]9-10] | PI (D30) | | | | | | | | | | | | | | | - | | | | | H | |
| | | | PI (D60) | | | | | | | | | | | | | | | | | | | | $\vdash$ | |
| | | 140 441 | PI (D90)<br>PI (D30) | | + | | | | | | | | | | | | | | | | | | H | |
| | | ]10-11] | PI (D30) | | + | | | | | | | | | | | | | | | | | | H | _ |
| | | | PI (D00) | | + | | | | | | | | | | | | | | | | | | H | _ |
| | | 144 401 | PI (D30) | | | | | | | | | | | | | | | | | | | | $\vdash$ | |
| | | ]11-12] | PI (D30) | | | | | | | | | | | | | | | | | | | | $\vdash$ | |
| | | | PI (D00) | | + | | | | | | | | | | | | | | | | | | H | _ |
| | | > 12 | PI (D90) | $\vdash$ | + | - | | + | + | | | | | $\dashv$ | | | - | + | - | | H | | H | |
| | | <i>&gt;</i> 12 | PI (D30) | H | + | - | | + | + | 1 | | | | $\dashv$ | | | + | - | - | 1 | $\vdash$ | | $\vdash$ | |
| | | | PI (D00) | $\vdash$ | + | - | - | - | + | | | | | - | | | + | + | | - | H | | H | |
| | | Total | PI (D90) | H | + | - | | + | + | 1 | | | | $\dashv$ | | | + | - | - | 1 | $\vdash$ | | $\vdash$ | |
| | | Total | PI (D30) | $\vdash$ | + | - | + | + | + | + | | | | - | | | + | + | | - | | | H | |
| | | | PI (D60) | | $\perp$ | - | | | $\perp$ | | | | | - | | | | + | - | | | | $\vdash$ | |

## 204812 (RSV F-021)

Statistical Analysis Plan Amendment 4 Final

| | | | | | < | 1 | ≥ | 1 | ≥: | 2 | ≥2 | .5 | ≥3 | | ≥4 | 1 | ≥6 | ≥ | ≥8 | ≥ | 10 | ≥′ | 11 | ≥′ |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Antibody | Group | Sub-group | Timing | N | | | | | | | | | n % | | | | | | | | | | | |
| | 120 PreF | <7 | PI (D30) | | | - | | - | | | | | | + | | | Ť | | | | | T | | |
| | 120 1 101 | • | PI (D60) | | | | | | | | 1 | | | | | | | t | | | | H | | r |
| | | | PI (D90) | | | | | | | | | | | $^{+}$ | | | | + | | | | H | | H |
| | | [7-8] | PI (D30) | | | | | | | | | | | | | | | | | | | H | | |
| | | [1-0] | PI (D60) | | | | | | | | | | | | | | | | | | | ╁ | | H |
| | | | PI (D00) | | _ | | | | | | | | | + | | - | | - | | | | ╁ | <u> </u> | ⊨ |
| | | 10.01 | | | | | | | | | | | | _ | | - | - | | | | | ₩ | | L |
| | | ]8-9] | PI (D30) | | | | | | | | | | | + | | - | | | | | | ╄ | _ | L |
| | | | PI (D60) | | | | | | | | | | | | | | | | | | | ╄ | | L |
| | | | PI (D90) | | | | | | | | | | | | | | | | | | | L | | L |
| | | ]9-10] | PI (D30) | | | | | | | | | | | | | | | | | | | L | | L |
| | | | PI (D60) | | | | | | | | | | | | | | | | | | | L | | L |
| | | | PI (D90) | | | | | | | | | | | | | | | | | | | L | L | L |
| | | ]10-11] | PI (D30) | | | | | | | | | | | | | | | | | | | L | | L |
| | | | PI (D60) | | | | | | | | | | | | | | | | | | | L | | L |
| | | | PI (D90) | | | | | | | | | | | | | | | | | | | | | |
| | | ]11-12] | PI (D30) | | | | | | | | | | | | | | | | | | | | | |
| | | | PI (D60) | | | | | | | | | | | | | | | | | | | | | |
| | | | PI (D90) | | | | | | | | | | | | | | | | | | | | | |
| | | > 12 | PI (D30) | | | | | | | | | | | | | | | | | | | | | |
| | | | PI (D60) | | | | | | | | | | | | | | | | | | | | | |
| | | | PI (D90) | | | | | | | | | | | | | | | | | | | T | | |
| | | Total | PI (D30) | | | | | | | | | | | | | | | | | | | T | | T |
| | | | PI (D60) | | | | | | | | | | | | | | | | | | | T | | |
| | | | PI (D90) | | | | | | | | | | | | | t | | | | | | + | | F |
| | Control | <7 | PI (D30) | | | | | | | | | | | | | t | | | | | | + | | F |
| | Control | ' | PI (D60) | | | | | | | | | | | | | | | | | | | <u> </u> | | - |
| | | | PI (D90) | | | | | | | | | | | | | | | | | | | H | | H |
| | | [7-8] | PI (D30) | | | | | | | | | | | | | | | | | | | H | | H |
| | | [1-0] | PI (D60) | | | | | | | | | | | + | | | + | + | | | | ╁ | _ | H |
| | | | PI (D00) | | | | | | | | | | | - | | | | | | | | ╁ | | - |
| | | 10.01 | PI (D30) | | _ | | | | | | | | | + | | - | | - | | | | ╁ | <u> </u> | ┝ |
| | | ]8-9] | | | | | | | | | | | | | | | | + | | | | ₽ | | L |
| | | | PI (D60) | | | | | | | | | | | + | | - | | | | | | ╄ | _ | |
| | | 10.401 | PI (D90) | | | | | | | | | | | | | | | | | | | ╄ | | _ |
| | | ]9-10] | PI (D30) | | | | | | | | | | | | | | | | | | | ╄ | | _ |
| | | | PI (D60) | | | | | | | | | | | | | | | | | | | Ļ | _ | |
| | | | PI (D90) | | | | | | | | | | | | | | | | | | | L | | L |
| | | ]10-11] | PI (D30) | | | | | | | | | | | | | | | | | | | L | | |
| | | | PI (D60) | | | | | | | | | | | | | | | | | | | L | L | |
| | | | PI (D90) | | | | | | | | | | | | | | | | | | | L | | |
| | | ]11-12] | PI (D30) | | | | | | | | | | | | | | | | | | | | | |
| | | | PI (D60) | | | | | | | | | | | | | | | | | | | | | |
| | | | PI (D90) | | | | | | | | | | | | | | | | | | | | | |
| | | > 12 | PI (D30) | | | | | | | | | | | | | | | | | | | | | |
| | | | PI (D60) | | | | | | | | | | | T | | | | | | | | | | |
| | | | PI (D90) | T | | | П | | П | | 1 | | | t | | | | | | T | | T | | Г |
| | | Total | PI (D30) | T | | | H | | H | | $\dagger$ | | $\dagger$ | t | | t | | t | | | | T | | T |
| | | | PI (D60) | | | | H | | H | | $\dagger$ | | + | $\dagger$ | + | t | 1 | t | 1 | | | T | | H |
| | | | PI (D90) | + | 1 | | H | | H | | $\dagger$ | | $\dashv$ | $\dagger$ | + | $^{\dagger}$ | + | t | | t | | + | | H |

## <each group>:

30 PreF = 30 μg PreF 60 PreF = 60 μg PreF 120 PreF = 120 μg PreF

120 Fiel = 120 µg Fiel

Control = Placebo

N = number of subjects with available results

204812 (RSV F-021)

Statistical Analysis Plan Amendment 4 Final

n/% = number/percentage of subjects with titer within the specified range PI(D30) = Post-vaccination at Day 30

PI(D60) = Post-vaccination at Day 60 PI(D90) = Post-vaccination at Day 90

204812 (RSV F-021) Statistical Analysis Plan Amendment 4 Final

## Template 45 Distribution of fold of anti-RSV-A neutralising antibody titer by cumulative pre-vaccination titer category (Per protocol set)

| Antibody | Graun | Sub- | Timing | | <1<br> 0/ | | 1 | | | 2.5 | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Antibody | Group | | ıımıng | N ľ | 1 % | n | 70 | לוו | oIn | 1 % | n | 70 | n ' | /0 | n ' | /0 | II ( | ∕o r | 1 70 | n | 70 | n | , |
| Anti-RSV A Neutralizing | 30 PreF | group<br><7 | PI(D30) | | | | | | | | | | | | | | | | | | | | ٢ |
| Antibody | | | PI(D60) | | | | | | | | | | | | | | | | | | | | F |
| | | | PI(D90) | | | | | | t | | | | | | | | | | t | | | H | ľ |
| | | ≥7 | PI(D30) | | | | | | | | | | | | | | | | | | | H | İ |
| | | _' | PI(D60) | | | Н | | | | | | | | | | | | | | | | H | ŀ |
| | | | PI(D90) | | | H | | | | | | | | | | | t | | | | | | |
| | | ≥8 | PI(D30) | | | H | | | | | | | | | | | t | | | | | | |
| | | _0 | PI(D60) | | | H | | | | | | | | | | | t | | | | | | |
| | | | PI(D90) | | | H | | | | | | | | | | | | | | | | H | Ì |
| | | ≥9 | PI(D30) | | | Н | | | | | | | | | | | | | | | | H | ŀ |
| | | _5 | PI(D60) | | | H | | | | | | | | | | | | | | | | H | İ |
| | | | PI(D90) | | | Н | | | | | | | | | | | | | | | | H | ŀ |
| | | ≥10 | PI(D30) | | | Н | | | | | | | | | | | | | | | | H | ŀ |
| | | =10 | PI(D60) | | | Н | | | | | | | | | | | | | | | | H | ŀ |
| | | | PI(D90) | | | H | | | | | | | | | | | + | | | | | H | ŀ |
| | | ≥11 | PI(D30) | | | Н | | | | | | | | | | - | | | | | | H | ı |
| | | -11 | PI(D60) | | | H | | | | | | | | | | | + | | | | | | |
| | | | PI(D90) | | | Н | | | | | | | | | | | | | | | | | |
| | | Total | PI(D30) | | | Н | | | | | | | | | | | | | | | | | |
| | | Total | PI(D60) | | | H | | | | | | | | | | | t | | | | | <u> </u> | |
| | | | PI(D90) | | | Н | | | | | | | | | | | | | | | | | |
| | 60 PreF | <7 | PI(D30) | | | H | | | | | | | | | | | t | | | | | <u> </u> | |
| | 001101 | 1 | PI(D60) | | | | | | | | | | | | | | 1 | | | | | | |
| | | | PI(D90) | | | | | | | | | | | | | | 1 | | | | | | |
| | | ≥7 | PI(D30) | | | H | | | | | | | | | | | t | | | | | <u> </u> | |
| | | _' | PI(D60) | | | H | | | | | | | | | | | t | | | | | <u> </u> | |
| | | | PI(D90) | | | Н | | | | | | | | | | | | | | | | | |
| | | ≥8 | PI(D30) | | | | | | + | | | | | | | | | | + | | | H | ı |
| | | _0 | PI(D60) | | | H | | | | | | | | | | | t | | | | | | |
| | | | PI(D90) | | | H | | | | | | | | | | | t | | | | | H | Ì |
| | | ≥9 | PI(D30) | | | | | | + | | | | | | | | | | + | | | H | ŀ |
| | | _0 | PI(D60) | | | H | | | | | | | | | | | t | | | | | H | Ì |
| | | | PI(D90) | | | H | | | | | | | | | | | | | | | | H | Ì |
| | | ≥10 | PI(D30) | | | | | | | | | | | | | | | | | | | H | Ì |
| | | _10 | PI(D60) | | | H | | | | | | | | | | | | | | | | | |
| | | | PI(D90) | | | | | | | | | | | | | | 1 | | | | | H | Ì |
| | | Total | PI(D30) | | | | | | | | | | | | | | | | | | | H | Ì |
| | | Total | PI(D60) | | | H | | | | | | | | | | | | | | | | H | Ì |
| | | | PI(D90) | | | | | | | | | | | | | | | | | | | H | ľ |
| | 120 | <7 | PI(D30) | | | | | | | | | | | | | | | | | | | | Ì |
| | PreF | | (200) | | | | | | | | | | | | | | | | | | | | l |
| | 1.101 | | PI(D60) | | | | | | | | | | | | | | | | | | | | ſ |
| | | | PI(D90) | | | | | | | | | | | | | | | | | | | | ĺ |
| | | ≥7 | PI(D30) | | | | | | | | | | | | | | | | | | | | ſ |
| | | - | PI(D60) | | | H | | | $\dagger$ | | | | | | | + | + | | 1 | | | Ħ | ĺ |
| | | | PI(D90) | | | H | | $\top$ | $\dagger$ | | | | | | | + | + | | | | | H | ĺ |
| | | ≥8 | PI(D30) | | | Ħ | | $\dagger$ | Ť | | | | 1 | | 1 | 1 | 1 | | 1 | | | Ħ | ı |
| | | - | PI(D60) | | | H | | $\dagger$ | Ť | | | | 1 | | 1 | 1 | 1 | | | | | Ħ | ı |
| | | | PI(D90) | | 1 | | | | + | + | $\vdash$ | | H | | + | _ | $\dashv$ | 1 | + | + | | | |

## 204812 (RSV F-021)

### Statistical Analysis Plan Amendment 4 Final

| | | | | | | | 4 | ,ai , | | <u> </u> | \ A | Ť | | Ť | | | • | | ^ - | | ·· | ÷ |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | - | 1 | | | <1 | ≥ | 1 | ≥2 | ≥ | 2.5 | ≥3 | | ≥4 | 2 | ≥6 | ≥ | ğ | ≥1 | 0 2 | ≥11 | 2 | :1 |
| Antibody | Group | Sub- | Timing | N r | ۱ % | n | % | n % | n | % | n % | σr | ۱ % | n | % | n | % | n | % r | ۱ % | n | 1 |
| | | group | | | | | | | | | | | | | | | | | | | | |
| | | ≥9 | PI(D30) | | | | | | | | | | | | | | | | | | | |
| | | | PI(D60) | | | | | | | | | | | | | | | | | | | |
| | | | PI(D90) | | | | | | | | | | | | | | | | | | | |
| | | ≥10 | PI(D30) | | | | | | | | | | | | | | | | | | | |
| | | | PI(D60) | | | | | | | | | | | | | | | | | | | |
| | | | PI(D90) | | | | | | | | | | | | | | | | | | | Ī |
| | | ≥11 | PI(D30) | | | | | | | | | | | | | | | | | | | Ī |
| | | | PI(D60) | | | | | | | | | | | | | | | | | | | Ī |
| | | | PI(D90) | | | | | | | | | | | | | | | | | | | 1 |
| | | Total | PI(D30) | | | | | | | | | | | | | | | | | | | 1 |
| | | | PI(D60) | | | | | | | | | | | | | | | | | | | |
| | | | PI(D90) | | | | | | | | | | | | | | | | | | | |
| | Control | <7 | PI(D30) | | | | | | | | | | | | | | | | | | | |
| | | | PI(D60) | | | | | | | | | | | | | | | | | | | |
| | | | PI(D90) | | | | | | | | | | | | | | | | | | | |
| | | ≥7 | PI(D30) | | | | | | | | | | | | | | | | | | | |
| | | | PI(D60) | | | | | | | | | | | | | | | | | | | |
| | | | PI(D90) | | | | | | | | | | | | | | | | | | | |
| | | ≥8 | PI(D30) | | | | | | | | | | | | | | | | | | | 1 |
| | | | PI(D60) | | | | | | | | | | | | | | | | | | | 1 |
| | | | PI(D90) | | | | | | | | | | | | | | | | | | | 1 |
| | | ≥9 | PI(D30) | | | | | | | | | | | | | | | | | | | 1 |
| | | | PI(D60) | | | П | | | | | | T | | | | | | | | | | 1 |
| | | | PI(D90) | | | П | | | | | | T | | | | | | | | | | 1 |
| | | ≥10 | PI(D30) | | | П | | | | | | T | | | | | | | | | | 1 |
| | | | PI(D60) | | | | | | | | | | | T | | | | T | | | T | 1 |
| | | | PI(D90) | | | Ħ | | | | | | T | | | | | | 1 | | | | 1 |
| | | Total | PI(D30) | | | Ħ | | | | | | T | | | | | | 1 | | | | 1 |
| | | | PI(D60) | | | Ħ | | | | | | T | | | | | | 1 | | | | t |
| | | | PI(D90) | | | H | | | t | | | t | | t | H | | | $\dagger$ | | | t | † |

30 PreF = 30 μg PreF

60 PreF = 60 µg PreF

120 PreF = 120 µg PreF

Control = Placebo

<7 = Log2 results are less than 7 at pre-vaccination

≥7 = Log2 results are ≥7 at pre-vaccination

≥8 = Log2 results are ≥8 at pre-vaccination

≥9 = Log2 results are ≥9 at pre-vaccination

≥10 = Log2 results are ≥10 at pre-vaccination

≥11 = Log2 results are ≥11 at pre-vaccination

Total = all subjects with pre-vaccination result available

N = number of subjects with available results

n/% = number/percentage of subjects with titre within the specified range

PI(D30) = Post-vaccination at Day 30

PI(D60) = Post-vaccination at Day 60

PI(D90) = Post-vaccination at Day 90

Statistical Analysis Plan Amendment 4 Final

Template 46 Reverse cumulative distribution curves for anti-RSV-A neutralising antibody titers in each group at <each time point> (Per protocol set)



30 PreF = 30  $\mu$ g PreF 60 PreF = 60  $\mu$ g PreF

120 PreF = 120 µg PreF

Control = Placebo

Note: This graph is provided as an example. The same graph will be provided for each time point and each assay comparing the values of the groups:30 PreF, 60 PreF, 120 PreF and Control.

204812 (RSV F-021)

Statistical Analysis Plan Amendment 4 Final

Template 47 Individual results of anti-RSV-A neutralising antibody titer at Day <30/60/90> versus pre-vaccination in <each group> and Control (Per protocol set)



## <each group>:

30 PreF = 30 μg PreF

60 PreF = 60 μg PreF 120 PreF = 120 μg PreF

Control = Placebo

Note: This graph is provided as an example. The same graph will be generated for each assay and each timepoint separately (Day 30, 60, 90):

204812 (RSV F-021)

Statistical Analysis Plan Amendment 4 Final

## Template 48 Vaccine response for anti-RSV-A neutralising antibody titer at each post-vaccination timepoint (Per protocol set)

| | | | | | | Vaccine | respon | se* |
|---|---|---|---|---|---|---|---|---|
| | | | | | | | 9 | 5% CI |
| Antibody | Group | Post-vaccination timing | Pre-vaccination category (log2) | N | n | % | LL | UL |
| <each<br>antibody&gt;</each<br> | <each group=""></each> | PI(D30) | <7 | | | | | |
| | | | [7-8] | | | | | |
| | | | ]8-10] | | | | | |
| | | | >10 | | | | | |
| | | | Total | | | | | |
| | | PI(D60) | <7 | | | | | |
| | | | [7-8] | | | | | |
| | | | ]8-10] | | | | | |
| | | | >10 | | | | | |
| | | | Total | | | | | |
| | | PI(D90) | <7 | | | | | |
| | | | [7-8] | | | | | |
| | | | ]8-10] | | | | | |
| | | | >10 | | | | | |
| | | | Total | | | | | |

### <each group>:

30 PreF = 30 µg PreF

60 PreF = 60 µg PreF

120 PreF = 120 µg PreF

Control = Placebo

Total = all subjects with pre-vaccination result available

\*Vaccine response defined as:

For subjects with pre-vaccination titer <7 log2: antibody titer at post-vaccination>= 4 fold the pre-vaccination antibody titer For subjects with pre-vaccination titer in [7-8] log2: antibody titer at post-vaccination >= 3 fold the pre-vaccination antibody titer For subjects with pre-vaccination titer in [8-10] log2: antibody titer at post-vaccination >= 2.5 fold the pre-vaccination antibody titer For subjects with pre-vaccination titer >10 log2: antibody titer at post-vaccination >= 1 fold the pre-vaccination antibody titer

N = number of subjects with both pre- and post-vaccination results available

n/% = number/percentage of responders

95% CI = exact 95% confidence interval, LL = Lower Limit, UL = Upper Limit

PI(D30) = Post-vaccination at Day 30

PI(D60) = Post-vaccination at Day 60

PI(D90) = Post-vaccination at Day 90

204812 (RSV F-021)

Statistical Analysis Plan Amendment 4 Final

## Template 49 Estimated GMTs and 95% CIs for anti-RSV-A neutralising antibody titre (Per protocol set)

| | | | | Est | imate | d GMT |
|---|---|---|---|---|---|---|
| | | | | | 9 | 5% CI |
| Antibody | Group | Timing | N | value | LL | UL |
| Anti-RSV-A | <each< td=""><td>PRE</td><td></td><td></td><td></td><td></td></each<> | PRE | | | | |
| Neutralizing | group> | | | | | |
| Antibody | | | | | | |
| • | | PI(D30) | | | | |
| | | PI(D60) | | | | |
| | | PI(D90) | | | | |

<each group>:

 $30 \text{ PreF} = 30 \mu \text{g PreF}$ 

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

GMT = geometric mean antibody titer estimated by the ANOVA model for repeated measures

N = Number of subjects with available results

95% CI = 95% confidence interval (ANOVA model); LL = lower limit, UL = upper limit

PRE= Pre-vaccination at Day 0

PI(D30) = Post-vaccination at Day 30

PI(D60) = Post-vaccination at Day 60

PI(D90) = Post-vaccination at Day 90

## Template 50 Exploratory comparisons (GMT ratios) between RSV groups with corresponding 95% confidence interval for anti-RSV A neutralizing antibody titre at Day 30 (Per protocol set)

| | | | | | | | | GI | /IT ratio | 0 | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | | Tukey's | 95% CI |
| Antibody | Timepoint | Group | N | <b>GMT</b> | Group | N | <b>GMT</b> | Ratio order | Value | LL | UL |
| | - | description | | | description | | | | | | |
| Anti-RSV A | PI(D30) | 120 PreF | | | 30 PreF | | | 120 PreF/30 PreF | | | |
| Neutralizing | , , | 120 PreF | | | 60 PreF | | | 120 PreF/60 PreF | | | |
| Antibody | | 60 PreF | | | 30 PreF | | | 60 PreF/30 PreF | | | |

30 PreF = 30 µg PreF

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

antibody titre estimated by the ANCOVA model

N = Number of subjects with pre-vaccination results available

Tukey's 95% CI = 95% confidence interval for the GMT ratio (ANCOVA model, Tukey's adjustment), LL = lower limit, UL = upper limit

Pvalue of ANCOVA model is xxxx

PI(D30) = Post-vaccination at Day 30

Statistical Analysis Plan Amendment 4 Final

Template 51 Individual kinetics of anti-neogenin antibody concentrations by group (Exposed set)



 $30 \text{ PreF} = 30 \mu \text{g PreF}$ 

60 PreF = 60 µg PreF

120 PreF = 120 µg PreF

Control = Placebo

Note: This graph is provided as an example. This graph will display the 4 groups and the 4 immuno timepoints: PRE, PI(D30), PI(D60) and PI(D90)

204812 (RSV F-021)

Statistical Analysis Plan Amendment 4 Final

# Template 52 GM of individual ratios (fold increase post over pre) and their 95% Cls for anti-RSV F IgG1 and IgG total antibody assays and each group, at <Day xx> (Per protocol set)



 $30 \text{ PreF} = 30 \mu \text{g PreF}$ 

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Control = Placebo

Note: this graph is provided as an example. It will be adapted to display IgG total and Ig1 only, and the 4 groups: 30 PreF, 60 PreF, 120 PreF, Control.

204812 (RSV F-021)

Statistical Analysis Plan Amendment 4 Final

# Template 53 Exploratory comparisons (GM ratios of fold increase post/pre) between RSV groups with corresponding 95% confidence interval for anti-RSV F antibody concentrations (IgG Total) at Day 30 (Per protocol set)

| | | | | | | | G | MF rati | 0 | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | | ukey s<br>05% CI |
| Antibody | Timepoint | Group description | N | Group description | N | GMF | Ratio order | Value | LL | UL |
| anti-RSV F antibody<br>(IgG Total) | PI(D30) | 120 PreF | | 60 PreF | | | 120 Pre/60<br>PreF | | | |
| , | | 120 PreF | | 30 PreF | | | 120 PreF/30<br>PreF | | | |
| | | 60 PreF | | 30 PreF | | | 60 PreF/30<br>PreF | | | |

30 PreF = 30 μg PreF

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 µg PreF

Antibody concentration estimated by the ANOVA model

GMF = Geometric mean of fold increase

N = Number of subjects with pre-vaccination results available

Tukey's 95% CI = 95% confidence interval for the GMF ratio (ANOVA model, Tukey's adjustment), LL = lower limit, UL = upper limit

Pvalue of ANOVA model at PI(D30) is: xxxx

PI(D30) = Post-vaccination at Day 30

204812 (RSV F-021)

Statistical Analysis Plan Amendment 4 Final

# Template 54 Comparisons of GM ratios with corresponding 95% confidence interval between anti-RSV F antibody concentrations (IgG Total) and anti-RSV-A neutralising antibody titers at pre-vaccination (Per protocol set)

| | | | | | | | | | GN | / rati | 0 |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | 959 | % CI | | 95% | 6 CI | | 95% | % CI |
| Timing | Group<br>description | N | IgG Total<br>GMC | LL | UL | RSV-A neut<br>GMT | LL | UL | Value | LL | UL |
| PRE(D0) | <each group=""></each> | | | | | | | | | | |
| PRE(D0) | | | | | | | | | | | |
| PRE(D0) | | | | | | | | | | | |
| PRE(D0) | | | | | | | | | | | |

<each group>:

30 PreF = 30 μg PreF

 $60 \text{ PreF} = 60 \mu \text{g PreF}$ 

120 PreF = 120 μg PreF

Control = Placebo

N = Number of subjects with available results at Day30 and pre-vaccination for IgG Total and RSV-A neut

GMC = Geometric mean antibody concentration calculated on all subjects for IgG Total

GMT = Geometric mean antibody titre calculated on all subjects for RSV-A neut

GM Ratio=Geometric mean of individual ratio of IgG Total to RSV-A neut for each group

95% CI = 95% confidence interval; LL = lower limit, UL = upper limit

PRE= Pre-vaccination at Day 0

204812 (RSV F-021)

Statistical Analysis Plan Amendment 4 Final

# Template 55 Exploratory comparisons (GM ratios of fold increase post/pre) with corresponding 95% confidence interval between anti-RSV F antibody concentrations (IgG Total) and anti-RSV-A neutralising antibody titers at Day 30 (Per protocol set)

| | | | | | | | | | GN | IF Rai | tio |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | | 95 | % CI |
| Timepoint | Group | N | IgG Total | 95% | CI | RSV-A neut | 95% | | Value | LL | UL |
| - | | | ĞMF | LL | UL | GMF | LL | UL | | | |
| PI(D30)/PRE | <each group=""></each> | | | | | | | | | | |
| PI(D30)/PRE | | | | | | | | | | | |
| PI(D30)/PRE | | | | | | | | | | | |
| PI(D30)/PRE | | | | | | | | | | | |

<each group>:

30 PreF = 30 μg PreF

60 PreF = 60 μg PreF

120 PreF = 120 µg PreF

Control = Placebo

N = Number of subjects with available results at the two considered time points for IgG Total and anti-RSV-A GMF = Geometric mean of fold increase

GMF Ratio= Geometric mean of individual ratio of fold increase for each group

95% CI = 95% confidence interval; LL = lower limit, UL = upper limit

PRE= Pre-vaccination at Day 0

PI(D30) = Post-vaccination at Day 30

204812 (RSV F-021)

Statistical Analysis Plan Amendment 4 Final

## Template 56 Desirability index of immunogenicity during the 30-day (Days 0-29) post-vaccination period (Per protocol set)

| Group | GMT | LL1 | DI1 | GMC | LL2 | DI2 | DI |
|---|---|---|---|---|---|---|---|
| <each< td=""><td></td><td></td><td></td><td></td><td></td><td></td><td></td></each<> | | | | | | | |
| group> | | | | | | | |

<each group>:

30 PreF = 30 μg PreF

60 PreF = 60 μg PreF

120 PreF = 120 µg PreF

Control = Placebo

GMT = estimated log2-scale GMT adjusted for pre-vaccination titres for neutralising anti-RSV-A

GMC = estimated log10-scale GMC adjusted for pre-vaccination concentrations for PCA

LL1 = estimated log2-scale lower limit adjusted for pre-vaccination titres for neutralising anti-RSV-A

LL2 = estimated log10-scale lower limit adjusted for pre-vaccination concentrations for PCA

DI1 = desirability index for neutralising anti-RSV-A

DI2 = desirability index for PCA concentrations

DI = immunogenicity index

## Template 57 Desirability index of reactogenicity during the 7-day (Days 0-6) post-vaccination period (Exposed set)

| Group | Incidence Rate<br>(I民 ) | Incidence Rate<br>(IR2) | DR1 | DR2 | DR |
|---|---|---|---|---|---|
| <each group=""></each> | | | | | |

<each group>:

30 PreF = 30 μg PreF

60 PreF = 60 μgPreF

120 PreF = 120 µg PreF

Control = Placebo

IR = incidence rate estimated by the model for any Grade 2/3 general AEs and any related SAEs

IR2 = incidence rate estimated by the model for Grade 2/3 fever

DR1 = desirability index for any Grade 2/3 general AEs and any related SAEs

DR2 = desirability index for Grade 2/3 fever

DR = reactogenicity index

204812 (RSV F-021)

Statistical Analysis Plan Amendment 4 Final

## Template 58 Desirability index based on reactogenicity and safety (Exposed set up to Day 7) and immunogenicity (Per protocol set up to Day 30)

| Group | Reactogenicity Index | | | Immunogenicity Index | | | Overall Desirability Index |
|---|---|---|---|---|---|---|---|
| | DR1 | DR2 | DR | DI1 | DI2 | DI | DR <sup>0.4</sup> * DI <sup>0.6</sup> |
| <each group=""></each> | | | | | | | |

<each group>:

30 PreF = 30 μg PreF

60 PreF = 60 μg PreF

120 PreF = 120 μg PreF

Control = Placebo

DR1 = desirability index for any Grade 2/3 general AEs and any related SAEs

DR2 = desirability index for Grade 2/3 fever

DR = reactogenicity index

DI1 = desirability index for neutralising anti-RSV-A

DI2 = desirability index for PCA concentrations

DI = immunogenicity index

204812 (RSV F-021)

Statistical Analysis Plan Amendment 4 Final

Template 59 Percentage of subjects reporting solicited local symptoms (any grade / grade 3) during the 7-day post-vaccination period (Exposed set)



30 PreF = 30 μg PreF 60 PreF = 60 μg PreF 120 PreF = 120 μg PreF Control = Placebo